

#### **CLINICAL PROTOCOL**

PROTOCOL NUMBER: LUM001-304

#### **ICONIC STUDY**

LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BLIND, PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN APICAL SODIUM-DEPENDENT BILE ACID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH ALAGILLE SYNDROME

Protocol Amendment 5.1: 08 February 2019

**Protocol** History

Protocol Amendment 5: 06 Nov 2017

Protocol Amendment 4: 28 Mar 2017

Protocol Amendment 3: 13 Nov 2015 Protocol Amendment 2:

08 May 2015

Protocol Amendment 1: 06 Mar 2015

Original Protocol: 20 Mar 2014

Mirum Pharmaceuticals, Inc. 70 Willow Road, Suite 200 Menlo Park, California 94025 **United States** 

#### CONFIDENTIAL

This document is a confidential communication of Mirum Pharmaceuticals, Inc. It is agreed that no unpublished information contained herein will be published or disclosed without prior approval from the sponsor. However, this document can be disclosed to an appropriate Independent Ethics Committee/Institutional Review Board (IEC/IRB) or authorized representatives of national regulatory authorities under the condition that they respect its confidential information.

#### **SPONSOR SIGNATURE PAGE**

## LUM001-304

### **ICONIC STUDY**

LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BLIND, PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN APICAL SODIUM-DEPENDENT BILE ACID TRANSPORTER INHIBITOR (ASBTI), IN PATIENTS WITH ALAGILLE SYNDROME

Protocol Amendment 5.1: 08 February 2019

**Protocol History** 

Protocol Amendment 5: 06 Nov 2017

Protocol Amendment 4: 28 Mar 2017

Protocol Amendment 3: 13 Nov 2015

Protocol Amendment 2: 08 May 2015

Protocol Amendment 1: 06 Mar 2015

Original Protocol: 20 Mar 2014

Sponsor: Mirum Pharmaceuticals, Inc.

70 Willow Road, Suite 200 Menlo Park, California 94025 USA

#### **TITLE PAGE**

Study Drug: LUM001

**Protocol Number:** LUM001-304

**Protocol Amendment:** 5.1

**Date:** 08 February 2019

**EudraCT No:** 2013-005373-43

Study Phase: 2

**Protocol Title:** Long-Term, Open-Label Study with a Double-Blind,

Placebo-Controlled, Randomized Drug Withdrawal Period of LUM001, an Apical Sodium-Dependent Bile Acid Transporter

Inhibitor (ASBTi), in Patients with Alagille Syndrome

**Sponsor:** Mirum Pharmaceuticals, Inc.

70 Willow Road, Suite 200 Menlo Park, California 94025

**USA** 

Medical Monitor: Cagil Ozen, MD

Premier Research

Office: +1 215 282 5406 Cell: +1 267 838 2380

Email: medmonitorLUM304@premier-research.com

Medical Lead: Thomas Jaecklin, MD

Mirum Pharmaceuticals AG Innere Margarethenstrasse 5

4051 Basel Switzerland

Phone: +41(0) 79 850 77 18

Email: tjaecklin@mirumpharma.com

Compliance Statement: This study will be conducted in accordance with all applicable

clinical research guidelines including the International Conference on Harmonization (ICH) Guidelines for current Good Clinical Practice (GCP). Study documents will be maintained in accordance with

applicable regulations.

Investigator's Name (Please print)

## CONFIDENTIAL

Page 4

08 February 2019

# PROTOCOL SIGNATURE PAGE

| Sponsor's (Mirum) | Approval | |
|---|---|---|
| Signature: Date: 10.2.2019 | | |
| Thomas Jaecklin, MI | | |
| SVP Clinical Develop | ent | |
| I agree to conduct thi and also in accordance | | equirements of this clinical study protocol |
| <ul> <li>Declaration of Helsinki (Oct 2008)</li> <li>Established principles of Good Clinical Practice (ICH E6; GCP) (Harmonized)</li> <li>US Code of Federal Regulations (CFR); Food and Drug Administration (FDA) (where applicable)</li> <li>European Union (EU) Directives and national laws (where applicable)</li> </ul> | | |
| Clinical Study Title: | | |
| CONTROLLED, RAAAPICAL SODIUM-D | | AWAL PERIOD OF LUM001, AN<br>NSPORTER INHIBITOR (ASBTi), IN |
| Protocol: | Amendment 5.1 | |
| Date: | 08 February 2019 | |
| EudraCT No: | 2013-005373-43 | |
| Sponsor: Mirum Pharmaceuticals, Inc. 70 Willow Road, Suite 200 Menlo Park, California 94025 | | |
| | USA | |
| As Agreed: | | |
| Investigator's Signa | ture | Date |

#### **EMERGENCY CONTACT INFORMATION**

In the event of a serious adverse event (SAE), the investigator must fax or e-mail the Premier Research Serious Adverse Event Form within 24 hours to the Premier Research Pharmacovigilance Department. Applicable fax numbers and e-mail address can be found on the form (sent under separate cover) and below.

# **Premier Research SAE Reporting:**

US and Canadian sites: fax 215-972-8765, or e-mail GlobalPV-US@premier-research.com

EU/ROW sites: fax +421 2 6820 3713 or e-mail PVDS-ROW@premier-research.com

For all urgent protocol- or safety-related issues during and outside of business hours, the investigator must contact the Premier Research Medical Monitor:

Cagil Ozen, MD, Medical Director

North America (US and Canada) sites:

Central phone number: +1 512 686 1256 (US)

**European and ROW sites:** 

Central phone number: +44 118 936 4096 (United Kingdom)

For non-emergencies, the Premier Research Medical Monitor may be contacted by e-mail: medmonitorLUM304@premier-research.com

## PRODUCT QUALITY COMPLAINTS

Investigators are required to report investigational product quality complaints to Mirum within 24 hours. This includes any instances wherein the quality or performance of a Mirum product (marketed or investigational) does not meet expectations (eg, inadequate or faulty closure, product contamination) or that the product did not meet the specifications defined in the application for the product (eg, wrong product such that the label and contents are different products). For instructions on reporting AEs related to product complaints, see Section 11.

Please use the information below as applicable to report the Product Quality Complaint:

| Origin of Product Quality Complaint | E-mail Address |
|-------------------------------------|-------------------------|
| North and South America | medinfo@mirumpharma.com |
| European Union and Rest of World | medinfo@mirumpharma.com |

Telephone numbers (provided for reference if needed):

Mirum, Menlo Park, CA (USA)

1-650-667-4085

# TABLE OF CONTENTS

| SPON | SOR SIGNATU | RE PAGE | 2 |
|---|---|---|---|
| TITLE | PAGE | | 3 |
| PROT | OCOL SIGNAT | TURE PAGE | 4 |
| PROD | UCT QUALITY | COMPLAINTS | 6 |
| TABL | E OF CONTEN | TS | 7 |
| LIST ( | OF TABLES | | 12 |
| LIST ( | OF FIGURES | | 13 |
| PROT | OCOL AMEND | MENT 5.1 SUMMARY OF CHANGES | 14 |
| 1 SY | YNOPSIS | | 17 |
| 2 LI | ST OF ABBRE | VIATIONS AND TERMS | 35 |
| 3 S7 | ГUDY OBJECT | IVES | 39 |
| 4 B | ACKGROUND | AND RATIONALE | 40 |
| 4.1 | Therapeu | tic Rationale | 40 |
| 4.2 | Alagille S | Syndrome | 41 |
| 4.3 | Pruritus. | | 41 |
| 4.4 | LUM001 | | 42 |
| | 4.4.1 Nonclin | nical Studies | 42 |
| | 4.4.1.1 | Pharmacology | 42 |
| | 4.4.1.2 | Pharmacokinetics | 43 |
| | 4.4.1.3 | Toxicology | 43 |
| | 4.4.2 Previou | s Clinical Experience | 44 |
| 4.5 | Rationale | e for Dose and Schedule of Administration | 45 |
| 5 IN | <b>VESTIGATION</b> | NAL PLAN | 48 |
| 5.1 | Study De | sign | 48 |
| 5.2 | Data Mor | nitoring Committee | 48 |
| 5.3 | Number | of Study Centers | 48 |
| 5.4 | Number | of Subjects | 48 |
| 5.5 | Overall S | Study Duration and Follow-up | 48 |
| | 5.5.1 Screeni | ng | 54 |
| | 5.5.2 Treatme | ent | 54 |
| | 5.5.2.1 | Dose Escalation Period | 55 |
| | 5.5.2.2 | Stable Dosing Treatment Period | 56 |
| | 5.5.2.3 | Double-blind Placebo-controlled Study Drug Withdrawal Period | 56 |
| | 5.5.2.4 | Long-term Exposure Period | 56 |
| | 5.5.2.5 | 52-week Optional Follow-up Treatment Period | 56 |

| | 5. | 5.2.6 Long-term Optional Follow-up Treatment Period | 57 |
|---|---|---|---|
| | 5.5.3 | Safety Follow-up Period | 58 |
| | 5.6 | End of Study | 58 |
| 6 | SUBJEC | T ENROLLMENT | 60 |
| | 6.1 | Screening | 60 |
| | 6.2 | Randomization | 60 |
| | 6.3 | Replacement of Subjects | 60 |
| | 6.4 | Unblinding of Treatment Assignment | 61 |
| 7 | SUBJEC | T ELIGIBILITY | 62 |
| | 7.1 | Inclusion Criteria | 62 |
| | 7.2 | Exclusion Criteria | 62 |
| 8 | STUDY | PROCEDURES | 65 |
| | 8.1 | Study Schedule | 65 |
| | 8.1.1 | Screening Period (Day -28 to Day -1) | 65 |
| | 8.1.2 | Dose Escalation Treatment Period (Day 0 to Week 6) | 65 |
| | 8.1.3 | Stable Dosing Treatment Period (Week 7 to Week 18) | 66 |
| | 8.1.4 | Double-blind, Placebo-controlled Study Withdrawal Period (Week 19 to Week 22) | 66 |
| | 8.1.5 | Long-term Exposure Period (Week 23 to Week 48) | 67 |
| | 8.1.6 | Week 48 | 67 |
| | 8.1.7 | Early Termination for Subjects without Participation in the 52-week Optional Follow-up Treatment Period | 68 |
| | 8.1.8 | 52-week Optional Follow-up Treatment Period | |
| | 8.1.9 | Long-term Optional Follow-up Treatment Period | |
| | 8.1.10 | End of Treatment or Early Termination | |
| | | Safety Follow-up Period | |
| | | Genetic Testing | |
| | 8.3 | Physical Examination, Weight and Height, Vital Signs | 73 |
| | | Laboratory Assessments | |
| | 8.5 | Pruritus and Quality of Life Assessments | 74 |
| | 8.5.1 | Itch Reported Outcome (ItchRO <sup>TM</sup> ) | 74 |
| | 8.5.2 | Clinician Scratch Scale | 75 |
| | 8.5.3 | Clinician Xanthoma Scale | 75 |
| | 8.5.4 | Pediatric Quality of Life Inventory (PedsQL) | 75 |
| | 8.5.5 | Patient Impression of Change | |
| | 8.5.6 | Caregiver Impression of Change | 76 |
| | 8.5.7 | Caregiver Global Therapeutic Benefit | 76 |
| | 8.5.8 | Palatability | 76 |

| | 8.6 Restriction on the Lifestyle of Subjects | 76 |
|----|------------------------------------------------------------------|----|
| | 8.6.1 Contraception Requirements | 76 |
| | 8.6.2 Fasting Requirements | 77 |
| 9 | STUDY DRUG | 78 |
| | 9.1 Study Drug Description | 78 |
| | 9.1.1 LUM001 | 78 |
| | 9.1.2 Placebo | 78 |
| | 9.2 Packaging and Labeling | 79 |
| | 9.3 Drug Accountability | 79 |
| 10 | TREATMENT OF SUBJECTS | 80 |
| | 10.1 Study Drug Administration | 80 |
| | 10.2 Treatment Compliance | 81 |
| | 10.3 Concomitant Medications | 81 |
| | 10.4 Other Protocol-required Drugs | 81 |
| | 10.5 Safety Monitoring Rules | 81 |
| | 10.5.1 General Monitoring Rules | 81 |
| | 10.5.2 Safety Monitoring Rules | 82 |
| | 10.5.2.1 Safety Monitoring for Liver Chemistry Tests | 83 |
| | 10.5.2.2 Stopping Rules for Liver Chemistry Elevations | 84 |
| | 10.5.2.3 Safety Monitoring for Triglycerides | 84 |
| | 10.5.2.4 Safety Monitoring for Fat Soluble Vitamins | 84 |
| | 10.5.2.5 Monitoring/Stopping Rules for Coagulation Panel Results | 84 |
| | 10.6 Adjustment of Dose | 84 |
| | 10.7 Withdrawal of Subjects from the Study | 85 |
| 11 | SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING | 86 |
| | 11.1 Regulatory Requirements | 86 |
| | 11.2 Definitions | 86 |
| | 11.2.1 Adverse Event | 86 |
| | 11.2.2 Adverse Reaction and Suspected Adverse Reaction | 87 |
| | 11.2.3 Serious Adverse Event (SAE) | 87 |
| | 11.3 Monitoring and Recording Adverse Events | 88 |
| | 11.3.1 Serious Adverse Events | 88 |
| | 11.3.2 Non-serious Adverse Events | 88 |
| | 11.3.3 Evaluation of Adverse Events (Serious and Non-Serious) | 89 |
| | 11.3.3.1 Relationship to the Study Drug | 89 |
| | 11.3.3.2 Severity | 89 |
| | 11.3.3.3 Action Taken with Study Drug | 90 |
| | 11.3.3.4 Treatment Given for Adverse Event | 90 |

| | 11.3 | .3.5 Outcome of the Adverse Event | 90 |
|---|---|---|---|
| | 11.4 Pr | ocedures for Handling Special Situations | 90 |
| | 11.4.1 I | Pregnancy Reporting | 91 |
| | 11.4.2 I | Oosing Errors | 91 |
| | 11.4.3 A | Abnormalities of Laboratory Tests | 91 |
| 12 | | CAL CONSIDERATIONS | |
| | 12.1 Sa | imple Size Considerations | 93 |
| | 12.2 Pc | ppulations | 93 |
| | 12.2.1 \$ | Safety Population | 93 |
| | 12.2.2 I | Efficacy Populations | 93 |
| | 12.2.3 \$ | Siblings 93 | |
| | 12.2.4 I | Demographic and Baseline Characteristics | 94 |
| | 12.2 | .4.1 Subject Disposition | 94 |
| | 12.2 | .4.2 Baseline Data | 94 |
| | 12.2.5 H | Efficacy Analyses | 94 |
| | 12.2 | .5.1 Efficacy Variables | 94 |
| | 12.2 | .5.2 Primary Efficacy Analysis | 96 |
| | 12.2 | | |
| | 12.2.6 \$ | Safety Analyses | 97 |
| | 12.2 | .6.1 Safety Assessments | 97 |
| | 12.2.7 I | Planned Method of Analysis | 97 |
| | 12.2.8 \$ | Safety Analysis | 97 |
| | 12.2 | .8.1 Adverse Events | 97 |
| | 12.2 | .8.2 Laboratory Tests | 98 |
| | 12.2 | .8.3 Physical Exams, Vital Signs and Weight/Height Measurements | 98 |
| | 12.2 | .8.4 Concomitant Medications | 98 |
| | 12.2 | .8.5 Study Drug Exposure | 99 |
| | 12.2 | .8.6 Serum Alpha-fetoprotein | 99 |
| | 12.2.9 I | Palatability Analyses | 99 |
| | 12.2.10 | Interim Analyses | 99 |
| | 12.2.11 | Additional Analyses | 99 |
| 13 | INVESTIG | ATOR'S REGULATORY OBLIGATIONS | 100 |
| | 13.1 In | formed Consent | 100 |
| | 13.2 St | udy Personnel | 100 |
| | 13.3 Et | hical Conduct of the Study | 101 |
| | 13.4 In | dependent Ethics Committee/Institutional Review Board | 101 |
| | 13.5 Co | onfidentiality | 101 |
| 14 | ADMINIST | FRATIVE AND LEGAL OBLIGATIONS | 103 |

| | 14.1 | Pre-study Documentation Required | .103 |
|---|---|---|---|
| | 14.2 | Protocol Amendments | .103 |
| | 14.3 | Study Termination | .103 |
| | 14.4 | Study Documentation and Storage | .104 |
| | 14.5 | Study Monitoring | .104 |
| | 14.6 | Language | .105 |
| | 14.7 | Compensation for Injury | .105 |
| 15 | REFER | ENCES | .106 |
| 16 | APPEN | DICES | .107 |
| | 16.1 | Schedule of Procedures | .108 |
| | 16.1. | 1 Schedule of Procedures A-D: Study Entry – Week 96 | .109 |
| | 16.1. | 2 Schedule of Procedures E-F: Rollover under Protocol Amendment 4 | .118 |
| | 16.1. | Schedule of Procedures G-I: Subject Re-Entry under Protocol Amendment 4 123 | |
| | 16.1. | 4 Schedule of Procedures J – Study Termination and End of Treatment Procedures | .130 |
| | 16.2 | List of Laboratory Analytes | .132 |
| | 16.3 | Alagille Syndrome Diagnostic Criteria | |
| | 16.4 | Itch Reported Outcome Instrument (ItchRO <sup>TM</sup> ) | |
| | 16.4. | 1 Patient Itch Reported Outcome Instrument, ItchRO(Pt) <sup>TM</sup> | |
| | 16.4. | 2 Observer Itch Reported Outcome Instrument, ItchRO(Obs) <sup>TM</sup> | .137 |
| | 16.5 | Clinician Scratch Scale | .139 |
| | 16.6 | Clinician Xanthoma Scale | .141 |
| | 16.7 | Pediatric Quality of Life Inventory (PedsQL <sup>TM</sup> ) | .142 |
| | 16.7. | Parent Report for Infants (1 to 12 months) | .143 |
| | 16.7. | 2 Parent Report for Infants (13 to 24 months) | .146 |
| | 16.7. | 3 Parent Report for Toddlers (ages 2-4) | .149 |
| | 16.7. | 4 Parent Report for Young Children (ages 5-7) | .151 |
| | 16.7. | 5 Parent Report for Children (ages 8-12) | .153 |
| | 16.7. | 6 Parent Report for Teenagers (ages 13-18) | .155 |
| | 16.7. | 7 Pediatric Quality of Life Inventory v 4.0 for Young Children (ages 5-7) | .157 |
| | 16.7. | 8 Pediatric Quality of Life Inventory for Children (ages 8-12) | .160 |
| | 16.7. | 9 Pediatric Quality of Life Inventory for Teenagers (ages 13-18) | .162 |
| | 16.7. | Multidimensional Fatigue Scale Parent Report for Toddlers (ages 2-4) 164 | |
| | 16.7. | Multidimensional Fatigue Scale Parent Report for Young Children | |
| | | (ages 5-7) | .166 |

| 16.7.12<br>8 | Multidimensional Fatigue Scale Parent Report for Children (ages 1-12) 168 | |
|---|---|---|
| 16.7.13 | Multidimensional Fatigue Scale Parent Report for Teenagers (age 3-18) 170 | S |
| 16.7.14 | Multidimensional Fatigue Scale Young Child Report (ages 5-7) | 172 |
| 16.7.15 | Multidimensional Fatigue Scale Child Report (ages 8-12) | 175 |
| 16.7.16 | Multidimensional Fatigue Scale Teen Report (ages 13-18) | 177 |
| 16.7.17 | Family Impact Module v 2.0 | 179 |
| 16.8 Pa | tient Impression of Change (PIC) | 182 |
| 16.9 Ca | regiver Impression of Change (CIC) | 183 |
| 16.10 Ca | regiver Global Therapeutic Benefit (CGTB) | 185 |
| 16.11 Co | ommon Terminology Criteria for Adverse Events (CTCAE) Version 4.0 | 186 |
| 16.12 Pa | latability Questionnaire | 267 |
| 16.13 Pro | otocol History | 269 |
| 16.13.1 | Protocol Amendment 5 Summary of Changes | 269 |
| 16.13.2 | Protocol Amendment 4 Summary of Changes | 271 |
| 16.13.3 | Protocol Amendment 3 Summary of Changes | 293 |
| 16.13.4 | Protocol Amendment 2 Summary of Changes | 306 |
| 16.13.5 | Protocol Amendment 1 Summary of Changes | 308 |
| | LIST OF TABLES | |
| Table 1: | Improvement in Biochemical Markers and Pruritus After Partial External Biliary Diversion in PFIC Disease and Alagille Syndrome Subjects | 42 |
| Table 2: | Sample Daily Exposure (mg/day) in Pediatric Subjects | 45 |
| Table 3: | GI-associated Adverse Events in Study 003 | |
| Table 4: | Composition of LUM001 1.0 mL Oral Solution | 78 |
| Table 5: | Composition of LUM001 0.5 mL Oral Solution | 78 |
| Table 6: | Composition of LUM001 0.25 mL Oral Solution | 78 |
| Table 7: | Composition of Placebo 1.0 mL Oral Solution | 79 |
| Table 8: | Composition of Placebo 0.5 mL Oral Solution | 79 |
| Table 9: | Composition of Placebo 0.25 mL Oral Solution | 79 |

# LIST OF FIGURES

| Figure 1: | Interruption of Enterohepatic Circulation with an ASBT/IBAT Inhibitor | 40 |
|---|---|---|
| Figure 2: | Serum Bile Salt Concentration and Degree of Itch | 42 |
| Figure 3: | Study Design for LUM001-304 (Day 0 – Week 48) | 49 |
| Figure 4: | 52-week Optional Follow-up Treatment Scheme (<7 days from last LUM001 dose) | 50 |
| Figure 5: | 52-week Optional Follow-up Treatment Scheme (≥7 days from last LUM001 dose) | 51 |
| Figure 6: | Long-term Optional Follow-up Treatment Scheme (≥7 days from Last LUM001 Dose between Protocol Amendment 3 and Protocol Amendment 4) | 52 |
| Figure 7: | Long-term Optional Follow-up Treatment Scheme, without Afternoon Dose Escalation (ADE) | 53 |
| Figure 8: | Long-term Optional Follow-up Treatment Scheme under Protocol<br>Amendment 4, with Afternoon Dose Escalation (ADE) | 54 |

**08 February 2019** 

#### PROTOCOL AMENDMENT 5.1 SUMMARY OF CHANGES

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BLIND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN API<u>C</u>AL S<u>O</u>DIUM-DEPE<u>N</u>DENT B<u>I</u>LE A<u>C</u>ID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 5.1

Date: 08 February 2019

The LUM001-304 protocol is being amended to reflect the change of sponsorship from Lumena Pharmaceuticals LLC (Lumena Pharmaceuticals LLC is an indirect wholly-owned subsidiary of Shire North American Group, Inc) to Mirum Pharmaceuticals, Inc.

The following changes have been made to the Protocol Amendment 5 (06 Nov 2017). Note that correction of typographical and grammatical errors are not captured in the below table.

| Section | | Description of Change |
|---|---|---|
| Cover page,<br>Sponsor;<br>Title Page, Sponsor;<br>Sponsor Signature<br>Page, Sponsor;<br>Protocol Signature<br>page, Sponsor | Changed from: | Lumena Pharmaceuticals LLC* 300 Shire Way Lexington, MA 02421 USA *Lumena Pharmaceuticals LLC is an indirect wholly-owned subsidiary of Shire North American Group, Inc |
| | То: | Mirum Pharmaceuticals, Inc. |
| | | 70 Willow Road, Suite 200<br>Menlo Park, California 94025<br>USA |
| Title Page, Medical | Changed from: | |
| Lead;<br>Protocol Signature<br>page, Sponsor<br>(Mirum) Approval | Medical Lead: | Thomas Jaecklin, MD, MSc Shire Zahlerweg 10 6300 Zug Switzerland Phone: +41(0) 79 850 77 18 Email: thomas.jaecklin@shire.com |
| | To: | |
| | Medical Lead: | Thomas Jaecklin, MD, MSc Mirum Pharmaceuticals AG Innere Margarethenstrasse 5 4051 Basel Switzerland Phone: +41(0) 79 850 77 18 Email: tjaecklin@mirumpharma.com |
| | Changed from: | |
| | Sponsor Medical<br>Monitor: | Susanne Schmidt, MD |
| | To: | |
| | Medical Monitor: | Cagil Ozen, MD |
| Emergency Contact<br>Information | Changed the Premier | Medical Monitor from Susanne Schmidt to Cagil Ozen. |

**08 February 2019** 

| Section | | Description of Change | : |
|---|---|---|---|
| Product Quality<br>Complaints | Changed from: | | |
| | | Origin of Product Quality<br>Complaint | E-mail Address |
| | | North and South America | PQC@shire.com |
| | | European Union and Rest of World | PQCROW@shire.com |
| | | Telephone numbers (provided for refe | erence if needed): |
| | | Shire, Lexington, MA (USA)<br>1-800-828-2088 | |
| | То: | Origin of Product Quality<br>Complaint | E-mail Address |
| | | North and South America | medinfo@mirumpharma.com |
| | | European Union and Rest of<br>World | medinfo@mirumpharma.com |
| | | Telephone numbers (provided for refe | erence if needed): |
| | | Mirum, Menlo Park, CA (USA)<br>1-650-667-4085 | |

# 1 SYNOPSIS

| Sponsor | Mirum Pharmaceuticals, Inc. |
|---|---|
| Protocol<br>Number | LUM001-304 |
| Protocol Title | Long-Term, Open-Label Study with a Double-Blind, Placebo-Controlled, Randomized Drug Withdrawal Period of LUM001, an Apical Sodium-Dependent Bile Acid Transporter Inhibitor (ASBTi), in Patients with Alagille Syndrome |
| Study Phase | 2 |
| Indication | Treatment of Patients with Alagille Syndrome (ALGS) |
| Objectives | <ul> <li>To evaluate the long-term safety and tolerability of LUM001 in children with ALGS.</li> <li>To evaluate the effect of LUM001 on serum bile acid levels in children with ALGS.</li> <li>To evaluate the effect of LUM001 on biochemical markers of cholestasis and liver disease in children with ALGS.</li> <li>To evaluate the effect of LUM001 on pruritus in children with ALGS.</li> <li>To evaluate the long-term effect of LUM001 in children with ALGS 48 weeks of treatment.</li> <li>Objectives of Long-term Optional Follow-up Treatment Period (After Week 48):</li> <li>To offer eligible subjects treated in the LUM001-304 study continued study treatment after Week 48 until the first of the following occurs: (i) the subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.</li> <li>To explore twice a day (BID) dosing regimen and higher daily dosing of LUM001.</li> <li>To obtain safety and efficacy data in subjects treated long term on LUM001 including genotyping characteristics.</li> <li>To assess the level of alpha-fetoprotein (AFP), a marker of hepatocellular carcinoma.</li> <li>To assess palatability of the LUM001 formulation.</li> </ul> |
| Study Design | This is a long-term, open-label study with a double-blind, placebo-controlled, randomized drug withdrawal period in children with ALGS designed to evaluate the safety and efficacy of LUM001. The study is divided into 6 parts: a 6-week open-label dose escalation period at doses up to 400 μg/kg/day, a 12-week open-label stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period at doses up to 400 μg/kg/day, a 52-week optional follow-up treatment period, and a long-term optional follow-up treatment period for eligible subjects who choose to stay on treatment with LUM001. During this long-term optional follow-up period, subjects may have their dose of LUM001 increased to a maximum of 800 μg/kg/day (400 μg/kg BID), based on efficacy (sBA level and ItchRO Observer [Obs] score) and safety assessment. Subjects' participation in the long-term optional follow-up treatment period will continue until the first of the following occurs: (i) the subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication. Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3. |
| Number of<br>Subjects | Approximately 30 subjects will be enrolled in this study. |
| Study<br>Population | Inclusion Criteria To participate in this study, subjects must meet all of the following criteria: |

- 1. Male or female between the ages of 12 months and 18 years inclusive.
- 2. Diagnosis of ALGS based on the diagnostic criteria.
- 3. Evidence of cholestasis (one or more of the following):
  - a. Total serum bile acid >3x ULN for age.
  - b. Conjugated bilirubin >1 mg/dL.
  - c. Fat soluble vitamin deficiency otherwise unexplainable.
  - d. GGT > 3x ULN for age.
  - e. Intractable pruritus explainable only by liver disease.
- 4. Females of childbearing potential must have a negative serum pregnancy test during Screening.
- 5. Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and for 30 days following the last dose of study drug, must agree to use acceptable contraception during the trial.
- 6. Subject is expected to have a consistent caregiver(s) for the duration of the study.
- 7. Informed consent and assent (per IRB/IEC) as appropriate.
- 8. Access to phone for scheduled calls from study site.
- 9. Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device during the study.
- 10. Caregivers (and age appropriate subjects) must digitally accept the licensing agreement in the eDiary software.
- 11. Caregivers (and age appropriate subjects) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period (maximum possible reports = 14 per week).
- 12. Average daily score >2 on the Itch Reported Outcome (ItchRO™) questionnaire (maximum possible daily score of 4) for two consecutive weeks in the screening period, prior to dosing. A daily score is the higher of the scores for the morning and evening ItchRO. The average daily score is the sum of all daily scores divided by the number of days the ItchRO was completed.

## Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

- 1. Chronic diarrhea requiring ongoing intravenous fluid or nutritional intervention.
- 2. Surgical interruption of the enterohepatic circulation.
- 3. Previous liver transplant.
- 4. Decompensated cirrhosis (ALT >15 x ULN, INR >1.5 [unresponsive to vitamin K therapy], albumin <3.0 g/dL, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy).
- 5. History or presence of other concomitant liver disease.
- 6. History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease).
- 7. History or presence of gallstones or kidney stones.
- 8. Known diagnosis of human immunodeficiency virus (HIV) infection.
- 9. Cancers, except for in situ carcinoma, or cancers treated at least 5 years prior to Screening with no evidence of recurrence.
- 10. Recent medical history or current status that suggests that the subject may be unable to

complete the study.

- 11. Any female who is pregnant or lactating or who is planning to become pregnant during the study period.
- 12. Known history of alcohol or substance abuse.
- 13. Administration of bile acid or lipid binding resins within 28 days prior to screening and throughout the trial.
- 14. Known hypersensitivity to LUM001 or any of its components.
- 15. Receipt of investigational drug, biologic, or medical device within 28 days prior to Screening, or 5 half-lives of the study agent, whichever is longer.
- 16. History of non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to non-adherence with the study protocol based upon investigator judgment.
- 17. Any other conditions or abnormalities which, in the opinion of the investigator or medical monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study.
- 18. Subjects weighing over 50 kg at screening.

<u>Protocol Amendment #3: Eligible subjects for the 52-week optional follow-up period:</u> Subjects will be considered eligible for the 52-week optional follow-up treatment period if they have:

- Completed the protocol through the Week 48 visit with no safety concerns. Subjects
  who were discontinued due to safety reasons can be rechallenged if blood tests are
  back to relatively normal values for this patient population and subject does not
  meet any of the protocol's stopping rules. The decision will be made by the
  investigator in consultation with the medical monitor.
- Subjects who have undergone a surgical disruption of the enterohepatic circulation will not be eligible to enter into the follow up treatment period.
- Subjects who were discontinued for other reasons will be considered for the 52-week optional follow-up treatment period on an individual basis. The decision will be made by the investigator in consultation with the medical monitor.

Protocol Amendment 4: Eligible subjects for the long-term optional follow-up period: Inclusion Criteria for subjects with LUM001 dosing interruption <7 days, or >7 days: Subjects will be considered eligible for the long-term optional follow-up treatment period if they meet the following criteria:

- 1. The subject has either:
  - Completed the protocol through the Week 48 visit with no major safety concerns

OR

- Discontinued due to safety reasons judged unrelated to the study drug, and laboratory results have returned to levels acceptable for this patient population or individual and subject does not meet any of the protocol's stopping rules at the time of entry into the follow-up period. The decision will be made by the investigator in consultation with the medical monitor. [Subjects who were discontinued for other reasons will be considered on an individual basis.]
- 2. Females of childbearing potential must have a negative urine or serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at the time of entry into the long-term optional follow-up treatment period.
- 3. Males and females of child-bearing potential who are sexually active, or are not

**08 February 2019** 

currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial.

- 4. Informed consent and assent (per IRB/EC) as appropriate.
- 5. Access to phone for scheduled calls from study site.
- 6. Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device during the study.

#### Exclusion Criteria for Subjects with LUM001 dosing interruption ≥7 days:

All exclusion criteria mentioned for the core study apply upon entry into the long-term optional follow-up period, with the exception of exclusion criterion #18.

# Treatment Groups

All subjects will receive LUM001 up to 400  $\mu g/kg/day$  or a maximum daily dose of 20 mg/day. After completion of the 12-week stable dosing period, subjects will be randomized 1:1 to either a 4-week double-blind study drug withdrawal period during the study or will remain on study drug. Subjects will then enter a 26-week long-term stable dosing period and all subjects will receive LUM001 up to 400  $\mu g/kg/day$  or a maximum daily dose of 20 mg/day. Subjects will be considered for a 52-week optional treatment period, if eligible, receiving up to 400  $\mu g/kg/day$ , or the highest tolerated dose below the 400  $\mu g/kg/day$  dose. Subjects will then be considered for the long-term optional follow-up treatment, if eligible, receiving up to 800  $\mu g/kg/day$  (given as twice daily doses of 400  $\mu g/kg$ ), or to a maximum possible daily dose of 50 mg/day.

#### Study Drug Dosage and Administration

## **Study Drug Administration**

Subjects will receive a grape-flavored solution containing LUM001, administered orally once a day (QD) or twice a day (BID) using the syringe provided. The first dose should be taken at least 30 minutes prior to the first meal of the day and the second dose, where applicable, should be taken at least 30 minutes prior to dinner (main evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the dose should be taken approximately at the same time each day for the duration of the treatment period.

#### **QD Dosing Regimen**

For QD dosing, the required dose will be delivered in 0.5 mL volume for subjects who weigh less than 10 kg and in 1.0 mL for subjects who weigh 10 kg or more.

#### **BID Dosing Regimen**

For BID dosing, the required dose is delivered in half the dosing volume: 0.25 mL BID for subjects who weigh less than 10 kg and 0.50 mL BID for subjects who weigh 10 kg or more.

For subjects weighing less than 10 kg at study entry, once a weight of 10 kg is reached while in the study, the subject will be moved from 0.5 mL maximum daily dosing volume (0.25 mL BID) to 1.0 mL maximum daily dosing volume (0.50 mL BID).

#### **Study Drug Dosage**

Initially, the LUM001 dose will be administered as a daily morning dose in either a 1.0 mL or 0.5 mL solution. The dose will be increased weekly over a 6-week period <u>up to 400 µg/kg/day QD</u> or a maximum daily dose of 20 mg/day QD as follows:

Week 1 Dose: 14 μg/kg/day QD Week 2 Dose: 35 μg/kg/day QD Week 3 Dose: 70 μg/kg/day QD Week 4 Dose: 140 μg/kg/day QD Week 5 Dose: 280 μg/kg/day QD Week 6 Dose: 400 µg/kg/day QD (maximum daily dose of 20 mg QD)

Subjects will continue dosing for another 12 weeks during the stable dosing period (to Week 18) using the dose administered at Week 6, which may be 400  $\mu$ g/kg/day or the highest tolerated dose below 400  $\mu$ g/kg/day.

At the Week 18 visit, subjects will be randomized 1:1 to continue to receive study drug or a corresponding placebo for 4 weeks (1:1 randomized double-blind withdrawal period).

Following the 4-week study drug randomized withdrawal period, subjects who received placebo will receive LUM001 dosed according to a dose escalation schedule that mirrors the initial escalation (ie, the LUM001 dose will be increased weekly over a 6-week period to the maximum tolerated dose up to 400  $\mu$ g/kg/day or 20 mg/day or the highest tolerated dose below the 400  $\mu$ g/kg/day dose). Subjects who were randomized to receive LUM001 will undergo a simulated dose escalation to maintain the blind in the randomized withdrawal period and will continue to receive LUM001 during the long-term exposure period, at the same dose administered at Week 22. Dosing with LUM001 will continue in a 26-week long-term exposure period to complete 48 weeks of study.

#### **Optional Follow-up Treatment Period**

At Week 48, all subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over into the 52-week optional follow-up treatment period. The 3 following possible scenarios may occur:

- Subjects who are eligible to roll over into the optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level.
- Subjects who are eligible to roll over into the optional follow-up treatment period with a LUM001 dosing interruption of ≥7 days will be dose escalated beginning at 35 μg/kg/day and up to a maximum of 400 μg/kg/day or highest tolerated dose.
- Subjects who do not wish to enter the follow-up treatment period will be contacted via telephone by the study site approximately 30 days after the last dose of study drug.

#### Long-term Optional Follow-up Treatment Period

Upon completion of the 52-week follow-up treatment period and/or implementation of this amendment, whichever occurs first, subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over (or enter) into the long-term optional, follow-up treatment period. The 3 following possible scenarios may occur:

Scenario 1: Subjects eligible to roll over into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days:

- Subjects with normal sBA level AND ItchRO(Obs) score <1.5 will be maintained at the same dose level and will continue morning dosing only.
- Subjects with sBA level above normal AND/OR ItchRO(Obs) score ≥1.5 will start BID dosing (afternoon dose escalation; ADE) as follows:
  - The morning dose will be continued at the same dose level, but the volume of the morning dose will be reduced by half at the same time that the afternoon dose is initiated.
  - The afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg.

# Scenario 2: Subjects eligible to roll over into the long-term optional follow-up treatment period with a LUM001 interruption of ≥7 days:

- First, the morning dose is escalated up to 400 μg/kg/day or highest tolerated dose following a 5-week dose escalation beginning at 35 μg/kg/day.
- Once the morning dose of 400 μg/kg or maximum tolerated dose is achieved, sBA and ItchRO(Obs) score will be evaluated.
  - Subjects with normal sBA AND ItchRO(Obs) score <1.5 after morning dose escalation will be maintained at the same dose level and will continue morning dosing only.
  - O Subjects with sBA above normal AND/OR ItchRO(Obs) score ≥1.5 will begin BID dosing (afternoon dose escalation) as follows:
    - The morning dose will be continued at the same dose level, but the volume of the morning dose will be reduced by half at the same time that the afternoon dose is initiated.
    - The afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg.

The following parameters apply to both dosing scenarios outlined above:

- The afternoon dose will only be initiated once the subject has been treated on stable morning doses for at least 4 weeks.
- The sBA value used for determination of ADE eligibility will be the most recent available value collected within the prior 16 weeks. The ItchRO(Obs) score used for ADE eligibility will be derived from the most recent available 7-day interval of ItchRO(Obs) collected within the prior 16 weeks.
- The maximum daily dose will be 400 μg/kg BID, ie, 800 μg/kg/day (up to a maximum possible daily dose of 50 mg/day).

# Scenario 3: Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3.

### Rationale for Dose and Schedule Selection

During the study, the study drug may be adjusted if there is a change of  $\geq 10\%$  in body weight since the screening visit or if there is a change of  $\geq 10\%$  in weight since the last weight based medication adjustment to maintain the target dose.

If a subject experiences intolerance due to gastrointestinal symptoms (eg, diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the medical monitor may lower the dose to a previously tolerated dose; later attempts to escalate the dose are permitted. If the subject is on a BID dosing regimen, dose lowering should first be attempted with the afternoon dose.

The dosage of LUM001 is based upon prior experience with this investigational product in healthy volunteers and adult and pediatric subjects with hypercholesterolemia. In these subjects, with normal bile flow and without liver disease, an increase in gastrointestinal (GI) adverse events (AEs) was observed in those receiving doses above 10 mg per day. These signs and symptoms were believed to be caused by increases in the concentration of free bile acids in the lower colon. Subjects with cholestatic liver disease have reduced bile flow compared to healthy volunteers and LUM001 is likely to produce a correspondingly smaller increase in free bile acids in the lower colon. There is evidence in subjects with cholestasis to suggest that ASBT expression may be upregulated and higher ASBTi concentrations may be

required to achieve the desired target inhibition.

Dosing in pediatric subjects will be based on the subject's weight. The appropriate dose of LUM001 for the lowering of bile acid concentrations and the reduction of pruritus in cholestatic populations is not known. Earlier studies in healthy volunteers and hypercholesterolemic subjects demonstrated that doses of 10 mg to 30 mg daily (equivalent to 140  $\mu$ g/kg/day to 400  $\mu$ g/kg/day for a 70 kg subject) led to a decrease in serum bile acids by >50% following 2 weeks of treatment.

In previous studies with LUM001, GI-associated AEs were generally recorded in the first weeks of LUM001 dosing and then at levels similar to those in the placebo group. In a 4-week dose finding study in healthy volunteers, a dose escalation regimen was evaluated to mitigate the risk of loose stools, diarrhea and abdominal pain or cramps. When the LUM001 dose was increased after each 7-day dosing period, to a maximum of 5 mg daily, the incidence of GI-associated AEs in the LUM001 treatment arm was comparable to the reported incidence in the placebo group.

To reduce the risk of loose stools, diarrhea and abdominal pain or cramps in this study, the LUM001 dose will be escalated over the first 6 weeks. Dosing will start at 14  $\mu$ g/kg/day, and will then be increased at 7 day intervals to a maximum dose of 400  $\mu$ g/kg/day (equivalent to approximately 20 mg daily dose in a 50 kg subject).

For subjects in the long-term optional follow-up treatment period with  $\geq 7$  days since the last dose of LUM001, dosing will start at 35  $\mu g/kg/day$ , and will then be increased over the first 5 weeks up to 400  $\mu g/kg/day$  or to the maximum tolerated dose. This escalation regimen is supported by the safety profile observed in completed and ongoing clinical studies of LUM001 and allows for subjects to reach 400  $\mu g/kg/day$  or a maximum tolerated dose within a 5-week period.

Under Protocol Amendment 4, an afternoon dose is introduced for eligible subjects in the long-term optional follow up treatment period. LUM001 doses will be escalated over a period of 4-8 weeks up to a maximum dose of 400  $\mu$ g/kg BID (or maximum tolerated dose). The afternoon dose is only initiated and escalated in subjects with elevated sBA and/or ItchRO(Obs)  $\geq$ 1.5 on the maximum (or maximum tolerated) morning dose.

This escalation regimen is supported by the safety profile observed in completed and ongoing clinical studies of LUM001. Twice daily dosing is used in this study based on the findings of a healthy volunteers study in adult males (Study SHP625-101), which demonstrated that bile acid levels in feces increase with escalating doses and twice-daily regimen of LUM001 (up to 100 mg QD and 50 mg BID). In this study, subjects who were randomized to LUM001 treatment, received 1 of 4 doses of LUM001 (10, 20, 50, 100 mg) during 7 days. No titration was used in this study. There was a dose-dependent increase in total fecal BA excretion. In addition, BID dosing (ie, 50 mg BID) led to a further increase in fecal BA excretion as compared to QD dosing (ie, 100 mg QD). It is therefore hypothesized that twice-daily dosing has the potential to allow for more complete target engagement throughout the day at the level of the distal ileum.

The higher dosing level is also supported by favorable results from a juvenile toxicity study conducted in rats administered LUM001 for 43 days (PND21 through PND63). As expected for a drug intentionally designed to be minimally absorbed, systemic LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies in adult rats. No adverse effects were observed on postnatal growth and development of offspring at the highest doses tested (200 mg/kg/day in males, 1000 mg/kg/day in females). This study was initiated in juvenile animals at PND21, which from a whole animal development perspective, is typically representative of a 2-year old child. However, given the fact that LUM001 is a minimally absorbed drug, of particular importance is the age at which the GI tract is considered functionally mature. In humans this is considered to have occurred by 12 months of age; likewise, postnatal maturation of the GI tract in rats occurs

during the first 3 weeks of life. Therefore, results from this study can be used to support the dosing levels proposed here for children 12 months of age and older.

### Study Visit Schedule and Procedures

Study activities will be conducted as described in the Schedule of Procedures.

The dosage and dosing regimen of concomitant drug therapy other than that specified by the protocol should not change during the first 22 weeks of the study, with the exception of weight-based study drug adjustments and vitamin supplementation. No new medications used to treat pruritus may be added during the first 22 weeks of the study.

Synopsis Figure 1: Study Design for LUM001-304 (Up to and including Week 48)



Screening Period (Day -28 to Day -1): After obtaining informed consent (and/or assent when appropriate), demographic data (gender, age, and race) will be collected and subjects will undergo a medical history and physical examination including body weight, height, and vital signs, compilation of concomitant medications, and have blood and urine samples taken for clinical laboratory testing. For subjects who do not have documentation of a JAGGED-1 or NOTCH2 mutation, a blood sample may be obtained for genotyping. The physician will provide an assessment of itch severity using the clinician scratch score during Screening. The eDiary for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the Screening visit. The patient/caregiver ItchROs will be completed twice daily during the Screening period to establish eligibility and a baseline score. Subjects 9 years of age and older will continue independent twice daily completion of their ItchRO. Subjects 5-8 years of age will continue twice daily completion of their ItchRO with the assistance of their caregivers, if needed. Caregivers will continue twice daily completion of their ItchRO. Caregivers (and age appropriate subjects) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period, (maximum possible reports = 14 per week). Subjects are required to discontinue bile acid resins for at least 28 days prior to screening and throughout the study. Females who are of childbearing potential will have a serum pregnancy test. Eligibility criteria will be reviewed to confirm a subject's eligibility 4-7 days prior to the Baseline Visit.

<u>Dose Escalation Treatment Period (Day 0 to Week 6)</u>: At the Baseline Visit (Day 0), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of bile acids and other cholestasis biochemical markers. Blood will also be collected for determination of

baseline fat-soluble vitamins and a plasma LUM001 drug level. Compliance with ItchRO will be assessed. The clinician scratch scale, xanthoma scale, and PedsQL questionnaires will be completed. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study medication for Weeks 1, 2, and 3 will be supplied at the Baseline Visit to eligible subjects. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the Dose-Escalation Treatment Period. Subjects will return to the clinic at Weeks 3 and 6 and follow-up phone calls will be made at Weeks 1, 2, 4, and 5. On clinic visit days, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Clinician scratch scale, adherence to study medication, and ItchRO compliance will be assessed. Concomitant medications and any adverse events will be recorded. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Weeks 3 and 6.

Stable Dosing Treatment Period (Week 7 to Week 18): Each subject will continue dosing with study drug during a 12-week Stable Dosing Treatment Period using the dose administered at Week 6, which may be 400 µg/kg/day or the highest tolerated dose below 400 μg/kg/day. Subjects 9 years of age and older will continue independent twice daily completion of their ItchRO. Subjects 5-8 years of age will continue twice daily completion of their ItchRO with the assistance of their caregivers, if needed. Caregivers will continue twice daily completion of their ItchRO. Subjects will receive a follow-up phone call at Week 9 and return to the clinic at Weeks 12 and 18. At the Week 12 and 18 visits, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fasting lipid panel, serum bile acids, fat soluble vitamins, and other cholestasis biochemical markers. Blood sampling for study drug determination may also be performed. After the baseline pharmacokinetic analysis, blood sampling for an additional pharmacokinetic analysis will be done at one additional time point at Week 12, 18, 38, or 48 – to be selected by the site/investigator (sample to be taken approximately 4 hours post-dosing). Clinician scratch scale, adherence to study medication, ItchRO compliance, and the PedsQL questionnaire will be assessed and concomitant medications and any adverse events will be recorded. In addition, at the Week 18 visit the Clinician Xanthoma Scale, Patient Impression of Change (PIC), Caregiver Impression of Change (CIC), and Caregiver Global Therapeutic Benefit (CGTB) assessments will be completed. At the Week 18 visit, subjects will also be randomized 1:1 to either continue to receive study drug or a corresponding placebo between Week 19 and Week 22. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Week 12 and study drug (or placebo) supplied at Week 18.

Double-Blind, Placebo-Controlled Study Drug Withdrawal Period (Week 19 to Week 22): Age appropriate subjects and caregivers will continue twice daily completion of their ItchRO. Subjects will receive a follow-up phone call at Week 20 and return to the clinic at Week 22. At the Week 22 visit, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fasting lipid panel, serum bile acids, fat soluble vitamins, and other cholestasis biochemical markers. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Week 22. Clinician scratch scale, adherence to study medication, ItchRO compliance, PIC, CIC, CGTB, and the PedsQL questionnaires will be assessed and concomitant medications and any adverse events will be recorded.

Long-Term Exposure Period (Week 23 to Week 48): Following the 4-week double-blind study drug withdrawal period, subjects who received placebo will once again receive LUM001 according to the schedule where the dose is increased weekly over a 6-week period up to  $400 \,\mu\text{g/kg/day}$  or a maximum daily dose of  $20 \,\text{mg/day}$ . Subjects who were randomized to receive LUM001 will undergo a simulated dose escalation to maintain the blind in the

randomized withdrawal period and will continue to receive LUM001 during the long-term exposure period, at the same dose administered at Week 22.

Subjects and caregivers will continue twice daily completion of their ItchRO throughout the long-term exposure period to the Week 48 clinic visit. Subjects will return to the clinic at Weeks 28, 38, and 48. At these visits, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fat soluble vitamins, as well as possible pharmacokinetic blood sampling for study drug determination (if not done previously at Week 12 or 18). Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Clinician scratch scale, adherence to study medication, and ItchRO compliance will be assessed. Subjects/caregivers will receive follow-up phone calls at the end of Weeks 23-27, 33, and 43. Concomitant medications and adverse events will be recorded at all clinic visits and at scheduled telephone contacts.

At the investigator's discretion, withdrawal of concomitant medications used for the treatment of pruritus may occur during the long-term exposure period. Additional study drug will be supplied at each clinic visit during the long-term exposure period.

Week 48: Subjects will be evaluated by the investigator to determine whether they are eligible to roll over into the optional follow-up treatment period. Eligible subjects must have documented consents in order to continue in the optional follow-up treatment period. A physical exam (including collection of vital signs, height and weight measurements) will be performed. Blood and urine samples will be taken for clinical laboratory testing, including a fasting lipid panel and determination of fat-soluble vitamins, bile acids, other cholestasis biochemical markers, and possibly LUM001 drug level analysis. Female subjects who are of childbearing potential will have a urine pregnancy test. The Clinician Scratch Scale, Clinician Xanthoma Scale, and PedsQL questionnaires will be completed. The PIC, the CIC, and the CGTB assessments will be completed. Concomitant medications and adverse events will be recorded. ItchRO and study drug compliance will be assessed and all remaining study drug and study supplies will be collected. eDiaries will be returned to the site and Study drug will be discontinued at this visit if the subject chooses not to participate in the optional follow-up treatment period.

Subjects who withdraw from the study prior to completion of all treatment period clinic visits should undergo the procedures specified for the Week 48/Study Termination visit.

<u>Follow-up Phone Call:</u> For subjects who do not roll over into the optional follow-up treatment period, a safety follow-up phone call will be made 30 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and adverse events noted during this phone call will be recorded.

Follow-up Treatment Period (post-Week 48):

**Subjects who are eligible to roll over into the follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days** will be maintained at the same dose level within the 52-week Optional Follow-Up Treatment period. During this period, subjects will return to the clinic at Weeks 60, 72, 84, 96, and 100; telephone contacts will occur at Weeks 64, 68, 76, 80, 88, and 92.



Subjects with ≥7 days since last dose of LUM001 will be dose escalated up to 400 μg/kg/day or to the highest tolerated dose. The dose escalation (DE) period will proceed as follows:

- Week DE-2 Clinic Visit: obtain consent, weight, and draw blood for laboratory analyses
- Week DE 0 Clinic Visit: investigator evaluates laboratory results, study drug is dispensed, and subject begins at 35 μg/kg/day dose level (if no safety concerns)
- Week DE 49 Telephone Contact: subject escalates to  $70 \,\mu g/kg/day$  dose level if prior dose level was tolerated
- Week DE 50 Telephone Contact: subject escalates to 140 μg/kg/day dose level if prior dose level was tolerated
- Week DE 51 Telephone Contact: subject escalates to 280 μg/kg/day dose level if prior dose level was tolerated
- Week DE 52 Clinic Visit: laboratory tests and dose escalates to 400 μg/kg/day dose (maximum daily dose of 20 mg), if prior dose level was tolerated

Synopsis Figure 3: 52-week Optional Follow-up Treatment (≥7 days from last LUM001 dose)



If any subject experiences intolerance, the investigator, in consultation with the medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period. At the investigator's discretion and in consultation with the medical monitor subjects who were previously down titrated may be rechallenged during the follow-up treatment period.

### **Long-term Optional Follow-up Treatment Period**

Upon completion of the additional 52-week follow up treatment period <u>and/or</u> implementation of this amendment, whichever occurs first, subjects who are eligible to roll over onto the long-term optional follow-up treatment period will continue to receive study drug until the first of the following occurs:

- i. The subjects are eligible to enter another LUM001 study,
- ii. LUM001 is commercially available, or
- iii. The sponsor stops the program or development of this indication.

Once Protocol Amendment 4 is implemented at the site, a determination about ADE will be made.

Subjects who are eligible to roll over from the 52-week follow up treatment period into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days prior to implementation of Protocol Amendment 4 will be consented and evaluated for eligibility for ADE. Once a determination about ADE has been made, the subject will then either initiate the ADE (Synopsis Figure 6) or continue receiving the same dose of LUM001 once a day (Synopsis Figure 5), depending on whether they meet criteria for initiating ADE.

Subjects with  $\geq$ 7 days since last dose of LUM001 prior to implementation of Protocol Amendment 4 who are eligible to enter the long-term optional follow-up treatment period will be dose escalated up to 400 µg/kg/day or to the highest tolerated dose beginning with 35 µg/kg/day, as outlined in Synopsis Figure 4.

The dose escalation (DE) period will proceed as follows:

- Protocol Amendment 4 DE-2 Clinic Visit: obtain consent, weight, and draw blood for laboratory analyses
- Protocol Amendment 4 DE Day 0 Clinic Visit: PI evaluates laboratory results, study drug is dispensed, and subject begins at 35 μg/kg/day dose level (if no safety concerns)
- Protocol Amendment 4 DE Week 1 Telephone Contact: subject escalates to 70 μg/kg/day dose level
- Protocol Amendment 4 DE Week 2 Telephone Contact: subject escalates to 140 μg/kg/day dose level if prior dose level was tolerated
- Protocol Amendment 4 DE Week 3 Telephone Contact: subject escalates to 280 μg/kg/day dose level if prior dose level was tolerated
- Protocol Amendment 4 DE Week 4 Clinic Visit: laboratory tests and dose escalates to 400 μg/kg/day dose (maximum daily dose of 20 mg), if prior dose level was tolerated
- Protocol Amendment 4 DE Week 8 Telephone Contact: eligibility for ADE will be determined.



Subjects not eligible for ADE (subjects with normal sBA level AND ItchRO(Obs) score <1.5), will be maintained at the same dose level and will continue morning dosing only. Subjects will have study activities repeated in repeating 12-week periods as follows, until study completion or termination:

- Repeating Period Week 4 (ie, beginning 4 weeks after consent to Protocol Amendment 4) Telephone Contact: Collection of concomitant medications and any adverse events.
- Repeating Period Week 8 Telephone Contact: Collection of concomitant medications and any adverse events.
- Repeating Period Week 12 Clinic Visit: Physical exam, body weight and height, vital signs, and blood samples for clinical laboratory testing including fasting lipid panel. Blood will also be collected for determination of baseline fat-soluble vitamins. Urine samples for clinical laboratory testing will be collected at every other visit. ItchRO compliance will be assessed, the electronic diary will be issued, the Clinician Scratch Scale and Clinician Xanthoma Scale will be administered, and the PedsQL questionnaire will be administered. Additionally, a palatability questionnaire will be completed. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and adverse events will be collected.
- Subjects who do not qualify for ADE may be assessed at a later time point on a case by case basis following discussions between the investigator and medical monitor. Such re-evaluations may only occur at the Week 12 visit of any Repeating Period beginning with RP2. If in the course of the ADE re-evaluation, a subject is found to qualify for ADE, then the subject will move into Schedule F or G, as outlined in Section 16.1. During the follow-up treatment period, subjects will return to the clinic every 3 months.



If the subject is eligible for ADE, ie, who have sBA level above normal AND/OR ItchRO(Obs) score ≥1.5, the subject will begin BID dosing (afternoon dose escalation; ADE) as follows:

- On ADE Day 0, morning dosing will continue at 400 µg/kg or the maximum tolerated dose. However, the volume of the morning dose will be reduced by half.
   Of note: Morning dosing must have been stable for ≥4 weeks prior to initiation of ADE.
- On ADE Day 0, the afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg.

The following procedures will occur during the ADE period:

- ADE Day 0 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician Xanthoma Scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and any adverse events will be collected.
- ADE Week 1 and Week 2 Telephone Contact: Collection of concomitant medications and any adverse events. Subject/caregiver will be reminded of dosing instructions.
- ADE Week 4 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician Xanthoma Scale, and the PedsQL questionnaire will be

administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and any adverse events will be collected.

- ADE Week 5 and Week 6 Telephone Contact: Collection of concomitant medications and any adverse events. Subject/caregiver will be reminded of dosing instructions.
- ADE Week 8 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician Xanthoma Scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and any adverse events will be collected.

# Synopsis Figure 6: Long-term Optional Follow-up Treatment, with Afternoon Dose Escalation (ADE)



If any subject experiences intolerance, the investigator, in consultation with the medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period; later attempts to escalate the dose are permitted. At the investigator's discretion, and in consultation with the medical monitor subjects who were previously down titrated may be rechallenged during the follow-up treatment period. If the subject is on a twice daily dosing regimen, dose lowering should be first attempted with the afternoon dose.

Safety and clinical laboratory evaluations and a physical exam (including collection of vital signs, height and weight measurements) will be completed at each clinic visit. In addition, the Clinician Scratch Scale, Clinician Xanthoma Scale, and PedsQL will be administered and study drug compliance will be assessed (PedsQL will not be performed at certain clinic visits – please refer to schedule of procedures). The PIC and CIC and the CGTB assessments will be completed at Weeks 84, 96, 100, and the End of Treatment (EOT)/Early Termination (ET)

visit. Palatability data will be collected at each clinic visit during the long-term optional follow up treatment period (including the EOT/ET visit), with the exception of the PA4 DE, and ADE visits. Plasma samples will be obtained for LUM001 pharmacokinetics at the ADE Day 0, ADE Week 4, and ADE Week 8 visits, and at the 3 scheduled clinic visits following completion of the ADE period. Subjects/caregivers will receive follow-up phone calls at Weeks 64, 68, 76, 80, 88, 92, as well as those outlined within the PA4 DE, ADE, and repeating 12-week periods. Concomitant medications and any AEs will be evaluated and recorded at all clinic visits and at scheduled telephone contacts.

Twice daily completion of the electronic diary will be required by caregivers and age appropriate subjects during the 2 weeks following the Week 60, 72, 84, 96 clinic visits, at PA4 DE Week 4, and every clinic visit within the repeating 12-week periods. Electronic diaries will be provided to subjects and caregivers at these visits and re-training on the use of the diary will occur, as appropriate.

At the physician investigator's discretion, withdrawal of concomitant medications used for the treatment of pruritus may occur during the long-term exposure period.

With the exception of the EOT/ET visit, additional study drug will be supplied at each clinic visit during the follow-up treatment period. Used and unused study drug will be collected at every visit.

Subjects will be encouraged to complete all study activities and visits. Any subject who withdraws from the study prior to completion of all treatment period clinic visits should undergo safety and clinical laboratory evaluations, including pharmacokinetic sampling of LUM001, determination of serum bile acids, other cholestasis biochemical markers, fat soluble vitamins, and AFP. In addition the following assessments should be completed: the Clinician Scratch Scale, the Clinician Xanthoma Scale, the PedsQL, the PIC, the CGTB, and the palatability questionnaire, as defined for ET. For subjects who complete the study, an EOT visit will be completed; the assessments performed at this visit will be identical to the assessments performed at the ET visit.

<u>Following completion of the Follow-up Treatment Period or early discontinuation:</u> a safety follow-up phone call will be made 30 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and adverse events noted during this phone call will be recorded.

#### Safety and Tolerability Evaluations

The safety and tolerability of LUM001 will be assessed by determining the incidence, relationship to study drug, and severity of treatment-emergent AEs, withdrawals due to AEs, and changes in vital signs, laboratory and other safety parameters. Alpha-fetoprotein (AFP), a marker of hepatocellular carcinoma, will be measured every 6 months throughout the long-term optional extension period.

A Data Monitoring Committee (DMC) will review serious adverse event data, and other key subject safety and study data at specified intervals for the duration of the study.

#### Safety Evaluations

The following assessments will be used to evaluate safety:

- Adverse events (AEs) and serious adverse events (SAEs).
- Clinical laboratory results, including alpha-fetoprotein (AFP) as a screening for hepatocellular carcinoma.
- Vital signs.
- Physical exam findings, including body weight and height.
- Concomitant medication usage.

**08 February 2019** 

# **Efficacy Evaluations**

The primary efficacy endpoints will be the mean change from Week 18 to 22 of fasting serum bile acid levels in subjects who previously responded to LUM001 treatment, as defined by a reduction in sBA  $\geq$ 50% from baseline to Week 12 or Week 18. A sensitivity analysis will also be conducted using subjects who experienced a reduction from baseline in serum bile acids of  $\geq$ 50% at the Week 48 measurement.

The secondary efficacy evaluations will include:

- Change from Week 18 to Week 22 in:
  - o Liver enzymes [alanine aminotransferase (ALT), alkaline phosphatase (ALP)] and bilirubin (total and direct).
  - Pruritus as measured by ItchRO (Observer ItchRO/patient ItchRO) in subjects who
    previously responded to LUM001 treatment, as defined by a reduction in ItchRO
    scale >1 point from baseline to Week 12 or Week 18.
- Change from baseline to Week 18 in:
  - o Fasting serum bile acid levels.
  - o Liver enzymes (ALT, ALP) and bilirubin (total and direct).
  - o Pruritus as measured by ItchRO (Observer ItchRO/patient ItchRO).

The following additional efficacy evaluations will be assessed:

- Change from baseline to Weeks 18, 22 48, and then every 12 weeks in:
  - o Fasting serum bile acid levels.
  - Liver enzymes (ALT, ALP) and bilirubin (total and direct).
     Pruritus as measured by the average daily ItchRO (Observer ItchRO/patient ItchRO).
  - Other biochemical markers of cholestasis [total cholesterol, low-density lipoprotein cholesterol (LDL-C)].
  - o Bile acid synthesis [serum  $7\alpha$ -hydroxy-4-cholesten-3-one ( $7\alpha$ C4)].
- Responder analysis at Weeks 18 and 48 in:
  - o Pruritus response rates as measured by ItchRO (Observer ItchRO/patient ItchRO).
  - o Clinician scratch score.
- Change from baseline for PedsQL at Week 18 and Week 48 and change from Week 18 to Week 22.
- PIC at Week 18 and 48 and change from Week 18 to Week 22.
- CIC at Week 18 and 48 and change from Week 18 to Week 22.
- CGTB assessment at Weeks 18 and 48 and change from Week 18 to Week 22.
- Change from Baseline (Day 0) to Week 48 in xanthomas, as measured by Clinician Xanthoma Scale.

Additional assessments of efficacy variables will occur during the 52-week and long-term optional treatment periods in 12 weekly intervals. Any of the above evaluations may also occur at clinic visits during the DE, PA4 DE, and ADE periods.

Additional exploration of evaluations of safety will be specified in the statistical analysis plan.

#### Palatability Data

Palatability data will be collected at each clinic visit in the follow up treatment period, with the exception of the PA4 DE, and ADE visits. A palatability questionnaire will be completed by the subject and/or caregiver (dependent on age). Assessment of change over time will be evaluated.

**08 February 2019** 

## Statistical Considerations

### Sample Size

The planned sample size of 30 evaluable subjects was based on practical considerations, rather than on statistical considerations and desired power for a pre-specified difference.

#### Safety

All safety analyses will be performed on the Safety Population, defined as all subjects who were assigned and received at least one dose of the study drug.

Safety measures including AEs, clinical laboratory tests, vital signs, physical exams, and concomitant medication usage will be summarized descriptively by study period and over the entire study duration (Weeks 0-EOT Visit). For quantitative variables, descriptive statistics including number of observations, mean, median, standard deviation and range will be given for the values themselves as well as for change from baseline at each study visit. Qualitative variables will be summarized using counts and percentages at each study visit.

#### Drug Level Analysis

Plasma concentrations of LUM001 will be examined descriptively by visit.

#### **Efficacy**

The main population for efficacy will be the modified intention-to-treat population (MITT), defined as all subjects who were enrolled, received study medication through Week 18, and had a reduction from baseline in serum bile acids of  $\geq 50\%$  at the Week 12 or Week 18 measurement. Subjects will be analyzed by assigned treatment.

Efficacy endpoints will be displayed by study visit, using summary statistics including the number of observations, the mean, median, standard deviation, and range for continuous measures and counts and percentages for categorical measures. Actual values as well as change from baseline will be presented. The change from baseline will be tested using the paired t-test, or comparable nonparametric measures if appropriate.

Examination of potential treatment effects by dose will be done if the sample sizes in the dose groups during the stable dosing phase of the study permit.

In addition to absolute change from baseline, a responder analysis will also be considered. The response definition and its appropriate analysis methodology will be outlined in the Statistical Analysis Plan (SAP) for the study.

Supportive and exploratory efficacy measures will be analyzed similarly as above. Details of the analysis methods will be outlined in the SAP.

#### Interim Analysis

There will be an interim analysis (IA) conducted after all subjects complete or discontinue the study after Week 48 to guide the future of the program. At the IA the study will be unblinded.

### Siblings

The enrollment of siblings is allowed. During the double-blind, placebo-controlled, randomized drug withdrawal period, siblings will be assigned in a blinded manner to the same treatment arm. The data from all enrolled participants (including siblings) will be used for the safety analysis. For the efficacy analysis, data from only one of the siblings will be used. The choice of which subject's data to use in the efficacy analysis will be done in a random fashion before the LUM001-304 study is unblinded. Details of the analysis methods will be outlined in the SAP.

All data will be included in data listings.

# 2 LIST OF ABBREVIATIONS AND TERMS

| Abbreviation | Definition |
|---|---|
| β-hCG | beta-sub-unit of human chorionic gonadotropin; pregnancy test |
| μg | microgram |
| μΜ | micromolar |
| 7αC4, C4 | $7\alpha$ -hydroxy-4-cholesten-3-one; an indirect method of bile acid synthesis |
| ac | before meals |
| ADE | afternoon dose escalation |
| ADME | absorption, distribution, metabolism, excretion |
| AE | adverse event |
| AFP | alpha-feto protein |
| ALGS | Alagille syndrome |
| ALP | alkaline phosphatase |
| ALT | alanine aminotransferase (SGPT) |
| ANA | antinuclear antibody |
| ANCOVA | analysis of covariance |
| aPTT | activated partial thromboplastin time |
| ASBT | apical sodium-dependent bile acid transporter |
| ASBTi | apical sodium-dependent bile acid transporter inhibitor |
| AST | aspartate aminotransferase (SGOT) |
| ATC | Anatomical Therapeutic Chemical; classification for drugs |
| ATX | autotaxin |
| BA | bile acid |
| BID | twice a day |
| BP | blood pressure |
| CBC | complete blood count |
| CFR | Code of Federal Regulations |
| CGTB | Caregiver Global Therapeutic Benefit questionnaire |
| cholesterol 7α-hydroxylase | rate-limiting enzyme in the synthesis of bile acid from cholesterol |
| CIC | Caregiver Impression of Change questionnaire |
| CRF | case report form |

| Abbreviation | Definition |
|---|---|
| CS | clinically significant |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CV | curriculum vitae |
| DE | dose escalation |
| dL | deciliter |
| DMC | Data Monitoring Committee |
| EC | Ethics Committee |
| eCRF | electronic case report form |
| EOT | End of Treatment |
| ET | Early Termination |
| EU | European Union |
| EudraCT | European Union Drug Regulating Authorities Clinical Trials |
| FDA | Food and Drug Administration |
| FGF-19 | fibroblast growth factor 19; regulates carbohydrate, lipid and bile acid metabolism |
| FGF-21 | fibroblast growth factor 21; modulates hepatic metabolism |
| g | gram |
| GCP | good clinical practices |
| GGT | gamma-glutamyltransferase |
| GGTP (γGTP) | gamma-glutamyl transpeptidase |
| GI | gastrointestinal |
| HDL | high-density lipoprotein |
| HDL-C | high-density lipoprotein cholesterol |
| HIV | human immunodeficiency virus |
| HMG-CoA reductase | 3-hydroxy-3-methyl-glutaryl-CoA reductase; rate-controlling enzyme of the pathway that produces cholesterol |
| HR | heart rate |
| HRQoL | health related quality of life |
| IAF | informed assent form |
| IB | investigator's brochure |
| IBAT | ileal bile acid transporter |
| Abbreviation | Definition |
|---------------------------|----------------------------------------------|
| IBATi | ileal bile acid transporter inhibitor |
| ICF | informed consent form |
| ICH | International Conference on Harmonization |
| IEC | independent ethics committee |
| INR | international normalized ratio |
| IRB | institutional review board |
| ItchRO <sup>TM</sup> | Itch Reported Outcome |
| ItchRO(Obs) <sup>TM</sup> | Itch Reported Outcome observer instrument |
| ItchRO(Pt) <sup>TM</sup> | Itch Reported Outcome patient instrument |
| ITT | intention-to-treat |
| IU | international unit(s) |
| IUD | intrauterine device |
| kg | kilogram |
| L | liter |
| LDL | low-density lipoprotein |
| LDL-C | low-density lipoprotein cholesterol |
| LPA | lysophosphatidic acid |
| MCH | mean corpuscular hemoglobin |
| MCHC | mean corpuscular hemoglobin concentration |
| MCV | mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | milligram |
| MITT | modified intention-to-treat |
| mL | milliliter |
| mmol | millimole |
| NBD | nasal biliary drainage |
| NCS | not clinically significant |
| ng | nanogram |
| ObsRO | observer reported outcome |
| PBC | primary biliary cirrhosis |
| PEBD | partial external biliary diversion |

| Abbreviation | Definition |
|---|---|
| PedsQL | Pediatric Quality of Life Inventory |
| PFIC | progressive familial intrahepatic cholestasis |
| PI | principal investigator |
| PIC | Patient Impression of Change questionnaire |
| PK | pharmacokinetic |
| PSC | primary sclerosing cholangitis |
| PND | post-natal day |
| Pt | patient |
| PT | prothrombin time |
| qAM | every morning |
| QD | once daily |
| q.s. | quantity sufficient |
| SAE | serious adverse event |
| SAP | statistical analysis plan |
| sBA | serum bile acid |
| SD-5613 | original designation for LUM001 |
| sec | second |
| SLC10A2 | solute carrier family 10 member 2; gene that encodes IBAT protein |
| SOC | system organ class |
| SUSAR | suspected unexpected serious adverse reaction |
| TG | triglycerides |
| TGR5 | a G protein-coupled receptor for bile acids |
| UDCA | ursodeoxycholic acid, ursodiol |
| ULN | upper limit of normal |
| US, USA | United States of America |
| WBC | white blood cell |
| WHO | World Health Organization |
| WMA | World Medical Association |
| yr(s) | year(s) |

### 3 STUDY OBJECTIVES

The objectives of this study (up to and including Week 48) are:

- To evaluate the long-term safety and tolerability of LUM001 in children with ALGS.
- To evaluate the effect of LUM001 on serum bile acid levels in children with ALGS.
- To evaluate the effect of LUM001 on biochemical markers of cholestasis and liver disease in children with ALGS.
- To evaluate the effect of LUM001 on pruritus in children with ALGS.
- To evaluate the long-term effect of LUM001 in children with ALGS during 48 weeks of treatment.

Objectives of Long-term Optional Follow-up Treatment Period (after Week 48):

- To offer eligible subjects treated in the LUM001-304 study continued study treatment at Week 48 until the first of the following occurs: (i) the subjects are eligible to enter another LUM001 study (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.
- To explore twice a day (BID) dosing regimen and higher daily dosing of LUM001.
- To obtain safety and efficacy data in subjects treated long term on LUM001 including genotyping characteristics.
- To assess the level of alpha-fetoprotein (AFP), a marker of hepatocellular carcinoma.
- To assess palatability of the LUM001 formulation.

### 4 BACKGROUND AND RATIONALE

LUM001 is an inhibitor of the ileal bile acid transporter/apical sodium-dependent bile acid transporter/soluble carrier family 10 member 2 (IBAT/ASBT/SLC10A2), initially developed as a lipid lowering agent (SD-5613). By virtue of its ability to inhibit bile acid absorption, LUM001 is being developed as a therapeutic agent for signs and symptoms of cholestatic liver disease.

### 4.1 Therapeutic Rationale

In patients with ALGS, impairment of the egress of bile acids from the liver leads to cholestasis, hepatocellular injury and damage, and progressive liver disease that may ultimately lead to the need for liver transplantation. Present in most patients with ALGS, Itch is the archetypal symptom of cholestasis, occurring at all stages of cholestatic liver disease, with or without jaundice.

Surgical interruption of the enterohepatic circulation in children with cholestatic liver disease has been shown to be beneficial. However, complications do occur and many patients and their families are reluctant to accept a permanent external ostomy in spite of the expected benefits. Pharmacological diversion of bile acids to the distal gut with an ASBTi/IBATi could be an attractive alternative to surgical intervention in ALGS.

LUM001 is a potent inhibitor of ASBT/IBAT. The ASBT/IBAT is present in lumen of the terminal 25% of the small intestine. This transporter mediates the uptake of conjugated bile acids across the brush border membrane of the enterocyte. Additional proteins and transporters carry bile acids from the enterocyte through the intestinal wall into the blood stream, where they are circulated to the liver via the portal vein and then re-secreted into the intestine in a system known as the enterohepatic circulation. Ninety-five percent of bile acids that enter the gut lumen are recycled to the gallbladder where they are stored for future release to the duodenum.

Figure 1: Interruption of Enterohepatic Circulation with an ASBT/IBAT Inhibitor



ASBT=apical sodium-dependent bile acid transporter.

ASBT/IBAT expression is under negative feedback regulation by bile acids; thus in the setting of cholestasis, ASBT/IBAT is maladaptively upregulated (Neimark et al., 2004; Hofmann, 2003). Therefore, inhibiting the reuptake of bile acids may represent an ideal treatment for cholestatic disease. In the current study, ALGS will serve as a model for generalized cholestasis. By inhibiting the intestinal reabsorption of bile acids, LUM001 could interrupt the enterohepatic circulation and mimic the effects of partial external biliary diversion of ileal exclusion (Figure 1).

## 4.2 Alagille Syndrome

Alagille syndrome (ALGS) is an autosomal dominant with variable penetration genetic multisystem disorder. The clinical diagnosis is based on the presence of intrahepatic bile duct paucity on liver biopsy in association with at least three of the major clinical features: chronic cholestasis, cardiac disease, skeletal abnormalities, ocular abnormalities and characteristic facial features. Fewer than 200 patients with ALGS are born each year in the United States. The estimated prevalence in the United States is 3 per 100,000. Elevations of serum bilirubin up to 30 times normal and serum bile salts up to 100 times normal are common. Levels of markers of bile duct damage, including gamma-glutamyltransferase (GGTP or GGT) and alkaline phosphatase (ALP), usually are significantly elevated. Cholesterol levels may also be elevated. Multiple xanthomas are common sequelae of severe cholestasis. The pruritus seen in patients with this condition is among the most severe of any chronic liver disease and it is present in most children by the third year of life. Although surgical interruption of the enterohepatic circulation has been successfully employed in the treatment of cholestasis and hypercholesterolemia in ALGS (Emerick and Whitington, 2002; Modi et al., 2007), the management of cholestasis in ALGS remains largely supportive at this time. As cholestasis tends to improve over the first 5 to 10 years, therapies that ameliorate the complications of cholestasis, without a commitment to liver transplantation, are highly desirable (Emerick et al., 1999).

### 4.3 Pruritus

Patients with ALGS and cholestatic liver disease frequently present with pruritus, which can be severe, even in the absence of jaundice. Elevation of serum bile acids is frequently accompanied by pruritus, and a causal association between pruritus and bile acids is suggested by the following: (1) pruritus can been induced in volunteers by applying topical unconjugated bile acids, deoxycholate and chenodeoxycholate to the skin; and (2) pruritus can be relieved by surgical interruption of the enterohepatic circulation, which dramatically lowers serum bile acids.

Intractable and pharmacologically recalcitrant pruritus is one of the major morbidities afflicting children with ALGS. Treatment with anti-pruritics and bile salt resins may provide partial relief of itching for children with ALGS, but currently available pharmacologic approaches are of limited value. It has been shown that removing bile with surgical procedures such as partial external biliary diversion (PEBD) and nasal biliary drainage (NBD) substantially reduces pruritus in ALGS (Emerick and Whitington, 2002), progressive familial intrahepatic cholestasis (PFIC) and primary biliary cholangitis (PBC). Almost complete resolution of pruritus has been observed in children with PFIC disease in a period of as little as two to four weeks following the procedure. The rapid resolution of itch in response to therapy can be seen in Figure 2 extracted

from the original description of this procedure by (Whitington and Whitington, 1988). Rapid lowering of bile acids, bilirubin, and ALT has also been observed (Table 1).

Figure 2: Serum Bile Salt Concentration and Degree of Itch



Patient SR- serum bile salt concentration and degree of itch over a 4-yr course. Nasoduodenal drainage (D) resulted in reduced serum bile salt concentration and itch. When medical management failed, a cholecystostomy tube was placed  $(S_1)$ , resulting in a reduction in serum bile salt concentration to normal and the disappearance of itching. When the cholecystostomy tube was accidentally pulled out (A), the serum bile salt concentration and itching increased rapidly. The construction of a permanent cholecystostomy  $(S_2)$  resulted in a quick return to normal, a state that has been maintained since (Whitington and Whitington, 1988).

Table 1: Improvement in Biochemical Markers and Pruritus After Partial External Biliary Diversion in PFIC Disease and Alagille Syndrome Subjects

| | Age at<br>Surgery | | Pruritus Score<br>(0-4 Scale)* Serum Bile Acids<br>(µM) | | Conjugated<br>Bilirubin<br>(µM) | | Alanine<br>Aminotransferase<br>(IU/L) | | |
|---|---|---|---|---|---|---|---|---|---|
| Diagnosis | (yrs) | Pre | Post | Pre | Post | Pre | Post | Pre | Post |
| PFIC | 3 | 4 | 0 | 226 | 2 | 24 | 0 | 140 | 30 |
| PFIC | 9 | 4 | 0 | 225 | 3 | 80 | 0 | 193 | 13 |
| PFIC | 3 | 4 | 0 | 275 | 9 | 17 | 0 | 155 | 69 |
| PFIC | 3 | 4 | 0 | 218 | 5 | 68 | 10 | 141 | 64 |
| Alagille | 12 | 4 | 1 - 2 | 153 | 37 | 164 | 77 | 198 | 168 |
| Alagille | 6 | 4 | 1 | 317 | 25 | 50 | 15 | 248 | 305 |

<sup>\* 0 =</sup> no itching; 4 = itching with cutaneous mutilation and bleeding (Whitington and Whitington, 1988)

### 4.4 **LUM001**

### 4.4.1 Nonclinical Studies

### 4.4.1.1 Pharmacology

LUM001 is a minimally-absorbed, potent selective inhibitor of the ileal apical sodium-dependent bile transporter, a transmembrane protein localized on the luminal surface of ileal enterocytes, commonly referred to as ASBT/IBAT. The drug is a competitive inhibitor for bile acid substrate

with a high affinity for the transporter. Nonclinical studies indicate that selective inhibition of ASBT by LUM001 results in increased fecal bile acid excretion, inhibition of the postprandial rise in serum bile acids, and decrease in serum total cholesterol. It also increases the activity of hepatic cholesterol  $7\alpha$ -hydroxylase and 3-hydroxy-3-methyl-glutaryl-CoA (HMG-CoA) reductase, consistent with inhibition of bile acid reabsorption as the mechanism of action.

### 4.4.1.2 Pharmacokinetics

Because of its large molecular weight and the presence of a quaternary nitrogen atom, LUM001 is poorly absorbed from the gut. In rats and dogs, oral bioavailability was < 0.4% at all doses tested. LUM001 is metabolically stable after oral administration. After intravenous administration, the majority of drug is excreted in the feces, with approximately 5% excretion in the urine.

# 4.4.1.3 Toxicology

A comprehensive assessment of LUM001 has been conducted in vitro and in animals. LUM001 is not toxic at doses much higher than those that are pharmacologically active in mice, rats, dogs, and monkeys. The most significant effect observed in rodents is a prolongation of coagulation time considered secondary to malabsorption of vitamin K, which in turn is related to inhibition of bile acid absorption, the pharmacologic effect of LUM001. Reversible prolongation of coagulation times was observed primarily in male rats that are especially sensitive to agents that alter vitamin K absorption and may not be an appropriate model for predicting vitamin K malabsorption in humans. Acute oral doses up to 200 mg/kg LUM001 were well tolerated in dogs, with emesis as the primary dose-limiting toxicity. There was no evidence of mutagenic activity in vitro and no clastogenic activity in vitro or in vivo. Results from rat and rabbit embryo/fetal development studies with doses up to 1000 and 250 mg/kg/day, respectively, showed no adverse effects on fetal growth and development.

To support the use of LUM001 in young children, a toxicity study in juvenile animals was completed. As expected for a drug intentionally designed to be minimally absorbed, LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies with adult rats. No adverse effects were observed on postnatal growth and development of offspring at a dose of 200 mg/kg/day in males and 1000 mg/kg/day in females, the highest doses tested. This study was initiated in juvenile animals at PND21, which from a whole animal development perspective is typically representative of a 2 year old child. However given the fact that LUM001 is a minimally absorbed drug, as evidenced by this and multiple other studies, of particular importance is the age at which the GI tract is considered functionally mature. In humans this occurs by 12 months of age; likewise, postnatal maturation of the GI tract in rats occurs during the first three weeks of birth. Therefore this study presented evidence to support the safety of LUM001 in future clinical trials in children 12 months of age and older. These trials have the promise to address a life-threatening clinical need in this patient population.

Additional toxicology information can be found in the investigator's brochure.

### 4.4.2 Previous Clinical Experience

Detailed information concerning the clinical studies conducted with LUM001 can be found in the investigator's brochure. A summary is included below.

The overall objective of the initial clinical development plan was to evaluate the safety and efficacy of chronic, oral administration of LUM001 (tablet and capsule formulations) for the reduction of serum LDL-C in subjects with hypercholesterolemia. The efficacy, pharmacokinetics, tolerability, and safety of LUM001 in humans have been evaluated in a total of 12 clinical studies, including 2 studies that also tested sustained release formulations. Phase 1 studies included a single and two multiple dose tolerability studies, an absorption, distribution, metabolism, and excretion (ADME) study, a statin co-administration study, a statin interaction study, and a food composition study. Phase 2 studies included two dose-ranging studies in adult subjects, a tolerability study in adolescents and children, and a multiple dose tolerability and efficacy study of three sustained release formulations, compared with the immediate release formulation. More than 1,400 human subjects have been exposed to LUM001 (immediate release) for up to 10 weeks.

In previous clinical studies, LUM001 inhibited the postprandial increase in serum total bile acids concentrations and increased fecal total bile acids excretion, consistent with the mechanism of action of inhibiting ASBT. LUM001 administration resulted in reductions of serum LDL-C in healthy volunteers and subjects with elevated cholesterol. These findings confirm that LUM001, a minimally absorbed inhibitor of ASBT, is effective in blocking enterohepatic recirculation of bile acids with the expected consequences on bile acid and cholesterol metabolism. With LUM001 administration, there was also a trend toward increases in high-density lipoprotein cholesterol (HDL-C) and total triglycerides relative to placebo.

Administration of LUM001 at doses up to 100 mg once daily over a four-week period was generally safe in healthy volunteers and at doses up to 40 mg once daily for up to 10 weeks in subjects with hypercholesterolemia. The most commonly reported adverse drug reactions in LUM001-treated subjects were abdominal cramping (pain) and diarrhea and loose stools. These GI AEs are also observed in patients who undergo biliary diversion, are believed to be mechanism-based, due to elevated bile acid concentrations in the colon. With the exception of a single serious adverse event of cholecystitis no other SAEs possibly related or related to LUM001 have been reported in the 12 studies conducted to date (over 1,400 subjects exposed).

The majority of orally administered LUM001 was excreted intact in the feces along with a few minor metabolites. LUM001 exposure in adolescents and children (Study 014) was low and consistent with a drug that is minimally absorbed. Pharmacokinetic parameters in adolescent and children subjects did not significantly differ from those seen in adult subjects.

No clinically significant laboratory abnormalities were documented in LUM001-treated subjects. LUM001 was associated with mild, often transient elevations of serum ALT in a small percentage of subjects. Clinically significant reductions of serum fat-soluble vitamin levels were not observed with LUM001 treatment in humans; however, levels of the carotenoid  $\beta$ -carotene were mildly reduced. No alterations in coagulation parameters were observed, indicating no

functional changes in vitamin K status. Fecal fat excretion was not increased compared to placebo after four weeks of LUM001 treatment at doses up to 100 mg.

### 4.5 Rationale for Dose and Schedule of Administration

The dosage of LUM001 chosen for the first studies in cholestatic subjects is based upon prior experience with this product in healthy volunteers and subjects with hypercholesterolemia. In these subjects, with normal bile flow and without liver disease, tolerability was limited above 10 mg daily by an increase in GI AEs. These signs and symptoms were believed to be related to increased bile acid excretion and an increased concentration of free bile acids in the lower colon. In patients with cholestatic liver disease it is likely that bile flow is reduced compared to healthy volunteers and hypercholesterolemic patients and LUM001 will produce a correspondingly smaller increase in free bile acids in the lower colon, and could potentially lead to the drug being better tolerated at the same dose level.

Ideally, dosing in pediatric subjects should be scaled from that in adults based on intestinal length, ie, mg of drug per cm of intestine. Differing relationships between intestinal mucosal surface area, age, and body weight have been reported in the literature (Weaver et al., 1991) provided data indicating that the average length of the small intestine increases with age from birth through 20 years; this relationship followed a curve that is similar to the height and weight growth curves (Weaver et al., 1991). However, a plateau had not been reached at the maximum age examined (20 years), precluding predictions of intestinal length for older adults and thus scaling to infants and children based on estimated intestinal length. An analysis of intestinal length as a function of age, weight, and height in adult cadavers was conducted by Hounnou et al (2002). Their analysis demonstrated that age had a negative correlation and body weight a positive correlation with intestinal length. Taken as a whole, the existing analyses are inconclusive with respect to the dependent variables that predict intestinal length. Consequently, the most reasonable approach is to calculate doses in a pediatric subject from those in adults based on using a direct mg/kg scaling. For reference in an average adult subject, weighing 70 kg, a 10 mg daily dose is equivalent to 140  $\mu$ g/kg/day.

Daily exposure (mg/day) across dose levels for subjects ranging in weight from 10-30 kg is depicted in Table 2.

Table 2: Sample Daily Exposure (mg/day) in Pediatric Subjects

| Weight | LUM001 | | | | | |
|---|---|---|---|---|---|---|
| (kg) | Dose Level 1 | Dose Level 2 | Dose Level 3 | Dose Level 4 | Dose Level 5 | Dose Level 6 |
| . 0/ | (14 µg/kg/day) | (35 µg/kg/day) | (70 μg/kg/day) | (140 μg/kg/day) | (280 μg/kg/day) | (560 μg/kg/day) |
| 10 | 0.14 | 0.35 | 0.70 | 1.40 | 2.80 | 5.60 |
| 15 | 0.21 | 0.53 | 1.05 | 2.10 | 4.20 | 8.40 |
| 20 | 0.28 | 0.70 | 1.40 | 2.80 | 5.60 | 11.20 |
| 25 | 0.35 | 0.88 | 1.75 | 3.50 | 7.00 | 14.00 |
| 30 | 0.42 | 1.05 | 2.10 | 4.20 | 8.40 | 16.80 |

In a previous study (Study 014), LUM001 was administered to 40 hyperlipidemic pediatric subjects (n=5, children ages 10-11; n=35 adolescents ages 12-17), up to a maximum tested dose of 5 mg/day for 14 days. The average subject weight in Study 014 was 60 kg and a 5 mg/day

dose of LUM001 was approximately equivalent to 83  $\mu$ g/kg/day. Plasma LUM001 exposure in adolescents and children was low (non-detectable <0.25cng/mL to 1.13 ng/mL) and consistent with a drug that is minimally absorbed. Detection of LUM001 in plasma samples was sporadic, both within and among subjects. In addition there does not appear to be a relationship with either subject age or gender. These data do not differ from the extensive pharmacokinetic data collected in adults to date. Although the bioavailability of LUM001 has not yet been characterized in children younger than 10 years of age, the GI systems are functionally mature in children by about 1 year of age (Walthall et al., 2005; van den Anker et al., 2011). This study will enroll children between the ages of 12 months and 18 years, inclusive.

In Study 014 no drug related serious AEs were observed. The most frequently reported AEs in all treatment groups (LUM001 and placebo) were diarrhea, abdominal pain, loose stools, and nausea. A total of 49 of 50 subjects completed 14 days of treatment. Most AEs were assessed with a probable or uncertain relationship to study medication and were generally characterized as mild or moderate in severity, except for those in six subjects who experienced severe nausea, diarrhea, or abdominal pain. These GI events usually resolved during continued treatment. It is noteworthy that the AEs were generally recorded in the first seven days of LUM001 dosing, and observed at a four-fold lower frequency from Day 8 to 14. This is consistent with the extensive adult dosing experience, where GI events were observed at levels similar to those in the placebo group after two weeks of continuous dosing.

To assess the effects of dose titration to mitigate dose-limiting adverse effects, LUM001 was evaluated in a 28-day once-daily dosing study in healthy volunteers (Study 003). In one arm, the dose was increased after each 7-day dosing period, to a maximum of 5 mg daily (equivalent to a dose of 67  $\mu$ g/kg/day, using the average subject weight). Using this dosing regimen, the incidence of GI-associated AEs was lower than those observed in the placebo group (Table 3) and in other treatment arms with constant dosing above and below 5 mg daily.

Table 3: GI-associated Adverse Events in Study 003

| GI Adverse Events | Placebo<br>(n=20) | 1 mg qAM<br>(n=8) | 2.5 mg qAM<br>(n=25) | 5 mg qAM<br>(n=26) | 0.5-5 mg<br>qAM*<br>(n=16) |
|---|---|---|---|---|---|
| Abdominal pain | 2 (10%) | 3 (37%) | 4 (16%) | 5 (17%) | 1 (6.3%) |
| Constipation | 2 (10%) | 0 | 3 (12%) | 0 | 0 |
| Diarrhea | 1 (5%) | 1 (12%) | 5 (20%) | 2 (7%) | 0 |
| Nausea | 0 | 0 | 1 (4%) | 1 (4%) | 0 |
| Pruritus Ani | 0 | 0 | 6 (24%) | 4 (15%) | 0 |

<sup>\*</sup>Escalation regimen: 0.5 mg qAM (7 μg/kg/day) on Days 1-7, 1 mg qAM (13 μg/kg/day) on Days 8-14, 2.5 mg qAM (33 μg/kg/day) on Days 15-21, 5 mg qAM (67 μg/kg/day) on Days 22-28. Average body weight 75 kg.

The appropriate efficacious dose of LUM001 for the lowering of bile acid concentrations and the reduction of pruritus in cholestatic populations is not known. However, earlier studies demonstrated that doses of 10 mg daily (equivalent to 140  $\mu$ g/kg/day for a 70 kg subject) led to a decrease in serum bile acids in healthy volunteers by >50% following 2 weeks of treatment. In

the PFIC population, there is some evidence that ASBT is upregulated, suggesting that higher doses may be required to saturate transporters and reach the desired effect in PFIC disease.

The doses explored in the current study (up to 400 µg/kg/day BID) in subjects with ALGS are supported by the safety profile observed in completed and ongoing clinical studies of LUM001. Twice daily dosing is used in this study based on the findings of a healthy volunteers study in adult males (Study SHP625-101), which demonstrated that bile acid levels in feces increase with escalating doses and twice-daily regimen of LUM001 (up to 100 mg QD and 50 mg BID, respectively). In this study, subjects who were randomized to LUM001 treatment, received 1 of 4 doses of LUM001 (10, 20, 50, 100 mg) during 7 days. No titration was used in this study. There was a dose-dependent increase in total fecal BA excretion. In addition, BID dosing (ie, 50 mg BID) led to a further increase in fecal BA excretion as compared to QD dosing (ie, 100 mg QD). It is therefore hypothesized that higher doses and twice-daily dosing both have the potential to allow for more complete target engagement throughout the day at the level of the distal ileum.

The higher dosing level is also supported by favorable results from a juvenile toxicity study conducted in rats administered LUM001 for 43 days (post-natal day, PND21 through PND63). As expected for a drug intentionally designed to be minimally absorbed, systemic LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies in adult rats. No adverse effects were observed on postnatal growth and development of offspring at the highest doses tested (200 mg/kg/day in males, 1000 mg/kg/day in females). This study was initiated in juvenile animals at PND21, which from a whole animal development perspective, is typically representative of a 2-year old child. However, given the fact that LUM001 is a minimally absorbed drug, of particular importance is the age at which the GI tract is considered functionally mature. In humans this is considered to have occurred by 12 months of age; likewise, postnatal maturation of the GI tract in rats occurs during the first 3 weeks of life. Therefore, results from this study can be used to support the dosing levels proposed here for children 12 months of age and older.

### 5 INVESTIGATIONAL PLAN

# 5.1 Study Design

This is a long-term open-label study with a double-blind, placebo-controlled, randomized drug withdrawal period in children with ALGS designed to evaluate the safety and efficacy of LUM001. The study is divided into 6 parts: a 6-week open-label, dose escalation period at doses up to 400  $\mu$ g/kg/day, a 12-week open-label stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period at doses up to 400  $\mu$ g/kg/day, a 52-week optional follow-up treatment period, and a long-term optional follow-up treatment period for eligible subjects who choose to stay on treatment with LUM001. During this long-term optional follow-up period, subjects may have their dose of LUM001 increased to a maximum of 800  $\mu$ g/kg/day (400  $\mu$ g/kg BID), based on efficacy (sBA level and ItchRO[Obs] score) and safety assessment. Subjects' participation in the long-term optional follow-up treatment period will continue until the first of the following occurs: i) the subjects are eligible to enter another LUM001 study, ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.

Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3.

# **5.2 Data Monitoring Committee**

A Data Monitoring Committee (DMC) will review serious adverse event data, other key subject safety and study data at specified intervals for the duration of the study. The DMC will be composed of several members who are otherwise independent from the conduct of the study: two or more physicians and one biostatistician. The DMC's primary responsibility is to review the progress of the study, particularly with regard to safety and risk/benefit, and make recommendations to stop or modify the study if safety concerns are identified. Further details regarding the structure, function and operation of the DMC will be detailed in the DMC charter.

### **5.3** Number of Study Centers

This will be a multi-center study in approximately 9 clinical sites.

### 5.4 Number of Subjects

Approximately 30 subjects will be enrolled in this study.

### 5.5 Overall Study Duration and Follow-up

For an individual subject, the study participation period will consist of a screening period of up to 4 weeks, a 48-week treatment period (including a 6-week, open-label dose escalation period, a 12-week open-label stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period) as well as a 52-week optional follow-up treatment period, and a long-term optional follow-up treatment period. A safety follow-up phone call will be made by the study site 30 days after the last dose of study drug.

Following screening, during the 48-week treatment period, subjects who meet all eligibility criteria will return to the clinic for 9 visits and will receive 14 telephone contacts from the study staff (see Figure 3). Subjects who complete 48 weeks of treatment may be eligible to receive further treatment during the 52-week optional follow-up treatment period and the long-term optional follow-up treatment period. Subjects' participation in the long-term optional follow-up treatment period will continue until the first of the following occurs: (i) the subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.

Study activities will be conducted as described in the Schedule of Procedures (Section 16.1).

400 μg/kg/day 280 μg/kg/day 70 μg/kg/day 35 μg/kg/day 14 μg/kg/day Placebo Randomized Open Label 26 Week Long-Term Exposure Withdrawal Follow-up **Dose Escalation** Stable Dose 1:1 Randomized Withdrawal 30 days 6 weeks 12 weeks 4 weeks Study 18 20 24 25 26 27 28 Week days = Clinic Visit = Phone Contact

Figure 3: Study Design for LUM001-304 (Day 0 – Week 48)

Figure 4: 52-week Optional Follow-up Treatment Scheme (<7 days from last LUM001 dose)

Applies to the following subject population:

• Subjects who experienced no interruption in LUM001 dosing, or interruption <7 days between Protocol Amendment 2 and Protocol Amendment 3.



<sup>\*\*</sup>In consultation with Medical Monitor, the dose may be lowered to a previously well-tolerated dose to address tolerability issues at any time during the study\*\*

\*\*At the Investigator's discretion, subjects who were previously down-titrated may be re-challenged during the follow-up period\*\*

Figure 5: 52-week Optional Follow-up Treatment Scheme (≥7 days from last LUM001 dose)

Applies to the following subject population:

• Subjects who experienced an interruption in LUM001 ≥7 days between Protocol Amendment 2 and Protocol Amendment 3.



Abbreviations: DE=dose escalation; FTP=follow-up treatment period.

Figure 6: Long-term Optional Follow-up Treatment Scheme (≥7 days from Last LUM001 Dose between Protocol Amendment 3 and Protocol Amendment 4)

Applies to the following subject population:

• Subjects who experienced an interruption in LUM001 ≥7 days between Protocol Amendment 3 and Protocol Amendment 4.



Abbreviations: ADE=afternoon dose escalation; DE=dose escalation; PA=protocol amendment; Wk=week.

Figure 7: Long-term Optional Follow-up Treatment Scheme, without Afternoon Dose Escalation (ADE)

Applies to the following subject population:

• Subjects deemed ineligible for ADE

# Without ADE



Abbreviations: EOT=end of treatment; ET=early termination; MTD=maximum tolerated dose; Wk=week.

Figure 8: Long-term Optional Follow-up Treatment Scheme under Protocol Amendment 4, with Afternoon Dose Escalation (ADE)

Applies to the following subject population:

• Subjects whose sBA levels have not normalized and/or whose ItchRO Obs score is  $\geq 1.5$  and therefore qualify for introduction of afternoon dosing.



Abbreviations: ADE=afternoon dose escalation; MTD=maximum tolerated dose; Wk=week.

# 5.5.1 Screening

Each subject who provides informed consent/assent will complete all screening activities in  $\leq$ 4 weeks.

### 5.5.2 Treatment

Study drug will be prepared for each individual subject by a central pharmacy based on the subject's weight at screening. Diluent will be added by the central pharmacy pharmacist prior to shipping study drug to the site. Study drug will be dispensed to subjects/caregivers. During the course of the study, it may be necessary to instruct the subject/caregiver to return to the site for an unscheduled dispensation of study drug. The appropriate amount of study drug will be dispensed at the Study Day 0 visit and daily dosing will begin on Study Day 1.

Subjects will receive a grape-flavored solution containing LUM001 administered orally once a day (QD) or twice a day (BID) using the syringe provided. The first dose should be taken at least 30 minutes prior to the first meal of the day and the second dose, where applicable, should be taken at least 30 minutes prior to dinner (main evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the dose should be taken approximately at the same time each day for the duration of the treatment period.

All subjects will receive LUM001, up to 400  $\mu g/kg/day$  or a maximum daily dose of 20 mg/day, during the initial open-label treatment period of the study. After completion of the 12-week stable dosing period, subjects will be randomized 1:1 to either a 4-week double-blind study drug withdrawal period during the study or will remain on study drug. Subjects will then enter a 26-week long-term stable dosing period and all subjects will receive LUM001, up to 400  $\mu g/kg/day$  or a maximum daily dose of 20 mg/day during the initial open-label treatment period of the study. Subjects will be considered for a 52-week optional treatment period, if eligible, receiving up to 400  $\mu g/kg/day$ , or the highest tolerated dose below the 400  $\mu g/kg/day$  dose. Subjects will then be considered for the long-term optional follow-up treatment, if eligible, receiving up to 800  $\mu g/kg/day$  (given as twice daily doses of 400  $\mu g/kg$ ), or a maximum possible daily dose of 50 mg/day.

During the study, the study drug may be adjusted if there is a change of  $\geq 10\%$  in body weight since the screening visit or if there is a change of  $\geq 10\%$  in weight since the last weight-based medication adjustment to maintain the target dose.

### **5.5.2.1 Dose Escalation Period**

Initially, the LUM001 dose will be administered as a daily morning dose in either a 1.0 mL or 0.5 mL solution. The dose will be increased weekly over a 6-week period up to 400  $\mu$ g/kg/day QD or a maximum daily dose of 20 mg/day QD as follows:

Week 1 Dose: 14 μg/kg/day QD Week 2 Dose: 35 μg/kg/day QD Week 3 Dose: 70 μg/kg/day QD Week 4 Dose: 140 μg/kg/day QD Week 5 Dose: 280 μg/kg/day QD

Week 6 Dose: 400 µg/kg/day QD (maximum daily dose of 20 mg QD)

Subjects should be administered study drug daily for at least 7 days at each dose level during the dose escalation period.

If a subject experiences intolerance due to gastrointestinal symptoms (eg, diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the medical monitor may lower the dose to a previously tolerated dose; later attempts to escalate the dose are permitted. In these circumstances, an unscheduled visit will occur and the appropriate

replacement study medication will be issued to the subject as quickly as possible. If the subject is on a BID dosing regimen, dose lowering should first be attempted with the afternoon dose.

# **5.5.2.2 Stable Dosing Treatment Period**

Subjects will continue dosing for another 12 weeks using the dose administered at Week 6, which may be 400 µg/kg/day or the highest tolerated dose below 400 µg/kg/day.

# 5.5.2.3 Double-blind Placebo-controlled Study Drug Withdrawal Period

At the Week 18 visit, eligible subjects will be randomized 1:1 to continue to receive study drug or a corresponding placebo for 4 weeks.

### 5.5.2.4 Long-term Exposure Period

Following the 4-week study drug randomized withdrawal period, subjects who received placebo will receive LUM001 dosed according to a dose escalation schedule that mirrors the initial escalation (ie, the LUM001 dose will be increased weekly over a 6-week period to the maximum tolerated dose up to 400  $\mu$ g/kg/day or 20 mg/day or the highest tolerated dose below the 400  $\mu$ g/kg/day dose). Subjects who were randomized to receive LUM001 during this period will continue to receive the same dose of LUM001 and, following Week 22, a simulated dose escalation will occur to maintain the blind in the randomized withdrawal period. Dosing with LUM001 will continue in a 26-week long-term exposure period to complete 48 weeks of study.

During the long-term exposure period, the dose may be adjusted to account for a change of  $\geq 10\%$  in weight since the screening visit (eg the amount of drug dosed may be increased to reflect the subject's weight increase).

# 5.5.2.5 52-week Optional Follow-up Treatment Period

At Week 48, all subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over into the 52-week optional follow-up treatment period. The 3 following possible scenarios may occur:

- Subjects who are eligible to roll over into the optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level.
- Subjects who are eligible to roll over into the optional follow-up treatment period with a LUM001 dosing interruption of ≥7 days will be dose escalated beginning at 35 µg/kg/day and up to a maximum of 400 µg/kg/day or highest tolerated dose (as detailed in Section 8.1.8.
- Subjects who do not wish to enter the follow-up treatment period will be contacted via telephone by the study site approximately 30 days after the last dose of study drug.

### 5.5.2.6 Long-term Optional Follow-up Treatment Period

Upon completion of the 52-week optional follow-up treatment period, and/or implementation of this amendment, whichever occurs first, subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over (or enter) the long-term optional treatment period. The 3 following possible scenarios may occur:

# Scenario 1: Subjects eligible to roll over into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 continuous days:

- Subjects with normal sBA level AND ItchRO(Obs) score <1.5 will be maintained at the same dose level and will continue morning dosing only.
- Subjects with sBA level above normal AND/OR ItchRO(Obs) score ≥1.5 will start BID dosing (afternoon dose escalation; ADE) as follows:
  - The morning dose will be continued at the same dose level, but the volume of the morning dose will be reduced by half at the same time that the afternoon dose is initiated.
  - $\circ$  The afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg.

# Scenario 2: Subjects eligible to roll over into the long-term optional follow-up treatment period with a LUM001 interruption of $\geq 7$ days:

- First, the morning dose is escalated up to 400  $\mu$ g/kg/day or highest tolerated dose following a 5-week dose escalation beginning at 35  $\mu$ g/kg/day.
- Once the morning dose of 400  $\mu$ g/kg or maximum tolerated dose is achieved, sBA and ItchRO(Obs) score will be evaluated.
  - Subjects with normal sBA AND ItchRO(Obs) score <1.5 after morning dose escalation will be maintained at the same dose level and will continue morning dosing only.
  - Subjects with sBA above normal AND/OR ItchRO(Obs) score ≥1.5 will begin BID dosing (ADE) as outlined as follows:
    - The morning dose will be continued at the same dose level, but the volume of the morning dose will be reduced by half at the same time that the afternoon dose is initiated
    - The afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg.

The following parameters apply to both dosing scenarios outlined above:

- The afternoon dose will only be initiated once the subject has been treated on stable morning doses for at least 4 weeks.
- The sBA value used for determination of ADE eligibility will be the most recent available value collected within the prior 16 weeks. The ItchRO(Obs) score used for ADE eligibility will be derived from the most recent available 7-day interval of ItchRO(Obs) collected within the prior 16 weeks.
- The maximum daily dose will be 400  $\mu$ g/kg BID, ie, 800  $\mu$ g/kg/day (up to a maximum possible daily dose of 50 mg/day).

Subjects will continue to receive study drug until they are eligible to enter another LUM001 study, or until LUM001 is available commercially, or until the sponsor stops the program or development in this indication, whichever occurs first.

If a subject experiences intolerance (eg, gastrointestinal symptoms such as diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the medical monitor may lower the dose for the remainder of the study; later attempts to escalate the dose are permitted. If the subject is on a BID dosing regimen, dose lowering should first be attempted with the afternoon dose.

# Scenario 3: Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3.

### 5.5.3 Safety Follow-up Period

A safety follow-up phone call will be made by the study site 30 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and any AEs noted during this phone call will be recorded. Subjects who complete the study or who discontinued early due to reasons other than safety may be eligible for participation in the long-term optional follow-up treatment period under Protocol Amendment 4.

Additional study drug will be supplied at each clinic visit during the follow-up treatment period. Used study drug will be collected at each clinic visit and dosing compliance will be assessed.

### 5.6 End of Study

For subjects who do not consent to the long-term optional follow-up treatment period, a subject is considered to have completed treatment if treatment was not permanently discontinued prior to the Week 48 visit. A follow-up phone contact is required for all subjects should the final visit occur earlier than 30 days from the final dose.

The subject is considered to have completed treatment and study period for the corresponding follow-up treatment period (when consented under Protocol Amendment 3 or Protocol

Amendment 4) if study treatment was not discontinued prior to completing Week 96 for Protocol Amendment 3 or completing the EOT visit in Schedule J under Protocol Amendment 4. Temporary drug interruption is not considered treatment discontinuation. A follow-up contact is required for all subjects should the final visit occur earlier than 30 days from the final dose.

The end of study for the purposes of regulatory reporting is the point at which the last contact with the last subject during the protocol-specified scheduled follow-up period is made.

### **6 SUBJECT ENROLLMENT**

# 6.1 Screening

Before subjects may be screened for eligibility to participate in the study, the sponsor, or designee, requires a copy of the appropriate written Independent Ethics Committee (IEC) approval of the protocol, informed consent/assent form(s) (ICF), and all other applicable subject information and/or recruitment material.

Following informed consent/assent, the subject will be considered enrolled into the study and will be assigned a unique subject identification number before any study procedures, including screening procedures, are performed. This number will be used to identify the subject throughout the study and must be used on all study documentation related to that subject. The subject identification number must remain constant throughout the entire study. In the event the subject is re-consented and rescreened, the subject must be given a new subject identification number. Subject identification numbers, once assigned, will not be reused.

Subjects will be enrolled in the optional follow-up treatment period based on the investigator's determination of meeting eligibility criteria outlined in Section 7. A subject will be considered enrolled in the long-term optional follow-up period under Protocol Amendment 4 after the subject consents and the investigator has determined the subject meets study entry eligibility criteria per Protocol Amendment 4. However, any subject who consents to Protocol Amendment 4 and does not meet criteria per the investigator is considered a screen failure for the long-term optional follow-up period under Protocol Amendment 4. Screen failures are eligible for rescreening (Section 8.1.1).

### 6.2 Randomization

Subjects begin the study at Day 0 and are treated in an open-label fashion from Week 1 to Week 18. Subjects will then be randomized 1:1 to continue to receive study drug or a corresponding placebo for 4 weeks between Week 19 and Week 22 at the start of the double-blind, placebo-controlled study drug withdrawal period (Week 19 to Week 22). This randomization will be stratified by response criteria where response is defined as a ≥50% reduction in serum bile acids between Baseline and Week 12 or Week 18. Serum bile acid results will remain blinded after baseline testing.

During the double-blind, placebo-controlled, randomized drug withdrawal period, siblings will be assigned in a blinded manner to the same treatment arm.

The sponsor (or designee) will prepare the randomization list; the pharmacist at a central pharmacy will be unblinded to treatment group. The study staff including the local site pharmacist (or qualified delegate) will remain blinded to the assignment.

### 6.3 Replacement of Subjects

A subject who withdraws from the study prior to completion of the stable dosing treatment period (Week 18) may be replaced at the discretion of the sponsor.

### **6.4** Unblinding of Treatment Assignment

Although subjects begin the study at Day 0 and are treated in an open-label fashion from Week 1 to Week 18, subjects will be randomized 1:1 to continue to receive study drug or a corresponding placebo for 4 weeks between Week 19 and Week 22 at the start of the double-blind, placebo-controlled study drug withdrawal period. The sponsor (or designee) will prepare the randomization list. All subjects, monitors, and study center personnel related to the study, except for the central pharmacist (or qualified designee) who prepares the study drug will be blinded to study treatment during the randomized withdrawal period (Weeks 19-22) and the long-term exposure period (Weeks 23-48) and to the subject's study drug withdrawal period treatment assignment.

After Week 48 the study will be unblinded to facilitate preparation of the interim analysis.

If in the event of an emergency situation when knowledge of the treatment assignment during the double-blind, randomized drug withdrawal period will impact the clinical management of the subject, the investigator will have the ability to unblind the treatment assignment for that subject. If a subject is unblinded by the investigator, the sponsor must be informed of the unblinding within 24 hrs. If the blinding is prematurely broken, it is the responsibility of the investigator to promptly document and explain any unblinding to the sponsor.

All subjects will receive LUM001, or LUM001 and placebo during this study. Breaking of the blind during the initial 48-week period of the study should not occur before all subjects either discontinue or complete Week 48, except in the event of a medical emergency where the identity of the drug must be known in order to properly treat the subject, or when causality must be determined prior to submitting a regulatory safety report for a serious adverse event (SAE) (as defined in Section 11.2.3).

Any unblinding event carried out in connection with submission of a regulatory safety report will be conducted by the sponsor (see Section 11.1).

Every reasonable attempt should be made to complete the Early Termination (ET) study procedures and observations (see Schedule of Procedures, Section 16.1) prior to unblinding, as knowledge of the treatment arm could influence subject assessment.

### 7 SUBJECT ELIGIBILITY

To be eligible to participate in this study, candidates must meet the following eligibility criteria before being assigned to study drug treatment.

### 7.1 Inclusion Criteria

To participate in this study subjects must meet all of the following criteria:

- 1. Male or female between the ages of 12 months and 18 years inclusive.
- 2. Diagnosis of ALGS based on the diagnostic criteria outlined in Section 16.3.
- 3. Evidence of cholestasis (one or more of the following):
  - a. Total serum bile acid > 3x ULN for age.
  - b. Conjugated bilirubin > 1 mg/dL.
  - c. Fat soluble vitamin deficiency otherwise unexplainable.
  - d. GGT > 3x ULN for age.
  - e. Intractable pruritus explainable only by liver disease.
- 4. Females of childbearing potential must have a negative serum pregnancy test during Screening.
- 5. Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial, as described in Section 8.6.1.
- 6. Subject is expected to have a consistent caregiver(s) for the duration of the study.
- 7. Informed consent and assent (per IRB/IEC) as appropriate.
- 8. Access to phone for scheduled calls from study site.
- 9. Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device during the study.
- 10. Caregivers (and age appropriate subjects) must digitally accept the licensing agreement in the eDiary software.
- 11. Caregivers (and age appropriate subjects) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period (maximum possible reports = 14 per week).
- 12. Average daily score >2 on the Itch Reported Outcome (ItchRO™) questionnaire (maximum possible daily score of 4) for two consecutive weeks in the screening period, prior to dosing. A daily score is the higher of the scores for the morning and evening ItchRO. The average daily score is the sum of all daily scores divided by the number of days the ItchRO was completed.

#### 7.2 Exclusion Criteria

Subjects will be excluded from the study if they meet any of the following criteria:

- 1. Chronic diarrhea requiring ongoing intravenous fluid or nutritional intervention.
- 2. Surgical interruption of the enterohepatic circulation.
- 3. Previous liver transplant.
- 4. Decompensated cirrhosis (ALT >15 x ULN, INR >1.5 [unresponsive to vitamin K therapy], albumin <3.0 g/dL, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy).
- 5. History or presence of other concomitant liver disease.
- 6. History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease).
- 7. History or presence of gallstones or kidney stones.
- 8. Known diagnosis of human immunodeficiency virus (HIV) infection.
- 9. Cancers, except for in situ carcinoma, or cancers treated at least 5 years prior to Screening with no evidence of recurrence.
- 10. Recent medical history or current status that suggests that the subject may be unable to complete the study.
- 11. Any female who is pregnant or lactating or who is planning to become pregnant during the study period.
- 12. Known history of alcohol or substance abuse.
- 13. Administration of bile acid or lipid binding resins within 28 days prior to screening and throughout the trial.
- 14. Known hypersensitivity to LUM001 or any of its components.
- 15. Receipt of investigational drug, biologic, or medical device within 28 days prior to screening, or 5 half-lives of the study agent, whichever is longer.
- 16. History of non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to non-adherence with the study protocol based upon investigator judgment.
- 17. Any other conditions or abnormalities which, in the opinion of the investigator or medical monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study.
- 18. Subjects weighing over 50 kg at screening.

### Protocol Amendment 3: Eligible subjects for the 52-week optional follow-up treatment period:

Subjects will be considered eligible for the 52-week optional follow-up treatment period if they have:

• Completed the protocol through the Week 48 visit with no safety concerns. Subjects who were discontinued due to safety reasons can be rechallenged if blood tests are back to relatively normal values for this patient population and subject does not meet any of the

- protocol's stopping rules. The decision will be made by the investigator in consultation with the medical monitor.
- Subjects who have undergone a surgical disruption of the enterohepatic circulation will not be eligible to enter into the follow up treatment period.
- Subjects who were discontinued for other reasons will be considered for the 52-week optional follow-up treatment period on an individual basis. The decision will be made by the investigator in consultation with the medical monitor.

Protocol Amendment 4: Eligible subjects for the long-term optional follow-up treatment period:

Inclusion Criteria for subjects with LUM001dosing interruption <7 days, or  $\ge 7$  days:

Subjects will be considered eligible for the long-term optional follow-up treatment period if they meet the following criteria:

- 1. The subject has either:
  - o completed the protocol through the Week 48 visit with no major safety concerns OR
    - o discontinued due to safety reasons judged unrelated to the study drug, and laboratory results have returned to levels acceptable for this patient population or individual and subject does not meet any of the protocol's stopping rules at the time of entry into the follow-up period. The decision will be made by the investigator in consultation with the medical monitor. [Subjects who were discontinued for other reasons will be considered on an individual basis.]
- 2. Females of childbearing potential must have a negative urine or serum pregnancy test (β-human chorionic gonadotropin [β-hCG]) at the time of entry into the long-term optional follow-up treatment period.
- 3. Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial, as described in Section 8.6.1.
- 4. Informed consent and assent (per IRB/EC) as appropriate.
- 5. Access to phone for scheduled calls from study site.
- 6. Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device during the study.

### Exclusion Criteria for Subjects with LUM001 dosing interruption>7 days:

All exclusion criteria mentioned in Section 7.2 apply upon entry into the long-term optional follow-up period, with the exception of exclusion criterion #18.

### 8 STUDY PROCEDURES

# 8.1 Study Schedule

The schedule of assessments for this study is provided in the Schedule of Procedures, Section 16.1. Subject-related events and activities including specific instructions, procedures, concomitant medications, dispensing of study drug, and descriptions of AEs should be recorded in the appropriate source documents and CRFs.

# 8.1.1 Screening Period (Day -28 to Day -1)

Screening evaluations will be performed from Day -28 to Day -1. In the absence of documented JAGGED1 or NOTCH2 mutation prior to screening, genetic testing may be performed for JAGGED1 and/or NOTCH2 (Spinner et al., 2000). The appropriate genetic counseling will be provided to subjects and their legal caregivers at a study visit following the receipt of results of genetic testing. Results of genetic screen will not impact continued participation in the study.

After obtaining informed consent (and/or assent when appropriate), demographic data (gender, age, and race) will be collected and subjects will undergo a medical history and physical examination including body weight, height, and vital signs, compilation of concomitant medications, and have blood and urine samples taken for clinical laboratory testing. For subjects who do not have documentation of a JAGGED-1 or NOTCH2 mutation, a blood sample may be obtained for genotyping. The physician will provide an assessment of itch severity using the clinician scratch score during Screening. The eDiary for assessing pruritus with the Itch Reported Outcome (ItchRO) instrument will be dispensed and subjects and caregivers will undergo training during the Screening visit. The patient/ caregiver ItchROs (ItchRO [Pt], ItchRO [Obs]) will be completed twice daily during the Screening period to establish eligibility and a baseline score. Subjects 9 years of age and older will continue independent twice daily completion of their ItchRO. Subjects 5-8 years of age will continue twice daily completion of their ItchRO with the assistance of their caregivers, if needed. Caregivers will continue twice daily completion of their ItchRO. Caregivers (and age appropriate subjects) must complete at least 10 eDiary reports (morning or evening) during each of two consecutive weeks of the screening period, (maximum possible reports = 14 per week). Subjects are required to discontinue bile acid resins for at least 28 days prior to screening and throughout the study. Females who are of childbearing potential will have a serum pregnancy test. Eligibility criteria will be reviewed to confirm a subject's eligibility 4-7 days prior to the Baseline Visit.

<u>Rescreening:</u> If a subject is unable to complete the screening procedures and meet eligibility criteria within the 28-day screening period, consideration may be given to rescreening at a later date. Screening procedures should be repeated at that time. Subject data pertaining to screening will be collected after the subject has been rescreened and determined to meet eligibility.

### 8.1.2 Dose Escalation Treatment Period (Day 0 to Week 6)

At the Baseline Visit (Day 0), subjects will be assessed to confirm continued study eligibility and undergo a physical examination including body weight, height, and vital signs, and have urine and blood samples taken for hematology, chemistry, fasting lipid panel, baseline levels of bile

acids and other cholestasis biochemical markers. Blood will also be collected for determination of baseline fat-soluble vitamins and a plasma LUM001 drug level. Compliance with ItchRO will be assessed. The Clinician Scratch Scale, Xanthoma Scale, and PedsQL questionnaires will be completed. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study medication for Weeks 1, 2, and 3 will be supplied at the Baseline Visit to eligible subjects. Subjects and caregivers will continue twice daily completion of their ItchRO throughout the Dose-Escalation Treatment Period. Subjects will return to the clinic at Weeks 3 and 6 and follow-up phone calls will be made at Weeks 1, 2, 4, and 5. On clinic visit days, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Clinician scratch scale, adherence to study medication, and ItchRO compliance will be assessed. Concomitant medications and any adverse events will be recorded. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Weeks 3 and 6.

# 8.1.3 Stable Dosing Treatment Period (Week 7 to Week 18)

Each subject will continue dosing with study drug during a 12-week Stable Dosing Treatment Period using the dose administered at Week 6, which may be 400 µg/kg/day or the highest tolerated dose below 400 µg/kg/day. Subjects 9 years of age and older will continue independent twice daily completion of their ItchRO. Subjects 5-8 years of age will continue twice daily completion of their ItchRO with the assistance of their caregivers, if needed. Caregivers will continue twice daily completion of their ItchRO. Subjects will receive a follow-up phone call at Week 9 and return to the clinic at Weeks 12 and 18. At the Week 12 and 18 visits, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fasting lipid panel, serum bile acids, fat soluble vitamins, and other cholestasis biochemical markers. Blood sampling for study drug determination may also be performed. After the baseline pharmacokinetic analysis, blood sampling for an additional pharmacokinetic analysis will be done at one additional time point - at Week 12, 18, 38, or 48 – to be selected by the site/investigator (sample to be taken approximately 4 hours post-dosing). Clinician scratch scale, adherence to study medication, ItchRO compliance, and the PedsQL questionnaire will be assessed and concomitant medications and any adverse events will be recorded. In addition, at the Week 18 visit the Clinician Xanthoma Scale, Patient Impression of Change (PIC), Caregiver Impression of Change (CIC), and Caregiver Global Therapeutic Benefit (CGTB) assessments will be completed. At the Week 18, visit subjects will also be randomized 1:1 to either continue to receive study drug or a corresponding placebo between Week 19 and Week 22. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Week 12 and study drug (or placebo) at Week 18.

# 8.1.4 Double-blind, Placebo-controlled Study Withdrawal Period (Week 19 to Week 22)

Age appropriate subjects and caregivers will continue twice daily completion of their ItchRO. Subjects will receive a follow-up phone call at Week 20 and return to the clinic at Week 22. At the Week 22 visit, safety and clinical laboratory evaluations will be performed, and a physical

exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fasting lipid panel, serum bile acids, fat soluble vitamins, and other cholestasis biochemical markers. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Study drug will be supplied at Week 22. Clinician Scratch Scale, adherence to study medication, ItchRO compliance, PIC, CIC, CGTB, and the PedsQL questionnaires will be assessed and concomitant medications and any adverse events will be recorded.

# 8.1.5 Long-term Exposure Period (Week 23 to Week 48)

Following the 4-week double-blind, study drug withdrawal period, subjects who received placebo will once again receive LUM001 according to the schedule where the dose is increased weekly over a 6-week period up to  $400~\mu g/kg/day$  or a maximum daily dose of 20~mg/day. Following the 4-week study drug withdrawal period, subjects who were randomized to receive LUM001 will undergo a simulated dose escalation to maintain the blind in the randomized withdrawal period and continue to receive LUM001 during the long-term exposure period, at the same dose administered at Week 22.

Subjects and caregivers will continue twice daily completion of their ItchRO throughout the long-term exposure period to the Week 48 clinic visit. Subjects will return to the clinic at Weeks 28, 38, and 48. At these visits, safety and clinical laboratory evaluations will be performed, and a physical exam will be performed (including collection of vital signs, height and weight measurements). Blood samples will be taken for fat soluble vitamins, as well as possible pharmacokinetic blood sampling for study drug determination (if not done previously at Week 12 or 18). Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study medication. Clinician scratch scale, adherence to study medication, and ItchRO compliance will be assessed. Subjects/caregivers will receive follow-up phone calls at the end of Weeks 23-27, 33, and 43. Concomitant medications and adverse events will be recorded at all clinic visits and at scheduled telephone contacts.

At the investigator's discretion, withdrawal of concomitant medications used for the treatment of pruritus may occur during the long-term exposure period. Additional study drug will be supplied at each clinic visit during the long-term exposure period.

### 8.1.6 Week 48

At Week 48, a physical exam (including collection of vital signs, height and weight measurements) will be performed. Blood and urine samples will be taken for clinical laboratory testing, including a fasting lipid panel and determination of fat-soluble vitamins, bile acids, other cholestasis biochemical markers, and possibly LUM001 drug level analysis. Females who are of childbearing potential will have a urine pregnancy test. The Clinician Scratch Scale, Clinician Xanthoma Scale, and PedsQL questionnaire will be completed. The PIC, the CIC, and the CGTB assessments will be completed. Concomitant medications and adverse events will be recorded. Study drug compliance will be assessed and all remaining study drug and study supplies will be collected. Study drug will be discontinued and eDiaries will be returned to the site at this visit.

Subjects will then be considered for a 52-week optional follow-up treatment, if eligible, to continue on their highest tolerated dose.

Subjects who withdraw from the study prior to completion of all treatment period clinic visits should undergo the procedures specified for the Week 48/Study Termination visit (Schedule of Procedures, 16.1).

# 8.1.7 Early Termination for Subjects without Participation in the 52-week Optional Follow-up Treatment Period

Any subject who withdraws from the study prior to completion of all treatment period clinic visits should undergo a physical examination, as well as have urine and blood samples taken for safety and clinical laboratory evaluations, lipid panel, bile acids, other cholestasis biochemical markers, fat soluble vitamins, and drug level. In addition the following assessments should be completed: the Clinician Scratch Scale, the Clinician Xanthoma Scale, the PedsQL, the PIC, the CIC, and the CGTB assessments, as defined for ET (see Schedule of Procedures, Section 16.1). For safety reasons, efforts must be made to follow subjects for at least 30 days following their last dose of study drug.

### 8.1.8 52-week Optional Follow-up Treatment Period

Subjects who are eligible to roll over into the 52-week optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level within the 52-week optional follow-up treatment period (Figure 4).

During this period, subjects will return to the clinic at Weeks 60, 72, 84, 96, and 100; telephone contacts will occur at Weeks 64, 68, 76, 80, 88, and 92.

Subjects with  $\geq$ 7 days since last dose of LUM001 will be dose escalated up to 400  $\mu$ g/kg/day or to the highest tolerated dose (see Figure 5). The dose escalation (DE) period will proceed as follows:

- Week DE-2 Clinic Visit: obtain consent, weight, and draw blood for laboratory analyses
- Week DE 0 Clinic Visit: PI evaluates laboratory results, study drug is dispensed, and subject begins at 35 µg/kg/day dose level (if no safety concerns)
- Week DE 49 Telephone Contact: subject escalates to 70 µg/kg/day dose level
- Week DE 50 Telephone Contact: subject escalates to 140 μg/kg/day dose level if prior dose level was tolerated
- Week DE 51 Telephone Contact: subject escalates to 280 μg/kg/day dose level if prior dose level was tolerated
- Week DE 52 Clinic Visit: laboratory tests and dose escalates to  $400 \mu g/kg/day$  dose, if prior dose level was tolerated

If any subject experiences intolerance, the investigator, in consultation with the medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period. At the investigator's discretion, and in consultation with the medical monitor, subjects who were previously down-titrated may be rechallenged during the follow-up treatment period.

### 8.1.9 Long-term Optional Follow-up Treatment Period

Upon completion of the additional 52-week optional follow-up treatment period <u>and/or</u> implementation of this amendment, whichever occurs first, subjects who are eligible to roll over onto the long-term optional follow-up treatment period will continue to receive study drug until the first of the following occurs:

- i. The subjects are eligible to enter another LUM001 study
- ii. LUM001 is available commercially, or
- iii. The sponsor stops the program or development in this indication

Once Protocol Amendment 4 is implemented at the site, a determination about Afternoon Dose Escalation (ADE) will be made.

Refer to Section 5.4 for schematics describing the flow of study visits within this period.

Subjects who are eligible to roll over from the 52-week optional follow up treatment period into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days prior to implementation of Protocol Amendment 4 will be consented and evaluated for eligibility for ADE. Once a determination about ADE has been made, the subject will then either initiate the ADE (see Figure 8) or continue receiving the same dose of LUM001 once a day (Figure 7), depending on whether they meet criteria for initiating ADE.

Screening evaluations for subjects with ≥7 days since last dose of LUM001 prior to implementation of Protocol Amendment 4 will be performed from Day -14 to Day -1. After obtaining informed consent (and/or assent when appropriate), subjects will undergo a physical examination including body weight, height, and vital signs, and have blood and urine samples taken for clinical laboratory testing. Females who are of childbearing potential will have a serum pregnancy test. Eligibility criteria will be confirmed prior to the Baseline Visit. The Clinician Scratch Scale and Clinician Xanthoma Scale will be completed. Concomitant medications and any adverse events will be recorded.

<u>Rescreening:</u> If a subject is unable to complete the screening procedures and meet eligibility criteria within the 14-day screening period, consideration may be given to rescreening at a later date. Screening procedures should be repeated at that time. Subject data pertaining to screening will be collected after the subject has been rescreened and determined to meet eligibility.

Subjects with  $\geq$ 7 days since last dose of LUM001 prior to implementation of Protocol Amendment 4 will be dose escalated up to 400  $\mu$ g/kg/day or to the highest tolerated dose beginning at Dose Level 2 (35  $\mu$ g/kg/day), as outlined in Figure 6.

The dose escalation (DE) period will proceed as follows:

- Protocol Amendment 4 DE Week -2 Clinic Visit: obtain consent, weight, and draw blood for laboratory analyses
- Protocol Amendment 4 DE Day 0 Clinic Visit: investigator evaluates laboratory results, study drug is dispensed, and subject begins at 35 μg/kg/day dose level (if no safety concerns)
- Protocol Amendment 4 DE Week 1 Telephone Contact: subject escalates to 70μg/kg/day dose level if prior dose level was tolerated
- Protocol Amendment 4 DE Week 2 Telephone Contact: subject escalates to 140 μg/kg/day dose level if prior dose level was tolerated
- Protocol Amendment 4 DE Week 3 Telephone Contact: subject escalates to 280 μg/kg/day dose, if prior dose level was tolerated
- Protocol Amendment 4 DE Week 4 Clinic Visit: laboratory tests and dose escalates to 400 µg/kg/day dose (maximum daily dose of 20 mg), if prior dose level was tolerated
- Protocol Amendment 4 DE Week 8 Telephone Contact: eligibility for ADE will be determined

**Subjects not eligible for the ADE (subjects with normal sBA level AND ItchRO[Obs] score** <1.5) will be maintained at the same dose level and will continue morning dosing only. Subjects will have study activities then repeated in repeating 12-week periods as follows, until study completion or termination (see Figure 7).

- Repeating Period Week 4 Telephone Contact (ie, beginning 4 weeks after consent to Protocol Amendment 4): Collection of concomitant medications and any adverse events.
- Repeating Period Week 8 Telephone Contact: Collection of concomitant medications and any adverse events.
- Repeating Period Week 12 Clinic Visit: Physical exam, body weight and height, vital signs, and blood samples for clinical laboratory testing including fasting lipid panel. Blood will also be collected for determination of baseline fat-soluble vitamins. Urine samples for clinical laboratory testing will be collected at every other visit. ItchRO compliance will be assessed, the electronic diary will be issued, the Clinician Scratch Scale and Clinician Xanthoma Scale will be administered, and the PedsQL questionnaire will be administered. Additionally, a palatability questionnaire will be completed. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and adverse events will be collected.
- Subjects who do not qualify for ADE may be assessed at a later time point on a case by case basis following discussions between the investigator and medical monitor. Such re-

evaluations may only occur at the Week 12 visit of any Repeating Period beginning with RP2. If in the course of the ADE re-evaluation, a subject is found to qualify for ADE, then the subject will move into Schedule F or G, as outlined in Section 16.1. During the follow-up treatment period, subjects will return to the clinic every 3 months.

Subjects eligible for ADE, (ie, who have sBA level above normal AND/OR ItchRO [Obs] score ≥1.5), will begin BID dosing (ADE) as follows (see Figure 8):

- On ADE Day 0, morning dosing will continue at 400 µg/kg or the maximum tolerated dose. However, the volume of the morning dose will be reduced by half. Of note: Morning dosing must have been stable for ≥4 weeks prior to initiation of ADE.
- On ADE Day 0, the afternoon dose will be initiated at 140  $\mu$ g/kg/day and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose then will be escalated up to 400  $\mu$ g/kg (ie, up to a maximum 800  $\mu$ g/kg/day or maximum tolerated dose).

The following procedures will occur during the ADE period:

- ADE Day 0 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician Xanthoma Scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed upon completion of other study procedures. Concomitant medications and any adverse events will be collected.
- ADE Week 1 and Week 2 Telephone Contact: Collection of concomitant medications and any adverse events. Subject/caregiver will be reminded of dosing instructions.
- ADE Week 4 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician Xanthoma Scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed upon completion of other study procedures. Concomitant medications and any adverse events will be collected.
- ADE Week 5 and Week 6 Telephone Contact: Collection of concomitant medications and any adverse events. Subject/caregiver will be reminded of dosing instructions.
- ADE Week 8 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The Clinician Scratch Scale, Clinician

Xanthoma Scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed upon completion of other study procedures. Concomitant medications and any adverse events will be collected.

Thereafter, subjects will have study activities repeated in repeating 12-week periods as described above, until study completion or termination (see Figure 8)

If any subject experiences intolerance, the investigator, in consultation with the medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period; later attempts to escalate the dose are permitted. At the investigator's discretion and in consultation with the medical monitor, subjects who were previously down-titrated may be rechallenged during the follow-up treatment period. If the subject is on a twice daily dosing regimen, dose lowering should first be attempted with the afternoon dose.

Safety and clinical laboratory evaluations and a physical exam (including collection of vital signs, height and weight measurements) will be completed at each clinic visit. In addition, the Clinician Scratch Scale, Clinician Xanthoma Scale, and PedsQL will be administered and study drug compliance will be assessed (PedsQL will not be performed at certain clinic visits - please refer to schedule of procedures). The PIC, CIC, and CGTB assessments will be completed at Weeks 84, 96, 100, and the End of Treatment (EOT) / ET visit. Palatability data will be collected at each clinic visit during the long-term optional follow up treatment period (including the EOT/ET visit), with the exception of the PA4 DE, and ADE visits. Plasma samples will be obtained for LUM001 pharmacokinetics at the ADE Day 0, ADE Week 4, and ADE Week 8 visits, and at the 3 scheduled clinic visits following completion of the ADE period. Subjects/caregivers will receive follow-up phone calls at Weeks 64, 68, 76, 80, 88, 92, as well as those outlined within the DE, PA4 DE, and repeating 12-week periods. Concomitant medications and any AEs will be evaluated and recorded at all clinic visits and at scheduled telephone contacts.

Twice daily completion of the electronic diary will be required by caregivers and age appropriate subjects during the 2 weeks following the Week 60, 72, 84, and 96 clinic visits, at PA4 DE Week 4, and at every clinic visit within the repeating 12-week periods. Electronic diaries will be provided to subjects and caregivers at these visits and re-training on the use of the diary will occur, as appropriate.

At the physician investigator's discretion, withdrawal of concomitant medications used for the treatment of pruritus may occur during the long-term exposure period.

With the exception of the EOT/ET visit, additional study drug will be supplied at each clinic visit during the follow-up treatment period. Unused study drug will be collected at every visit.

Subjects will be encouraged to complete all study activities and visits. Any subject who withdraws from the study prior to completion of all treatment period clinic visits should undergo safety and clinical laboratory evaluations, including pharmacokinetic sampling of LUM001, determination of serum bile acids, other cholestasis biochemical markers, fat soluble vitamins,
and AFP. In addition the following assessments should be completed: the Clinician Scratch Scale, Clinician Xanthoma Scale, the PedsQL, the PIC, the CIC, the CGTB, and the palatability questionnaire, as defined for ET (see Schedule of Procedures, Section 16.1). For subjects who complete the study, the assessments performed at the EOT visit will be identical to the assessments performed at the ET visit.

### 8.1.10 End of Treatment or Early Termination

Any subject who completes or withdraws from the study should undergo all procedures specified for the EOT/ET visit (see Schedule J). The following assessments are to be completed at the EOT/ET visit: safety and clinical laboratory evaluations, including determination of serum bile acids, lipid panel, other cholestasis biochemical markers, fat soluble vitamins and AFP. Female subjects who are of childbearing potential will have a urine pregnancy test. Study drug compliance will be assessed. Concomitant medications and adverse events will be collected. In addition, the following assessments should be completed: the Clinician Scratch Scale, Clinician Xanthoma Scale, the PedsQL, the PIC, the CIC, and the CGTB assessments, as defined for the ET visit (see Schedule of Procedures, Section 16.1).

### 8.1.11 Safety Follow-up Period

A safety follow-up phone call will be made 30 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and adverse events noted during this phone call will be recorded.

### 8.2 Genetic Testing

JAGGED1 and NOTCH2 mutations can be predictive of ALGS. For ALGS subjects who meet clinical diagnostic criteria for ALGS (see Section 16.3) but do not have documentation of a JAGGED1 or NOTCH2 mutation, the clinical diagnosis of ALGS may be confirmed by genotyping. Genetic counseling, as appropriate, will be provided to subjects and their legal caregivers. Subjects for whom prior genotyping was performed may need to have an optional repeat analysis performed if the original information collected at screening was insufficient for complete documentation of the diagnosis of ALGS including the type of mutation recorded. For those participants for which the type of the mutation cannot be documented, genetic testing may be conducted and the results recorded.

## 8.3 Physical Examination, Weight and Height, Vital Signs

A physician investigator will conduct a physical examination on each subject at screening and at every study clinic visit. In addition, body weight, height, and vital signs, including body temperature, blood pressure, respiration and pulse, will be determined at every study clinic visit.

#### **8.4** Laboratory Assessments

Laboratory analyte samples will be collected throughout the study. A list of planned tests is compiled in Section 16.2.

The investigator is responsible for reviewing and signing all laboratory reports. The clinical significance of each value outside of the reference range will be assessed and documented as either not clinically significant (NCS) or clinically significant (CS). See Section 11.4.3 regarding laboratory abnormalities.

### 8.5 Pruritus and Quality of Life Assessments

### 8.5.1 Itch Reported Outcome (ItchRO<sup>TM</sup>)

Pruritus will be assessed using the Itch caregiver and patient reported outcome measures (ItchRO) administered as a twice daily electronic diary. Caregivers for all subjects will complete the Observer instrument: ItchRO(Obs)<sup>TM</sup>. Children ≥9 years of age will independently complete the patient instrument: ItchRO(Pt)<sup>TM</sup>. Children between the ages of 5 and 8 years will complete the patient instrument with the assistance of their caregiver: ItchRO(Pt), if needed. Age at screening will be used as the age for the determination of the appropriate ItchRO instrument to be used for the study and this same instrument will be used for the duration of the study (regardless of subsequent birthdays after the screening visit). The primary measure of pruritus will be made using the ItchRO(Obs).

Subjects and caregivers will be trained in the use of the electronic diary during the screening visit. Beginning with the screening period, pruritus will be assessed and recorded twice daily by caregivers and subjects (ItchRO), as described in Section 16.4.

To be eligible for study entry, caregivers must complete at least 10 eDiary reports (morning and/or evening) during each of two consecutive weeks of the screening period and have an average daily score of >2 for 2 consecutive weeks prior to study start. In addition, subjects ≥9 years of age must complete at least 10 eDiary reports (morning and/or evening) during each of two consecutive weeks of the screening period. Subjects are required to discontinue bile acid resins for at least 28 days prior to screening and throughout the study.

ALGS subjects/caregivers will be required to submit twice daily assessments using the electronic diary for the duration of the study. Electronic diaries will be returned to the study site at the Week 48 clinic visit (or sooner if the subject has withdrawn from the study before the Week 48 visit). For subjects who enter the 52-week and long-term optional follow-up treatment periods, completion of the diary will occur as outlined in the Schedule of Procedures in Section 16.1.

Both the morning and evening ItchRO reports have a minimum score of 0 and a maximum score of 4, with 4 representing more severe itching. The highest score between the morning and evening reports will represent the daily score: a measure of the worst itching over the previous 24-hour period. In the event that either the morning or evening report is not completed within the allowed reporting window, whichever report has been completed will represent the daily score. In the event that a subject/caregiver failed to complete both the morning and evening reports, the daily score for that day will be treated as missing data. The handling of missing data on the daily ItchRO score will be outlined in the SAP for the study.

#### 8.5.2 Clinician Scratch Scale

A clinician's assessment of pruritus made by the principal investigator or appropriate designee using the clinician scratch scale (Section 16.5) will be recorded at screening, Day 0 (baseline), Weeks 3, 6, 12, 18, 22, 28, 38, and 48. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the clinician scratch scale will also be administered at clinic visits as outlined in the Schedule of Procedures in Section 16.1.

The clinician's assessment of the subject's pruritus is focused on scratching and visible damage to the skin as a result of scratching as observed by the physician. The clinician scratch scale uses a 5-point scale, in which 0 designates no evidence of scratching and 4 designates cutaneous mutilation with bleeding, hemorrhage and scarring. Whenever possible, the same individual should make the assessments for a subject's visits.

#### 8.5.3 Clinician Xanthoma Scale

A clinician's assessment of xanthomatosis will be made by the principal investigator or appropriate designee using the Clinician Xanthoma Scale (Section 16.6). This assessment will be completed at Baseline (Day 0) and at Weeks 18, and 48. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the Clinician Xanthoma Scale will be recorded as outlined in the Schedule of Procedures in Section 16.1.

The clinician's assessment of the subject's xanthomatosis is focused on the number of lesions present and the degree to which the subject's lesions interfere or limit his or her activities. The clinician xanthoma scale uses a 5-point scale, in which 0 represents no evidence of xanthomatosis, 1 represents fewer than 20 scattered individual lesions, 2 represents more than 20 lesions that do not interfere with or limit activities, 3 represents large numbers of lesions that by their large numbers or size cause distortion of the face or extremities, and 4 represents xanthomas that interfere with function (such as hand use or ability to walk) because of excess size or number (Emerick and Whitington, 2002).

## 8.5.4 Pediatric Quality of Life Inventory (PedsQL)

The PedsQL™ is a questionnaire that will be administered to subjects and/or caregivers at the Week 0 (baseline), 18, 22, and 48. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the PedsQL will be administered as outlined in the Schedule of Procedures in Section 16.1. For subjects with interruptions in LUM001 dosing of ≥7 days, the PedsQL will also be administered at DE Day 0. The PedsQL is a validated, modular instrument designed to measure health-related quality of life (HRQoL) in children and adolescents (Varni et al., 2001). In addition to the core generic PedsQL module, the multidimensional fatigue and family impact questionnaire will also be administered at the Week 0 (baseline), 18, 22, and Week 48 using the age-appropriate module (see Section 16.7). Age at baseline will be used as the age for the determination of the appropriate module to be used for the study and this same module will be used for the duration of the study (regardless of subsequent birthdays after the baseline visit). For subjects who enter the 52-week and long-term optional follow-up treatment periods, the multidimensional fatigue and family impact questionnaire will be administered as outlined in the Schedule of Procedures in Section 16.1.

## 8.5.5 Patient Impression of Change

The PIC is designed to assess the subject's perception of his/her itching after various points of study drug treatment compared to his/her itching prior to the start of treatment with study drug. The PIC will be completed, by subjects who were 9 years of age or older at the Week 18, 22, and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the PIC will be completed by subjects who were 9 years of age or older at clinic visits as outlined in the Schedule of Procedures in Section 16.1.

### 8.5.6 Caregiver Impression of Change

The CIC is designed to assess the caregiver's perception of the subject's itch related symptoms and xanthoma severity after various points of study drug treatment compared to his/her itch related symptoms and xanthoma severity prior to the start of treatment with study drug. The CIC will be completed by all caregivers at the Week 18, 22, and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the CIC will be completed as outlined in the Schedule of Procedures in Section 16.1.

## 8.5.7 Caregiver Global Therapeutic Benefit

The CGTB questionnaire is designed to assess the caregiver's perception of the treatment benefits on the subject's itching compared to the side effects experienced with study drug. The CGTB will be completed by all caregivers at the Week 18, 22, and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the CGTB will be completed as outlined in the Schedule of Procedures in Section 16.1.

### 8.5.8 Palatability

A palatability questionnaire (see Section 16.12) will be completed by the subject and/or caregiver (dependent on age) at clinic visits at time points as outlined in the Schedule of Procedures in Section 16.1.

## 8.6 Restriction on the Lifestyle of Subjects

#### **8.6.1** Contraception Requirements

Sexually active female subjects of childbearing potential must continue to use acceptable contraception with their partners, or refrain from sexual activity, from the time of screening, throughout the study period and for 30 days following the last dose of study drug.

If hormonal contraceptives are used they should be administered according to the package insert.

Females of child-bearing potential who are not currently sexually active must agree to use acceptable contraception, as defined below, if they become sexually active during the period of the study and 30 days following the last dose of the IP.

Acceptable methods of contraception are:

- a. Hormonal contraceptives (eg, oral contraceptive pill, depot, patch, intramuscular implant or injection, or vaginal ring), stabilized for at least 30 days if first use, plus condoms; and/or
- b. Barrier method, eg, (i) condom (male or female) or (ii) diaphragm, with spermicide; or
- c. Intrauterine device (IUD).
- d. or a sexual partner who is surgically sterilized.

## Male Contraception:

Contraception is required for all sexually-active male subjects and their partners. All male subjects agree not to donate sperm, and to use 1 of the following approved methods of contraception until 30 days following study discharge:

- a. Male condom with spermicide
- b. Intrauterine device with spermicide (use by female sexual partner)
- c. Female condom with spermicide (use by female sexual partner)
- d. Contraceptive sponge with spermicide (use by female sexual partner)
- e. Intravaginal system (eg, vaginal ring with spermicide, a diaphragm with spermicide, or a cervical cap with spermicide) (use by female sexual partner)
- f. Oral, implantable, transdermal, or injectable hormonal contraceptive (use by female sexual partner).

## **8.6.2** Fasting Requirements

On study days in which blood samples are collected for the lipid panel and/or cholestasis biomarkers, all subjects will be required to fast for at least 4 hours (only water is permitted) before blood sample collection. On these visit days study drug should be administered as usual (1 mL, 5 mL, or 0.25 qAM, ac), in the morning 30 minutes before breakfast. After breakfast only water should be consumed until the scheduled clinic visit.

#### 9 STUDY DRUG

## 9.1 Study Drug Description

### 9.1.1 LUM001

LUM001 is a powder that is to be dissolved with an appropriate diluent in order to administer the study drug as an oral solution. The compositions of LUM001 study drug 1.0 mL, 0.5 mL, and 0.25 mL oral solutions are described, respectively, in Table 4, Table 5, and Table 6.

Table 4: Composition of LUM001 1.0 mL Oral Solution

| Component | Function | Quantity per 1.0 mL |
|-----------------------|---------------------|---------------------|
| LUM001 | Active Ingredient | up to 50.0 mg |
| Propylene Glycol | Co-solvent | 250.0 mg |
| Sucralose | Sweetener | 7.5 mg |
| Grape Flavoring Agent | Taste Masking Agent | 5.0 mg |
| Water | Vehicle | q.s. to 1.0 mL |

q.s = quantity sufficient

**Table 5:** Composition of LUM001 0.5 mL Oral Solution

| Component | Function | Quantity per 0.5 mL |
|-----------------------|---------------------|---------------------|
| LUM001 | Active Ingredient | up to 25.0 mg |
| Propylene Glycol | Co-solvent | 125.0 mg |
| Sucralose | Sweetener | 3.75 mg |
| Grape Flavoring Agent | Taste Masking Agent | 2.5 mg |
| Water | Vehicle | q.s. to 0.5 mL |

q.s = quantity sufficient

Table 6: Composition of LUM001 0.25 mL Oral Solution

| Component | Function | Quantity per 0.25 mL |
|-----------------------|---------------------|----------------------|
| LUM001 | Active Ingredient | up to 12.5 mg |
| Propylene Glycol | Co-solvent | 62.5 mg |
| Sucralose | Sweetener | 1.875 mg |
| Grape Flavoring Agent | Taste Masking Agent | 1.25 mg |
| Water | Vehicle | q.s. to 0.25 mL |

q.s = quantity sufficient

#### 9.1.2 Placebo

The matching placebo contains the diluent with no active ingredient. The compositions of placebo 1.0 mL, 0.5 mL, and 0.25 mL study drug oral solutions are described, respectively, in Table 7, Table 8, and Table 9.

Table 7: Composition of Placebo 1.0 mL Oral Solution

| Component | Function | Quantity per 1.0 mL |
|-----------------------|---------------------|---------------------|
| Propylene Glycol | Co-solvent | 250 mg |
| Sucralose | Sweetener | 7.5 mg |
| Grape Flavoring Agent | Taste Masking Agent | 5 mg |
| Water | Vehicle | q.s. to 1.0 mL |

q.s = quantity sufficient

**Table 8:** Composition of Placebo 0.5 mL Oral Solution

| Component | Function | Quantity per 0.5 mL |
|-----------------------|---------------------|---------------------|
| Propylene Glycol | Co-solvent | 125 mg |
| Sucralose | Sweetener | 3.75 mg |
| Grape Flavoring Agent | Taste Masking Agent | 2.5 mg |
| Water | Vehicle | q.s. to 0.5 mL |

q.s = quantity sufficient

Table 9: Composition of Placebo 0.25 mL Oral Solution

| Component | Function | Quantity per 0.5 mL |
|-----------------------|---------------------|---------------------|
| Propylene Glycol | Co-solvent | 62.5 mg |
| Sucralose | Sweetener | 1.875 mg |
| Grape Flavoring Agent | Taste Masking Agent | 1.25 mg |
| Water | Vehicle | q.s. to 0.25 mL |

q.s = quantity sufficient

### 9.2 Packaging and Labeling

The sponsor will provide the investigator with packaged study drug labeled in accordance with specific country regulatory requirements. Standard syringes will be provided for oral administration of study drug.

### 9.3 Drug Accountability

Study staff is required to document the receipt, dispensing and return/destruction of study drug supplies provided by the sponsor.

At the conclusion of the study, any unused drugs (including placebo), as well as original containers (even if empty), will be returned to the sponsor or handled according to written instructions from the sponsor, following approval by the sponsor.

#### 10 TREATMENT OF SUBJECTS

## 10.1 Study Drug Administration

The dose of study drug (LUM001 or placebo) in this study is based on weight. The subject's weight determined at the screening visit will be used to calculate the administered dose of study drug for the first 22 weeks of the study. During the study, the study drug may be adjusted if there is a change of  $\geq 10\%$  in weight since the screening visit or if there is a change of  $\geq 10\%$  in weight since the last weight-based medication adjustment to maintain the target dose ( $\mu g/kg/day$ ). The dose may also be down-titrated, at the investigator's discretion and in consultation with the medical monitor, for subjects experiencing intolerance (eg, gastrointestinal symptoms such as diarrhea, abdominal pain, cramping) to a given dose. If the subject is on twice daily dosing regimen, dose reduction should first be attempted with the afternoon dose. Subjects who were previously down-titrated may be rechallenged during the long-term exposure period.

Study drug will be prepared for each subject by a central pharmacy based on the subject's weight at screening. Grape flavored diluent will be added by the central pharmacy pharmacist prior to shipping study drug to the site. Once study drug has been added to the diluent the resulting solution is stable at temperatures ranging from 4-8°C to room temperature for at least 12 months.

Subjects will receive a grape-flavored solution containing LUM001. Each subject dose will be administered orally once a day (QD) or twice a day (BID) using the syringe provided. The first dose should be taken at least 30 minutes prior to the first meal of the day and the second dose, where applicable, should be taken at least 30 minutes prior to dinner (evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the doses should be taken approximately at the same time each day for the duration of the treatment period. See Section 5.5.2 for information regarding dosing during the treatment periods, respectively.

### **QD Dosing Regimen**

For QD dosing, the required dose will be delivered in 0.5 mL volume for subjects who weigh less than 10 kg and in 1.0 mL for subjects who weigh 10 kg or more.

### **BID Dosing Regimen**

For BID dosing, the required dose is delivered in half the dosing volume: 0.25 mL BID for subjects who weigh less than 10 kg and 0.50 mL BID for subjects who weigh 10 kg or more.

For subjects weighing less than 10 kg at study entry, once a weight of 10 kg is reached while in the study, the subject will be moved from 0.5 mL maximum daily dosing volume (0.25 mL BID) to 1.0 mL maximum daily dosing volume (0.50 mL BID).

Please refer to the Study Drug Manual provided by the sponsor for more detailed instructions for study drug preparation, administration and storage.

### **10.2** Treatment Compliance

Compliance with treatment dosing will be monitored and recorded by the study center staff. Subjects and/or caregivers will be asked to complete a paper drug dosing diary indicating when they took their study medication and when they ate breakfast and, for subjects who receive a BID regimen, when they ate dinner (evening meal).

#### 10.3 Concomitant Medications

A concomitant medication is any non-protocol specified drug or substance (including over-the-counter medications, herbal medications and vitamin supplements) administered during participation in the study (the period from the first day of screening through the last contact.

All subjects will have fat soluble vitamin levels monitored; blood samples for fat soluble vitamins should be obtained before the daily dose of vitamins is administered, and approximately 4 hours after any food or formula.

All medications (other than study drug) taken by subjects during the course of the study will be recorded and reviewed by the principal investigator (PI)/investigator's designee. Concomitant medication will be coded using the World Health Organization (WHO) Drug Dictionary (release date 01 Sep 2008, or more recent version if available). AEs related to administration of these medications must also be documented.

Subjects are required to discontinue bile acid resins for at least 28 days prior to screening and for duration of the study. The dosage and dosing regimen of concomitant drug therapy other than that specified by the protocol should not change during the first 22 weeks of study, with the exception of weight-based dose adjustments and vitamin supplementation. No new medications used to treat pruritus may be added during the first 22 weeks of the study. All modifications to a subject's concomitant drug therapy, including weight-based dose adjustments and vitamin supplementation regimen must be carefully documented in the relevant case report forms. If drug therapy other than that specified by the protocol is taken, a joint decision will be made by the investigator or investigator's designee and sponsor to continue or discontinue the subject.

### 10.4 Other Protocol-required Drugs

There are no other protocol required drugs. Subjects are expected to maintain a stable dose and administration schedule for all permitted concomitant medications throughout the course of the study.

## 10.5 Safety Monitoring Rules

### **10.5.1** General Monitoring Rules

In the evaluation of adverse events and the potential relationship to study drug it is important to note that due to their liver disease many patients with ALGS have abnormal liver enzyme levels (eg ALT, ALP) and total bilirubin at baseline. If an individual subject exhibits a CTCAE Grade 3 treatment emergent laboratory abnormality, with the exception of the specific rules outlined

below (Sections 10.5.2), dosing can be suspended or continued as per the investigator's judgment and following discussion with the medical monitor. If suspended the investigator and medical monitor will evaluate the subject's safety data and make a decision to either restart dosing at the same level, restart dosing at a lower dose level, or discontinue dosing.

To ensure subject safety, if 6 or more subjects at a dose level lower, suspend or stop study medication or exhibit treatment emergent toxicity of CTCAE Grade 3 or greater in the same system organ class (SOC), with the exception of the specific rules outlined below, further dosing of subjects at that dose level and any higher dose levels will be halted until a safety assessment is completed. Study visits and completion of the ItchRO diaries, for all randomized subjects, will continue during the assessment period. After review a decision will be made whether to restart dosing at the same dose level, restart dosing at a lower dose level, or discontinue the subjects from the study. The Data Monitoring Committee (DMC) will be notified of any SAE as specified in the DMC charter.

## **10.5.2** Safety Monitoring Rules

The following guidelines are provided for the monitoring of selected parameters chosen based on preclinical and clinical observations.

<u>Confirmation Guidance</u>: At any time during the study, the initial clinical laboratory results exceeding the safety monitoring criteria presented below **must be confirmed** by performing measurements on new specimens. Of note: the INR re-test should be conducted by the central laboratory, but may also be conducted at a local laboratory on an as needed basis. All new specimen collections should take place as soon as possible, ideally within 48 to 72 hours of the notification of the laboratory result. It may be difficult for some subjects who live far from the study site to return to the study site promptly. In this case, the subjects should be retested locally, but normal laboratory ranges should be recorded, results should be made available to study investigators and medical monitors immediately, and the data should be included in the case reports.

Stopping Rule Guidance: Subject dosing must be suspended until the retest results are available. If any of the stopping criteria described below (see Section 10.5.2.2 and Section 10.5.2.5) is confirmed, the physician investigator (PI) in consultation with the medical monitor (or appropriately qualified designee) will permanently discontinue the subject from further treatment with study drug (LUM001 or placebo). The subject will be evaluated as outlined below and will be encouraged to complete the ET study procedures (Week 48 visit). Subjects who do not meet the stopping rules based on retest may continue dosing and the investigator and the medical monitor (or appropriately qualified designee) should confer as to whether additional close monitoring of the subject is appropriate. The investigator should also assess the need to capture an AE, its severity according to the CTCAE directives and potential causality. These assessments should also include an evaluation of whether criteria for an SAE are fulfilled (see Section 11.2.3), in particular whether the event should be considered as an important medical event, ie, an event that would have met one of the other seriousness criteria in the absence of appropriate medical interventions.

### **10.5.2.1** Safety Monitoring for Liver Chemistry Tests

Safety monitoring criteria take into consideration the subject's baseline ALT and total bilirubin levels. The baseline will be defined as the last evaluation before dosing with study drug (Day 0).

If at any time in the study an ALT or total bilirubin result meets the criteria shown in the table below, in relation to the subject's baseline level, the initial measurement(s) should be confirmed within 48 to 72 hours of notification of the laboratory result.

| Baseline ALT | ALT |
|--------------|---------------------------------------|
| ≤ULN | > 5 x ULN |
| > ULN | > 3 x baseline <u>and</u> $>$ 5 x ULN |

| Baseline Total Bilirubin | Total Bilirubin |
|----------------------------|-----------------|
| Total Bilirubin 1-10 mg/dL | 3 mg increase |
| Total Bilirubin >10 mg/dL | 5 mg increase |

<u>Frequency of Repeat Measurements</u>: Subjects with a confirmed ALT or total bilirubin level that is continuing to rise should have their liver chemistry tests (ALT, ALP, INR and total bilirubin) retested as clinically indicated, until levels stabilize or begin to recover.

<u>Further Investigation into Liver Chemistry Elevations</u>: Based on the inclusion criteria for this study the population to be enrolled will have pre-existing baseline liver disease and will be closely monitored by the investigators with experience in the management of pediatric hepatic diseases. For subjects with a confirmed elevation in ALT or total bilirubin level as described above, the following evaluations should be performed as clinically indicated:

- Close and frequent monitoring of liver enzyme and serum bilirubin tests as clinically indicated. Frequency of retesting can decrease if abnormalities stabilize or the study drug has been discontinued and the subject is asymptomatic. If the appropriate frequency of monitoring is not feasible study drug administration will be suspended.
- Obtain a detailed history of symptoms and prior and concurrent diseases.
- Obtain comprehensive history for concomitant drug use (including nonprescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets.
- Obtain a history for exposure to environmental chemical agents and travel.
- Serology for viral hepatitis (HAV IgM, HBsAg, HCV antibody, CMV IgM, and EBV antibody panel).
- Serology for autoimmune hepatitis [eg, antinuclear antibody (ANA)].

Additional liver evaluations, including gastroenterology/hepatology consultations, hepatic CT or MRI scans, may be performed at the discretion of the investigator, in consultation with the medical monitor.

## 10.5.2.2 Stopping Rules for Liver Chemistry Elevations

In the event of confirmed laboratory results exceeding the following criteria, and the event is without an alternative explanation as discussed with the medical monitor, discontinuation of dosing of a subject with study drug (LUM001 or placebo) will be considered if:

| Baseline Tests | Change Observed |
|---|---|
| ALT (any level) | ALT ≥ 20 x ULN |
| Total Bilirubin 1-10 mg/dL | 5 mg increase and a 2 x increase over baseline level |
| Total Bilirubin >10 mg/dL | 2 x increase over baseline level |

## 10.5.2.3 Safety Monitoring for Triglycerides

In the event of a confirmed laboratory result for fasting total triglyceride >500 mg/dL, the investigator and the medical monitor may consider a temporary interruption of study drug. Dosing may resume when the triglyceride level returns to <300 mg/dL or to the subject's baseline level.

### 10.5.2.4 Safety Monitoring for Fat Soluble Vitamins

Vitamin status will be assessed per the schedule of procedures (see Section 16.1), and blood samples will be obtained at the study visits before the daily dose of vitamins is administered. In the event of a confirmed laboratory result that falls either below or above the normal range for a vitamin (25-hydroxy vitamin D, retinol, retinol binding protein, tocopherol  $[\alpha]$ ), or for an elevated INR (as a proxy for vitamin K status), the investigator should make the appropriate modification to the subject's vitamin supplementation regimen.

The response to the change in regimen will be assessed by relevant follow up blood work one month later. Changes will continue to be made until the levels are in the desired range. Adjustments may be discontinued outside of the desired range if there is agreement between the investigator and medical monitor that vitamin sufficiency cannot be reasonably expected.

#### 10.5.2.5 Monitoring/Stopping Rules for Coagulation Panel Results

In the event of a confirmed laboratory result for INR >1.5 that is unresponsive to vitamin K therapy, the investigator and the medical monitor may consider a temporary interruption of study drug. Dosing may resume when the INR falls below 1.5 or returns to the subject's baseline level.

### 10.6 Adjustment of Dose

Gastrointestinal intolerance, as evidenced by diarrhea/loose stools, abdominal pain/cramping and nausea, is expected to be the most frequent manifestation of a lack of tolerability to study drug. If an individual subject exhibits a treatment emergent CTCAE Grade 2 or greater drug-related GI

toxicity, study drug dose may be lowered to a previously well tolerated dose; later attempts to escalate the dose are permitted. If the subject is on a twice daily dosing regimen, dose lowering should first be attempted with the afternoon dose. This decision should be made in consultation with the medical monitor. A requirement for intravenous fluids as treatment for diarrhea will lead to discontinuation of study drug.

## 10.7 Withdrawal of Subjects from the Study

Subjects have the right to withdraw from the study at any time and for any reason without prejudice to his or her future medical care by the physician or the institution. Any subject who withdraws consent to participate in the study will be removed from further treatment and/or study observation immediately upon the date of the request.

Any investigator decision to withdraw a subject from the study must first be discussed with the medical monitor prior to withdrawal. The investigator will provide the reason for withdrawal on the appropriate eCRF.

For any subject who requests to stop study treatment or has withdrawn from study treatment at the request of the legal caregiver, investigator or sponsor before completion of the protocol-specified treatment period, and has received >1 dose of study drug, every effort should be made to complete the assessments scheduled for the ET visit (see Section 16.1), provided the subject has not withdrawn full consent. The ET visit should be scheduled within 7 days of the last study drug dose. The eDiary must also be retrieved.

For safety reasons, efforts must be made to follow subjects for at least 28 days following their last dose of study drug. If a subject withdraws due to an AE, the investigator should arrange for the subject to have follow-up visit(s) until the AE has resolved or stabilized.

Subjects must be withdrawn from the study for any of the following reasons:

- Withdrawal of consent/assent by the subject or legal caregiver.
- Pregnancy.
- An AE (including disease progression) that leads the investigator to decide that the subject should be withdrawn. If a subject suffers an AE that, in the judgment of the investigator or the sponsor, presents an unacceptable consequence or risk to the subject, the subject must be discontinued from the study.
- Significant protocol deviation (eg., medication or treatment that is prohibited by the protocol).
- At the discretion of the investigator if deemed not medically acceptable to continue study treatment.
- Noncompliance, including failure to adhere to the study requirements as stated in the study protocol.
- Administrative decision by the investigator or sponsor.

#### 11 SERIOUS AND NON-SERIOUS ADVERSE EVENT REPORTING

All AEs, whether observed by the investigator, reported by the subject or the subject's caregiver, from laboratory findings, or other means, will be recorded on the AE eCRF and medical record.

Safety information will be collected, reviewed, and evaluated by the sponsor or designee throughout the conduct of the study.

### 11.1 Regulatory Requirements

The sponsor or designee is responsible for regulatory submissions and reporting to the investigators of serious adverse events (SAEs) including suspected unexpected serious adverse reactions (SUSARs) per the International Conference on Harmonisation (ICH) guidelines E2A and ICH E6. Country-specific regulatory requirements will be followed in accordance with local country regulations and guidelines.

The investigator should immediately report all SAEs to the sponsor or designee. It is essential to report SAEs in a timely manner to the sponsor, or designee, along with completed documentation of adverse events to allow the sponsor, or designee, to identify potential study-related, study drug- or dose-related adverse events.

The sponsor is responsible for reporting any suspected adverse reaction that is both serious and unexpected to the applicable regulatory authorities. The sponsor or designee will evaluate the available information and decide if there is a reasonable possibility that the study drug caused the AE and, therefore, meets the definition of a SUSAR.

Additionally, Independent Ethics Committees (IEC)/Institutional Review Boards (IRB) will be notified of any SAE according to applicable regulations. The Data Monitoring Committee (DMC) will be notified of any SAE as specified in the DMC charter.

Appropriate personnel at the sponsor or designee will unblind SUSARs for the purposes of regulatory reporting. The sponsor or designee will submit SUSARs to regulatory agencies in blinded or unblinded fashion according to local law. The sponsor or designee will submit SUSARs to investigators in a blinded fashion.

#### 11.2 Definitions

#### 11.2.1 Adverse Event

An adverse event (AE) is any unfavorable and unintended sign (including a clinically significant abnormal laboratory finding, for example), symptom, or disease temporally associated with the study or use of investigational drug product, whether or not the AE is considered related to the investigational drug product.

An adverse event does not include the following:

• Continuous persistent disease/symptom present before the start of study drug, which does not unexpectedly progress, or change in severity following drug administration.

- Disease being studied and/or signs and symptoms associated with the disease, such as jaundice or itching, or abnormalities in liver enzymes already present during the screening period or at the baseline visit.
- Treatment failure or lack of efficacy.

## 11.2.2 Adverse Reaction and Suspected Adverse Reaction

An <u>adverse reaction</u> is any adverse event caused by the study drug.

A <u>suspected adverse reaction</u> is any adverse event for which there is a reasonable possibility that the drug caused the adverse event. A suspected adverse reaction implies a lesser degree of certainty about causality than an adverse reaction.

## 11.2.3 Serious Adverse Event (SAE)

A serious adverse event is any adverse event that in the view of either the investigator or sponsor, meets any of the following criteria:

- Results in death.
- Is life-threatening: that is, poses an immediate risk of death at the time of the event.
- An AE or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the subject at immediate risk of death. It does not include an AE or suspected adverse reaction that, had it occurred in a more severe form, might have caused death.
- Requires inpatient hospitalization or prolongation of existing hospitalization.
- Hospitalization is defined as an admission of greater than 24 hours to a medical facility and
  does not always qualify as an AE. Hospitalization for elective treatment or a pre-existing
  condition that did not worsen during the clinical investigation is not considered an AE.
  Hospitalization or nursing home admission for the purpose of caregiver respite is not
  considered an AE.
- Complications that occur during hospitalization are AEs, and if a complication prolongs hospitalization, the event is considered serious. Treatment in a hospital emergency room is not a hospitalization. Admission to the hospital is the criterion that defines "serious," not the duration of hospital stay.
- Results in a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions.
- Results in congenital anomaly or birth defect in the offspring of the subject (whether the subject is male or female).
- Important medical events that may not result in death, are not life-threatening, or do not require hospitalization may also be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at

home, blood dyscrasias or convulsions that do not result in inpatient hospitalization, or the development of drug dependency or drug abuse.

### 11.3 Monitoring and Recording Adverse Events

Any pre-existing conditions or signs and/or symptoms present in a subject prior to the start of the study (ie, before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. In addition, AEs that occur while the subject is not enrolled in the study during a gap period will be collected as medical history unless the AE started within 30 days of last dose. Symptoms of the disease under study should not be classed as AEs as long as they are within the normal day-to-day fluctuation or expected progression of the disease and are part of the efficacy data to be collected in the study; however, significant worsening of the symptoms should be recorded as an AE. The investigator should always group signs and symptoms into a single term that constitutes a single unifying diagnosis if possible.

Subjects should be questioned in a general way, without asking about the occurrence of any specific symptom. Following questioning and evaluation, all AEs, whether believed by the investigator to be related or unrelated to the study drug, must be documented in the subject's medical records, in accordance with the investigator's normal clinical practice, and on the AE eCRF. Each AE is to be evaluated for seriousness, causal relationship to the study drug, intensity, action taken, any treatment given, outcome, and duration. It should be noted that the term "severe" used to grade intensity is not synonymous with the term "serious."

#### 11.3.1 Serious Adverse Events

In the interest of subject safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to study drug) should be reported to the sponsor or designee within 24 hours of the study center's first knowledge of the event. The collection of SAEs will begin after the subject signs the informed consent/assent form and stop 30 days after the last dose of study drug.

When the investigator is reporting by telephone, it is important to speak to someone in person versus leaving a message. An initial report of the SAE should be completed and a copy should be transmitted to the sponsor or designee.

Detailed information should be actively sought and provided to the sponsor or designee as soon as additional information becomes available. All SAEs will be followed until resolution. SAEs that remain ongoing past the subject's last protocol-specified follow-up visit will be evaluated by the investigator and sponsor. If the investigator and sponsor agree the subject's condition is unlikely to resolve, the investigator and sponsor will determine the follow-up requirement.

#### 11.3.2 Non-serious Adverse Events

The recording of non-serious AEs will begin after the subject signs the informed consent/assent form and will stop 30 days after the last dose of study drug. The investigator will monitor each subject closely and record all observed or volunteered AEs on the Adverse Event Case Report Form.

#### 11.3.3 Evaluation of Adverse Events (Serious and Non-Serious)

The following should be documented on the Adverse Event Case Report Form.

### 11.3.3.1 Relationship to the Study Drug

The investigator will document his/her opinion of the relationship of the AE to treatment with study drug using the following criteria:

Related: There is clear evidence that the event is related to the use of study drug (eg, confirmation by positive rechallenge test).

Possible: The event cannot be explained by the subject's medical condition, concomitant therapy, or other causes, and there is a plausible temporal relationship between the event and study drug administration.

Unlikely/Remote: An event for which an alternative explanation is more likely (eg, concomitant medications or ongoing medical conditions) or the temporal relationship to study drug administration and/or exposure suggests that a causal relationship is unlikely (for reporting purposes, Unlikely/Remote will be grouped together with Not Related).

Not Related: The event can be readily explained by the subject's underlying medical condition, concomitant therapy, or other causes, and therefore, the investigator believes no relationship exists between the event and study drug.

### **11.3.3.2** Severity

The Common Terminology Criteria for Adverse Events (CTCAE) grade of the event should be reported according to CTCAE Version 4.0 (Section 16.11). If the CTCAE does not have a grading for a particular adverse event, the severity of the event should be reported based on the following:

- Mild (Grade 1): The event is easily tolerated by the subject and does not affect the subject's usual daily activities.
- Moderate (Grade 2): The event causes the subject more discomfort and interrupts the subject's usual daily activities.
- Severe (Grade 3): The event is incapacitating and causes considerable interference with the subject's usual daily activities.

Specific definitions will be provided for designated GI events expected to occur in this study, in order to aid investigators with determination of event severity.

Please also refer to Section 10.5.2 regarding specific safety monitoring for liver chemistry tests given that subjects with ALGS may have abnormal liver enzymes at baseline.

If the event is an SAE, then all applicable <u>seriousness criteria</u> must be indicated (criteria listed in Section 11.2.3).

### 11.3.3.3 Action Taken with Study Drug

Action taken with study drug due to the event is characterized by one of the following:

- None: No changes were made to study drug administration and dose.
- Permanently Discontinued: Study drug was discontinued and not restarted.
- Temporarily Interrupted, restarted same dose: Dosing was temporarily interrupted or delayed due to the AE and restarted at the same dose.
- Reduced dose: Dosing was reduced, temporarily interrupted or delayed due to the AE and restarted at the next lower dose.

#### 11.3.3.4 Treatment Given for Adverse Event

Any treatment (eg medications or procedures) given for the AE should be recorded on the AE eCRF (treatment should also be recorded on the concomitant treatment or ancillary procedures CRF as appropriate).

#### 11.3.3.5 Outcome of the Adverse Event

If the event is a non-serious AE then the event's outcome is characterized by one of the following:

- AE Persists: Subject terminates from the study and the AE continues.
- Recovered: Subject recovered completely from the AE.
- Became Serious: The event became serious (the date that the event became serious should be recorded as the Resolution Date of that AE and the Onset Date of the corresponding SAE).
- Change in Severity (if applicable): AE severity changed.

If the event is an SAE then the event's outcome is characterized by one of the following:

- Ongoing: SAE continuing.
- Persists (as non-serious AE): Subject has not fully recovered but the event no longer meets serious criteria and should be captured as an AE on the non-serious AE eCRF (the SAE resolution date should be entered as the date of onset of that AE).
- Recovered: Subject recovered completely from the SAE (the date of recovery should be entered as the SAE resolution date).
- Fatal: Subject died (the date of death should be entered as the SAE resolution date).

## 11.4 Procedures for Handling Special Situations

The following categories of medical events that could occur during participation in a clinical study must be reported within 24 hours.

• Serious adverse event (SAE; see Section 11.3.1)

- Pregnancy
- Dosing errors
- Treatment unblinding for any reason (see Section 6.4)

## 11.4.1 Pregnancy Reporting

If a subject becomes pregnant or a pregnancy is suspected during the study, the study center staff must be informed immediately. The sponsor or designee should be notified within 24 hours of first learning of the occurrence of pregnancy. Follow-up information including delivery or termination should be reported within 24 hours.

If pregnancy is suspected during the study (including follow-up), a pregnancy test will be performed. A subject with a confirmed pregnancy will be immediately withdrawn from treatment with study drug. However, the subject will be encouraged to complete the ET procedures to the extent that study procedures do not interfere with the pregnancy. Regardless of continued study participation, the study physician will assist the subject in getting obstetrical care and the progress of the pregnancy will be followed until the outcome of the pregnancy is known (ie, delivery, elective termination, or spontaneous abortion). If the pregnancy results in the birth of a child, the study center and sponsor may require access to the mother and infant's medical records for additional follow-up after birth.

Payment for all aspects of obstetrical care, child or related care will be the subject's responsibility.

## 11.4.2 Dosing Errors

Study drug dosing errors should be documented as protocol deviations. A brief description should be provided in the deviation, including whether the subject was symptomatic (list symptoms) or asymptomatic, and if the event was accidental or intentional.

Dosing details should be captured on the appropriate eCRF. If the subject takes a dose of study drug that exceeds protocol specifications and the subject is symptomatic, then the symptom(s) should be documented as an AE and be reported per Section 11.3.

Should an overdose occur, the investigator or designee should refer to the Guidance to investigator's section of the investigator's brochure and contact the sponsor or designee within 24 hours.

### 11.4.3 Abnormalities of Laboratory Tests

Clinically significant abnormal laboratory test results may, in the opinion of the investigator, constitute or be associated with an AE. Examples of these include abnormal laboratory results that are associated with symptoms, or require treatment (eg, bleeding due to thrombocytopenia, tetany due to hypocalcemia, or cardiac arrhythmias due to hyperkalemia). Whenever possible, the underlying diagnosis should be listed in preference to abnormal laboratory values as AEs. Clinically significant abnormalities will be monitored by the investigator until the parameter returns to its baseline value or until agreement is reached between the investigator and medical

monitor. Laboratory abnormalities deemed not clinically significant (NCS) by the investigator should not be reported as AEs. Similarly, laboratory abnormalities reported as AEs by the investigator should not be deemed NCS on the laboratory sheet.

The investigator is responsible for reviewing and signing all laboratory reports. The signed clinical laboratory reports will serve as source documents.

#### 12 STATISTICAL CONSIDERATIONS

This section presents a summary of the planned statistical analyses. A statistical analysis plan (SAP) will be written for the study that contains detailed descriptions of the analyses to be performed. The SAP will be finalized prior to unblinding of the data.

Continuous variables will be summarized using descriptive statistics including n, mean, median, standard deviation, range (eg, minimum and maximum). Qualitative variables will be summarized using counts and percentages. Summaries will be provided overall, as well as by phase, dose level, and treatment group as appropriate. Unless otherwise specified, statistical analyses will be performed using SAS Version 9 or higher. Where appropriate, statistical tests will be conducted at the 0.05 significance level using two-tailed tests and p-values will be reported if applicable. Given the rare nature of ALGS, the statistical power of any comparisons is limited. As such the analysis will be largely descriptive in nature.

## 12.1 Sample Size Considerations

Alagille syndrome is a rare disease. The planned sample size of 30 evaluable ALGS subjects is based on practical considerations, rather than a desired power for a pre-specified difference.

### 12.2 Populations

## **12.2.1** Safety Population

The Safety Population is defined as all subjects who were enrolled and received at least one dose of the study drug. The Safety Population will be used for all safety analyses. Subjects will be analyzed by the treatment they received.

### 12.2.2 Efficacy Populations

The main population for efficacy will be the modified intention-to-treat population (MITT), defined as all subjects who were enrolled, received study medication through Week 18, and had a reduction from baseline in serum bile acids of ≥50% at the Week 12 or Week 18 measurement. Subjects will be analyzed by assigned treatment.

The intention-to-treat (ITT) Population includes all subjects who were enrolled and received at least one dose of the study medication. Subjects will be analyzed by assigned treatment.

Membership in the analysis populations will be determined before study unblinding.

## 12.2.3 Siblings

The enrollment of siblings is allowed. During the double-blind, placebo-controlled, randomized drug withdrawal period, siblings will be assigned in a blinded manner to the same treatment arm. The data from all enrolled participants (including siblings) will be used for the safety analysis. For the efficacy analysis, data from only one of the siblings will be used. The choice of which subject's data to use in the efficacy analysis will be done in a random fashion before the LUM001-304 study is unblinded. Details of the analysis methods will be outlined in the SAP.

### 12.2.4 Demographic and Baseline Characteristics

## 12.2.4.1 Subject Disposition

Subject disposition will be summarized descriptively. The number and percentage of subjects enrolled, completed, and withdrawing, along with reasons for withdrawal, will be tabulated overall, and by study phase and treatment group. For purposes of analysis, there will be 3 study phases: Dose escalation/stable dose (Weeks 0-18), Randomized Withdrawal (Weeks 19-22) and Long-Term Exposure (Weeks 23-48 and 23-100).

The number of subjects in each analysis population will be reported. Line listings will be prepared for all subjects not following the planned dosing schedule, showing all doses and dose changes occurring.

Other disposition and study conduct information, including major protocol violations will be listed. Duration of the follow-up period will be summarized.

#### 12.2.4.2 Baseline Data

The following baseline data will be used to describe the study population:

- Demographic variables, including age, gender and race/ethnicity.
- Medical history.
- Baseline disease characteristics (eg, genotyping results, pruritus scores, liver biochemistries).
- Prior medications of interest (eg, ursodiol [UDCA], rifampicin) and concomitant medications.

Demographic and baseline characteristics will be summarized descriptively overall, by dose group (as appropriate), responder group and treatment group.

Treatment group comparisons will be made using analysis of variance for continuous measures and the chi-square test for categorical measures. Adjustment for responder stratification will be made as appropriate. These analyses will be conducted on the Safety Population.

Medical history information will be presented in listings.

### 12.2.5 Efficacy Analyses

The primary analysis population for the efficacy analysis will be the MITT population defined in Section 12.2.2. Analyses for the primary and secondary efficacy outcome variables will also be done on the ITT population. No adjustment for multiplicity will be made. All data will be included in data listings.

#### 12.2.5.1 Efficacy Variables

The primary efficacy endpoint will be the mean change from Week 18 to 22 of fasting serum bile acid levels in subjects who previously responded to LUM001 treatment, as defined by a reduction in sBA  $\geq$ 50% from baseline to Week 12 or Week 18. A sensitivity analysis will also be

conducted using subjects who experienced a reduction from baseline in serum bile acids of ≥50% at the Week 48 measurement.

Secondary efficacy endpoints include mean change from Week 18 to Week 22 in liver enzymes (ALP, ALT, and bilirubin [total and direct]) and pruritus as measured by ItchRO (Observer ItchRO/patient ItchRO), in subjects who previously responded to LUM001 treatment, as defined by a reduction in ItchRO scale >1 point from baseline to Week 12 or Week 18. Secondary efficacy endpoints also include mean change from baseline to Week 18 in fasting serum bile acid levels, liver enzymes (ALP, ALT, and bilirubin [total and direct]) and pruritus as measured by ItchRO (Observer ItchRO/Patient ItchRO).

The assessment of pruritus in this study will be the ItchRO assessment from the eDiary. Given the age range of this population and the small sample size, the ItchRO score will be derived from the ItchRO(Obs) instrument. The itch score from the ItchRO(Pt) will be analyzed separately. Subjects 9 years of age or older will complete the ItchRO(Pt) independently. Subjects between the ages of 5 and 8 years of age or where the investigator has expressed concern about the subject's ability to reliably complete the data (eg, due to developmental delay) will complete the ItchRO(Pt) with the help of the caregiver. There will be no ItchRO(Pt) report for subjects under the age of 5.

For this instrument the caregiver and/or subject will indicate the itch severity in the morning and in the evening each day for the duration of the study (baseline to Week 48). The daily score will be assessed as outlined in Section 16.4 and will have a range from 0-4, with the higher score indicating increasing itch severity. A daily score is defined as the higher of the scores from the morning and evening ItchRO, representing the most severe itch over the 24 hour period. For the change from baseline calculation in average daily ItchRO score, baseline is defined as the average daily ItchRO score in the week consisting of the 7 days immediately prior to Day 0. The average daily score will be the average of the daily scores over a defined study week consisting of the 7 days prior to the visit.

In addition, an analysis for a daily score defined as an average of morning and evening scores will be conducted.

If a caregiver is not compliant with the ItchRO(Obs) during the week prior to a study visit, the average daily score from the most recent, previous compliant week will be used in a Last Observation Carried Forward format. On study compliance for the ItchRO(Obs) will be defined as having at least 4 of the 7 daily ItchRO(Obs) scores for a 7-day period. Similar methods will be used for the ItchRO(Pt). Missing data imputation will not be done for other efficacy endpoints.

The additional questions included in the ItchRO(Obs/Pt) that are not scored, will be tabulated overall and by treatment group.

The following additional efficacy evaluations will be assessed:

- Change from baseline to Weeks 18, 22, 48 and then every 12 weeks in:
  - o Fasting serum bile acid levels

- o Liver enzymes (ALT, ALP) and bilirubin (total and direct)
- o Pruritus as measured by the average daily ItchRO (Observer ItchRO/patient ItchRO)
- Other biochemical markers of cholestasis [total cholesterol, low-density lipoprotein cholesterol (LDL-C)]
- O Bile acid synthesis [serum  $7\alpha$ -hydroxy-4-cholesten-3-one ( $7\alpha$ C4)]
- Responder analysis at Weeks 18, 48, 60, 72, 84, 96, and 100 in:
  - o Pruritus response rates as measured by ItchRO (Observer ItchRO/patient ItchRO)
  - Clinician scratch scale
- Change from baseline for PedsQL at Week 18, 22, 48, 60, 72, 84, 96, and 100 and change from Week 18 to Week 22
- PIC at Week 18, 22, 48, 84, 96, and 100 and change from Week 18 to Week 22
- CIC at Week 18, 22, 48, 84, 96, and 100 and change from Week 18 to Week 22
- CGTB assessment at Weeks 18, 22, 48, 84, 96, and 100 and change from Week 18 to Week 22
- Change from Baseline (Day 0) to Week 48 in xanthomas, as measured by Clinician Xanthoma Scale

Additional assessments of efficacy variables will occur during the 52-week and long-term optional treatment periods in 12-week intervals. Any of the above evaluations may also occur at clinic visits during the DE, PA4 DE, and ADE periods. Additional exploration of evaluations will be specified in the statistical analysis plan.

A number of sensitivity analyses will be performed to assess the robustness of the results as well as consider the time course of the efficacy assessments. Details of these analyses will be outlined in the SAP for the study.

### 12.2.5.2 Primary Efficacy Analysis

The change from baseline in serum bile acid will be displayed for each treatment group during the randomized withdrawal phase using summary statistics including the number of observations, the mean, median, standard deviation, minimum and maximum. Differences from baseline will be calculated and summarized as above, with a 95% confidence interval for the mean.

The difference between treatment groups in change from Week 18 to Week 22 in serum bile acid will be evaluated using an ANCOVA model with treatment group as a factor, and Week 18 serum bile acid as a covariate. Treatment group differences within responder groups as well as the potential interaction between responder group and treatment group will also be examined where possible.

## 12.2.5.3 Secondary, Exploratory and Other Efficacy Analyses

Secondary and exploratory efficacy variables that are continuous measures will be analyzed similarly to the primary efficacy analyses. Where sample size allows, treatment effects over time will be examined using methods appropriate for repeated observations.

Exploratory efficacy measures that are categorical will be analyzed using the chi-square test or Fisher's Exact test as appropriate based on sample sizes. Additionally, the Cochran-Mantel-Haenszel test will be used to adjust for response group. Exploratory efficacy measures will be summarized by frequencies and percents, overall, and by phase and treatment group. This includes the responder definition for pruritus, which will be outlined in the SAP. P-values from the secondary and exploratory efficacy analyses will be considered nominal.

The sensitivity of the results for pruritus to missing data assumptions will be explored as outlined in the SAP for the study. The sensitivity analyses may include analyses using observed cases as well as various assumptions for missing data from subjects who terminate from the study early.

Additional exploratory analyses may be performed and will be defined and outlined in the SAP for the study.

### 12.2.6 Safety Analyses

Safety analyses will be performed on the Safety Population.

### 12.2.6.1 Safety Assessments

The following assessments will be used to monitor safety:

- Adverse events (AEs) and SAEs
- Clinical laboratory results
- Vital signs
- Physical exam findings, including body weight and height
- Concomitant medication usage
- Serum alpha-fetoprotein (AFP)

### 12.2.7 Planned Method of Analysis

Safety data, including AEs, clinical laboratory tests, vital signs, physical examinations, and concomitant medication usage will be summarized descriptively overall, by phase (Section 12.2.4.1) and by treatment group for the Safety Population. Summaries may also be provided by dose group if appropriate. Individual subject listings will be prepared for all safety data.

### 12.2.8 Safety Analysis

Safety data, including AEs, clinical laboratory tests, vital signs, physical examinations, and concomitant medication usage will be summarized descriptively for the Safety population. Individual subject listings will be prepared for all safety data.

## 12.2.8.1 Adverse Events

Frequencies (number and percentage) of subjects with one or more treatment emergent AEs will be summarized by dose group and/or treatment group, by system organ class and preferred term

according to the Medical Dictionary for Regulatory Activities (MedDRA<sup>TM</sup>) terminology. All treatment emergent AEs, all treatment emergent AEs potentially related to study drug, all treatment emergent SAEs and all treatment emergent SAEs potentially related to study drug will be summarized. Specific AEs of special interest, particularly GI related AEs, will be outlined in the SAP and summarized. AEs will be summarized over the entire study and then separately for the dose escalation/stable dose periods (weeks 0-18), randomized withdrawal, and long-term exposure periods of the study.

The incidence of AEs, and their severity, as well as the incidence of subjects who withdraw due to an AE will be tabulated. A subject listing of all treatment emergent AEs, and AEs causing study discontinuation will be presented.

### 12.2.8.2 Laboratory Tests

Clinical laboratory (chemistry panel, complete blood count (CBC) with differential, coagulation, lipid panel, cholestasis biomarkers, fat soluble vitamins, and urinalysis parameters) test parameters will be listed for individual subjects and summarized using descriptive statistics by study visit and treatment group. Change from baseline for the safety variables will also be presented over time after study drug administration, as appropriate. Percent change from baseline will be added for laboratory values as outlined in the SAP. Baseline for clinical laboratory parameters will be defined as the last evaluation before dosing with study drug (Day 0).

A separate listing will present laboratory values of all subjects who change from normal to abnormal or from abnormal to normal during the course of the study, where normal ranges for this population are outlined in the SAP. Changes within a treatment group for selected safety measures will be assessed at Weeks 3, 6, 12, 18, 22, 28, 38, 48, 60, 72, 84, 96 and at additional time points during the 52-week and long-term optional treatment periods and final study evaluation visit using methods to be specified in the SAP prior to unblinding the data.

The effect of LUM001 on fat soluble vitamin levels will be assessed. These laboratory values will be summarized as above and listed for individual subjects. A separate listing presenting laboratory values of all subjects who change from sufficient to insufficient or from insufficient to sufficient during the course of the study will be created.

### 12.2.8.3 Physical Exams, Vital Signs and Weight/Height Measurements

Changes in physical exam findings after baseline will be listed for individual subjects.

Vital signs, weight and height (both weight and height are to be measured as an absolute number and as a z-score for age and gender) will be listed for individual subjects and summarized using descriptive statistics by study visit and treatment group. Changes from baseline for all visits after the baseline visit will be included in the summary table. Baseline for vital signs will be defined as the last evaluation before dosing with study drug. In general this will be the Day 0 visit.

### 12.2.8.4 Concomitant Medications

Concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary and summarized descriptively by Anatomical Therapeutic Chemical (ATC) class,

using counts and percentages. Medications started prior to the first dose of study medication will be indicated in the data listing. A separate listing for medications taken for pruritus will be given that clearly indicates the phase of the study.

### 12.2.8.5 Study Drug Exposure

Due to poor absorption of LUM001 very low systemic exposure and plasma drug levels are expected. The key measurement will be the pharmacodynamic effect on serum bile acid levels. However, exposure to study drug will be measured approximately 4 hours post dose at baseline and one other visit during the study as determined by the investigator. Data will be summarized and listed across the treatment period. Average daily dose, total drug exposure, and total subject days of exposure to study medication will be summarized descriptively overall and by phase and treatment group.

### 12.2.8.6 Serum Alpha-fetoprotein

Assessments of serum AFP will be listed for individual subjects and summarized using descriptive statistics by study visit.

## 12.2.9 Palatability Analyses

Palatability data will be collected at each clinic visit in the follow up treatment period, with the exception of the DE, PA4 DE, and ADE visits. A palatability questionnaire will be completed by the subject and/or caregiver (dependent on age). Data will be listed for individual subjects and summarized using descriptive statistics by study visit. Assessment of change over time will be evaluated. Baseline will be defined as the first recorded evaluation.

### 12.2.10 Interim Analyses

There will be an interim analysis (IA) conducted after all subjects complete or discontinue the study after Week 48 to guide the future of the program. At the IA the study will be unblinded.

### 12.2.11 Additional Analyses

Additional analyses may be performed to explore both safety and efficacy measures collected in this study. The precise methods and analyses will be determined after the database is locked and the blind is broken. Thus all such analyses will be interpreted cautiously and not used for formal inference, although inferential statistics may be used as part of the data summary.

#### 13 INVESTIGATOR'S REGULATORY OBLIGATIONS

#### 13.1 Informed Consent

The written informed consent/assent documents should be prepared in the languages of the potential patient population, based on an English template version provided by the sponsor or designee.

The investigator is responsible for obtaining written informed consent/assent from the subject and/or their legally acceptable representative(s). Before any screening tests or assessments are performed, an adequate explanation of the aims, methods, anticipated benefits, and potential hazards of the study will be provided to the subject and/or legally acceptable representative. The subject and/or legally acceptable representative must be given sufficient time to consider whether to participate in the study and be assured that withdrawal from the study may be requested at any time without jeopardizing medical care related to or required as a result of study participation.

Subjects and/or their legally acceptable representative(s) will be required to read, sign, and date an IEC approved informed consent/assent form (ICF/IAF) summarizing the discussion at screening. Since this is a pediatric study, in addition to the written informed consent, the assent of the child must also be obtained. The person who conducted the informed consent discussion (not necessarily an investigator) should also sign and date the ICF/IAF. The original signed ICF/IAF should be retained in accordance with institutional policy. Subjects and/or their legally acceptable representative(s) will be given a copy of their ICF/ IAF.

The subject's and/or legal representative's agreement and the acquisition of informed consent should be documented in the subject's medical record. When the study is completed and the CRF has been monitored, the ICF/IAF will be kept in the investigator's central study file. Regulatory authorities may check the existence of the signed ICF/IAF in this central study folder if not done so during the performance of the study.

Over the course of the study, the ICF/IAF may be modified, as appropriate (eg, due to a protocol amendment or significant new safety information). The resulting IEC-approved ICF/IAF will be used for all subjects subsequently entering the study or those already enrolled and still actively participating in the study.

## 13.2 Study Personnel

Prior to the start of this study, the investigator must supply the sponsor or designee with a list of the names of the site's investigator(s) for the study and other possible participants, their professional background (eg, investigator, coordinator, technician) and their role in the study. The investigator should ensure that all appropriately qualified persons to whom he/she has delegated study duties are recorded on a sponsor-approved Delegation of Site Responsibilities Form.

### 13.3 Ethical Conduct of the Study

The Guidelines of the World Medical Association (WMA) Declaration of Helsinki dated October 2008, the applicable regulations and guidelines of current Good Clinical Practice (GCP) as well as the demands of national drug and data protection laws and other applicable regulatory requirements will be strictly followed.

## 13.4 Independent Ethics Committee/Institutional Review Board

A copy of the protocol, proposed informed consent/assent forms, other written subject information, and any proposed advertising material must be submitted to the IEC/IRB for written approval. A copy of the written approval of the protocol and informed consent/assent forms must be received by the sponsor or designee before recruitment of subjects into the study and shipment of study drug. A copy of the written approval of any other items/materials that must be approved by the study center or IEC/IRB must also be received by the sponsor or designee before recruitment of subjects into the study and shipment of study drug. The investigator's Brochure must be submitted to the IEC/IRB for acknowledgement.

The investigator must submit and, where necessary, obtain approval from the IEC/IRB for all subsequent protocol amendments and changes to the informed consent/assent documents. The investigator should notify the IEC/IRB of deviations from the protocol in accordance with ICH GCP Section 4.5.2. The investigator should also notify the IEC/IRB of serious adverse events occurring at the study center and other adverse event reports received from the sponsor or designee, in accordance with local procedures.

The investigator will be responsible for obtaining annual IEC/IRB approval/renewal throughout the duration of the study. Copies of the investigator's reports, all IEC/IRB submissions and the IEC/IRB continuance of approval must be sent to the sponsor or designee.

### 13.5 Confidentiality

The investigator must ensure that the subject's confidentiality is maintained. On the case report forms or other documents submitted to the sponsor or designee, subjects should be identified by unique initials and a subject study number only. Documents that are not for submission to the sponsor or designee (eg, signed informed consent/assent forms) should be kept in strict confidence by the investigator.

In compliance with federal and local regulations/ICH GCP Guidelines, it is required that the investigator and institution permit authorized representatives of the sponsor, regulatory agency(ies), and the IEC/IRB direct access to review subjects' original medical records for verification of study-related procedures and data. Direct access includes examining, analyzing, verifying, and reproducing any records and reports that are important to the evaluation of the study. The investigator is obligated to inform and obtain the consent of the subject and/or their legally acceptable representative to permit named representatives to have access to his/her study-related records without violating the confidentiality of the subject.

All information concerning this study and which was not previously published is considered confidential information. This confidential information shall remain the sole property of Mirum Pharmaceuticals, Inc.; it shall not be disclosed to others without written consent of Mirum Pharmaceuticals, Inc.; and shall not be used except in the performance of this study.

The information compiled during the conduct of this clinical study is also considered confidential and may be disclosed and/or used only by Mirum Pharmaceuticals, Inc., as they deem necessary. To allow the use of the information derived from this clinical study and to ensure compliance to current federal regulations, the investigator is obliged to furnish Mirum Pharmaceuticals, Inc., with the complete test results and all data compiled in this study.

#### 14 ADMINISTRATIVE AND LEGAL OBLIGATIONS

## 14.1 Pre-study Documentation Required

The investigator must provide the sponsor or designee with the following documents (copies should be kept by the investigator in the site's regulatory document binder):

- Signed and dated Protocol Signature Page.
- Completed and signed statement of investigator (Form FDA 1572/financial disclosure form) (where applicable).
- Curriculum vitae (CV) of the investigator and sub-investigators (where applicable, all persons listed on Form FDA 1572).
- Letter of approval from the IEC/IRB for both protocol and consent/assent forms.
- Copy of the IEC/IRB-approved written informed consent/assent forms, and any other written information and/or advertisement to be used.
- IEC/IRB membership list or compliance certification letter.
- Name and location of the laboratory utilized for laboratory assays, and other facilities conducting tests, including a copy of the laboratory certificate (where applicable).
- In case a laboratory certification is not available, a written statement as to how the laboratory complies with quality assurance should be provided. The sponsor's monitor must be notified if the laboratory is changed.
- List of normal laboratory values (where applicable).

In addition, in advance of enrollment of subjects, study staff are required to complete all required training.

### 14.2 Protocol Amendments

Protocol amendments must be made only with the prior approval of the sponsor or designee. Agreement from the investigator must be obtained for all protocol amendments and amendments to the informed consent/assent documents. The regulatory authority and IEC/IRB must be informed of all amendments and give approval for any amendments likely to affect the safety of the subjects or the conduct of the study. The investigator must send a copy of the approval letter from the IEC/IRB to the sponsor or designee. Amendments to the protocol will not be implemented until written IEC/IRB approval has been received.

### 14.3 Study Termination

Both the sponsor or designee and the investigator reserve the right to terminate the study at the investigator's site, according to the terms of the study contract. The investigator/sponsor or designee should notify the IEC/IRB in writing of the study's completion or ET and send a copy of the notification to the sponsor or designee.

The sponsor or designee reserves the right to terminate the study overall.

## 14.4 Study Documentation and Storage

Source documents are original documents, data, and records from which the subject's case report form data are obtained. These include but are not limited to hospital records, clinical and office charts, laboratory and pharmacy records, diaries, imaging, and correspondence. All original source documents supporting entries in the case report forms must be maintained and be readily available.

The investigator and the study center staff are responsible for maintaining a comprehensive and centralized filing system of all study-related (essential) documentation in accordance with Section 8 of the ICH Guidelines (E6), suitable for inspection at any time by representatives from the sponsor or designee and/or applicable regulatory authorities. The clinical site's regulatory document binder essential elements should include:

- Subject files containing completed case report forms (eCRFs), informed consents/assents, and supporting copies of source documentation.
- Study files containing the protocol with all amendments, investigator's brochure, copies of
  pre-study documentation and all correspondence to and from the IEC/IRB and the sponsor or
  designee.
- If drug supplies are maintained at the study center, documentation for proof of receipt, study drug accountability records, return of study drug for destruction, final study drug product reconciliation statement, and all drug-related correspondence.

No study document should be destroyed without prior written agreement between the sponsor or designee and the investigator. Should the investigator wish to assign the study records to another party or move them to another location, he/she must notify the sponsor or designee.

### 14.5 Study Monitoring

The sponsor representative and regulatory authority inspectors are responsible for contacting and visiting the investigator for the purpose of inspecting the facilities and, upon request, inspecting the various records of the study (eg, case report forms and other pertinent data) provided that subject confidentiality is respected. Quality control audits may be performed at the sponsor's discretion.

Throughout the course of the study, a study monitor will make frequent contacts with the investigator and/or study staff. This will include telephone calls and on-site visits. During the on-site visits, the CRFs will be reviewed for completeness and adherence to the protocol, accuracy, consistency of the data, and adherence to local regulations on the conduct of clinical research. The monitor will need access to subject medical records and other study-related records needed to verify the entries on the case report forms. The study monitor will also perform drug accountability checks and review the clinical site's regulatory document binder to assure completeness of documentation in all respects of clinical study conduct. On completion of the

study, the study monitor will arrange for a final review of the study files after which the files should be secured for the appropriate time period.

The investigator or appointed delegate will receive the study monitor during these on-site visits and will cooperate in providing the documents for inspection and respond to inquiries. In addition, the investigator will permit inspection of the study files by authorized representatives of the regulatory agencies.

### 14.6 Language

Case report forms must be completed in English. Generic names for concomitant medications should be recorded in English if possible, unless it is a combination drug, then record the trade name in English.

All written information and other material to be used by subjects and investigative staff must use vocabulary and language that are clearly understood.

### 14.7 Compensation for Injury

The sponsor maintains appropriate insurance coverage for clinical studies and will follow applicable local compensation laws. Subjects will be treated and/or compensated for any study-related illness/injury in accordance with the information provided in the Informed Consent document.

### 15 REFERENCES

- Emerick, K. M., Rand, E. B., Goldmuntz, E., Krantz, I. D., Spinner, N. B. & Piccoli, D. A. 1999. Features of Alagille syndrome in 92 patients: frequency and relation to prognosis. *Hepatology*, 29, 822-9.
- Emerick, K. M. & Whitington, P. F. 2002. Partial external biliary diversion for intractable pruritus and xanthomas in Alagille syndrome. *Hepatology*, 35, 1501-6.
- Hofmann, A. F. 2003. Inappropriate ileal conservation of bile acids in cholestatic liver disease: homeostasis gone awry. *Gut*, 52, 1239-41.
- Hounnou, G., Destrieux, C., Desme, J., Bertrand, P. & Velut, S. 2002. Anatomical study of the length of the human intestine. *Surg Radiol Anat*, 24, 290-4.
- Modi, B. P., Suh, M. Y., Jonas, M. M., Lillehei, C. & Kim, H. B. 2007. Ileal exclusion for refractory symptomatic cholestasis in Alagille syndrome. *J Pediatr Surg*, 42, 800-5.
- Neimark, E., Chen, F., Li, X. & Shneider, B. L. 2004. Bile acid-induced negative feedback regulation of the human ileal bile acid transporter. *Hepatology*, 40, 149-56.
- Spinner, N., Hutchinson, A., Krantz, I. & Kamath, B. 2000. *Alagille Syndrome* [Online]. Seattle, WA. Available: http://www.ncbi.nlm.nih.gov/pubmed/20301450 2000].
- Van Den Anker, J., Schwab, M. & Kearns, G. 2011. Developmental Pharmacokinetics. *In:* Seyberth, H., Rane, A. & Schwab, M. (eds.) *Pediatric Clinical Pharmacology*
- Varni, J. W., Seid, M. & Kurtin, P. S. 2001. PedsQL 4.0: reliability and validity of the Pediatric Quality of Life Inventory version 4.0 generic core scales in healthy and patient populations. *Medical care*, 39, 800-12.
- Walthall, K., Cappon, G. D., Hurtt, M. E. & Zoetis, T. 2005. Postnatal development of the gastrointestinal system: a species comparison. *Birth Defects Res B Dev Reprod Toxicol*, 74, 132-56.
- Weaver, L. T., Austin, S. & Cole, T. J. 1991. Small intestinal length: a factor essential for gut adaptation. *Gut*, 32, 1321-3.
- Whitington, P. F. & Whitington, G. L. 1988. Partial external diversion of bile for the treatment of intractable pruritus associated with intrahepatic cholestasis. *Gastroenterology*, 95, 130-6.

# 16 APPENDICES

## 16.1 Schedule of Procedures

## **Overall Scheme and Corresponding Schedule of Procedures**

The following schematic shows the study flow and corresponding Schedule of Procedures (A - I).

Study Termination and End of Treatment Procedures are outlined in Schedule J.



<sup>\*</sup> If eligible for ADE at or after RP2 W12, in consultation with Medical Monitor
# 16.1.1 Schedule of Procedures A-D: Study Entry – Week 96

Schedule of Procedures A – Screening – Week 22

| Schedule of Procedures <u>A</u> – So | 3 | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | Screening | Baseline | | | Dose Es | calation <sup>i</sup> | i | | s | Stable Dos | se | | omized<br>Irawal |
| Study Week | | | 1 | 2 | 3 | 4 | 5 | 6 | 9 | 12 | 18 | 20 | 22 |
| Study Day | Day -28 to -1 | Day 0 | 7 | 14 | 21 | 28 | 35 | 42 | 63 | 84 | 126 | 140 | 154 |
| Window (in days) | | | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±5) | (±5) | (±5) | (±5) | (±5) |
| Informed Consent | X | | | | | | | | | | | | |
| Eligibility Assessment/<br>Medical History | X | X | | | | | | | | | | | |
| Demographics | X | | | | | | | | | | | | |
| Physical Exam | X | X | | | X | | | X | | X | X | | X |
| Body Weight & Height | X | X | | | X | | | X | | X | X | | X |
| Randomization to Placebo vs.<br>LUM001 | | | | | | | | | | | X | | |
| Vital Signs <sup>a</sup> | X | X | | | X | | | X | | X | X | | X |
| CBC with Differential <sup>b</sup> | X | X | | | X | | | X | | X | X | | X |
| Coagulation <sup>b</sup> | X | X | | | X | | | X | | X | X | | X |
| Chemistry Panel <sup>b</sup> | X | X | | | X | | | X | | X | X | | X |
| Lipid Panel <sup>b,c</sup> | | X | | | | | | | | X | X | | X |
| Cholestasis Biomarkers <sup>b,c</sup> | | X | | | | | | | | X | X | | X |
| Total Serum bile acids <sup>c</sup> | X <sup>k</sup> | X | | | | | | | | X | X | | X |
| Fat Soluble Vitamins <sup>b,c</sup> | | X | | | | | | | | X | X | | X |
| JAGGED1/NOTCH2 Genotyping <sup>d</sup> (if needed) | X | | | | | | | | | | | | |
| Plasma Sample for LUM001 | | $X^{j}$ | | | | | | | | $X^{j}$ | $X^{j}$ | | |
| Urinalysis <sup>b</sup> | X | Xg | | | Xg | | | Xg | | X | X | | X |
| Serum or Urine Pregnancy Test<br>(if indicated) <sup>e</sup> | X | X | | | X | | | X | | X | X | | Х |
| Subject eDiary/Caregiver eDiary (ItchRO) | X <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> | Xh | Xh | Xh | X <sup>h</sup> | Xh | X <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> |
| Clinician Scratch Scale | X | X | | | X | | | X | | X | X | | X |
| Clinician Xanthoma Scale | | X | | | | | | | | | X | | |
| PedsQL | | X | | | | | | | | | X | | X |
| Patient/Caregiver Impression of Change | | | | | | | | | | | X | | X |

Schedule of Procedures A – Screening – Week 22

| Schedule of Flocedules A – St | , | | | Treatment Period | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | Screening | Baseline | | | Dose Es | calationi | i | | S | table Dos | se | Rando<br>Withd | mized<br>Irawal |
| Study Week | | | 1 | 2 | 3 | 4 | 5 | 6 | 9 | 12 | 18 | 20 | 22 |
| Study Day | Day -28 to -1 | Day 0 | 7 | 14 | 21 | 28 | 35 | 42 | 63 | 84 | 126 | 140 | 154 |
| Window (in days) | | | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±5) | (±5) | (±5) | (±5) | (±5) |
| Caregiver Global Therapeutic Benefit | | | | | | | | | | | X | | X |
| Enrollment | | X | | | | | | | | | | | |
| Study Drug Supplied | | X | | | X | | | X | | X | X | | X |
| Review Study Diaries & Assess<br>Compliance | | X | | | X | | | X | | X | X | | X |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Phone Contact <sup>f</sup> | | | X | X | | X | X | | X | | | X | |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes. Blood samples for analysis of fat soluble vitamins should be drawn prior to administration of vitamin supplementation.
- Subjects are required to fast at least 4 hrs (only water permitted prior to collection).
- d Optional genotype sample will be performed to provide a full characterization and the associated documentation of the mutation in support of the diagnosis of ALGS.
- <sup>e</sup> For females of childbearing potential, result must be reviewed prior to dispensing study drug.
- Subjects must be available to receive a phone call from study staff.
- At the indicated visits during the treatment period, oxalate will be part of the urinalysis.
- b During screening and throughout the study, the eDiary (ItchRO) will be completed twice daily (AM & PM). Compliance will be assessed at each visit/phone contact.
- Subjects should be dosed for at least 7 days at each dose level.
- Pharmacokinetic analysis will be done at Baseline, and then approximately 4 hours post-dosing at one additional time point at Week 12, 18, 38, or 48 (to be selected by site/investigator).

| k | Sub | jects are NOT required to fast prior to sample collection at the screening visit |
|---|---|---|
| | | Clinic Visit |
| | | Phone Contact |

Schedule of Procedures **B** – Long-term Exposure: Week 23–Week 48

| | | | | Treatme | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | | | | Long- | Term Ex | posure | | | | | Follow Up |
| Study Week | 23 | 24 | 25 | 26 | 27 | 28 | 33 | 38 | 43 | Week 48<br>(or Early<br>Termination <sup>f</sup> ) | |
| Study Day | 161 | 168 | 175 | 182 | 189 | 196 | 231 | 266 | 301 | 336 | 30 days after final dose |
| Window (in days) | (±2) | (±2) | (±2) | (±2) | (±2) | (±5) | (±5) | (±5) | (±5) | (±14) | (±5) |
| Physical Exam | | | | | | X | | X | | X | |
| Body Weight & Height | | | | | | X | | X | | X | |
| Vital Signs <sup>a</sup> | | | | | | X | | X | | X | |
| CBC with Differential <sup>b</sup> | | | | | | X | | X | | X | |
| Coagulation <sup>b</sup> | | | | | | X | | X | | X | |
| Chemistry Panel <sup>b</sup> | | | | | | X | | X | | X | |
| Lipid Panel <sup>b,c</sup> | | | | | | | | | | X | |
| Total Serum bile acids <sup>c</sup> | | | | | | | | | | X | |
| Cholestasis Biomarkers <sup>b,c</sup> | | | | | | | | | | X | |
| Fat Soluble Vitamins <sup>b,c</sup> | | | | | | X | | X | | X | |
| Plasma Sample for LUM001 | | | | | | | | $X^{i}$ | | $X^{i}$ | |
| Urinalysis <sup>b</sup> | | | | | | X | | X | | Xg | |
| Urine Pregnancy Test (if indicated) <sup>d</sup> | | | | | | X | | X | | X | |
| Clinician Scratch Scale | | | | | | X | | X | | X | |
| Clinician Xanthoma Scale | | | | | | | | | | X | |
| Subject eDiary/Caregiver eDiary (ItchRO) | $X^h$ | $X^h$ | $X^h$ | $X^h$ | $X^h$ | $X^h$ | $X^h$ | $X^h$ | $X^h$ | X <sup>h</sup> | |
| PedsQL | | | | | | | | | | X | |
| Patient & Caregiver Impression of Change | | | | | | | | | | X | |
| Caregiver Global Therapeutic Benefit | | | | | | | | | | X | |
| Study Drug Supplied | | | | | | X | | X | | $\mathbf{X}^{\mathrm{j}}$ | |
| Review Study Diaries & Assess Compliance | | | | | | X | | X | | X | |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X |
| Phone Contact <sup>e</sup> | X | X | X | X | X | | X | | X | | X |

Phone Contact

Schedule of Procedures **B** – Long-term Exposure: Week 23–Week 48

| | | Treatment Period (cont'd) | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | | Long-Term Exposure | | | | | | | | | Follow Up |
| | | | | | | | | | | Week 48 | |
| | | | | | | | | | | (or Early | |
| Study Week | 23 | 24 | 25 | 26 | 27 | 28 | 33 | 38 | 43 | Termination <sup>f</sup> ) | |
| | | | | | | | | | | | 30 days after |
| Study Day | 161 | 168 | 175 | 182 | 189 | 196 | 231 | 266 | 301 | 336 | final dose |
| Window (in days) | (±2) | (±2) | (±2) | (±2) | (±2) | (±5) | (±5) | (±5) | (±5) | (±14) | (±5) |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- See Section 16.2 for detailed list of laboratory analytes. Blood samples for analysis of fat soluble vitamins should be drawn prior to administration of vitamin supplementation.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted prior to collection).
- For females of childbearing potential, result must be reviewed prior to dispensing study drug.
- e Subjects must be available to receive a phone call from study staff.
- Subjects who withdraw early should complete all evaluations at this visit.
- At the indicated visits during the treatment period, oxalate will be part of the urinalysis.
- b During screening and throughout the study, the eDiary (ItchRO) will be completed twice daily (AM and PM). Compliance will be assessed at each visit/phone contact.
- Pharmacokinetic analysis will be done at Baseline, and then approximately 4 hours post-dosing at one additional time point at Week 12, 18, 38, or 48 (to be selected by site/investigator).

| j | For subjects entering optional Follow-up Treatment Period, once corresponding consent is signed. |
|---|---|
| | Clinic Visit |

Schedule of Procedures <u>C</u> – 52-week Optional Follow-up Treatment Period (FTP): Week 48-96 for Those Subjects <7 Days from the Last Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen.

| from the Last Dose of LUMI001 | . Includ | ies evaiu | auon or e | engivini | y lur bi | D dosing | g regime | <del>.</del> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | | 52-week FTP | | | | | | | | | | |
| Study Week | 52 | 56 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| Study Day | 364 | 392 | 420 | 448 | 476 | 504 | 532 | 560 | 588 | 616 | 644 | 672 |
| Window (in days) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) |
| Informed Consent/Assent for PA4g | | | X | | | X | | | X | | | X |
| Afternoon Dose Escalation (ADE) eligibility assessment followed by shift in visit schedule <sup>h</sup> | X <sup>h</sup> | X <sup>h</sup> | $X^{h}$ | X <sup>h</sup> | X <sup>h</sup> | $X^h$ | X <sup>h</sup> | $X^h$ | $X^h$ | X <sup>h</sup> | $X^h$ | $X^h$ |
| Physical Exam | | | X | | | X | | | X | | | X |
| Body Weight & Height | | | X | | | X | | | X | | | X |
| Vital Signs <sup>a</sup> | | | X | | | X | | | X | | | X |
| CBC with Differential <sup>b</sup> | | | X | | | X | | | X | | | X |
| Coagulation <sup>b</sup> | | | X | | | X | | | X | | | X |
| Chemistry Panel <sup>b</sup> | | | X | | | X | | | X | | | X |
| Lipid Panel <sup>b,c</sup> | | | X | | | X | | | X | | | X |
| Cholestasis Biomarkers <sup>b,c</sup> | | | X | | | X | | | X | | | X |
| Fat Soluble Vitamins <sup>b,c</sup> | | | X | | | X | | | X | | | X |
| Optional Genotyping <sup>d</sup> | | | X | | | | | | | | | |
| Urinalysis <sup>b</sup> | | | X | | | X | | | X | | | X |
| Urine Pregnancy Test (if indicated) <sup>e</sup> | | | X | | | X | | | X | | | X |
| Clinician Scratch Scale | | | X | | | X | | | X | | | X |
| Clinician Xanthoma Scale | | | X | | | X | | | X | | | X |
| Subject eDiary/Caregiver eDiary (ItchRO) | | | Xi | X <sup>i</sup> to<br>Week<br>62 | | Xi | X <sup>i</sup> to<br>Week<br>74 | | Xi | Xi to<br>Week<br>86 | | Xi |
| PedsQL | | | X | | | X | | | X | | | X |
| Patient & Caregiver Impression of Change | | | | | | | | | X | | | X |
| Caregiver Global Therapeutic Benefit | | | | | | | | | X | | | X |
| Study Drug Supplied | | | X | | | X | | | X | | | X |
| Review Study Diaries & Assess<br>Compliance | | | X | | | X | | | X | | | X |

Schedule of Procedures <u>C</u> – 52-week Optional Follow-up Treatment Period (FTP): Week 48-96 for Those Subjects <7 Days from the Last Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen.

| II OIII THE LAST DOSE OF LONIOUT | · Includ | ics crain | ation of C | ingibilit | y ioi Di | i dosing | , regime | U11• | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | | 52-week FTP | | | | | | | | | | |
| Study Week | 52 | 56 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| Study Day | 364 | 392 | 420 | 448 | 476 | 504 | 532 | 560 | 588 | 616 | 644 | 672 |
| Window (in days) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) |
| Concomitant Medications | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X |
| Phone contact <sup>f</sup> | X | X | | X | X | | X | X | | X | X | |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes. Blood samples for analysis of fat soluble vitamins should be drawn prior to administration of vitamin supplementation.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted prior to collection).
- d Genotyping sample will be drawn at Week 60 or at the time of re-consent for the optional follow-up treatment period; sample will be used to provide a full characterization and documentation of the mutation type in support of the diagnosis of ALGS.
- For females of childbearing potential, result must be reviewed prior to dispensing study drug.
- Subjects must be available to receive a phone call from study staff.
- Once necessary approvals are received for Protocol Amendment 4 and associated consent/assent documents are available, site will consent/assent patient for Protocol Amendment 4 at the next clinic visit.
- Once the Protocol Amendment 4 consent/assent has been signed, site will assess subject eligibility for Protocol Amendment 4 and ADE. Depending on the outcome of ADE eligibility assessment, subject will move into either Schedule of Procedures E or F. Of note: It is possible that subject will not necessarily complete up through Week 96 before they move to Schedule of Procedures E or F. ADE eligibility assessments may occur any time between Week 52 and Week 100.

| aily completion of the study |
|------------------------------|

| Clinic Visit |
|---------------|
| Phone Contact |

Schedule of Procedures  $\underline{D}$  – 52-week Optional Follow-up Treatment Period: DE -2 – Week 96 for Those Subjects  $\geq$ 7 Days from the Last Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen.

| from the Last L | Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen. Treatment Period (cont'd) | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | FT | | | | FTP | | | | | | | | | |
| Study Period | | Dos | se Escal | ation (D | E) | | | | | FII | | | | | | |
| FTP Study Week DE Study Day | <b>DE</b> - 2 | <b>DE 0</b> | DE<br>49<br>343 a | DE<br>50<br>350 a | DE<br>51<br>357 a | DE<br>52<br>364 a | 60<br>420 a | <b>64</b><br>448 <sup>a</sup> | 68<br>476 a | 72<br>504 <sup>a</sup> | 76<br>532 a | <b>80</b> 560 a | <b>84</b> 588 a | 88<br>616 a | 92<br>644 a | <b>96</b> 672 a |
| Window<br>(in days) | (±14) | (±2) | (±2) | (±2) | (±2) | (±2) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) |
| Informed<br>Consent/Assent for<br>study re-entry under<br>PA3 | X | | | | | | | | | | | | | | | |
| Eligibility Assessment for study re-entry | X | | | | | | | | | | | | | | | |
| Informed<br>Consent/Assent for<br>PA4 <sup>h</sup> | | | | | | | X | | | X | | | X | | | X |
| Afternoon Dose<br>Escalation (ADE)<br>eligibility<br>assessment followed<br>by shift in visit<br>schedule <sup>i</sup> | | | | | | | Xi | Xi | Xi | X <sup>i</sup> | Xi | Xi | Xi | Xi | Xi | Xi |
| Physical Exam | X | X | | | | X | X | | | X | | | X | | | X |
| Body Weight &<br>Height | X | X | | | | X | X | | | X | | | X | | | X |
| Vital Signs <sup>b</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| CBC with<br>Differential <sup>c</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Coagulation <sup>c</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Chemistry Panel <sup>c</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Lipid Panel <sup>c,d</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Cholestasis<br>Biomarkers <sup>c,d</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Fat Soluble<br>Vitamins <sup>c,d</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Optional<br>Genotyping <sup>e</sup> | X | | | | | | | | | | | | | | | |
| Urinalysis <sup>c</sup> | X | X | | | | X | X | | | X | | | X | | | X |
| Urine Pregnancy<br>Test <sup>f</sup> | X | X | | | | X | X | | | X | | | X | | | X |

Schedule of Procedures <u>D</u> – 52-week Optional Follow-up Treatment Period: DE -2 – Week 96 for Those Subjects ≥7 Days from the Last Dasa of LUM001. Includes evaluation of eligibility for BID design regimen

| from the Last D | Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen. Treatment Period (cont'd) | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | - | | | | | Trea | tment Per | riod (cont'd) | | | | | | |
| Study Period | | Dos | FT<br>se Escal | | E) | | | FTP | | | | | | | | |
| FTP Study Week | DE - | DE 0 | DE<br>49 | DE<br>50 | DE 51 | DE 52 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| DE Study Day<br>Window<br>(in days) | -14<br>(±14) | (±2) | 343 a (±2) | 350 a (±2) | 357 a (±2) | 364 a (±2) | 420 a (±14) | 448 <sup>a</sup> (±7) | 476 a (±7) | 504 a (±14) | 532 a (±7) | 560 a (±7) | 588 a (±14) | 616 <sup>a</sup> (±7) | 644 a (±7) | 672 a (±14) |
| Clinician Scratch<br>Scale | X | X | | | | X | X | | | X | | | X | | | X |
| Clinician Xanthoma<br>Scale | | X | | | | X | X | | | X | | | X | | | X |
| Subject<br>eDiary/Caregiver<br>eDiary | | | | | | | $\mathbf{X}^{\mathrm{j}}$ | x <sup>j</sup><br>to Week<br>62 | | X <sup>j</sup> | X <sup>j</sup><br>to Week<br>74 | | Xª | X <sup>j</sup><br>to<br>Week<br>86 | | Xª |
| PedsQL | | X | | | | | X | | | X | | | X | | | X |
| Patient & Caregiver<br>Impression of<br>Change | | | | | | | | | | | | | X | | | X |
| Caregiver Global<br>Therapeutic Benefit | | | | | | | | | | | | | X | | | X |
| Study Drug<br>Supplied | | X | | | | X | X | | | X | | | X | | | |
| Review Study<br>Diaries & Assess<br>Compliance | | | | | | X | X | | | X | | | X | | | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Phone Contact <sup>g</sup> | | | X | X | X | | 1 1 6 | X | X | | X | X | | X | X | |

<sup>&</sup>lt;sup>a</sup> Calculation of Study Day includes subject's participation through the first 48 weeks.

b Blood pressure (BP), heart rate (HR), temperature, respiration rate.

See Section 16.2 for detailed list of laboratory analytes. Blood samples for analysis of fat soluble vitamins should be drawn prior to administration of vitamin d supplementation.

d Subjects are required to fast at least 4 hrs (only water permitted prior to collection).

Optional genotype sample will be performed to provide a full characterization and the associated documentation of the mutation type in support of the diagnosis of ALGS. Females of childbearing potential, result must be reviewed prior to dispensing study drug.

For females of childbearing potential, result must be reviewed prior to dispensing study drug.

Subjects must be available to receive a phone call from study staff.

Once necessary approvals are received for Protocol Amendment 4 and associated consent/assent documents are available, site will consent/assent subject for Protocol Amendment 4 at the next clinic visit.

Schedule of Procedures  $\underline{D}$  – 52-week Optional Follow-up Treatment Period: DE -2 – Week 96 for Those Subjects  $\geq$ 7 Days from the Last Dose of LUM001. Includes evaluation of eligibility for BID dosing regimen.

| II om the Last L | JUSC UI | se of Bowloot. Includes evaluation of engionity for BID dosing regimen. | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | Trea | atment Pe | riod (cont'd) | | | | | | |
| Study Period | | FTP Dose Escalation (DE) FTP | | | | | | | | | | | | | | |
| Study 1 criou | | | l Betti | | | | | | | | | | | | | |
| | DE - | | DE | DE | DE | DE | | | | | | | | | | |
| FTP Study Week | 2 | DE 0 | 49 | 50 | 51 | 52 | 60 | 64 | 68 | 72 | 76 | 80 | 84 | 88 | 92 | 96 |
| DE Study Day | -14 | 0 | 343 a | 350 a | 357 a | 364 a | 420 a 448 a 476 a 504 a 532 a 560 a 588 a 616 a 644 a 672 a | | | | | | | 672 a | | |
| Window | | | | | | | | | | | | | | | | |
| (in days) | (±14) | (±2) | (±2) | (±2) | (±2) | (±2) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) | (±7) | (±7) | (±14) |

Once the Protocol Amendment 4 consent/assent has been signed, site will assess subject eligibility for Protocol Amendment 4 and ADE. Depending on the outcome of ADE eligibility assessment, subject will move into either Schedule of Procedures E or F. Of note: It is possible that subject will not necessarily complete up through Week 96 before they move to Schedule of Procedures E or F. ADE eligibility assessments may occur any time between Week 60 and Week 100.

During the Follow-up Treatment Period, daily completion of the study diary for 2 consecutive weeks following Week 68, Week 96, and Week 120 visits.



## 16.1.2 Schedule of Procedures E-F: Rollover under Protocol Amendment 4

Schedule of Procedures  $\underline{E}$  – Extension of Long-term Optional Follow-up Treatment Period, for subjects <u>ineligible</u> for ADE, applicable as follows:

- Subject did not yet complete the long-term optional follow up treatment period as outlined under Protocol Amendment 3 and is able to consent to Protocol Amendment 4 activities without an interruption in LUM001 dosing, OR
- Subject completed long-term optional follow up treatment period as outlined under PA3 and dosing interruption was <7 days.
- Subject deemed ineligible for ADE.

| | Below study activities | repeat in repeating | 12-week periods <sup>h</sup> |
|---|---|---|---|
| Repeating Period Week (RPx) | RPx Week 4 | RPx Week 8 | RPx Week 12 |
| Scheduling Considerations | 4 weeks after consent<br>under PA4 | | |
| Window (in days) | (±7) | (±7) | (±14) |
| Physical Exam | | | X |
| Body Weight & Height | | | X |
| Vital Signs <sup>a</sup> | | | X |
| CBC with Differential <sup>b</sup> | | | X |
| Coagulation <sup>b</sup> | | | X |
| Chemistry Panel <sup>b</sup> | | | X |
| Lipid Panel <sup>b,c</sup> | | | X |
| Cholestasis Biomarkers <sup>b,c</sup> | | | X |
| Fat Soluble Vitamins <sup>b,c,d</sup> | | | X |
| Urinalysis <sup>b</sup> | | | $\mathbf{X}^{\mathrm{j}}$ |
| AFP Sample | | | Xi |
| Serum or Urine Pregnancy Test (if indicated) <sup>e</sup> | | | X |
| Clinician Scratch Scale | | | X |
| Clinician Xanthoma Scale | | | X |
| Caregiver ItchRO/ | | | X |
| Patient ItchRO | | | (collected for 2 |
| | | | week period |
| | | | following this |
| | | | visit) |

| | Below study activitie | s repeat in repeating | 12-week periodsh |
|---|---|---|---|
| Repeating Period Week (RPx) | RPx Week 4 | RPx Week 8 | RPx Week 12 |
| Scheduling Considerations | 4 weeks after consent<br>under PA4 | | |
| Window (in days) | (±7) | (±7) | (±14) |
| PedsQL | | | X |
| Palatability Questionnaire | | | X |
| Study Drug Supplied <sup>f</sup> | | | X |
| Assess Compliance | | | X |
| Concomitant Medications | X | X | X |
| Adverse Events | X | X | X |
| Follow-up Phone Contactg | X | X | |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- d Blood samples must be drawn before administration of vitamin supplementation.
- <sup>e</sup> Females of childbearing potential, result must be reviewed prior to dispensing study drug.
- f Study drug may be dispensed at unscheduled clinic visits.
- g Subjects must be available to receive a phone call from study staff.
- Study visits will continue in the same pattern until the first of the following occur: (i) subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.
- Sample will be drawn at every other clinic visit starting with RP1 Week 12.
- At indicated visits during treatment period, oxalate will be part of the urinalysis.



Schedule of Procedures  $\underline{F}$  – Extension of Long-term Optional Follow-up Treatment Period, for subjects <u>eligible</u> for ADE, applicable as follows:

- Subject did not yet complete the long-term optional follow up treatment period as outlined under Protocol Amendment 3 (PA3) and is able to consent to Protocol Amendment 4 activities without an interruption in LUM001 dosing OR
- Subject completed the long-term optional follow up treatment period as outlined under PA3 and dosing interruption was <7 days.
- Subject deemed eligible for ADE.

| Study Period | | | Afternoo | v-up Treatm<br>on Dose Esca | Study activities repeat in repeating 12-week periods after completion of the ADE period <sup>h</sup> | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | ADE<br>Day 0 | ADE<br>Week 1 | ADE<br>Week 2 | ADE<br>Week 4 | ADE<br>Week 5 | ADE<br>Week 6 | ADE<br>Week 8 | Week 4 | Week 8 | Week 12 |
| Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | Week I | Week 2 | WCCR 4 | WEEK 3 | WEER | Week o | The initial Week 4 contact will be scheduled 4 weeks following ADE Week 8. | Week o | Week 12 |
| Window (in days) | N/A – see<br>above | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±7) | (±7) | (±14) |
| Physical Exam | X | () | () | X | () | () | X | () | () | X |
| Body Weight &<br>Height | X | | | X | | | X | | | X |
| Vital Signs <sup>a</sup> | X | | | X | | | X | | | X |
| CBC with Differential <sup>b</sup> | X | | | X | | | X | | | X |
| Coagulation <sup>b</sup> | X | | | X | | | X | | | X |
| Chemistry Panel <sup>b</sup> | X | | | X | | | X | | | X |
| Lipid Panel <sup>b,c</sup> | X | | | X | | | X | | | X |
| Cholestasis<br>Biomarkers <sup>b,c</sup> | X | | | X | | | X | | | X |
| Fat Soluble<br>Vitamins <sup>b,c,d</sup> | X | | | X | | | X | | | X |

| Study Period | | | | v-up Treatn<br>on Dose Esc | | | Study activities repeat in repeating 12-week periods after completion of the ADE period <sup>h</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | ADE<br>Day 0 | ADE<br>Week 1 | ADE<br>Week 2 | ADE<br>Week 4 | ADE<br>Week 5 | ADE<br>Week 6 | ADE<br>Week 8 | Week 4 | Week 8 | Week 12 |
| Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | Week I | Week 2 | WCCK 4 | week 3 | WEER O | WEEK 8 | The initial Week 4 contact will be scheduled 4 weeks following ADE Week 8. | WEEK | Week 12 |
| Window (in | N/A – see | (12) | (12) | (12) | (12) | (12) | (12) | (17) | (17) | (114) |
| <b>days)</b> Urinalysis <sup>b</sup> | above<br>X | (±2) | (±2) | (±2)<br>X | (±2) | (±2) | (±2)<br>X | (±7) | (±7) | (±14)<br>X <sup>k</sup> |
| AFP Sample | Λ | | | Λ | | | Λ | | | X <sup>i</sup> |
| Plasma Sample<br>for LUM001 <sup>j</sup> | X | | | X | | | X | | | X <sup>j</sup> |
| Serum or Urine<br>Pregnancy Test<br>(if indicated) <sup>e</sup> | X | | | X | | | X | | | Х |
| Clinician Scratch<br>Scale | X | | | X | | | X | | | X |
| Clinician<br>Xanthoma Scale | X | | | X | | | X | | | X |
| Caregiver<br>ItchRO/<br>Patient ItchRO | | | | | | | | | | X (collected for 2 week period following this visit) |
| PedsQL | X | | | X | | | X | | | X |
| Palatability<br>Questionnaire | | | | | | | | | | X |
| Study Drug<br>Supplied <sup>f</sup> | X | | | X | | | X | | | X |
| Assess<br>Compliance | X | | | X | | | X | | | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X |

**08 February 2019** 

| Study Period | | | | v-up Treatn<br>on Dose Esca | | repeat in repeating<br>mpletion of the AD | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Week | ADE<br>Day 0 | ADE<br>Week 1 | ADE<br>Week 2 | ADE<br>Week 4 | ADE<br>Week 5 | ADE<br>Week 8 | Week 4 | Week 8 | Week 12 | |
| Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | | | | | | | The initial Week 4<br>contact will be<br>scheduled 4 weeks<br>following ADE<br>Week 8. | | |
| Window (in days) | N/A – see<br>above | (±2) | (±2) | (±2) | (±2) | (±2) | (±2) | (±7) | (±7) | (±14) |
| Adverse Events | X | X | X | X | X | X | X | X | X | X |
| Follow-up Phone Contact <sup>g</sup> | | X | X | | X | X | | X | X | |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- d Blood samples must be drawn before administration of vitamin supplementation.
- Females of childbearing potential, result must be reviewed prior to dispensing study drug.
- Study drug may be dispensed at unscheduled clinic visits.
- g Subjects must be available to receive a phone call from study staff.
- Study visits will continue in the same pattern until the first of the following occur: (i) subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.
- Sample will be drawn at every other clinic visit starting with RP1 Week 12.
- Pharmacokinetic sample will additionally be collected at the three scheduled clinic visits following completion of the afternoon dose escalation period.
- At indicated visits during treatment period, oxalate will be part of the UA.

| Clinic Visit |
|---------------|
| Phone Contact |

# 16.1.3 Schedule of Procedures G-I: Subject Re-Entry under Protocol Amendment 4

Schedule of Procedures  $\underline{G}$  – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, applicable as follows:

- Subject previously completed (or early terminated from) the long-term optional follow up treatment period as defined under Protocol Amendment 3 and has subsequently experienced an interruption in LUM001 dosing ≥7days.
- Subject is considered eligible for study re-entry under Protocol Amendment 4.
- Subject eligibility will be assessed for afternoon dose escalation at Protocol Amendment 4 DE Week 8 shown in the table below.
  - o If subject is found to be ineligible for ADE, subject will move from Schedule G to Schedule H.
  - o If subject is found to be eligible for ADE, subject will move from Schedule G to Schedule I.

| Study Period | | | | ment 4 Follow-up Ti<br>Dose Escalation (DE) | | | |
|---|---|---|---|---|---|---|---|
| PA4 DE Study<br>Week | PA4<br>DE -2 | PA4<br>DE<br>Day 0 | PA4<br>DE<br>Week 1 | PA4<br>DE<br>Week 2 | PA4<br>DE<br>Week 3 | PA4<br>DE<br>Week 4 | PA4<br>DE<br>Week 8 |
| Scheduling<br>Considerations | -14 | 0 | | | | | |
| Window (in days) | (±14) | (±2) | (±2) | (±2) | (±2) | (±2) | (±14) |
| Informed<br>Consent/Assent | X | | | | | | |
| Assess Eligibility for study re-entry | X | X | | | | | |
| Assess Eligibility for ADE | | | | | | | X |
| Physical Exam | X | X | | | | X | |
| Body Weight &<br>Height | X | X | | | | X | |
| Vital Signs <sup>a</sup> | X | X | | | | X | |
| CBC with<br>Differential <sup>b</sup> | X | X | | | | X | |
| Coagulation <sup>b</sup> | X | X | | | | X | |
| Chemistry Panel <sup>b</sup> | X | X | | | | X | |
| Lipid Panel <sup>b,c</sup> | X | X | | | | X | |
| Cholestasis<br>Biomarkers <sup>b,c</sup> | X | X | | | | X | |

| Study Period | | | | dment 4 Follow-up To<br>Dose Escalation (DE) | | | |
|---|---|---|---|---|---|---|---|
| PA4 DE Study<br>Week | PA4<br>DE -2 | PA4<br>DE<br>Day 0 | PA4<br>DE<br>Week 1 | PA4<br>DE<br>Week 2 | PA4<br>DE<br>Week 3 | PA4<br>DE<br>Week 4 | PA4<br>DE<br>Week 8 |
| Scheduling<br>Considerations | -14 | 0 | | | | | |
| Window (in days) | (±14) | (±2) | (±2) | (±2) | (±2) | (±2) | (±14) |
| Fat Soluble<br>Vitamins <sup>b,c,d</sup> | X | X | | | | X | |
| Urinalysis <sup>b</sup> | X | X | | | | X | |
| Serum or Urine<br>Pregnancy Test (if<br>indicated) <sup>e</sup> | X | X | | | | X | |
| Clinician Scratch<br>Scale | X | X | | | | X | |
| Clinician Xanthoma<br>Scale | X | X | | | | X | |
| Caregiver ItchRO/<br>Patient ItchRO | | | | | | X<br>(collected for 2<br>week period<br>following this visit) | |
| PedsQL | | X | | | | · · | |
| Study Drug Supplied <sup>f</sup> | | X | | | | X | |
| Assess Compliance | | | | | | X | |
| Concomitant<br>Medications | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X |
| Follow-up Phone<br>Contact <sup>g</sup> | | | X | X | X | | X |

- Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- d Blood samples must be drawn before administration of vitamin supplementation.
- <sup>e</sup> Females of childbearing potential, result must be reviewed prior to dispensing study drug.
- Study drug may be dispensed at unscheduled clinic visits.
- Subjects must be available to receive a phone call from study staff.



# Schedule of Procedures $\underline{\mathbf{H}}$ – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, subject ineligible for ADE

| | Below study | activities repeat in r | epeating 12-week periods <sup>h</sup> |
|---|---|---|---|
| Repeating Period Week Scheduling Considerations | Week 4 The Week 4 visit of the first repeating period will take place 4 weeks after PA4 DE Week 8 | Week 8 | Week 12 |
| Window (in days) | (±7) | (±7) | (±14) |
| Physical Exam | | | X |
| Body Weight & Height | | | X |
| Vital Signs <sup>a</sup> | | | X |
| CBC with Differential <sup>b</sup> | | | X |
| Coagulation <sup>b</sup> | | | X |
| Chemistry Panel <sup>b</sup> | | | X |
| Lipid Panel <sup>b,c</sup> | | | X |
| Cholestasis Biomarkers <sup>b,c</sup> | | | X |
| Fat Soluble Vitamins <sup>b,c,d</sup> | | | X |
| Urinalysis <sup>b</sup> | | | $\mathbf{X}^{\mathrm{j}}$ |
| AFP Sample | | | X <sup>i</sup> |
| Serum or Urine Pregnancy Test (if indicated) <sup>e</sup> | | | X |
| Clinician Scratch Scale | | | X |
| Clinician Xanthoma Scale | | | X |
| Caregiver ItchRO/<br>Patient ItchRO | | | X (collected for 2 week period following this visit) |
| PedsQL | | | X |
| Palatability Questionnaire | | | X |
| Study Drug Supplied <sup>f</sup> | | | X |
| Assess Compliance | | | X |
| Concomitant Medications | X | X | X |
| Adverse Events | X | X | X |
| Follow-up Phone Contactg | X | X | |

| | Below study | Below study activities repeat in repeating 12-week periods <sup>h</sup> | |
|---|---|---|---|
| Repeating Period Week | Week 4 | Week 8 | Week 12 |
| | The Week 4 visit of | | |
| | the first repeating | | |
| | period will take place<br>4 weeks after PA4 DE | | |
| Scheduling Considerations | Week 8 | | |
| Window (in days) | (±7) | (±7) | (±14) |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- Blood samples must be drawn before administration of vitamin supplementation.
- <sup>e</sup> Females of childbearing potential, result must be reviewed prior to dispensing study drug.
- Study drug may be dispensed at unscheduled clinic visits.
- Subjects must be available to receive a phone call from study staff.
- Study visits will continue in the same pattern until the first of the following occur: (i) subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.
- Sample will be drawn at every other clinic visit starting with RP1 Week 12
- At indicated visits during treatment period, oxalate will be part of the UA.



# Schedule of Procedures <u>I</u> – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, subject

| eligible for A | <u> Մ</u> ե | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Study Period | | | | w-up Treatm<br>on Dose Esca | | 1 | | Study activities repeating in repeating 12-week periods after completion of the ADE period <sup>h</sup> | | |
| FTP Study | ADE | ADE | ADE | ADE | ADE | ADE | ADE | | | |
| Week | Day 0 | Week 1 | Week 2 | Week 4 | Week 5 | Week 6 | Week 8 | Week 4 | Week 8 | Week 12 |
| Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | | | | | | | The initial Week 4<br>contact will be<br>scheduled 4 weeks<br>following ADE<br>Week 8. | | |
| Window (in days) | N/A – see<br>above | (±2) | (±2) | (±2) | | (±2) | (±2) | (±7) | (±7) | (±14) |
| Physical Exam | X | (±2) | (±2) | X | | (±2) | X | (±1) | (±1) | X |
| Body Weight &<br>Height | X | | | X | | | X | | | X |
| Vital Signs <sup>a</sup> | X | | | X | | | X | | | X |
| CBC with<br>Differential <sup>b</sup> | X | | | X | | | X | | | X |
| Coagulation <sup>b</sup> | X | | | X | | | X | | | X |
| Chemistry Panel <sup>b</sup> | X | | | X | | | X | | | X |
| Lipid Panel <sup>b,c</sup> | X | | | X | | | X | | | X |
| Cholestasis<br>Biomarkers <sup>b,c</sup> | X | | | X | | | X | | | X |
| Fat Soluble<br>Vitamins <sup>b,c,d</sup> | X | | | X | | | X | | | X |
| Urinalysis <sup>b</sup> | X | | | X | | | X | | | $X^k$ |
| AFP Sample | | | | | | | | | | Xi |
| Plasma Sample<br>for LUM001 <sup>j</sup> | X | | | X | | | X | | | X <sup>j</sup> |
| Serum or Urine<br>Pregnancy Test<br>(if indicated) <sup>e</sup> | X | | | X | | | X | | | X |
| Clinician Scratch<br>Scale | X | | | X | | | X | | | X |

| Study Period | Follow-up Treatment Period<br>Afternoon Dose Escalation (ADE) | | | | | | Study activities repeating in repeating 12-week periods after completion of the ADE period <sup>h</sup> | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| FTP Study | ADE | ADE | ADE | ADE | ADE | ADE | ADE | | | |
| Scheduling<br>Considerations | Day 0 To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | Week 1 | Week 2 | Week 4 | Week 5 | Week 6 | Week 8 | Week 4 The initial Week 4 contact will be scheduled 4 weeks following ADE Week 8. | Week 8 | Week 12 |
| Window (in | N/A – see | | | | | | | | | |
| days) Clinician | above | (±2) | (±2) | (±2) | | (±2) | (±2) | (±7) | (±7) | (±14) |
| Xanthoma Scale | X | | | X | | | X | | | X |
| Caregiver<br>ItchRO/<br>Patient ItchRO | | | | | | | | | | X (collected for 2 week period following this visit) |
| PedsQL | X | | | X | | | X | | | X |
| Palatability<br>Questionnaire | | | | | | | | | | X |
| Study Drug<br>Supplied <sup>f</sup> | X | | | X | | | X | | | X |
| Assess<br>Compliance | X | | | X | | | X | | | X |
| Concomitant<br>Medications | X | X | X | X | X | X | X | X | X | X |
| Adverse Events | X | X | X | X | X | X | X | X | X | X |
| Follow-up Phone<br>Contact <sup>g</sup> | | X | X | | X | X | | X | X | |

| Study Period | Follow-up Treatment Period<br>Afternoon Dose Escalation (ADE) | | | | | | epeating in repeating ompletion of the ADI | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| FTP Study | ADE | ADE | ADE | ADE | ADE | ADE | ADE | | | |
| Week | Day 0 | Week 1 | Week 2 | Week 4 | Week 5 | Week 6 | Week 8 | Week 4 | Week 8 | Week 12 |
| Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | | | | | | | The initial Week 4<br>contact will be<br>scheduled 4 weeks<br>following ADE<br>Week 8. | | |
| Window (in | N/A – see | | | | | | | THE CONTROL | | |
| days) | above | (±2) | (±2) | (±2) | | (±2) | (±2) | (±7) | (±7) | (±14) |

- <sup>a</sup> Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- b See Section 16.2 for detailed list of laboratory analytes.
- <sup>c</sup> Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- d Blood samples must be drawn before administration of vitamin supplementation.
- <sup>e</sup> Females of childbearing potential, result must be reviewed prior to dispensing study drug.
- f Study drug may be dispensed at unscheduled clinic visits.
- Subjects must be available to receive a phone call from study staff.
- Study visits will continue in the same pattern until the first of the following occur: (i) subjects are eligible to enter another LUM001 study, or (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication.
- Sample will be drawn at every other clinic visit starting with RP1 Week 129.
- Pharmacokinetic sample will additionally be collected at the three scheduled clinic visits following completion of the afternoon dose escalation period.
- At indicated visits during treatment period, oxalate will be part of the UA.



# 16.1.4 Schedule of Procedures <u>J</u> – Study Termination and End of Treatment Procedures

# Schedule of Procedures $\underline{J}$ – End of Treatment (EOT) / Early Termination (ET) Visit and Post-Treatment Safety Follow Up

| Scheduling Considerations | EOT / ET To take place upon completion of study <sup>g</sup> or at the time of early withdrawal | Safety Follow Up Minimum of 30 days after final dose |
|---|---|---|
| Physical Exam | X | |
| Body Weight & Height | X | |
| Vital Signs <sup>a</sup> | X | |
| CBC with Differential <sup>b</sup> | X | |
| Coagulation <sup>b</sup> | X | |
| Chemistry Panel <sup>b</sup> | X | |
| Lipid Panel <sup>b,c</sup> | X | |
| Cholestasis Biomarkers <sup>b,c</sup> | X | |
| Fat Soluble Vitamins <sup>b,c,d</sup> | X | |
| Urinalysis <sup>b</sup> | X <sup>h</sup> | |
| AFP Sample | X | |
| Serum or Urine Pregnancy<br>Test (if indicated) <sup>e</sup> | X | |
| Clinician Scratch Scale | X | |
| Clinician Xanthoma Scale | X | |
| PedsQL | X<br>X<br>X | |
| Patient/Caregiver<br>Impression of Change | | |
| Caregiver Global Therapeutic Benefit | X | |
| Palatability Questionnaire | X | |
| Assess Compliance | X | |
| Concomitant Medications | X | X |
| Adverse Events | X | X |
| Follow-up Phone Contact <sup>f</sup> | | X |

# Schedule of Procedures $\underline{J}$ – End of Treatment (EOT) / Early Termination (ET) Visit and Post-Treatment Safety Follow Up

| | EOT / ET | Safety Follow Up |
|---|---|---|
| <b>Scheduling Considerations</b> | To take place upon | |
| | completion of study <sup>g</sup> or at | |
| | the time of early | Minimum of 30 days after final |
| | withdrawal | dose |

- Blood pressure (BP), heart rate (HR), temperature, respiration rate.
- See Section 16.2 for detailed list of laboratory analytes.
- Subjects are required to fast at least 4 hrs (only water permitted) prior to collection.
- Blood samples must be drawn before administration of vitamin supplementation.
- Females of childbearing potential.
- Subjects must be available to receive a phone call from study staff.

  Will take place when the first of the following occur: (i) subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) or the sponsor stops the program or development in
- At indicated visits during treatment period, oxalate will be part of the urinalysis.

| Clinic Visit |
|---------------|
| Phone Contact |

## 16.2 List of Laboratory Analytes

| Screening Tests | Clinical Chemistry | Lipid Panela | <u>Urinalysis</u> |
|---|---|---|---|
| JAGGED1/NOTCH2 | Sodium | Total cholesterol | pH |
| Genotyping | Potassium | LDL-C (direct) | Specific gravity |
| (if indicated) | Chloride | HDL-C | Protein |
| Serum βhCG (if indicated) | Bicarbonate | Triglycerides (TG) | Glucose |
| CBC with Differential | Total protein | Cholestasis Biomarkers <sup>1</sup> | Ketones |
| Red blood cells | Albumin | Serum bile acids | Bilirubin |
| Hemoglobin | Calcium | 7α hydroxy-4-cholesten-3- | Occult blood and cells |
| Hematocrit | Phosphorus | one (C4) | Nitrite |
| MCV, MCH, MCHC | Glucose | Fat Soluble Vitaminsb | Urobilinogen |
| Platelets | BUN | 25-hydroxy vitamin D | Leukocyte esterase |
| White blood cells | Creatinine | Retinol | Microscopic examination <sup>c</sup> |
| WBC Differential | Uric Acid | Retinol binding protein | Oxalate <sup>d</sup> |
| (% and absolute) | Total bilirubin | Tocopherol (α) | <b>LUM001 Drug Levels</b> |
| <ul> <li>Neutrophils</li> </ul> | Direct bilirubin | | LUM001 in plasma |
| • Eosinophils | Alkaline phosphatase (ALP) | Marker of hepatocellular carcinoma | |
| <ul> <li>Basophils</li> </ul> | AST (SGOT) | alpha-fetoprotein (AFP) | |
| <ul> <li>Lymphocytes</li> </ul> | ALT (SGPT) | | |
| <ul> <li>Monocytes</li> </ul> | GGT | | |
| Coagulation | 001 | | |
| aPTT (sec) | | | |
| PT (sec) | | | |
| INR | | | |

- <sup>a</sup> Other biomarkers [eg, autotaxin, lysophosphatidic acid (LPA), FGF-19, FGF-21] may be measured at the discretion of the sponsor, samples will be collected and appropriately stored for subsequent analysis, as needed.
- b Blood samples for the analysis of fat soluble vitamins should be drawn prior to administration of vitamin supplementation and approximately 4 hours after food or formula.
- <sup>c</sup> Will be performed on abnormal findings unless otherwise specified.
- d At the specified time points on the Schedule of Procedures (Section 16.1), oxalate will be part of the urinalysis.

# 16.3 Alagille Syndrome Diagnostic Criteria

Major clinical criteria/features for ALGS include: cholestasis, consistent cardiac, renal, vascular, ocular, skeletal involvement, or characteristic "Alagille" facies.

| ALGS Family History <sup>a</sup> | Paucity | JAGGED1 or<br>NOTCH2 Mutation | # Major Clinical<br>Criteria Needed for Diagnosis |
|---|---|---|---|
| Present or Absent | Present | Identified <sup>b</sup> | Any or no features |
| None (proband) | Absent or unknown | Identified | 1 or more features |
| None (proband) | Present | Not identified <sup>c</sup> | 3 or more features |
| None (proband) | Absent or unknown | Not identified | 4 or more features |
| Present | Absent or unknown | Identified | Any or no features |
| Present | Present | Not identified | 1 or more features |
| Present | Absent or unknown | Not identified | 2 or more features |

<sup>&</sup>lt;sup>a</sup> Family history = ALGS present in a first degree relative.

b Identified = JAGGED1 or NOTCH2 mutation identified in clinical laboratory.

Not identified = Not identified on screening, or not screened for.

**08 February 2019** 

## 16.4 Itch Reported Outcome Instrument (ItchRO<sup>TM</sup>)

Many of the ALGS subjects in this study are expected to be between the ages of 2 and 10, necessitating reliance upon an observer-reported outcome instrument (ObsRO) to evaluate a pruritus endpoint.

The ItchRO instrument is being developed both as a patient reported outcome (PRO) instrument for pediatric subjects (9 years of age and older) and an ObsRO for caregivers/parents. The ItchRO will be completed using an electronic diary (eDiary) twice daily (morning and evening) for both the PRO and ObsRO.

### 16.4.1 Patient Itch Reported Outcome Instrument, ItchRO(Pt)<sup>TM</sup>

A screen shot from the ItchRO(Pt) **morning report** is show below. The score associated with each response option is indicated in red text (these will not be shown on the eDiary). The minimum ItchRO(Pt) morning report score is 0 and the maximum score is 4.



If the patient selects "I didn't feel itchy at all" the diary is complete, if not the following screens will be shown on the eDiary:



A screen shot from the ItchRO(Pt) **evening report** is shown below. The score associated with each response option is indicated in red text (these will not be shown on the eDiary). The minimum ItchRO(Pt) evening report score is 0 and the maximum score is 4.



If the patient selects "I didn't feel itchy" the diary is complete, if not the following screen will be shown on the eDiary:



### 16.4.2 Observer Itch Reported Outcome Instrument, ItchRO(Obs)<sup>TM</sup>

A screen shot from the ItchRO(Obs) **morning report** is shown below. The score associated with each response option is indicated in red text (these will not be shown on the eDiary). The minimum ItchRO(Obs) morning report score is 0 and the maximum score is 4.



If the caregiver selects "None observed or reported" the diary is complete, if not the following screen will be shown on the eDiary:



All caregivers will also be required to answer the following question on the ItchRO(Obs) **morning report**:



A screen shot from the ItchRO(Obs) **evening report** is shown below. The score associated with each response option is indicated in red text (these will not be shown on the eDiary). The minimum ItchRO(Obs) evening report score is 0 and the maximum score is 4.



If the caregiver selects "None observed or reported" the diary is complete, if not the following screen will be shown on the eDiary:

| Child reported itching |
|-----------------------------------------------------------------------------|
| Observed difficulty falling asleep<br>or staying asleep (sleep disturbance) |
| Observed rubbing or scratching |
| Observed new or worsening marks or<br>the skin due to rubbing or scratching |
| Observed fussiness or irritability |

All caregivers will also answer the following question on the ItchRO(Obs) evening report:



#### 16.5 Clinician Scratch Scale

This scoring scale was originally developed to assess pruritus before and after surgical intervention in children with ALGS and PFIC (Whitington and Whitington, 1988).

The clinician will rate the subject's pruritus, as evidenced by scratching, according to the following scale:

| Score | Description |
|-------|------------------------------------------------------|
| 0 | None |
| 1 | Rubbing or mild scratching when undistracted |
| 2 | Active scratching without evident skin abrasions |
| 3 | Abrasion evident |
| 4 | Cutaneous mutilation hemorrhage and scarring evident |

#### 16.6 Clinician Xanthoma Scale

This scoring scale was originally developed to assess xanthomas before and after surgical intervention in children with ALGS (Emerick and Whitington, 2002).

The clinician will rate the subject's degree of xanthomatosis according to the following scale:

| Score | Description |
|-------|-------------|
| 0 | None |
| 1 | Minimal |
| 2 | Moderate |
| 3 | Disfiguring |
| 4 | Disabling |

In the study in which this scale was used to assess xanthomas before and after surgical intervention in children with ALGS (Emerick and Whitington, 2002), "minimal" xanthomas represented fewer than 20 scattered individual lesions, "moderate" represented more than 20 lesions that did not interfere with or limit activities, "disfiguring" represented large numbers of lesions that by their large numbers or size caused distortion of the face or extremities, and "disabling" represented xanthomas that interfered with function (such as hand use of ability to walk) because of excess size or number.

**08 February 2019** 

## 16.7 Pediatric Quality of Life Inventory (PedsQL<sup>TM</sup>)

The PedsQL Generic Cores Scale is composed of 23 items to assess pediatric HRQoL measurements across 4 domains: Physical Functioning (8 items), Emotional Functioning (5 items), Social Functioning (5 items), and School Functioning (5 items). Each item consists of a 5-level Likert item survey (0-4). Each PedsQL<sup>TM</sup> age-appropriate form should take less than four minutes to complete.

Pediatric HRQoL measurement instruments must be sensitive to cognitive development and must include both child self-report and parent proxy-report. Accordingly, the PedsQL consists of developmentally appropriate forms for children ages 1-12 months and 13-24 months, and 2-4, 5-7, 8-12, and 13-18 years. Pediatric self-report is measured in children and adolescents ages 5-18 years, and parent proxy-report of child HRQOL is measured for children and adolescents ages 2-18 years. Subjects will continue to fill out the same questionnaire used at baseline for continuity of data collection, regardless of subsequent birthdays after the baseline visit.

Quality of life will be assessed using the appropriate PedsQL<sup>TM</sup> module(s) provided below.

## 16.7.1 Parent Report for Infants (1 to 12 months)

| ID# |
|-------|
| Date: |



PARENT REPORT for INFANTS (ages 1-12 months)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for your child. Please tell us how much of a problem each one has been for your child during the past ONE month by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

In the past ONE month, how much of a problem has your child had with .

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Low energy level | 0 | 1 | 2 | 3 | 4 |
| Difficulty participating in active play | 0 | 1 | 2 | 3 | 4 |
| Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling tired | 0 | 1 | 2 | 3 | 4 |
| 5. Being lethargic | 0 | 1 | 2 | 3 | 4 |
| 6. Resting a lot | 0 | 1 | 2 | 3 | 4 |

| PHYSICAL SYMPTOMS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Having gas | 0 | 1 | 2 | 3 | 4 |
| Spitting up after eating | 0 | 1 | 2 | 3 | 4 |
| Difficulty breathing | 0 | 1 | 2 | 3 | 4 |
| 4. Being sick to his/her stomach | 0 | 1 | 2 | 3 | 4 |
| 5. Difficulty swallowing | 0 | 1 | 2 | 3 | 4 |
| Being constipated | 0 | 1 | 2 | 3 | 4 |
| 7. Having a rash | 0 | 1 | 2 | 3 | 4 |
| 8. Having diarrhea | 0 | 1 | 2 | 3 | 4 |
| 9. Wheezing | 0 | 1 | 2 | 3 | 4 |
| 10. Vomiting | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 3. Crying or fussing when left alone | 0 | 1 | 2 | 3 | 4 |
| 4. Difficulty soothing himself/herself when upset | 0 | 1 | 2 | 3 | 4 |
| Difficulty falling asleep | 0 | 1 | 2 | 3 | 4 |
| 6. Crying or fussing while being cuddled | 0 | 1 | 2 | 3 | 4 |
| 7. Feeling sad | 0 | 1 | 2 | 3 | 4 |
| 8. Difficulty being soothed when picked up or held | 0 | 1 | 2 | 3 | 4 |
| 9. Difficulty sleeping mostly through the night | 0 | 1 | 2 | 3 | 4 |
| 10. Crying a lot | 0 | 1 | 2 | 3 | 4 |
| 11. Feeling cranky | 0 | 1 | 2 | 3 | 4 |
| 12. Difficulty taking naps during the day | 0 | 1 | 2 | 3 | 4 |

PedsQL™ Infant Scales 1-12 months Not to be reproduced without permission Copyright © 1998 JW Varni, Ph.D. All rights reserved 1/10
PedsQL 3

## In the past ONE month, how much of a problem has your child had with ...

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Not smiling at others | 0 | 1 | 2 | 3 | 4 |
| Not laughing when tickled | 0 | 1 | 2 | 3 | 4 |
| 3. Not making eye contact with a caregiver | 0 | 1 | 2 | 3 | 4 |
| Not laughing when cuddled | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Not imitating caregivers' actions | 0 | 1 | 2 | 3 | 4 |
| 2. Not imitating caregivers' facial expressions | 0 | 1 | 2 | 3 | 4 |
| 3. Not imitating caregivers' sounds | 0 | 1 | 2 | 3 | 4 |
| 4. Not able to fix his/her attention on objects | 0 | 1 | 2 | 3 | 4 |

#### 16.7.2 Parent Report for Infants (13 to 24 months)

| ID# | _ |
|-------|---|
| _ | |
| Date: | |

# PedsQL Pediatric Quality of Life Inventory Infant Scales

PARENT REPORT for INFANTS (ages 13-24 months)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**. Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

0 if it is never a problem
1 if it is almost never a problem
2 if it is sometimes a problem
3 if it is often a problem
4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

In the past **ONE month**, how much of a **problem** has your child had with ...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Low energy level | 0 | 1 | 2 | 3 | 4 |
| Difficulty participating in active play | 0 | 1 | 2 | 3 | 4 |
| 3. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling tired | 0 | 1 | 2 | 3 | 4 |
| 5. Being lethargic | 0 | 1 | 2 | 3 | 4 |
| 6. Resting a lot | 0 | 1 | 2 | 3 | 4 |
| 7. Feeling too tired to play | 0 | 1 | 2 | 3 | 4 |
| 8. Difficulty walking | 0 | 1 | 2 | 3 | 4 |
| Difficulty running a short distance without falling | 0 | 1 | 2 | 3 | 4 |

| PHYSICAL SYMPTOMS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Having gas | 0 | 1 | 2 | 3 | 4 |
| 2. Spitting up after eating | 0 | 1 | 2 | 3 | 4 |
| 3. Difficulty breathing | 0 | 1 | 2 | 3 | 4 |
| 4. Being sick to his/her stomach | 0 | 1 | 2 | 3 | 4 |
| 5. Difficulty swallowing | 0 | 1 | 2 | 3 | 4 |
| 6. Being constipated | 0 | 1 | 2 | 3 | 4 |
| 7. Having a rash | 0 | 1 | 2 | 3 | 4 |
| 8. Having diarrhea | 0 | 1 | 2 | 3 | 4 |
| 9. Wheezing | 0 | 1 | 2 | 3 | 4 |
| 10. Vomiting | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| Crying or fussing when left alone | 0 | 1 | 2 | 3 | 4 |
| Difficulty soothing himself/herself when upset | 0 | 1 | 2 | 3 | 4 |
| 5. Difficulty falling asleep | 0 | 1 | 2 | 3 | 4 |
| Crying or fussing while being cuddled | 0 | 1 | 2 | 3 | 4 |
| 7. Feeling sad | 0 | 1 | 2 | 3 | 4 |
| Difficulty being soothed when picked up or held | 0 | 1 | 2 | 3 | 4 |
| Difficulty sleeping mostly through the night | 0 | 1 | 2 | 3 | 4 |
| 10. Crying a lot | 0 | 1 | 2 | 3 | 4 |
| 11.Feeling cranky | 0 | 1 | 2 | 3 | 4 |
| 12. Difficulty taking naps during the day | 0 | 1 | 2 | 3 | 4 |

PedsQL™ Infant Scales 13-24 months Not to be reproduced without permission Copyright © 1998 JW Varni, Ph.D. All rights reserved 1/10

PedsQL 3

In the past **ONE month**, how much of a **problem** has your child had with ...

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Not smiling at others | 0 | 1 | 2 | 3 | 4 |
| Not laughing when tickled | 0 | 1 | 2 | 3 | 4 |
| Not making eye contact with a caregiver | 0 | 1 | 2 | 3 | 4 |
| Not laughing when cuddled | 0 | 1 | 2 | 3 | 4 |
| 5. Being uncomfortable around other children | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Not imitating caregivers' actions | 0 | 1 | 2 | 3 | 4 |
| Not imitating caregivers' facial expressions | 0 | 1 | 2 | 3 | 4 |
| Not imitating caregivers' sounds | 0 | 1 | 2 | 3 | 4 |
| 4. Not able to fix his/her attention on objects | 0 | 1 | 2 | 3 | 4 |
| 5. Not imitating caregivers' speech | 0 | 1 | 2 | 3 | 4 |
| 6. Difficulty pointing to his/her body parts when asked | 0 | 1 | 2 | 3 | 4 |
| 7. Difficulty naming familiar objects | 0 | 1 | 2 | 3 | 4 |
| Difficulty repeating words | 0 | 1 | 2 | 3 | 4 |
| Difficulty keeping his/her attention on things | 0 | 1 | 2 | 3 | 4 |

#### 16.7.3 Parent Report for Toddlers (ages 2-4)

| ID# |
|-------|
| Date: |



Version 4.0 - Language (Country)

#### PARENT REPORT for TODDLERS (ages 2-4)

#### DIRECTIONS

On the following page is a list of things that might be a problem for your child. Please tell us how much of a problem each one has been for your child during the past ONE month by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2
In the past **ONE month**, how much of a **problem** has your child had with ...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. Walking | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| Participating in active play or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Bathing | 0 | 1 | 2 | 3 | 4 |
| 6. Helping to pick up his or her toys | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying | 0 | 1 | 2 | 3 | 4 |

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Playing with other children | 0 | 1 | 2 | 3 | 4 |
| 2. Other kids not wanting to play with him or her | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other children | 0 | 1 | 2 | 3 | 4 |
| Not able to do things that other children his or her age can do | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up when playing with other children | 0 | 1 | 2 | 3 | 4 |

\*Please complete this section if your child attends school or daycare

| SCHOOL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Doing the same school activities as peers | 0 | 1 | 2 | 3 | 4 |
| Missing school/daycare because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| Missing school/daycare to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

#### 16.7.4 Parent Report for Young Children (ages 5-7)

| ID# |
|-------|
| Date: |



Version 4.0

#### PARENT REPORT for YOUNG CHILDREN (ages 5-7)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for your child. Please tell us how much of a problem each one has been for your child during the past ONE month by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2
In the past **ONE month**, how much of a **problem** has your child had with ...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Walking more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| Participating in sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a bath or shower by him or herself | 0 | 1 | 2 | 3 | 4 |
| 6. Doing chores, like picking up his or her toys | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying about what will happen to him or her | 0 | 1 | 2 | 3 | 4 |

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Getting along with other children | 0 | 1 | 2 | 3 | 4 |
| 2. Other kids not wanting to be his or her friend | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other children | 0 | 1 | 2 | 3 | 4 |
| Not able to do things that other children his or her age can do | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up when playing with other children | 0 | 1 | 2 | 3 | 4 |

| SCHOOL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Paying attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. Forgetting things | 0 | 1 | 2 | 3 | 4 |
| Keeping up with school activities | 0 | 1 | 2 | 3 | 4 |
| 4. Missing school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. Missing school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

PedsQL 4.0 - Parent (5-7)  $\,$  Not to be reproduced without permission  $01/00\,$ 

Copyright © 1998 JW Varni, Ph.D. All rights reserved

#### 16.7.5 Parent Report for Children (ages 8-12)

| ID# |
|-------|
| Date: |



Version 4.0

#### PARENT REPORT for CHILDREN (ages 8-12)

#### DIRECTIONS

On the following page is a list of things that might be a problem for your child. Please tell us how much of a problem each one has been for your child during the past ONE month by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

 $$\operatorname{PedsQL}\ 2$$  In the past **ONE month**, how much of a **problem** has your child had with ...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Walking more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| 3. Participating in sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a bath or shower by him or herself | 0 | 1 | 2 | 3 | 4 |
| 6. Doing chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying about what will happen to him or her | 0 | 1 | 2 | 3 | 4 |

| SOCIAL FUNCTIONING (problems with) | | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Getting along with other children | 0 | 1 | 2 | 3 | 4 |
| Other kids not wanting to be his or her friend | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other children | 0 | 1 | 2 | 3 | 4 |
| Not able to do things that other children his or her age can do | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up when playing with other children | 0 | 1 | 2 | 3 | 4 |

| SCHOOL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Paying attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. Forgetting things | 0 | 1 | 2 | 3 | 4 |
| Keeping up with schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. Missing school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. Missing school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

PedsQL 4.0 - Parent (8-12)  $\,$  Not to be reproduced without permission 01/00  $\,$ 

Copyright © 1998 JW Varni, Ph.D. All rights reserved

#### 16.7.6 Parent Report for Teenagers (ages 13-18)

| ID# |
|-------|
| Date: |



Version 4.0

#### PARENT REPORT for TEENS (ages 13-18)

#### DIRECTIONS

On the following page is a list of things that might be a problem for your teen. Please tell us how much of a problem each one has been for your teen during the past ONE month by circling:

0 if it is never a problem
1 if it is almost never a problem
2 if it is sometimes a problem
3 if it is often a problem
4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

In the past **ONE month**, how much of a **problem** has your teen had with ...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Walking more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. Running | 0 | 1 | 2 | 3 | 4 |
| 3. Participating in sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. Lifting something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a bath or shower by him or herself | 0 | 1 | 2 | 3 | 4 |
| 6. Doing chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. Having hurts or aches | 0 | 1 | 2 | 3 | 4 |
| 8. Low energy level | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. Feeling sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling angry | 0 | 1 | 2 | 3 | 4 |
| 4. Trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. Worrying about what will happen to him or her | 0 | 1 | 2 | 3 | 4 |

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Getting along with other teens | 0 | 1 | 2 | 3 | 4 |
| 2. Other teens not wanting to be his or her friend | 0 | 1 | 2 | 3 | 4 |
| Getting teased by other teens | 0 | 1 | 2 | 3 | 4 |
| 4. Not able to do things that other teens his or her age can do | 0 | 1 | 2 | 3 | 4 |
| 5. Keeping up with other teens | 0 | 1 | 2 | 3 | 4 |

| SCHOOL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Paying attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. Forgetting things | 0 | 1 | 2 | 3 | 4 |
| Keeping up with schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. Missing school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| Missing school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

#### 16.7.7 Pediatric Quality of Life Inventory v 4.0 for Young Children (ages 5-7)



Version 4.0 - Language (Country)

YOUNG CHILD REPORT (ages 5-7)

Instructions for interviewer:

I am going to ask you some questions about things that might be a problem for some children. I want to know how much of a problem any of these things might be for you.

Show the child the template and point to the responses as you read.

If it is not at all a problem for you, point to the smiling face

If it is sometimes a problem for you, point to the middle face

If it is a problem for you a lot, point to the frowning face

I will read each question. Point to the pictures to show me how much of a problem it is for you. Let's try a practice one first.

| | Not at all | Sometimes | A lot |
|-----------------------------------------|------------|-----------|---------|
| Is it hard for you to snap your fingers | $\odot$ | <u>:</u> | $\odot$ |

Ask the child to demonstrate snapping his or her fingers to determine whether or not the question was answered correctly. Repeat the question if the child demonstrates a response that is different from his or her action.

PedsQL 2

# Think about how you have been doing for the last few weeks. Please listen carefully to each sentence and tell me how much of a problem this is for you.

After reading the item, gesture to the template. If the child hesitates or does not seem to understand how to answer, read the response options while pointing at the faces.

| PHYSICAL FUNCTIONING (problems with) | Not at all | Some-<br>times | A lot |
|---|---|---|---|
| Is it hard for you to walk | 0 | 2 | 4 |
| 2. Is it hard for you to run | 0 | 2 | 4 |
| Is it hard for you to play sports or exercise | 0 | 2 | 4 |
| 4. Is it hard for you to pick up big things | 0 | 2 | 4 |
| 5. Is it hard for you to take a bath or shower | 0 | 2 | 4 |
| 6. Is it hard for you to do chores (like pick up your toys) | 0 | 2 | 4 |
| 7. Do you have hurts or aches (Where?) | 0 | 2 | 4 |
| Do you ever feel too tired to play | 0 | 2 | 4 |

Remember, tell me how much of a problem this has been for you for the last few weeks.

| EMOTIONAL FUNCTIONING (problems with) | Not at all | Some-<br>times | A lot |
|---|---|---|---|
| Do you feel scared | 0 | 2 | 4 |
| 2. Do you feel sad | 0 | 2 | 4 |
| Do you feel mad | 0 | 2 | 4 |
| Do you have trouble sleeping | 0 | 2 | 4 |
| 5. Do you worry about what will happen to you | 0 | 2 | 4 |

| SOCIAL FUNCTIONING (problems with) | Not at all | Some-<br>times | A lot |
|---|---|---|---|
| Is it hard for you to get along with other kids | 0 | 2 | 4 |
| 2. Do other kids say they do not want to play with you | 0 | 2 | 4 |
| Do other kids tease you | 0 | 2 | 4 |
| Can other kids do things that you cannot do | 0 | 2 | 4 |
| Is it hard for you to keep up when you play with other kids | 0 | 2 | 4 |

| SCHOOL FUNCTIONING (problems with) | Not at all | Some-<br>times | A lot |
|---|---|---|---|
| Is it hard for you to pay attention in school | 0 | 2 | 4 |
| 2. Do you forget things | 0 | 2 | 4 |
| Is it hard to keep up with schoolwork | 0 | 2 | 4 |
| 4. Do you miss school because of not feeling good | 0 | 2 | 4 |
| Do you miss school because you have to go to the doctor's or hospital | 0 | 2 | 4 |

PedsQL 3

## How much of a problem is this for you?

Not at all



Sometimes



A lot



PedsQL 4.0 - (5-7)

PedsQL-4.0-Core - United States/English - Mapi. PedsQL-4.0-Core-YC\_eng-USorl.doc Not to be reproduced without permission

Copyright © 1998 JW Varni, Ph.D. All rights reserved

#### 16.7.8 Pediatric Quality of Life Inventory for Children (ages 8-12)

| ID#_ |
|-------|
| Date: |



Version 4.0 - Language (Country)

CHILD REPORT (ages 8-12)

#### DIRECTIONS

On the following page is a list of things that might be a problem for you. Please tell us how much of a problem each one has been for you during the past ONE month by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

## In the past **ONE month**, how much of a **problem** has this been for you ...

| ABOUT MY HEALTH AND ACTIVITIES (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard for me to walk more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to run | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to do sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to lift something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard for me to take a bath or shower by myself | 0 | 1 | 2 | 3 | 4 |
| 6. It is hard for me to do chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. I hurt or ache | 0 | 1 | 2 | 3 | 4 |
| 8. I have low energy | 0 | 1 | 2 | 3 | 4 |

| ABOUT MY FEELINGS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. I feel sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. I feel angry | 0 | 1 | 2 | 3 | 4 |
| 4. I have trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. I worry about what will happen to me | 0 | 1 | 2 | 3 | 4 |

| How I GET ALONG WITH OTHERS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I have trouble getting along with other kids | 0 | 1 | 2 | 3 | 4 |
| 2. Other kids do not want to be my friend | 0 | 1 | 2 | 3 | 4 |
| 3. Other kids tease me | 0 | 1 | 2 | 3 | 4 |
| 4. I cannot do things that other kids my age can do | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard to keep up when I play with other kids | 0 | 1 | 2 | 3 | 4 |

| ABOUT SCHOOL (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard to pay attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. I forget things | 0 | 1 | 2 | 3 | 4 |
| 3. I have trouble keeping up with my schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. I miss school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. I miss school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

#### 16.7.9 Pediatric Quality of Life Inventory for Teenagers (ages 13-18)

| ID# |
|-------|
| Date: |



Version 4.0 - Language (Country)

TEEN REPORT (ages 13-18)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for you. Please tell us **how much of a problem** each one has been for you during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

## In the past **ONE month**, how much of a **problem** has this been for you ...

| ABOUT MY HEALTH AND ACTIVITIES (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard for me to walk more than one block | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to run | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to do sports activity or exercise | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to lift something heavy | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard for me to take a bath or shower by myself | 0 | 1 | 2 | 3 | 4 |
| 6. It is hard for me to do chores around the house | 0 | 1 | 2 | 3 | 4 |
| 7. I hurt or ache | 0 | 1 | 2 | 3 | 4 |
| 8. I have low energy | 0 | 1 | 2 | 3 | 4 |

| ABOUT MY FEELINGS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel afraid or scared | 0 | 1 | 2 | 3 | 4 |
| 2. I feel sad or blue | 0 | 1 | 2 | 3 | 4 |
| 3. I feel angry | 0 | 1 | 2 | 3 | 4 |
| 4. I have trouble sleeping | 0 | 1 | 2 | 3 | 4 |
| 5. I worry about what will happen to me | 0 | 1 | 2 | 3 | 4 |

| HOW I GET ALONG WITH OTHERS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I have trouble getting along with other teens | 0 | 1 | 2 | 3 | 4 |
| 2. Other teens do not want to be my friend | 0 | 1 | 2 | 3 | 4 |
| 3. Other teens tease me | 0 | 1 | 2 | 3 | 4 |
| 4. I cannot do things that other teens my age can do | 0 | 1 | 2 | 3 | 4 |
| 5. It is hard to keep up with my peers | 0 | 1 | 2 | 3 | 4 |

| ABOUT SCHOOL (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard to pay attention in class | 0 | 1 | 2 | 3 | 4 |
| 2. I forget things | 0 | 1 | 2 | 3 | 4 |
| 3. I have trouble keeping up with my schoolwork | 0 | 1 | 2 | 3 | 4 |
| 4. I miss school because of not feeling well | 0 | 1 | 2 | 3 | 4 |
| 5. I miss school to go to the doctor or hospital | 0 | 1 | 2 | 3 | 4 |

#### 16.7.10 Multidimensional Fatigue Scale Parent Report for Toddlers (ages 2-4)

| ID# |
|-------|
| Date: |



Standard Version

#### PARENT REPORT for TODDLERS (ages 2-4)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**. Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

In the past **ONE month**, how much of a **problem** has this been for your child ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling tired | 0 | 1 | 2 | 3 | 4 |
| Feeling physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling too tired to do things that he/she likes to do | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling too tired to spend time with his/her friends | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| 6. Trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. Sleeping a lot | 0 | 1 | 2 | 3 | 4 |
| Difficulty sleeping through the night | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling tired when he/she wakes up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. Resting a lot | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a lot of naps | 0 | 1 | 2 | 3 | 4 |
| 6. Spending a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Difficulty keeping his/her attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. Difficulty remembering what people tell him/her | 0 | 1 | 2 | 3 | 4 |
| 3. Difficulty remembering what he/she just heard | 0 | 1 | 2 | 3 | 4 |
| 4. Difficulty thinking quickly | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble remembering what he/she was just thinking | 0 | 1 | 2 | 3 | 4 |
| 6. Trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

# 16.7.11 Multidimensional Fatigue Scale Parent Report for Young Children (ages 5-7)

| ID#_ | - |
|-------|---|
| Date: | |



Standard Version

#### PARENT REPORT for YOUNG CHILDREN (ages 5-7)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**. Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

0 if it is never a problem
1 if it is almost never a problem
2 if it is sometimes a problem
3 if it is often a problem
4 if it is almost always a problem

There are no right or wrong answers. If you do not understand a question, please ask for help.

PedsQL 2

In the past **ONE month**, how much of a **problem** has this been for your child ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling tired | 0 | 1 | 2 | 3 | 4 |
| Feeling physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling too tired to do things that he/she likes to do | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling too tired to spend time with his/her friends | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| Trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Sleeping a lot | 0 | 1 | 2 | 3 | 4 |
| Difficulty sleeping through the night | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling tired when he/she wakes up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. Resting a lot | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a lot of naps | 0 | 1 | 2 | 3 | 4 |
| 6. Spending a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Difficulty keeping his/her attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. Difficulty remembering what people tell him/her | 0 | 1 | 2 | 3 | 4 |
| 3. Difficulty remembering what he/she just heard | 0 | 1 | 2 | 3 | 4 |
| Difficulty thinking quickly | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble remembering what he/she was just thinking | 0 | 1 | 2 | 3 | 4 |
| 6. Trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

#### 16.7.12 Multidimensional Fatigue Scale Parent Report for Children (ages 8-12)

| ID# |
|-------|
| Date: |



Standard Version

#### PARENT REPORT for CHILDREN (ages 8-12)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**. Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

#### In the past **ONE month**, how much of a **problem** has this been for your child ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling tired | 0 | 1 | 2 | 3 | 4 |
| Feeling physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling too tired to do things that he/she likes to do | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling too tired to spend time with his/her friends | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| 6. Trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Sleeping a lot | 0 | 1 | 2 | 3 | 4 |
| Difficulty sleeping through the night | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling tired when he/she wakes up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. Resting a lot | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a lot of naps | 0 | 1 | 2 | 3 | 4 |
| Spending a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| C | OGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|---|
| 1. | Difficulty keeping his/her attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. | Difficulty remembering what people tell him/her | 0 | 1 | 2 | 3 | 4 |
| 3. | Difficulty remembering what he/she just heard | 0 | 1 | 2 | 3 | 4 |
| 4. | Difficulty thinking quickly | 0 | 1 | 2 | 3 | 4 |
| 5. | Trouble remembering what he/she was just thinking | 0 | 1 | 2 | 3 | 4 |
| 6. | Trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

#### 16.7.13 Multidimensional Fatigue Scale Parent Report for Teenagers (ages 13-18)

| ID# |
|-------|
| Date: |



Standard Version

PARENT REPORT for TEENS (ages 13-18)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for **your child**. Please tell us **how much of a problem** each one has been for **your child** during the **past ONE month** by circling:

0 if it is never a problem
1 if it is almost never a problem
2 if it is sometimes a problem
3 if it is often a problem
4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2

In the past ONE month, how much of a problem has this been for your child ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Feeling tired | 0 | 1 | 2 | 3 | 4 |
| Feeling physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling too tired to do things that he/she likes to do | 0 | 1 | 2 | 3 | 4 |
| 4. Feeling too tired to spend time with his/her friends | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| Trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. Sleeping a lot | 0 | 1 | 2 | 3 | 4 |
| Difficulty sleeping through the night | 0 | 1 | 2 | 3 | 4 |
| 3. Feeling tired when he/she wakes up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. Resting a lot | 0 | 1 | 2 | 3 | 4 |
| 5. Taking a lot of naps | 0 | 1 | 2 | 3 | 4 |
| 6. Spending a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Difficulty keeping his/her attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. Difficulty remembering what people tell him/her | 0 | 1 | 2 | 3 | 4 |
| 3. Difficulty remembering what he/she just heard | 0 | 1 | 2 | 3 | 4 |
| Difficulty thinking quickly | 0 | 1 | 2 | 3 | 4 |
| 5. Trouble remembering what he/she was just thinking | 0 | 1 | 2 | 3 | 4 |
| 6. Trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

#### 16.7.14 Multidimensional Fatigue Scale Young Child Report (ages 5-7)

| ID#_ |
|-------|
| Date: |



Standard Version

YOUNG CHILD REPORT (ages 5-7)

Instructions for interviewer:

I am going to ask you some questions about things that might be a problem for some children. I want to know how much of a problem any of these things might be for you.

Show the child the template and point to the responses as you read.

If it is not at all a problem for you, point to the smiling face

If it is sometimes a problem for you, point to the middle face

If it is a problem for you a lot, point to the frowning face

I will read each question. Point to the pictures to show me how much of a problem it is for you. Let's try a practice one first.

| | Not at all | Sometimes | A lot |
|-----------------------------------------|------------|-----------|-------|
| Is it hard for you to snap your fingers | $\odot$ | <u></u> | 8 |

Ask the child to demonstrate snapping his or her fingers to determine whether or not the question was answered correctly. Repeat the question if the child demonstrates a response that is different from his or her action.

Do you have trouble starting things

PedsQL 2

# Think about how you have been doing for the past few weeks. Please listen carefully to each sentence and tell me how much of a problem this is for you.

After reading the item, gesture to the template. If the child hesitates or does not seem to understand how to answer, read the response options while pointing at the faces.

| General Fatigue (PROBLEMS WITH) | NOT AT<br>ALL | SOME-<br>TIMES | A LOT |
|---|---|---|---|
| Do you feel tired | 0 | 2 | 4 |
| Do you feel physically weak (not strong) | 0 | 2 | 4 |
| Do you feel too tired to do things that you like to do | 0 | 2 | 4 |
| Do you feel too tired to spend time with your friends | 0 | 2 | 4 |
| 5 Do you have trouble finishing things | 0 | 2 | 4 |

Remember, tell me how much of a problem this has been for you for the last few weeks.

| Sleep/Rest Fatigue (PROBLEMS WITH) | | SOME- | A LOT |
|---------------------------------------------------|-----|-------|-------|
| , | ALL | TIMES | |
| Do you sleep a lot | 0 | 2 | 4 |
| Is it hard for you to sleep through the night | 0 | 2 | 4 |
| Do you feel tired when you wake up in the morning | 0 | 2 | 4 |
| 4. Do you rest a lot | 0 | 2 | 4 |
| 5. Do you take a lot of naps | 0 | 2 | 4 |
| Do you spend a lot of time in bed | 0 | 2 | 4 |

| Cognitive Fatigue (PROBLEMS WITH) | | SOME-<br>TIMES | A LOT |
|---|---|---|---|
| Is it hard for you to keep your attention on things | 0 | 2 | 4 |
| Is it hard for you to remember what people tell you | 0 | 2 | 4 |
| Is it hard for you to remember what you just heard | 0 | 2 | 4 |
| 4. Is it hard for you to think quickly | 0 | 2 | 4 |
| 5. Do you have trouble remembering what you were just thinking | 0 | 2 | 4 |
| Do you have trouble remembering more than one thing at a time | 0 | 2 | 4 |

0

PedsQL 3

# How much of a problem is this for you?

Not at all



A lot







PedsQL (5-7) Fatigue Not to be reproduced without permission 05/01 PedsQL TM Multidimensional Fatigue Scale - Young child (5-7) - United States/English PedsQcL-Fatigue-YC-NU4 Beng-USonq Not to be reproduced without permission

Copyright © 1998 JWVarni, Ph.D. All rights reserved

#### 16.7.15 Multidimensional Fatigue Scale Child Report (ages 8-12)

| Γ | ID# |
|---|-------|
| | Date: |



Standard Version

CHILD REPORT (ages 8-12)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for you. Please tell us **how much of a problem** each one has been for you during the **past ONE month** by circling:

0 if it is never a problem
1 if it is almost never a problem
2 if it is sometimes a problem
3 if it is often a problem
4 if it is almost always a problem

There are no right or wrong answers. If you do not understand a question, please ask for help.

PedsQL 2

### In the past ONE month, how much of a problem has this been for you ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. I feel tired | 0 | 1 | 2 | 3 | 4 |
| 2. I feel physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. I feel too tired to do things that I like to do | 0 | 1 | 2 | 3 | 4 |
| 4. I feel too tired to spend time with my friends | 0 | 1 | 2 | 3 | 4 |
| 5. I have trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| 6. I have trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. I sleep a lot | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to sleep through the night | 0 | 1 | 2 | 3 | 4 |
| 3. I feel tired when I wake up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. I rest a lot | 0 | 1 | 2 | 3 | 4 |
| 5. I take a lot of naps | 0 | 1 | 2 | 3 | 4 |
| 6. I spend a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard for me to keep my attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to remember what people tell me | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to remember what I just heard | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to think quickly | 0 | 1 | 2 | 3 | 4 |
| 5. I have trouble remembering what I was just thinking | 0 | 1 | 2 | 3 | 4 |
| I have trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

#### 16.7.16 Multidimensional Fatigue Scale Teen Report (ages 13-18)

| ID# |
|-------|
| Date: |



Standard Version

TEEN REPORT (ages 13-18)

#### **DIRECTIONS**

On the following page is a list of things that might be a problem for you. Please tell us **how much of a problem** each one has been for you during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

2 if it is sometimes a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers. If you do not understand a question, please ask for help.

PedsQL 2

## In the past ONE month, how much of a problem has this been for you ...

| GENERAL FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. I feel tired | 0 | 1 | 2 | 3 | 4 |
| 2. I feel physically weak (not strong) | 0 | 1 | 2 | 3 | 4 |
| 3. I feel too tired to do things that I like to do | 0 | 1 | 2 | 3 | 4 |
| 4. I feel too tired to spend time with my friends | 0 | 1 | 2 | 3 | 4 |
| 5. I have trouble finishing things | 0 | 1 | 2 | 3 | 4 |
| I have trouble starting things | 0 | 1 | 2 | 3 | 4 |

| SLEEP/REST FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. I sleep a lot | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to sleep through the night | 0 | 1 | 2 | 3 | 4 |
| 3. I feel tired when I wake up in the morning | 0 | 1 | 2 | 3 | 4 |
| 4. I rest a lot | 0 | 1 | 2 | 3 | 4 |
| 5. I take a lot of naps | 0 | 1 | 2 | 3 | 4 |
| 6. I spend a lot of time in bed | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FATIGUE (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| 1. It is hard for me to keep my attention on things | 0 | 1 | 2 | 3 | 4 |
| 2. It is hard for me to remember what people tell me | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to remember what I just heard | 0 | 1 | 2 | 3 | 4 |
| 4. It is hard for me to think quickly | 0 | 1 | 2 | 3 | 4 |
| 5. I have trouble remembering what I was just thinking | 0 | 1 | 2 | 3 | 4 |
| I have trouble remembering more than one thing at a time | 0 | 1 | 2 | 3 | 4 |

#### 16.7.17 Family Impact Module v 2.0

| ID#_ |
|-------|
| Date: |



Version 2.0

#### PARENT REPORT

#### DIRECTIONS

Families of children sometimes have special concerns or difficulties because of the child's health. On the following page is a list of things that might be a problem for **you**. Please tell us **how much of a problem** each one has been for **you** during the **past ONE month** by circling:

0 if it is never a problem

1 if it is almost never a problem

 $\boldsymbol{2}$  if it is  $\boldsymbol{sometimes}$  a problem

3 if it is often a problem

4 if it is almost always a problem

There are no right or wrong answers.

If you do not understand a question, please ask for help.

PedsQL 2 In the past **ONE month**, as a result of your child's health, how much of a problem have **you** had with...

| PHYSICAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel tired during the day | 0 | 1 | 2 | 3 | 4 |
| I feel tired when I wake up in the morning | 0 | 1 | 2 | 3 | 4 |
| I feel too tired to do the things I like to do | 0 | 1 | 2 | 3 | 4 |
| I get headaches | 0 | 1 | 2 | 3 | 4 |
| I feel physically weak | 0 | 1 | 2 | 3 | 4 |
| I feel sick to my stomach | 0 | 1 | 2 | 3 | 4 |

| EMOTIONAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel anxious | 0 | 1 | 2 | 3 | 4 |
| 2. I feel sad | 0 | 1 | 2 | 3 | 4 |
| 3. I feel angry | 0 | 1 | 2 | 3 | 4 |
| I feel frustrated | 0 | 1 | 2 | 3 | 4 |
| I feel helpless or hopeless | 0 | 1 | 2 | 3 | 4 |

| SOCIAL FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel isolated from others | 0 | 1 | 2 | 3 | 4 |
| I have trouble getting support from others | 0 | 1 | 2 | 3 | 4 |
| It is hard to find time for social activities | 0 | 1 | 2 | 3 | 4 |
| I do not have enough energy for social activities | 0 | 1 | 2 | 3 | 4 |

| COGNITIVE FUNCTIONING (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| It is hard for me to keep my attention on things | 0 | 1 | 2 | 3 | 4 |
| It is hard for me to remember what people tell me | 0 | 1 | 2 | 3 | 4 |
| It is hard for me to remember what I just heard | 0 | 1 | 2 | 3 | 4 |
| It is hard for me to think quickly | 0 | 1 | 2 | 3 | 4 |
| 5. I have trouble remembering what I was just thinking | 0 | 1 | 2 | 3 | 4 |

| COMMUNICATION (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I feel that others do not understand my family's situation | 0 | 1 | 2 | 3 | 4 |
| It is hard for me to talk about my child's health with others | 0 | 1 | 2 | 3 | 4 |
| 3. It is hard for me to tell doctors and nurses how I feel | 0 | 1 | 2 | 3 | 4 |
PedsQL 3 In the past **ONE month**, as a result of your child's health, how much of a problem have **you** had with...

| WORRY (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| I worry about whether or not my child's medical treatments are working | 0 | 1 | 2 | 3 | 4 |
| I worry about the side effects of my child's medications/medical treatments | 0 | 1 | 2 | 3 | 4 |
| I worry about how others will react to my child's condition | 0 | 1 | 2 | 3 | 4 |
| I worry about how my child's illness is affecting<br>other family members | 0 | 1 | 2 | 3 | 4 |
| I worry about my child's future | 0 | 1 | 2 | 3 | 4 |

## DIRECTIONS

Below is a list of things that might be a problem for your family. Please tell us how much of a problem each one has been for your family during the past ONE month.

In the past **ONE month**, as a result of your child's health, how much of a problem has **your family** had with...

| DAILY ACTIVITIES (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Family activities taking more time and effort | 0 | 1 | 2 | 3 | 4 |
| Difficulty finding time to finish household tasks | 0 | 1 | 2 | 3 | 4 |
| Feeling too tired to finish household tasks | 0 | 1 | 2 | 3 | 4 |

| FAMILY RELATIONSHIPS (problems with) | Never | Almost<br>Never | Some-<br>times | Often | Almost<br>Always |
|---|---|---|---|---|---|
| Lack of communication between family members | 0 | 1 | 2 | 3 | 4 |
| Conflicts between family members | 0 | 1 | 2 | 3 | 4 |
| Difficulty making decisions together as a family | 0 | 1 | 2 | 3 | 4 |
| Difficulty solving family problems together | 0 | 1 | 2 | 3 | 4 |
| Stress or tension between family members | 0 | 1 | 2 | 3 | 4 |

# 16.8 Patient Impression of Change (PIC)

The Patient Impression of Change (PIC) is designed to assess the subject's perception of his/her itching at the end of study drug treatment compared to his/her itching prior to the start of treatment with study drug. The PIC will be completed by subjects who were 9 years of age or older at the Week 18, 22 and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the CIC will be completed as outlined in the Schedule of Procedures in Section 16.1.

The questionnaire is designed for self-administration and uses a 7-point scale in which 1 designates the best outcome and 7 designate the worst outcome.

# **PIC**

| <br>y | <i>B B</i> , | , , , | <i>j</i> | · |
|---|---|---|---|---|
| Much better (1) | | | | |
| Better (2) | | | | |
| A little better (3) | | | | |
| No change (4) | | | | |
| A little worse (5) | | | | |
| Worse (6) | | | | |
| Much worse (7) | | | | |

How much has your itching changed, if at all, since you started this study?

# 16.9 Caregiver Impression of Change (CIC)

The Caregiver Impression of Change (CIC) is designed to assess the caregiver's perception of the subject's itch related symptoms and xanthoma severity at the end of study drug treatment compared to his/her itch related symptoms and xanthoma severity prior to the start of treatment with study drug. The CIC will be completed by all caregivers at the Week 18, 22 and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the CIC will be completed as outlined in the Schedule of Procedures in Section 16.1.

The questionnaire is designed for self-administration and uses a 7-point scale in which 1 designates the best outcome and 7 designates the worst outcome.

# **CIC**

How would you rate the change in your child's itch related symptoms since the start of the study?

| Much better (1) |
|---------------------|
| Better (2) |
| A little better (3) |
| No change (4) |
| A little worse (5) |
| Worse (6) |
| Much worse (7) |

Much worse (7)

**08 February 2019** 

| How | would you rate the change in your child's xanthoma severity since the start of the study? |
|---|---|
| П | Much better (1) |
| 同 | Better (2) |
| | A little better (3) |
| $\Box$ | No change (4) |
| 一 | A little worse (5) |
| | Worse (6) |

# 16.10 Caregiver Global Therapeutic Benefit (CGTB)

The Caregiver Global Therapeutic Benefit (CGTB) questionnaire is designed to assess the caregiver's perception of the treatment benefits on the subject's itching compared to the side effects experienced with study drug. The CGTB will be completed by all caregivers at the Week 18, 22 and 48 visits. For subjects who enter the 52-week and long-term optional follow-up treatment periods, the CIC will be completed as outlined in the Schedule of Procedures in Section 16.1.

The questionnaire is designed for self-administration and uses a 5-point scale in which 1 designates the best outcome and 5 designates the worst outcome.

# **CGTB**

Considering all aspects of your child's treatment, do you feel that the benefits of this treatment outweigh the side-effects?

| Definitely (1) |
|--------------------|
| Somewhat (2) |
| About the same (3) |
| Maybe not (4) |
| Definitely not (5) |

**08 February 2019** 

# 16.11 Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

Adverse events should be graded by severity based using CTCAE Version 4.0 [Published: May 28, 2009 (v4.03: June 14, 2010)].

# Common Terminology Criteria for Adverse Events (CTCAE)

# Version 4.0

Published: May 28, 2009 (v4.03: June 14, 2010)

### U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES

National Institutes of Health National Cancer Institute

# Common Terminology Criteria for Adverse Events v4.0 (CTCAE) Publish Date: May 28, 2009

### Quick Reference

The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term.

### Components and Organization

### SO

System Organ Class, the highest level of the MedDRA hierarchy, is identified by anatomical or physiological system, etiology, or purpose (e.g., SOC Investigations for laboratory test results), CTCAE terms are grouped by MedDRA Primary SOCs. Within each SOC, AEs are listed and accompanied by descriptions of severity (Grade).

#### CTCAFTermo

An Adverse Event (AE) is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medical treatment or procedure that may or may <u>not</u> be considered related to the medical treatment or procedure. An AE is a term that is a unique representation of a specific event used for medical documentation and scientific analyses. Each CTCAE v4.0 term is a MedDRA LLT (Lowest Level Term).

### Definitions

A brief definition is provided to clarify the meaning of each AE term.

### Grades

Grade refers to the severity of the AE. The CTCAE displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline:

- Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
- Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL\*.
- Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL\*\*.
- Grade 4 Life-threatening consequences; urgent intervention indicated.
- Grade 5 Death related to AE.

A Semi-colon indicates 'or' within the description of the grade.

A single dash (-) indicates a grade is not available.

Not all Grades are appropriate for all AEs. Therefore, some AEs are listed with fewer than five options for Grade selection.

### Grade 5

Grade 5 (Death) is not appropriate for some AEs and therefore is not an option.

### Activities of Daily Living (ADL)

\*Instrumental ADL refer to preparing meals, shopping for groceries or clothes, using the telephone, managing money, etc.

\*\*Self care ADL refer to bathing, dressing and undressing, feeding self, using the tollet, taking medications, and not bedridden.

<sup>\*</sup> CTCAE v4.0 incorporates certain elements of the MedDRA terminology. For further details on MedDRA refer to the MedDRA MSSO Web site (http://www.meddramsso.xom).

## CONTENTS

| SOC | Page |
|---------------------------------------------------------------------|------|
| Blood and lymphatic system disorders | - 3 |
| Cardiac disorders | -4 |
| Congenital, familial and genetic disorders | 7 |
| Ear and labyrinth disorders | 8 |
| Endocrine disorders | 19 |
| Eye disorders | 10 |
| Gastrointestinal disorders | 12 |
| General disorders and administration site conditions | 22 |
| Hepatobiliary disorders | 24 |
| Immune system disorders | 26 |
| Infections and infestations | 27 |
| Injury, poisoning and procedural complications | 34 |
| Investigations | 41 |
| Metabolism and nutrition disorders | 44 |
| Musculoskeletal and connective tissue disorders | 46 |
| Neoplasms benign, malignant and unspecified (incl cysts and polyps) | - 50 |
| Nervous system disorders | 51 |
| Pregnancy, puerperium and perinatal conditions | 56 |
| Psychiatric disorders | 57 |
| Renal and urinary disorders | 59 |
| Reproductive system and breast disorders | 61 |
| Respiratory, thoracic and mediastinal disorders | 65 |
| Skin and subcutaneous tissue disorders | 71 |
| Social circumstances | 75 |
| Surgical and medical procedures | 76 |
| Vascular disorders | 77 |

| | | lood and lymphatic syst | elli disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | á |
| Anemia | Hemoglobin (Hgb) <lln -="" 10.0<br="">g/dL; <lln -="" -<br="" 6.2="" <lln="" l;="" mmol="">100 g/L</lln></lln> | Hgb <10.0 - 8.0 g/dL; <6.2 - 4.9<br>mmol/L; <100 - 80g/L | Hgb <8.0 g/dL; <4.9 mmol/L;<br><80 g/L; transfusion indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by an reduction in the amount<br>h, palpitations of the heart, soft sys | | | ay include pallor of the skin and n | nucous |
| Bone marrow hypocellular | Mildly hypocellular or <=25%<br>reduction from normal cellularity<br>for age | cellularity for age | <=75% reduction cellularity from<br>normal for age | Aplastic persistent for longer than 2 weeks | Death |
| Definition: A disorder character | ized by the inability of the bone man | row to produce hematopoietic ele | ments. | 1 | |
| Disseminated intravascular<br>coagulation | - | Laboratory findings with no bleeding | Laboratory findings and bleeding | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by systemic pathological activa<br>is depleted of platelets and coagula | the second secon | which results in clot formation thre | oughout the body. There is an inc | rease in the |
| Febrila neutropenia | | | ANC <1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >38 degrees C (100.4 degrees F) for more than one hour. | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character<br>degrees F) for more than one h | ized by an ANC <1000/mm3 and a our. | single temperature of >38.3 degre | es C (101 degrees F) or a sustain | ed temperature of >=38 degrees ( | (100,4 |
| Hemolysis | Laboratory evidence of<br>hemolysis only (e.g., direct<br>antiglobulin test; DAT; Coombs';<br>schistocytes; decreased<br>haptoglobin) | Evidence of hemolysis and S=2 gm decrease in hemoglobin. | Transfusion or medical intervention indicated (e.g., steroids) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by laboratory test results that in | ndicate widespread erythrocyte ce | Il membrane destruction. | | |
| Hemolytic uremic syndrome | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| Definition: A disorder character | ized by a form of thrombotic microa | ngiopathy with renal failure, hemo | lytic anemia, and severe thromboo | ytopenia. | |
| Leukocytosis | | | >100,000/mm3 | Clinical manifestations of<br>leucostasis; urgent intervention<br>indicated | Death |
| Definition: A disorder character | ized by laboratory test results that in | ndicate an increased number of w | nite blood cells in the blood | | |
| Lymph node pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | |
| Definition: A disorder character | ized by a sensation of marked disco | omfort in a lymph node. | | | |
| Spleen disorder | incidental findings (e.g., Howell-<br>Jolly bodies); mild degree of<br>thrombocytosis and<br>leukocytosis | Prophylactic antibiotics indicated | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder of the spli | een, | | | | |
| Thrombotic thrombocytopenic<br>purpura | Evidence of RBC destruction<br>(schistocytosis) without clinical<br>consequences | | Laboratory findings with clinical consequences (e.g., renal insufficiency, petechiae) | Life-threatening consequences,<br>(e.g., CNS hemorrhage or<br>thrombosis/embolism or renal<br>failure) | Death |
| | ized by the presence of microangion<br>sual disturbances. It is an acute or s | | cytopenic purpura, fever, renal abr | normalities and neurological abno | malities su |
| Blood and lymphatic system<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| | T | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | ā |
| Acule coronary syndrome | | Symptomatic, progressive<br>angina; cardiac enzymes<br>normal; hemodynamically stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>stable | Symptomatic, unstable angina<br>and/or acute myocardial<br>infarction, cardiac enzymes<br>abnormal, hemodynamically<br>unstable | Death |
| | zed by signs and symptoms related<br>nunstable angina to myocardial inf | | fium secondary to coronary artery | disease. The clinical presentation | covers a |
| Aortic valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate regurgitation or stenosis by imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Dife-threatening consequences,<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteria | zed by a defect in aortic valve func | tion or structure. | | | |
| Asystole | Periods of asystole; non-urgent medical management indicated | * | | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a dysrhythmia without cardi | ac electrical activity. Typically, this | is accompanied by cessation of t | he pumping function of the heart. | |
| Atrial fibrillation | Asymptomatic, intervention not indicated | Non-urgent medical intervention<br>indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characterial<br>originates above the ventricles. | zed by a dysrhythmia without disce | mible P waves and an irregular ve | intricular response due to multiple | reentry circuits. The rhythm distu | rbance |
| Atrial flutter | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker), or ablation | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria<br>atria. | zed by a dysrhythmia with organize | ed rhythmic strial contractions with | a rate of 200-300 beats per minu | te. The rhythm disturbance origina | tes in the |
| Atrioventricular block complete | | Non-urgent intervention<br>indicated | Symptomatic and incompletely<br>controlled medically, or<br>controlled with device (e.g.,<br>pacemaker) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a dysrhythmia with complet | e failure of atrial electrical impulse | conduction through the AV node | to the ventricles | |
| Atrioventricular block first<br>degree | Asymptomatic, intervention not indicated | Non-urgent intervention<br>indicated | | | + |
| | zed by a dysrhythmia with a delay i<br>t interval greater than 200 milliseco | | tion of an electrical impulse through | gh the atrioventricular (AV) node b | eyond 0.2 |
| Cardiac arrest | - | 7 | - | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteris | zed by cessation of the pumping fu | nction of the heart. | | | |
| Chest pain - cardiac | Mild pain | Moderate pain; limiting instrumental ADL | Pain at rest, limiting self care<br>ADL | | 2 |
| Definition: A disorder characteris | zed by substernal discomfort due to | o insufficient myocardial oxygenati | on. | | |
| Conduction disorder | Mild symptoms; intervention not indicated | Moderate symptoms | Severe symptoms; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| The second secon | zed by pathological irregularities in | the cardiac conduction system. | | | |
| Constrictive pericarditis | | | Symptomatic heart failure or<br>other cardiac symptoms,<br>responsive to intervention | Refractory heart failure or other<br>poorly controlled cardiac<br>symptoms | Death |
| Definition: A disorder characteris | zed by a thickened and fibrotic peri | cardial sac: these fibrotic changes | | | e action. |
| Heart failure | Asymptomatic with laboratory<br>(e.g., BNP [B-Natriuretic<br>Peptide ]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or<br>with minimal activity or exertion;<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic | Death |

| | 1 | Cardiac disord | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Left ventricular systolic<br>dysfunction<br>Definition: A disorder characteri | zed by failure of the (eft ventricle to | produce adequate output despit | Symptomatic due to drop in<br>ajection fraction responsive to<br>intervention e an increase in distending pressur | Refractory or poorly controlled<br>heart failure due to drop in<br>ejection fraction; intervention<br>such as ventricular assist<br>device, intravenous vasopressor<br>support, or heart transplant<br>indicated<br>e and in end-diastolic volume. Clin | Death |
| | onea, orthopnea, and other signs ar | | The state of the s | | |
| Mitral valvė disėase | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate<br>regurgitation or stenosis by<br>imaging | Symptomatic: severe<br>regurgitation or stenosis by<br>imaging, symptoms controlled<br>with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder characteri | zed by a defect in mitral valve func | tion or structure. | | | |
| Mobitz (type) II atrioventricular<br>block | Asymptomatic, intervention not indicated | Symptomatic; medical<br>intervention indicated | Symptomatic and incompletely<br>controlled medically, or<br>controlled with device (e.g.,<br>pacemaker) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by a dysrhythmia with relatively<br>atrioventricular (AV) node to the ve | | block of an atrial impulse. This is t | he result of intermittent failure of a | trial electri |
| Mobitz type I | Asymptomatic, intervention not indicated | Symptomatic; medical intervention indicated | Symptomatic and incompletely controlled medically, or controlled with device (e.g., pacemaker) | Life-threatening consequences; urgent intervention indicated | Death |
| | zed by a dysthythmia with a progre<br>ion through the atrioventricular (AV | | rior to the blocking of an atrial impu | ulse. This is the result of intermitter | nt failure o |
| Myocardial infarction | | Asymptomatic and cardiac<br>enzymes minimally abnormal<br>and no evidence of ischemic<br>ECG changes | Severe symptoms; cardiac<br>enzymes abnormal;<br>hemodynamically stable; ECG<br>changes consistent with<br>infarction | Life-threatening consequences;<br>hemodynamically unstable | Death |
| Definition: A disorder characteri | zed by gross necrosis of the myors | ardium; this is due to an interrupti | on of blood supply to the area. | | |
| Myocarditis | Asymptomatic with laboratory<br>(e.g., BNP B-Natriuretic<br>Peptide ) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe with symptoms at rest or with minimal activity or exertion; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., continuous IV therapy or<br>mechanical hemodynamic<br>support) | Death |
| Definition: A disorder characteri | zed by inflammation of the muscle | tissue of the heart. | - | - | _ |
| Palpitations | Mild symptoms; intervention not indicated | | | | |
| | zed by an unpleasant sensation of | Tari Victor Tari | T | | |
| Paroxysmal atrial tachycardia | Asymptomatic, intervention not indicated | Symptomatic; medical<br>management indicated | IV medication indicated | Life-threatening consequences;<br>incompletely controlled<br>medically; cardioversion<br>indicated | Death |
| Definition: A disorder characterioriginates in the atria. | zed by a dysrhythmia with abrupt o | nset and sudden termination of a | trial contractions with a rate of 150 | -260 beats per minute: The rhythm | disturban |
| Pericardial effusion | P | Asymptomatic effusion size small to moderate | Effusion with physiologic consequences | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by fluid collection within the pe | ricardial sac, usually due to inflan | nmation. | | |
| Pericardial tamponade | 1 | | 1 | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an increase in intrapericard | al pressure due to the collection | of blood or fluid in the pericardium | | |
| Pericarditis | Asymptomatic, EOG or physical findings (e.g., rub) consistent with pericarditis | Symptomatic pericarditis (e.g., chest pain) | Pericarditis with physiologic consequences (e.g., pericardial constriction) | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | · · | Cardiac disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 1 | 4 | 5 |
| Pulmonary valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis by imaging | Asymptomatic; moderate<br>regurgitation or stenosis by<br>imaging | Symptomatic; severe<br>regurgitation or stenosis by<br>imaging; symptoms controlled<br>with medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| | ized by a defect in pulmonary valve | function or structure | | - | |
| Restrictive cardiomyopathy | | | Symptomatic heart failure or other cardiac symptoms, responsive to intervention | Refractory heart failure or other<br>poorly controlled cardiac<br>symptoms | Death |
| | ized by an inability of the ventricles | to fill with blood because the myo | | | 1 |
| Right ventricular dysfunction | Asymptomatic with laboratory<br>(e.g., BNP [8-Natriuretic<br>Peptide]) or cardiac imaging<br>abnormalities | Symptoms with mild to moderate activity or exertion | Severe symptoms, associated<br>with hypoxemia, right heart<br>failure; oxygen indicated | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., ventricular assist device);<br>heart transplant indicated | Death |
| Definition: A disorder character | ized by impairment of right ventricul | ar function associated with low eje | ection fraction and a decrease in I | motility of the right ventricular wall. | |
| Sick sinus syndrome | Asymptomatic, intervention not<br>indicated | Non-urgent intervention<br>indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with alternati | ng periods of bradycardia and atri | al tachycardia accompanied by sy | ncope, fatigue and dizziness. | ß. |
| Sinus bradycardia | Asymptomatic, intervention not<br>indicated | Symptomatic, medical<br>intervention indicated | Severe, medically significant,<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart i | ate less than 60 beats per minute | that originates in the sinus node. | | ř |
| Sinus tachycardia | Asymptomatic, intervention not<br>indicated | Symptomatic; non-urgent<br>medical intervention indicated | Urgent medical intervention indicated | | |
| Definition: A disorder character | ized by a dysrhythmia with a heart i | ale greater than 100 beats per mi | nute that originates in the sinus ri | ode, | |
| Supraventricular tachycardia | Asymptomatic, intervention not<br>indicated | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart i | ale greater than 100 beats per mi | nute that originates above the ver | ntricles. | _ |
| Tricuspid valve disease | Asymptomatic valvular<br>thickening with or without mild<br>valvular regurgitation or<br>stenosis | Asymptomatic; moderate<br>regurgitation or stenosis by<br>imaging | Symptomatic; severe<br>regurgitation or stenosis;<br>symptoms controlled with<br>medical intervention | Life-threatening consequences;<br>urgent intervention indicated<br>(e.g., valve replacement,<br>valvuloplasty) | Death |
| Definition: A disorder character | ized by a defect in tricuspid valve fu | nction or structure. | | | |
| Ventricular arrhythmia | Asymptomatic, intervention not<br>indicated | Non-urgent medical intervention<br>indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia that originate | s in the ventricles. | , | | |
| Ventricular fibrillation | | | | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder character<br>ventricles | ized by a dysrhythmia without disce | mible ORS complexes due to rapi | d repetitive excitation of myocard | lial fibers without coordinated contr | action of th |
| Ventricular tachycardia | | Non-urgent medical intervention indicated | Medical intervention indicated | Life-threatening consequences;<br>hemodynamic compromise;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a dysrhythmia with a heart r | ate greater than 100 beats per mi | nute that originates distal to the b | undle of His. | |
| Wolff-Parkinson-White<br>syndrome | Asymptomatic, intervention not indicated | Non-urgent medical intervention<br>indicated | Symptomatic and incompletely<br>controlled medically or<br>controlled with procedure | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by the presence of an accesso | ry conductive pathway between th | | uses premature ventricular activation | n: |
| Cardiac disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences; urgent intervention indicated | Death |

| | Co | ngenital, familial and ge | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event Congenital, familial and genetic disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling: limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | fi<br>Death |

| | | Ear and labyrinth dis | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | -1 | 2 | 3 | 4 | 5 |
| Ear pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | L |
| Definition: A disorder character | rized by a sensation of marked disco | mfort in the ear. | | | |
| External ear inflammation | External obtis with erythema or<br>dry desquamation | External otitis with moist<br>desquamation, edema,<br>enhanced cerumen or<br>discharge; tympanic membrane<br>perforation; tympanostomy | External otitis with mastoiditis;<br>stenosis or osteomyelitis;<br>necrosis of soft tissue or bone | Urgent operative intervention indicated | Death |
| Definition: A disorder character | rized by inflammation, swelling and r | edness to the outer ear and ear c | anal. | | - |
| External ear pain | Mild pain | Moderate pain: limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | P |
| Definition: A disorder characte | rized by a sensation of marked disco | mfort in the external ear region. | | | |
| Hearing impaired | Adults enrolled on a Monitoring Program (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift of 15 - 25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: subjective change in itearing in the absence of documented hearing loss. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 8 kHz in at least one sar. | Adults enrolled in Monitoring Program (on a 1, 2, 3, 4, 6 and 6 kHz audiogram): Threshold shift of >25 dB averaged at 2 contiguous test frequencies in at least one ear. Adults not enrolled in Monitoring Program: hearing loss but hearing aid or intervention not indicated; limiting instrumental ADL. Pediatric (on a 1, 2, 3, 4, 6 and 8 kHz audiogram): Threshold shift >20 dB at 4 kHz and above in at least one ear. | Adults enrolled in Monitoring<br>Program (on a 1, 2, 3, 4, 6 and<br>8 kHz audiogram): Threshold<br>shift of >25 dB averaged at 3<br>contiguous test frequencies in at<br>least one ear; therapeutic<br>intervention indicated. Adults not enrolled in Monitoring<br>Program: hearing loss with<br>hearing aid or intervention<br>indicated; limiting self care ADL. Pediatric (on a 1, 2, 3, 4, 8 and<br>8 kHz audiogram): hearing loss<br>sufficient to indicate therapeutic<br>intervention, including hearing<br>aids; threshold shift >20 dB at 3<br>kHz and above in at least one<br>ear; additional speech-language<br>related services indicated. | Pediatric: Audiologic Indication<br>for cochlear implant and | |
| Definition: A disorder characte<br>Middle ear inflammation | Serous otitis | e ability to detect or understand s<br>Serous otitis, medical<br>intervention indicated | ounds resulting from damage to e<br>Mastoiditis; necrosis of canal<br>soft tissue or bone | ar structures. Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | rized by inflammation (physiologic re | sponse to irritation), swelling and | redness to the middle ear. | | |
| Tinnitus | Mild symptoms; Intervention not<br>indicated | instrumental ADL | Severe symptoms; limiting self care ADL | * | €. |
| | ized by noise in the ears, such as ri | | an and an | 7 | |
| Vertigo Definition: A disorder character | Mild symptoms. | Moderate symptoms; limiting<br>instrumental ADL<br>I world were revolving around the | Severe symptoms; limiting self<br>care ADL<br>patient (objective vertigo) or as if | he himself were revolving in space | e (subjecti |
| vertigo). | | | | | |
| Vestibular disorder | | Symptomatic; limiting instrumental ADL | Severe symptoms: limiting self care ADL | • | |
| Definition: A disorder character | ized by dizziness, imbalance, nause | | | | |
| Ear and tabyrinth disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADI. | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | W. | Endocrine disord | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | |
| Adrenal insufficiency | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Severe symptoms;<br>hospitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rs when the adrenal cortex does no<br>ison's disease or primary adrenal in | | cortisol and in some cases, the ho | ormone aldosterone. It may be due | to a disor |
| Cushingaid | Mild symptoms, intervention not<br>indicated | Moderate symptoms; medical intervention indicated | Severe symptoms, medical<br>intervention or hospitalization<br>indicated | | e) |
| Definition: A disorder character<br>osteoporosis, usually due to ex | rized by signs and symptoms that re<br>rogenous corticosteroids. | semble Cushing's disease or syn | drome: buffalo hump obesity, striat | tions, adiposity, hypertension, diab | etes, and |
| Delayed puberfy | | No breast development by age<br>13 yrs for females; testes<br>volume of <3 cc or no Tanner<br>Stage 2 development by age<br>14.5 yrs for males | No breast development by age<br>14 yrs for females; no increase<br>in testes volume or no Tanner<br>Stage 2 by age 16 yrs for<br>males; hormone replacement<br>indicated | | F |
| Growth accelerated | rized by unusually late sexual matur | >= +2 SD (standard deviation)<br>above mid parental height or<br>target height | - | 5 | + |
| Definition: A disorder characte | ized by greater growth than expects | | | | 1 |
| Hyperparathyroidism | Mild symptoms; intervention not<br>indicated<br>rized by an increase in production of | Moderate symptoms, medical intervention indicated | thyroid glands. This results in hyp | ercalcemia (abnormally high levels | of calciur |
| the blood). | | V-10-12-12-13-13-13-13-13-13-13-13-13-13-13-13-13- | | | |
| Hyperthyroidism | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; thyroid<br>suppression therapy indicated;<br>limiting instrumental ADL | Severe symptoms; limiting self care ADL; hospitalization indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by excessive levels of thyroid t | normone in the body. Common ca | uses include an overactive thyroid | gland or thyroid hormone overdos | se. |
| Hypoparathyroidism | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; medical intervention indicated | Severe symptoms, medical<br>intervention or hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by a decrease in production of | parathyroid hormone by the parat | thyroid glands. | | |
| Hypothyroidism | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; thyroid<br>replacement indicated; limiting<br>instrumental ADL | Severe symptoms: limiting self-<br>care ADL, hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by a decrease in production of | thyroid harmone by the thyroid gl | and. | I - | |
| Precocious puberty | Physical signs of puberty with<br>no biochemical markers for<br>females <8 years and males <9<br>years | Physical signs and biochemical<br>markers of puberty for females<br><8 years and males <9 years | | | |
| Definition: A disorder character<br>9 for boys. | rized by unusually early developmen | nt of secondary sexual features; th | ne onset of sexual maturation begin | ns usually before age 8 for girls an | d before a |
| Virilization | Mild symptoms; intervention not<br>indicated | Moderate symptoms; medical intervention indicated | | ( ) | 200 |
| Definition: A disorder character | rized by inappropriate masculinization | on occurring in a female or prepub | ertal male. | | |
| Endocrine disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | W. Control | Eye di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Blurred vision | Intervention not indicated | Symptomatic: limiting instrumental ADL | Limiting self care ADL | | - |
| Definition: A disorder charac | terized by visual perception of u | nclear or luzzy images. | | | Ť. |
| Cataract | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, moderate decrease in visual acuity (20/40 or better) | Symptomatic with marked decrease in visual acuity (worse than 20/40 but better than 20/200); operative intervention indicated (e.g., cataract surgery) | Blindness (20/200 or worse) in the affected eye | |
| Definition: A disorder characteristics. | terized by partial or complete op | acity of the crystalline lens of | one or both eyes. This results in | n a decrease in visual acuity an | nd eventual blindness if |
| Conjunctivitis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; topical intervention indicated (e.g., antibiotics); limiting instrumental ADL | Limiting self care ADL | | |
| Definition: A disorder charac | terized by inflammation, swelling | and redness to the conjunctiv | a of the eye. | | |
| Comeat ulcer | | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Limiting self care ADL;<br>declining vision (worse than<br>20/40 but better than 20/200) | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | - |
| Definition: A disorder charac | terized by an area of epithelial ti | ssue loss on the surface of the | cornea. It is associated with in | flammatory cells in the comea | and anterior chamber. |
| Dry eye | Asymptomatic; clinical or<br>diagnostic observations only;<br>mild symptoms relieved by<br>lubricants | Symptomatic; multiple<br>agents indicated; limiting<br>instrumental ADL | Decrease in visual acuity<br>(<20/40); limiting self care<br>ADL | | * |
| Definition: A disorder charac | terized by dryness of the cornea | and conjunctiva. | | | 1 |
| Extraocular muscle paresis | Asymptomatic; clinical or<br>diagnostic observations only | Symptomatic: limiting instrumental ADL | Limiting self care ADL;<br>disabling | - | * |
| Definition: A disorder charac | terized by incomplete paralysis | of an extraocular muscle. | | | T |
| Eye pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care ADL | 7 | • |
| Eyelld function disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, nonoperative intervention indicated; limiting instrumental ADL | Limiting self care ADL;<br>operative intervention<br>indicated | | |
| A Life Box 10 Co. | terized by impaired eyelid functi | | Charling and same ADC | 1,00 | - |
| Flashing lights | Symptomatic but not limiting ADL | | Limiting self care ADL | | • |
| | terized by a sudden or brief burs | | Climitian Authoriti Action Action | | |
| Floaters | Symptomatic but not limiting ADL | | Limiting self care ADL | | |
| | terized by an individual seeing s | I STATE OF THE STA | TYTY E E CO | THE RESERVE THE PROPERTY OF THE PERSON NAMED IN COLUMN TWO IN COLUMN TO THE PERSON NAMED IN COLU | or or lens. |
| Glaucoma | Elevated intraocular<br>pressure (EIOP) with single<br>topical agent for intervention;<br>no visual field deficit | limiting instrumental ADL | EIOP causing marked visual<br>field deficits (e.g., involving<br>both superior and inferior<br>visual fields); operative<br>intervention indicated;<br>limiting self care ADL | Blindness (20/200 or worse)<br>in the affected eye | |
| Definition: A disorder charac | terized by an increase in pressu | re in the eyeball due to obstru | ction of the aqueous humor out | flaw. | |
| Keratitis | | Symptomatic; medical intervention indicated (e.g., topical agents); limiting instrumental ADL | Decline in vision (worse than<br>20/40 but better than<br>20/200); limiting self care<br>ADL | Perforation or blindness<br>(20/200 or worse) in the<br>affected eye | |
| | terized by inflammation to the co | | Wagning and a second | A. D. C. | 1 |
| Night blindness | Symptomatic but not limiting<br>ADL | Limiting instrumental ADL | Limiting self care ADL | Blindness (20/200 or worse) in the affected eye | - |

| | Eye disorders | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Optic nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only | Limiting vision of the affected<br>eye (20/40 or better) | Limiting vision in the affected<br>eye (worse than 20/40 but<br>better than 20/200) | Blindness (20/200 or worse) in the affected eye | • |
| Definition: A disorder chara | acterized by involvement of the op | tic nerve (second cranial nerve | 0). | | |
| Papilledema | Asymptomatic; no visual field defects | vision; visual field defect<br>present sparing the central<br>20 degrees | Marked visual field defect<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse) in the affected eye | |
| Photophobia | Symptomatic but not limiting ADL | Limiting instrumental ADL | Limiting self care ADL | - | š |
| Definition: A disorder chara | acterized by fear and avoidance o | Flight. | , | | |
| Relinal detachment | Asymptomatic | Exudative and visual acuity<br>20/40 or better | Rhegmatogenous or<br>exudative detachment:<br>operative intervention<br>indicated; decline in vision<br>(worse than 20/40 but better<br>than 20/200) | Blindness (20/200 or worse)<br>in the affected eye | ٠ |
| Definition: A disorder chara | acterized by the separation of the | inner retina layers from the uni | derlying pigment epithelium. | | |
| Retinal tear | | Laser therapy or<br>pneumopexy indicated | Vitroretinal surgical repair indicated | Blindness (20/200 or worse) in the affected eye | - |
| Definition: A disorder chara | acterized by a small laceration of t | he retina, this occurs when the | vitreous separates from the re | tina. Symptoms include flashes | and floaters |
| Retinal vascular disorder | | Topical medication indicated | intravitreal medication;<br>operative intervention<br>indicated | | 1 |
| Definition: A disorder chara | acterized by pathological retinal bl | ood vessels that adversely affe | ects vision. | | |
| Retinopathy | Asymptomatic; clinical or diagnostic observations only | Symptomatic with moderate decrease in visual acuity (20/40 or better); limiting instrumental ADL | Symptomatic with marked<br>decrease in visual acuity<br>(worse than 20/40);<br>disabling; limiting self care<br>ADL | Blindness (20/200 or worse) in the affected eye | |
| Definition: A disorder invol- | ving the retins | | 7,000 | | |
| Scleral disorder | Asymptomatic; clinical or diagnostic observations only | Symptomatic, limiting instrumental ADL; moderate decrease in visual acuity (20/40 or better). | Symptomatic, limiting self care ADL; marked decrease in visual acuity (worse than 20/40) | Blindness (20/200 or worse)<br>in the affected eye | ā |
| Definition: A disorder chara | acterized by involvement of the sc | lera of the eye | | | |
| Úveitis | Asymptomatic; clinical or<br>diagnostic observations only | Anterior uveitis; medical intervention indicated | Posterior or pan-uveitis | Blindness (20/200 or worse) in the affected eye | 1 |
| Definition: A disorder chara | acterized by inflammation to the u | vea of the eye. | | | |
| Vitreous hemorrhage | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only | Symptomatic; limiting<br>instrumental ADL | Limiting self care ADL;<br>vitrectomy indicated | Blindness (20/200 or worse)<br>in the affected eye | - |
| Definition: A disorder chara | acterized by blood extravasation in | nto the vitreous humor | | | |
| Watering eyes | Intervention not indicated | Intervention indicated | Operative intervention indicated | | 7 |
| Definition: A disorder of ex | cessive tearing in the eyes; it can | be caused by overproduction | of tears or impaired drainage of | the tear duct. | |
| Eye disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate: minimal, local or<br>noninvasive intervention<br>indicated, limiting age-<br>appropriate instrumental<br>ADL | Severe or medically<br>significant but not<br>immediately sight-<br>threatening; hospitalization<br>or protongation of existing<br>hospitalization indicated;<br>disabling; limiting self care<br>ADL | Sight-threatening<br>consequences, urgent<br>intervention indicated;<br>blindness (20/200 or worse)<br>in the affected eye | • |

| | - 10 | Gastrointestinal di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abdominal distension | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting<br>instrumental ADL | Severe discomfort; limiting self<br>care ADL | | Y |
| Definition: A disorder charac | terized by swelling of the abdomen. | Tr. | To the second se | 1 | |
| Abdominal pain Definition: A disorder charac | Mild pain terized by a sensation of marked disc | Moderate pain; limiting instrumental ADL omfort in the abdominal region. | Severe pain; limiting self care<br>ADL | | 3 |
| Anal fistule | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an abnormal communication | n between the opening in the ana | I canal to the perianal skin. | | |
| Anal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated. | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the anal regi | on. | | | |
| Anal mucositis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by inflammation of the mucous | s membrane of the anus. | 1 | | |
| Anal necrosis | | | TPN or hospitalization indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | terized by a necrotic process occurrin | | Boundary Building St. | - | |
| Anal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | - |
| Definition: A disorder charac | terized by a sensation of marked disc | omfort in the anal region. | | | E |
| Anal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; non-<br>emergent operative intervention<br>indicated: TPN or hospitalization<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen o | f the anal canal | | | |
| Anal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a circumscribed, inflammat | ory and necrotic erosive lesion on | the mucosal surface of the anal ca | mal. | |
| Asoites | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, medical<br>intervention indicated | Severe symptoms; invasive<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by accumulation of serous or I | nemorrhagic fluid in the peritonea | cavity. | | |
| Bloating | No change in bowel function or<br>oral intake | Symptomatic, decreased oral<br>intake; change in bowel function | | ÷ | + |
| Definition: A disorder charac | terized by subject-reported feeling of | uncomfortable fullness of the abd | onien: | | |
| Cecal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>andoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the cecum. | | | | |
| Cheilitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms, limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL; intervention indicated | • | € |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Colitis | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated<br>erized by inflaromation of the colon. | Abdominal pain; mucus or blood<br>in stool | Severe abdominal pain; change<br>in bowel habits; medical<br>intervention indicated;<br>peritoneal signs | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Colonic fistula | Asymptomatic; clinical or | Symptomatic; altered Gi | Severely altered GI function: | Life threatening contraction can | Death |
| Colonic risula | diagnostic observations only;<br>intervention not indicated | function | bowel rest, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the large intestine and a | enother organ or anatomic site. | | |
| Colonic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the colon. | | | | |
| Colonic obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Hospitalization indicated;<br>elective operative intervention<br>indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by blockage of the normal flow | of the intestinal contents in the co | lon, | | |
| Colonic perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by a rupture in the colonic wall | | p- | | |
| Colonic stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function:<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a narrowing of the lumen of | the colon | | | , |
| Colonic ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic: altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a circumscribed, inflammate | ory and necrotic erosive lesion on t | he mucosal surface of the colon. | | ^ |
| Constipation | Occasional or intermittent<br>symptoms; occasional use of<br>stool softeners, laxatives,<br>dietary modification, or enema | Persistent symptoms with<br>regular use of laxatives or<br>enemas; limiting instrumental<br>ADL | Obstipation with manual<br>evacuation indicated; limiting<br>selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by irregular and infrequent or o | difficult evacuation of the bowels. | | | |
| Dental caries | One or more dental caries, not involving the root | Dental caries involving the root | Dental caries resulting in pulpitis<br>or periapical abscess or<br>resulting in tooth loss | | - |
| Definition: A disorder charact | erized by the decay of a tooth, in which | ch it becomes softened, discolored | and/or porous. | | , |
| Diarrhea | increase of <4 stools per day<br>over baseline; mild increase in<br>ostomy output compared to<br>baseline | Increase of 4 - 6 stools per day<br>over baseline; moderate<br>increase in ostorny output<br>compared to baseline | Increase of >= 7 stools per day<br>over baseline; incontinence;<br>hospitalization indicated; severe<br>increase in ostomy output<br>compared to baseline; limiting<br>self care ADL | Life-threatening consequences; urgent intervention indicated | Death |
| Definition, A disorder charact | erized by frequent and watery bowel | movements, | | | |
| Dry mouth | Symptomatic (e.g., dry or thick saliva) without significant dielary alteration; unstimulated saliva flow >0.2 ml/min | Moderate symptoms; oral intake, alterations (e.g., copious water, other lubricants, diet limited to purees and/or soft, moist foods); unstimulated saliva 0.1 to 0.2 ml/min | Inability to adequately aliment<br>orally, tube feeding or TPN<br>indicated; unstimulated saliva<br><0.1 ml/min | * | 5 |

| Gastrointestinal disorders | | | | | |
|---|---|---|---|---|---|
| | | T | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Duodenal fistule | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: altered GI function | Severely altered GI function;<br>tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the duodenum and and | other organ or anatomic site. | 1 | |
| Duodenal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the duadenur | n. | | | |
| Duodenal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Hospitalization or elective<br>operative intervention indicated;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| And the second s | erized by blockage of the normal flow | | The state of the s | | |
| Duodenal perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Duodenal steriosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a narrowing of the lumen of | the duodenum | All the second | | |
| Duodenal ülcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Severely altered GI function:<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabiling | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a circumscribed, inflammate | ory and necrotic erosive lesion on | A CONTRACTOR OF THE PARTY OF TH | nal wall. | |
| Dyspepsia | Mild symptoms, intervention not indicated | | Severe symptoms; surgical intervention indicated | 8 | + |
| | erized by an uncomfortable, often pai | nful feeling in the stomach, resulti | ng from impaired digestion. Sympl | loms include burning stomach, blo | ating, |
| heartburn, nauses and vomit | 113 | English of the same | Samuel Action | Ive a second | latinu. |
| Dysphagia | Symptomatic, able to eat<br>regular diet | Symptomatic and altered<br>eating/swallowing | Severely altered<br>eating/swallowing; tube feeding<br>or TPN or hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by difficulty in swallowing. | | | | |
| Enterocolitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Abdominal pain; mucus or blood<br>in stool | Severe or persistent abdominal<br>pain; fever; lieus; peritoneal<br>signs | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by inflammation of the small ar | nd large intestines. | | | |
| Enterovesical fistula | Asymptometic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; noninvasive intervention indicated | Severe, medically significant;<br>medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the unnary bladder and | the intestine. | | |
| Esophageal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, altered GI function | Severely altered GI function;<br>tube feeding. TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the esophagus and an | other organ or anatomic site. | | |
| Esophageal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | | Gastrointestinal di | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Esophageal necrosis | | | Inability to aliment adequately<br>by GI tract; radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact<br>Esophageal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | g in the esophageal wall. Symptomatic; altered Gifunction; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL; | Life-threatening consequences; urgent intervention indicated | Death |
| | | and the second second second second | disabling | | |
| Definition: A disorder charac | terized by blockage of the normal flow | of the contents in the esophagus | | | |
| Esophageal pain | Mild pain | Moderate pain; limiting<br>Instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | - |
| Definition: A disorder charac | terized by a sensation of marked disc | omfort in the esophageal region. | | | |
| Esophageal perforation | | Symptomatic, medical<br>intervention indicated | Severe symptoms, elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a rupture in the wall of the | esophagus. | 1- | | 6 |
| Esophageal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a narrowing of the lumen of | fthe esophagus, | 1 | | |
| Esophageal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function: limiting instrumental<br>ADL | Severely attered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by a circumscribed, inflammat | ory and necrotic erosive lesion on | Control of the Contro | ageal wall. | |
| Esophageal varices<br>hemorrhage | | Self-limited; intervention not indicated | Transfusion, radiologic, endoscopic, or elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from esophageal v | varices. | (-63-41-41-41-41-41-41-41-41-41-41-41-41-41- | | |
| Esophagitis | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Symptomatic; altered<br>eating/swallowing; oral<br>supplements indicated | Severely altered<br>eating/swallowing; tube feeding,<br>TPN or hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by inflammation of the esopha | geal wall. | | | |
| Fecal incontinence | Occasional use of pads required | | Severe symptoms, elective<br>operative intervention indicated | | |
| Definition: A disorder charac | terized by inability to control the escap | pe of stool from the rectum. | | | |
| Flatulence | Mild symptoms; intervention not<br>indicated | psychosocial sequelae | | | S |
| | terized by a state of excessive gas in | | 1 | | |
| Gastric fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely attered GI function;<br>bowel rest, tube feeding, TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charac | terized by an abnormal communication | n between the stomach and anoth | her organ or anatomic site. | | |
| Gastric hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by bleeding from the gastric w | The state of the s | A PACIFIC COMPANY OF THE PACIFIC COMPANY | | |
| Gastric necrosis | ÷. | * | Inability to aliment adequately<br>by GI tract, radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Gastric perforation | | Symptomatic: medical<br>intervention indicated | Severe symptoms, elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a rupture in the stomach wa | (I) | | | |
| Gastric stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding; hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | erized by a narrowing of the lumen of | the stomach. | 7 7 7 77 1 | | |
| Gastric ulcer | Asymptomatic; clinical or diagnostic observations only, intervention not indicated | Symptomatic; altered Gl<br>function; medical intervention<br>indicated; limiting instrumental<br>ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>self care ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a circumscribed, inflammato | ory and necrolic erosive lesion on | the mucosal surface of the stomac | th. | |
| Gastritis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, altered GI function, medical intervention indicated | Severely altered eating or<br>gastric function; TPN or<br>hospitalization indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | erized by inflammation of the stomach | ACRES AND THE RESERVE OF THE PARTY OF THE PA | Fr. Avenues a S.C. | | |
| Gastroesophageal reflux<br>disease | Mild symptoms; intervention not<br>indicated | Moderate symptoms, medical<br>intervention indicated | Severe symptoms, surgical<br>intervention indicated | | |
| | erized by reflux of the gastric and/or d<br>by result in injury to the esophageal m | the state of the s | | nd usually caused by incompetent | e of the l |
| Gastrointestinal fistule | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function:<br>tube feeding, TPN or<br>hospitalization indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between any part of the gastroin | testinal system and another organ | or anatomic site: | , |
| Gastrointestinal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| Definition: A disorder character | erized by a sensation of marked disco | omfort in the gastrointestinal region | n. | | |
| Gastroparesis | Mild nausea, early satiety and<br>bloating, able to maintain caloric<br>intake on regular diet | Moderate symptoms; able to<br>maintain nutrition with dietary<br>and lifestyle modifications; may<br>need pharmacologic<br>intervention | Weight loss; refractory to<br>medical intervention; unable to<br>maintain nutrition orally | | E |
| Definition: A disorder characte | erized by an incomplete paralysis of t | he muscles of the stomach wall re | sulting in delayed emptying of the | gastric contents into the small inte | estine. |
| Gingival pain | Mild pain | Moderate pain interfering with<br>oral intake | Severe pain; inability to aliment<br>orally | | 4 |
| | erized by a sensation of marked disco | | Tour Parley in Calcul | Continue to the continue to | 6 4 |
| Hemorrhoidal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>lurgent intervention indicated | Death |
| Definition: A disorder character | erized by bleeding from the hemorrho | ids, | | | |
| Hemorrhoids | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; banding or medical intervention indicated | Severe symptoms, radiologic,<br>endoscopic or elective operative<br>intervention indicated | | 1 |
| Definition: A disorder characte | erized by the presence of dilated vein | s in the rectum and surrounding a | rea. | | |
| lleaí fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely aftered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the ileum and another | organ or anatomic site. | | |
| lisal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor | Transfusion, radiologic, endoscopic, or elective | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | Y | Gastrointestinal di | sorders | | |
|---|---|---|---|---|---|
| | 1 | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Real obstruction | Asymptomatic, clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of the intestinal contents in the il | eum. | | |
| lieal perforation | | Symptomatic; medical intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | ized by a rupture in the iteal wall. | V | 1 | 122 N 12 | |
| leal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | ized by a narrowing of the lumen o | | 1 | | |
| lleal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a circumscribed, inflammat | ory and necrotic erosive lesion on | the mucosal surface of the ileum. | Y | |
| lléus | | Symptomatic; altered GI function; bowel rest indicated | Severely altered GI function;<br>TPN indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by failure of the ileum to transp | port intestinal contents. | 12 | | |
| Intra-abdominal hemorrhage | | Medical intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding in the abdominal o | savity. | | | |
| Jejunal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: altered GI function | Severely altered GI function:<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an abnormal communication | n between the jejunum and anoth | er organ or anatomic site. | | |
| Jejunal hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the jejunal w | ell. | | | |
| Jejunal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI<br>function; limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of the intestinal contents in the j | ojunum. | | |
| Jejunal perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a rupture in the jejunal wall | | | | |
| Jejunal stenosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a narrowing of the lumen o | f the jejunum. | | | |
| Jejunal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function | Severely altered GI function:<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a circumscribed, inflammat | ory and necrotic erosive lesion on | the mucosal surface of the jejunun | 0. | |
| Lip pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | ÷ | € |

| | 1 | Gastrointestinal dis | e-co-co-co-co-co-co-co-co-co-co-co-co-co- | | |
|---|---|---|---|---|---|
| | | | Grade | , | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Lower gastrointestinal<br>hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | erized by bleeding from the lower gas | strointestinal tract (small intestine, | large intestine, and anus). | | |
| Malabsorption | * | Altered diet; oral intervention<br>indicated | Inability to aliment adequately;<br>TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by inadequate absorption of no | utrients in the small intestine. Sym | ptoms include abdominal marked | discomfort, bloating and diarrhea. | |
| Mucositis oral | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Moderate pain; not interfering<br>with oral intake; modified diet<br>indicated | Severe pain; interfering with oral intake | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | erized by inflammation of the oral mu | cosal. | IT. | 1 | |
| Nausea | Loss of appetite without<br>alteration in eating habits | Oral intake decreased without<br>significant weight loss,<br>dehydration or malnutrition | Inadequate oral caloric or fluid<br>intake; tube feeding, TPN, or<br>hospitalization indicated | | |
| Definition: A disorder character | erized by a queasy sensation and/or | the urge to vomit. | P | | |
| Obstruction gastric | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | erized by blockage of the normal flow | of the contents in the stomach. | | | |
| Oral cavity fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | erized by an abnormal communicatio | n between the oral cavity and and | ther organ or anatomic site | | |
| Oral dysesthesia | Mild discomfort; not interfering with oral intake | Moderate pain; interfering with<br>oral intake | Disabling pain; tube feeding or<br>TPN indicated | * | + |
| Definition: A disorder character | erized by a burning or tingling sensat | ion on the lips, tangue or entire m | outh. | | |
| Oral hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | erized by bleeding from the mouth. | | | | |
| Oral pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 2. | 2 |
| Definition: A disorder character | erized by a sensation of marked disc | omfort in the mouth, tongue or lip: | | | |
| Pancreatic duct stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Ufe-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | erized by a narrowing of the lumen of | f the pancreatic duct. | | | |
| Pancreatic fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: attered GI function | Severely altered GI function:<br>tube feeding or TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | erized by an abnormal communication | n between the pancreas and anot | her organ or anatomic site. | | |
| Pancreatic hemorrhage | Mild; intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | erized by bleeding from the pancreas | i, | | | |
| Pancreatic necrosis | | 4- | Tube feeding or TPN indicated<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | erized by a necrotic process occurring | g in the pancreas. | | | |
| Pancreatitis | | Enzyme elevation or radiologic findings only | Severe pain; vomiting; medical intervention indicated (e.g., | Life-threatening consequences; urgent intervention indicated | Death |

| | 1 | Gastrointestinal dis | e-colesce. | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | erized by inflammation of the pancrea | s. | | | |
| Periodonial diseas€ | Gingival recession or gingivitis,<br>limited bleeding on probing; mild<br>local bone loss | Moderate gingival recession or<br>gingivitis; multiple sites of<br>bleeding on probing; moderate<br>bone loss | Spontaneous bleeding; severe<br>bone loss with or without tooth<br>loss; osteonecrosis of maxilla or<br>mandible | | - |
| Definition: A disorder in the gi | ngival tissue around the teeth. | | | | |
| Peritoneal necrosis | 1 | 1 | Tube feeding or TPN indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a necrotic process occurring | in the peritoneum. | | | |
| Proctitis | Rectal discomfort, intervention not indicated | Symptoms (e.g., rectal<br>discomfort, passing blood or<br>mucus); medical intervention<br>indicated; limiting instrumental<br>ADL | Severe symptoms; fecal<br>urgency or stool incontinence;<br>limiting self care ADL. | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by inflammation of the rectum. | | | | - |
| Rectal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Severely altered GI function;<br>TPN or hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an abnormal communication | between the rectum and anothe | r organ or anatomic site. | | |
| Rectal hemorrhage | Mild, intervention not indicated | Moderate symptoms; medical<br>intervention or minor<br>cauterization indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by bleeding from the rectal wall | and discharged from the anus. | | | |
| Rectal mucositis | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by inflammation of the mucous | membrane of the rectum. | | | |
| Rectal necrosis | | | Tube feeding or TPN indicated:<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a necrotic process occurring | in the rectal wall. | | | |
| Rectal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered Gl<br>function: limiting instrumental<br>ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self-care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by blockage of the normal flow | of the intestinal contents in the re | ectum. | | |
| Rectal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain, limiting self care<br>ADL | | r |
| | erized by a sensation of marked disco | | E-man | log more and a second | E |
| Rectal perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms, elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a rupture in the rectal wall. | | | | |
| Rectal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: altered GI function | Severely altered GI function;<br>tube feeding or hospitalization<br>indicated; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | erized by a narrowing of the lumen of | the rectum. | | | |
| Rectal ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function (e.g. altered dietary habits, vomiting, diarrhea) | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | · · | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Retroperitoneal hemorrhage | ized by bleeding from the retroperit | Self-limited; intervention indicated | Transfusion, medical, radiologic,<br>andoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | Tuesday and the same of the sa | | A Department of the Post of the Contractions | (ck-st-section) | N |
| Salivary duet inflammation | Slightly thickened saliva; slightly altered taste (e.g., metallic) | Thick, ropy, sticky saliva;<br>markedly altered taste;<br>alteration in diet indicated;<br>secretion-induced symptoms;<br>limiting instrumental ADL | Acute salivary gland necrosis;<br>severe secretion-induced<br>symptoms (e.g., thich saliva/oral<br>secretions or gagging); tube<br>feeding or TPN indicated;<br>limiting self care ADL; disabling | Ufe-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by inflammation of the salivary | | | | |
| Salivary gland fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; tube feeding indicated | Severely altered GI function;<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by an abnormal communication | between a salivary gland and an | other organ or anatomic site. | | |
| Small intestinal mucositis. | Asymptomatic or mild<br>symptoms; intervention not<br>indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | Severe pain; interfering with oral<br>intake; tube feeding, TPN or<br>hospitalization indicated; limiting<br>self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation of the mucous | membrane of the small intestine. | | | |
| Small intestinal obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Hospitalization indicated;<br>elective operative intervention<br>indicated; limiting self care ADL;<br>disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of the intestinal contents. | | | |
| Small intestinal perforation | | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a rupture in the small intesti | ne wall. | | | |
| Small intestinal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function | Symptomatic and severely<br>altered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a narrowing of the lumen of | the small Intestine. | | | |
| Small intestine ulcer | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; altered GI function; limiting instrumental ADL | Severely altered GI function;<br>TPN indicated; elective<br>operative or endoscopic<br>intervention indicated; limiting<br>selfcare ADL; disabling | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a circumscribed, inflammato | ory and necrotic erosive lesion on | the mucosal surface of the small in | testine. | |
| Stomach pain | Mild pain | Moderate pain: limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 8 |
| Definition: A disorder character | ized by a sensation of marked disco | omfort in the stomach. | | | |
| Tooth development disorder | Asymptomatic; hypoplasis of tooth or enamel | Impairment correctable with oral surgery | Maldévelopment with<br>impairment not surgically<br>correctable; disabling | | ì |
| Definition: A disorder character | ized by a pathological process of th | e teeth occurring during tooth dev | elopment. | | |
| Tooth discoloration | Surface steins | * | • | | - |
| Definition: A disorder character | ized by a change in tooth hue or tin | t. | | | |
| Toothache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | - |

| minutes) in 24 hrs tube feeding, a urgent intervention indicated TPN or hospitalization indicated Definition: A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth. Gastrointestinal disorders - Asymptomatic or mild Moderate; minimal, local or Severe or medically significant Life-threatening consequences; Death | | | Gastrointestinal dis | orders | | |
|---|---|---|---|---|---|---|
| Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritorneal signs Definition: A disorder characterized by inflaromation of the cecum: Upper gastrointestinal hemorrhage Mild; intervention not indicated intervention or minor cauterization indicated Definition: A disorder characterized by bleeding from the upper gastrointestinal read (oral cavity, pharynx, esophagus, and stomach). Vomiting 1 · 2 episodes (separated by 5 minutes) in 24 hrs Definition: A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth. Gastrointestinal disorders Other, specify Asymptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritorneal signs Uffe-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Use threatening consequences; urgent intervention indicated Death Womiting 1 · 2 episodes (separated by 5 minutes) in 24 hrs TPN or hospitalization indicated Definition: A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth. Gastrointestinal disorders Other, specify Asymptomatic or mild symptoms; (clinical or diagnostic observations only; intervention indicated intervention indicated) Moderate; minimal, local or or minor | | | | Grade | | |
| Definition: A disorder characterized by bleeding from the upper gastrointestinal tract (oral cavity, pharymx, esophagus, and stomach). | | | | Symptomatic (e.g., abdominal pain, fever, change in bowel habits with ileus); peritoneal | Ufe-threatening consequences; urgent operative intervention | |
| intervention or minor cauterized by bleeding from the upper gastrointestinal tract (oral cavity, pharymx, esophagus, and stomach). //omiting | Definition: A disorder characte | erized by inflammation of the cecum. | | | | |
| 1 - 2 episodes (separated by 5 minutes) in 24 hrs 3 - 5 episodes (separated by 5 minutes) in 24 hrs 3 - 5 episodes (separated by 5 minutes) in 24 hrs 2 + 6 episodes (separated by 5 minutes) in 24 hrs 2 + 6 episodes (separated by 5 minutes) in 24 hrs 2 + 6 episodes (separated by 5 minutes) in 24 hrs 2 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 + 6 + 6 episodes (separated by 5 minutes) in 24 hrs, tube feeding, TPN or hospitalization indicated 2 + 6 + | nemorrhage | | intervention or minor<br>cauterization indicated | endoscopic, or elective operative intervention indicated | | Death |
| minutes) in 24 hrs turbe feeding, TPN or hospitalization indicated Definition: A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth. Gastrointestinal disorders - Other, specify symptoms; clinical or diagnostic observations only; intervention not indicated symptoms and indicated; limiting age appropriate instrumental ADL prolongation of existing hospitalization indicated; | Definition: A disorder character | erized by bleeding from the upper gas | strointestinal tract (oral cavity, pha | rynx, esophagus, and stomach). | | |
| Other, specify symptoms; clinical or diagnostic noninvasive intervention but not immediately life urgent intervention indicated threatening; hospitalization of existing hospitalization indicated; limiting age appropriate instrumental ADL hospitalization indicated; | <b>Jomiting</b> | | | minutes) in 24 hrs, tube feeding, | | Death |
| Other, specify symptoms; clinical or diagnostic noninvasive intervention but not immediately life urgent intervention indicated threatening; hospitalization or prolongation of existing hospitalization indicated; | Jefinition: A disorder characte | erized by the reflexive act of ejecting | the contents of the stomach throu | gh the mouth. | | |
| | | symptoms; clinical or diagnostic observations only; intervention | noninvasive intervention indicated; limiting age- | but not immediately life-<br>threataning; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | | Death |

| | General | disorders and administra | ation site conditions | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Chills | Mild sensation of cold;<br>shivering; chattering of teeth | Moderate tremor of the entire body; narcotics indicated | Severe or prolonged, not responsive to narcotics | | 1 |
| Definition: A disorder charac | terized by a sensation of cold that ofte | en marks a physiologic response to | sweating after a fever. | | |
| Death neonatal | - | | - | 1 | Death |
| Definition: A disorder charac | terized by cessation of life occurring d | luring the first 28 days of life. | | | |
| Death NOS | + | * | + | € | Death |
| Definition: A cessation of life | that cannot be attributed to a CTCAE | term associated with Grade 5. | | | |
| Edema face | Localized facial edema | Moderate localized facial edema; limiting instrumental ADL | Severe swelling; limiting self care ADL | | ň |
| Definition: A disorder charac | terized by swelling due to excessive fi | uid accumulation in facial tissues. | | | |
| Edema limbs | 5 - 10% inter-limb discrepancy in volume or circumference at point of greatest visible difference; swelling or obscuration of anatomic architecture on close inspection | >10 - 30% inter-fimb<br>discrepancy in volume or<br>circumference at point of<br>greatest visible difference;<br>readily apparent obscuration of<br>anatomic architecture;<br>obiteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour, limiting<br>instrumental ADL | >30% inter-limb discrepancy in<br>volume; gross deviation from<br>normal anatomic contour;<br>limiting self care ADL | ÷ | K |
| Definition: A disorder charac | cterized by swelling due to excessive fi | uid accumulation in the upper or lo | ower extremities. | | |
| Edema trunk | Swelling or obscuration of<br>anatomic architecture on slose<br>inspection | Readily apparent obscuration of<br>anatomic architecture;<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic confour; limiting<br>instrumental ADL | Gross deviation from normal<br>anatomic contour; limiting self<br>care ADL | | S |
| Definition: A disorder charac | sterized by swelling due to excessive fi | uid accumulation in the trunk area | | | 7. |
| Facial pain | Mild pain | Moderate pain: limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | 1 |
| Definition: A disorder charac | sterized by a sensation of marked disc | omfort in the face. | | | - |
| Fatigue | Fatigue relieved by rest | Fatigue not relieved by rest:<br>limiting instrumental ADL | Fatigue not relieved by rest,<br>limiting self care ADL | | e |
| Definition: A disorder charac | terized by a state of generalized weak | ness with a pronounced inability to | summon sufficient energy to acc | omplish daily activities. | |
| Fever | 38.0 - 39.0 degrees C (100.4 - 102.2 degrees F) | >39.0 - 40.0 degrees C (102.3 -<br>104.0 degrees F) | >40.0 degrees C (>104.0<br>degrees F) for <=24 hrs | >40.0 degrees C (>104.0<br>degrees F) for >24 hrs | Death |
| | derized by elevation of the body's tem | | | | |
| | Mild flu-like symptoms present<br>derized by a group of symptoms simila | Moderate symptoms; limiting<br>instrumental ADL<br>ir to those observed in patients wit | Severe symptoms; limiting self<br>care ADL<br>h the flu it includes fever, chills, b | ody aches, malaise, loss of appeti | ite and dry |
| cough. | Manager of the same of the sam | On the head of the second | Michigan Bally and Ann | | |
| Gait disturbance | Mild change in gait (e.g., wide-<br>based, limping or hobbling) | Moderate change in gait (e.g.,<br>wide-based, limping or<br>hobbling); assistive device<br>indicated; limiting instrumental<br>ADL | Disabling; limiting self care ADL | | |
| Definition: A disorder charac | derized by walking difficulties. | | | | |
| Hypothermia | × | 35 - >32 degrees C: 95 - >89.6<br>degrees F | 32 ->28 degrees C; 89.6 -<br>>82.4 degrees F | <=28 degrees C; 82.4 degrees<br>F; life-threatening<br>consequences (e.g., coma,<br>hypotension, pulmonary edema,<br>acidemia, ventricular fibrillation) | Death |

| | 1 | disorders and administra | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4: | 5 |
| Infusion related reaction | Mild transient reaction; infusion<br>interruption not indicated;<br>intervention not indicated | Therapy or infusion interruption<br>indicated but responds promptly<br>to symptomatic treatment (e.g.,<br>antihistamines, NSAIDS.<br>narcotics, IV fluids); prophylactic<br>medications indicated for <=24<br>hrs. | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteris | zed by adverse reaction to the infu | sion of pharmacological or biologic | al substances | | , |
| Infusion site extravasation | | Erythema with associated symptoms (e.g., edema, pain, induration, phlebibs) | Ulceration or necrosis; severe<br>tissue damage; operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by leakage of a pharmacologic<br>sation and marked discomfort at th | | nfusion site into the surrounding ti | ssue. Signs and symptoms includ | e induratio |
| Injection site reaction | Tenderness with or without associated symptoms (e.g., warmth, erythema, itching) | Pain; lipodystrophy; edema;<br>phlebitis | Ulceration or necrosis; severe tissue damage; operative intervention indicated | Life-threatening consequences, urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an intense adverse reaction | (usually immunologic) developing | at the site of an injection. | | |
| irritability | Mild; easily consolable | Moderate; limiting instrumental<br>ADL; increased attention<br>indicated | Severe abnormal or excessive<br>response, limiting self care ADL,<br>inconsolable | | ę |
| Definition: A disorder characteric<br>condition: | zed by an abnormal responsivenes | ss to stimuli or physiological arous | al: may be in response to pain, frig | ht, a drug, an emotional situation | or a medic |
| Localized edema | Localized to dependent areas,<br>no disability or functional<br>impairment | Moderate localized edema and<br>intervention indicated; limiting<br>instrumental ADL | Severe localized edema and<br>intervention indicated; limiting<br>self care ADL | - | - |
| | zed by swelling due to excessive fl | 17 | omic site. | 1 | |
| Maldise | Uneasiness or lack of well being | Uneasiness or lack of well<br>being, limiting instrumental ADL | | - | Ī |
| Definition: A disorder characteris | zed by a feeling of general discomi | fort or uneasiness, an out-of-sorts | feeling. | | |
| Multi-organ failure | | | Shock with azotemia and acid-<br>base disturbances; significant<br>coagulation abnormalities | Life-threatening consequences<br>(e.g., vasopressor dependent<br>and oliguric or anuric or<br>ischemic colitis or lactic<br>acidosis) | Death |
| Definition: A disorder characteris | zed by progressive deterioration of | the lungs, liver, kidney and clottin | g mechanisms. | | |
| Neck edema | Asymptomatic localized neck edema | Moderate neck edema; slight obliteration of anatomic landmarks; limiting instrumental ADL: | Generalized neck edema (e.g.,<br>difficulty in turning neck);<br>limiting self care ADL | •1 | * |
| Definition: A disorder characteria | zed by swelling due to an accumula | ation of excessive fluid in the neck | | | |
| Non-cardiac chest pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | ě. | S |
| Definition: A disorder characteris | zed by discomfort in the chest unre | elated to a heart disorder. | | | |
| Pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | ų. | +0 |
| Definition: A disorder characteris | zed by the sensation of marked dis | | h 47 | | - |
| Sudden death NOS | | | 4 | 2 | Death |
| | ation of life that cannot be attributed | d to a CTCAE term associated with | Grade 5 | | 2.500 |
| General disorders and<br>administration site conditions -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate: minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | | Hepatobiliary disc | rders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | - 6 |
| Bile duct stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated<br>erized by a narrowing of the lumen o | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Severely altered GI function;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Biliary fistula | and the state of t | Symptomatic and intervention not indicated | Severely altered GI function:<br>TPN indicated; endoscopic<br>intervention indicated; elective<br>operative intervention indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the bile ducts and anoth | her organ or anatomic site. | | _ |
| Cholecystitis | | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | erized by inflammation involving the | | | In a market and the second | la car |
| Gallbladder fistula | Asymptomatic clinical or<br>diagnostic observations only,<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Symptomatic or severely altered<br>Gl function: TPN indicated;<br>radiologic, endoscopic or<br>elective operative intervention<br>indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by an abnormal communication | n between the gallbladder and and | other organ or anatomic site | | |
| Gallbladder necrosis | | | | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charact | erized by a necrotic process occurrin | g in the gallbladder. | | | |
| Gallbladder obstruction | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; altered GI function; IV fluids indicated <24 hrs | Symptomatic and severely<br>aftered GI function; tube<br>feeding, TPN or hospitalization<br>indicated; non-emergent<br>operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by blockage of the normal flow | of the contents of the gallbladder | | | |
| Gallbladder pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | €. | * |
| Definition: A disorder charact | erized by a sensation of marked disc | omfort in the gallbladder region. | T . | 1 | - |
| Gallbladder perforation | | | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by a rupture in the gallbladder | wall. | | | |
| Hepatic failure | | · | Asterixis: mild encephalopathy;<br>limiting self care ADL | Moderate to severe<br>encephalopathy; coma; life-<br>threatening consequences | Death |
| Definition: A disorder charact<br>dehydrogenase, and alkaline | erized by the inability of the liver to m<br>phosphatase. | etabolize chemicals in the body. L | aboratory test results reveal abno | rmal plasma levels of ammonia, bi | lirubin, lac |
| Hepatic hemorrhage | Mild; intervention not indicated | Symptomatic; medical intervention indicated | Transfusion indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the liver. | | | 11 | |
| Hepatic necrosis | | + | | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| | erized by a necrotic process occurrin | | | | |
| Hepatic pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| The second second | erized by a sensation of marked disc | omfart in the liver region. | I | | - |
| Perforation bile duct | - | * | Rediclogic, endoscopic or<br>elective operative intervention | Life-threatening consequences;<br>urgent operative intervention | Death |

| ad by an increase in blood pressured by the formation of a thrombus Asymptomatic or mild symptoms; clinical or diagnostic observations only, intervention not indicated | Intervention not indicated (blood clot) in the portal vein. Moderate: minimal, local or | Grade Reversal/retrograde portal vein flow; associated with varices and/or ascites Medical intervention indicated Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; disabiling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
|---|---|---|---|---|
| ad by an increase in blood pressu<br>ad by the formation of a thrombus<br>Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention | Decreased portal vein flow use in the portal venous system. Intervention not indicated s (blood clot) in the portal vein. Moderate; minimal, local or noninvasive intervention indicated; limiting age. | Reversal/retrograde portal vein flow; associated with varices and/or ascites Medical intervention indicated Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; | Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| ad by an increase in blood pressured<br>by the formation of a thrombus<br>Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention | Intervention not indicated (blood clot) in the portal vein. Moderate; minimal, local or noninvasive intervention indicated; limiting age | flow; associated with varices and/or ascites Medical intervention indicated Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; | Life-threatening consequences; urgent intervention indicated Life-threatening consequences; urgent intervention indicated | Death |
| ad by the formation of a thrombus<br>Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention | Intervention not indicated (blood clot) in the portal vein. Moderate; minimal, local or noninvasive intervention indicated; limiting age- | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | urgent intervention indicated Life-threatening consequences; urgent intervention indicated | |
| Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age- | but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | urgent intervention indicated | Death |

| | | | Grade | | 1 2 |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | |
| Allergic reaction | Transient flushing or rash, drug<br>fever <38 degrees C (<100.4<br>degrees F); intervention not<br>indicated | Intervention or infusion interruption indicated; responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, narcotics); prophylactic medications indicated for <=24 hrs. | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment pulmonary infiltrates) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an adverse local or general | response from exposure to an alle | ergen. | | |
| Anaphylexis | rized by an acute inflammatory reac | | Symptomatic bronchospasm,<br>with or without urticaria;<br>parenteral intervention<br>indicated; allergy-related<br>adema/angioedema;<br>hypotension | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | rized by an acute inhammatory read<br>t presents with breathing difficulty, di | | | Section of a section of the section | rypersensitivity |
| Autoimmune disorder | Asymptomatic, serologic or other evidence of autoimmune reaction, with normal organ function; intervention not indicated | Evidence of autoimmune reaction involving a non-<br>essential organ or function (e.g., hypothyroidism) | Autoimmune reactions involving major organ (e.g., colitis, anemia, myocarditis, kidney) | Actual Contract of the Contrac | Death |
| Definition: A disorder resulting<br>tissue constituents. | from loss of function or tissue destri | uction of an organ or multiple orga | ns, arising from humoral or cellula | r immune responses of the individ | ual to his own |
| Cytokine release syndrome | Mild reaction; infusion<br>interruption not indicated;<br>intervention not indicated | Therapy or infusion interruption indicated but responds promptly to symptomatic treatment (e.g., antihistamines, NSAIDS, nercotics, IV fluids); prophylactic medications indicated for <=24 hrs | Prolonged (e.g., not rapidly responsive to symptomatic medication and/or brief interruption of infusion); recurrence of symptoms following initial improvement; hospitalization indicated for clinical sequelae (e.g., renal impairment, pulmonary infiltrates) | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | Death |
| Definition: A disorder characte | rized by nausea, headache, tachyca | rdia bypotension rash and short | | release of cytokines from the cells | |
| Serum sickness | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate arthralgia; fever, rash,<br>urticaria, antihistamines<br>indicated | | Life-threatening consequences;<br>pressor or ventilatory support<br>indicated | Death |
| | rized by a delayed-type hypersensiti<br>the foreign antigen. Symptoms inclu | The same of the sa | the second secon | | |
| Immune system disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling, limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | - | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | -5 |
| Abdominal infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>jurgent intervention indicated | Death |
| | erized by an infectious process invo | | Die sole sole sol | I was not to be a second and | |
| Anorectal infection | Localized; local intervention<br>indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungat, or<br>antiviral intervention indicated<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | erized by an infectious process invo | lving the anal area and the rectum: | 7- | | |
| Appendicitis | | | IV antibiotic antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| V | - acute inhammation to the | vermiform appendix caused by a po | | Tife theretesia a vaccourant | Donth |
| Appendicitis perforated | | Symptomatic, medical<br>intervention indicated | Severe symptoms, elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by acute inflammation to the | vermiform appendix caused by a pa | (1.0 | | the |
| | | se of inflammatory and bacterial cor | | | - |
| Arteritis infective | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invo | olving an artery. | | | |
| Biliary tract infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invo | lving the billiary tract. | Tour Carrier a contrain- | | |
| Bladder infection | 1. | Oral intervention indicated (e.g., | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| | | antibiotic, antifungal, antiviral) | antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | urgent intervention indicated | |
| Definition: A disorder characte | erized by an infectious process invo | olving the bladder. | | | |
| Bone infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte<br>Breast infection | erized by an infectious process invo | Local infection with moderate | Severe infection, axillary | Life-threatening consequences; | Death |
| activity intopholi | | symptoms; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | adenitis; IV antibacterial,<br>antifungal, or antiviral<br>intervention indicated | urgent intervention indicated | Douth |
| Definition: A disorder characte | erized by an infectious process invo | lving the breast. | | | |
| Bronchial infection | • | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antiblotic, antifungal, antiviral) | IV antibiotic antifungal, or<br>antiviral intervention indicated,<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process invo | lving the bronchi | A | | |
| Catheter related infection | | Localized; local intervention<br>indicated; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by an infectious process that | | ALL MANAGEMENT AND | | ^ |
| Cecal infection | * | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | 1 | Infections and infes | | | |
|---|---|---|---|---|---|
| Andrews Work | Grade 1 2 3 4 | | | | |
| Adverse Event | | | 1 | 4 | 5 |
| Definition: A disorder characteris | zed by an infectious process in | | I A TO A TO A TO A TO A TO A TO A TO A T | | 2.77 |
| Dervicitis infection Definition: A disorder characteris | and by an infectious process is | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Conjunctivitis infective | Lea by an interioral process in | Localized; local intervention | IV antibiotic, antifungal, or | Life-threatening consequences; | Death |
| onjunctivitis inrective | | indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by an infectious process in | ivolving the conjunctiva. Clinical manif | estations include pink or red color | in the eyes. | |
| Comeal infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder characteris | zed by an infectious process in | volving the cornea. | | | |
| Cranial nerve infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteris | zed by an infectious process in | volving a cranial nerve. | | | |
| Device related infection | | 1 | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition, A disorder characteric | zed by an Infectious process in | volving the use of a medical device. | | | h. |
| Duodenal infection | 8 | Moderate symptoms; medical intervention indicated (e.g., oral antibiotics) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by an infectious process in | volving the duodenum. | 10.00.00.00.00.00.00.00.00.00.00.00.00.0 | | 1 |
| Encephalitis infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>severe changes in mental<br>status; self-limited seizure<br>activity; focal neurologic<br>abnormalities | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteris | zed by an infectious process in | evolving the brain tissue. | | | |
| Encephalomyelitis infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by an infectious process in | volving the brain and spinal cord tissu | es. | | |
| Endocardibs infective | ŧ. | V | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by an infectious process in | nvolving the endocardial layer of the he | eart. | (************************************* | |
| Definition: A disorder characteria | | Local intervention indicated | Systemic intervention or | Blindness (20/200 or worse) | F |

| - | -1 | Infections and infes | A STATE OF THE PARTY OF THE PAR | | |
|---|---|---|---|---|---|
| | | T | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Enterocolitis infectious | | Passage of >3 unformed stools.<br>per 24 hrs or duration of illness<br>>48 hrs; moderate abdominal<br>pain | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated;<br>profuse watery diarrhea with<br>signs of hypovolemia; bloody<br>diarrhea, fever; severe<br>abdominal pain; hospitalization<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invol | ving the small and large intestines. | | | |
| Esophageal infection | | Local intervention indicated<br>(e.g., oral antibiotic, antifungal,<br>antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | terized by an infectious process invol- | | A Complete Company (Co.) | wine have been a | 2 |
| Eye infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated;<br>enucleation | Death |
| Definition: A disorder charact | terized by an infectious process invol- | ving the eye. | | | |
| Gallbladder infection | erized by an infectious process Invol | and the callbladder | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | | A second second | Two ships and a contract of | Maritan State Commission Commissi | Loren |
| Gum infection | Local therapy indicated (swish<br>and swallow) | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invol | ving the gums. | | | |
| Hepatic infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | terized by an infectious process invol | ving the liver. | <b>6</b> | Account to the control of | D |
| Hepatitis viral | Asymptomatic, treatment not<br>indicated: | | Symptomatic liver dysfunction;<br>fibrosis by biopsy; compensated<br>cirrhosis; reactivation of chronic<br>hepatitis | Decompensated liver function<br>(e.g., ascites, coagulopathy,<br>encephalopathy, coma) | Death |
| Definition: A disorder charact | terized by a viral pathologic process i | nvolving the liver parenchyma. | | | |
| Infective myositis | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invol | ving the skeletal muscles. | | | |
| Joint infection | | Localized; local intervention<br>indicated; oral intervention<br>indicated (e.g., antibiotic,<br>antifungal, antiviral); needle<br>aspiration indicated (single or<br>multiple) | Arthroscopic intervention<br>indicated (e.g., drainage) or<br>arthrotomy (e.g., open surgical<br>drainage) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | terized by an infectious process invol | ving a joint | | | |
| Kidney infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | - Y | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Laryngilis<br>Definition: A disorder charac | derized by an inflammatory process | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Lip infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | | |
| Definition: A disorder charac | sterized by an infectious process inve | olving the lips. | | | |
| Lung infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| a | terized by an infectious process inve | | 2222 | 113 | |
| Lymph gland infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic;<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | cterized by an infectious process inve | olving the lymph nodes. | , | | |
| Mediastinal infection | | 8 | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process inve | olving the mediastinum. | | | |
| Meningitis | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated; focal<br>neurologic deficit | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by acute inflammation of the | meninges of the brain and/or spinal | cord. | | |
| Mucosal infection. | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process invo | olving a mucosal surface. | T | | 1 |
| Nail infection | Localized, local intervention<br>indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | | F |
| Definition: A disorder charac | terized by an infectious process inve | olving the nail. | | | |
| Otitis externa | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | sterized by an infectious process invo<br>ymptoms include fullness, itching, sw | | | ve water exposure (swimmer's ea | r infection |
| Otitis media | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an infectious process inve | olving the middle ear. | 17 | | |
| Ovarian infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pancreas infection Definition: A disorder charact | erized by an infectious process involv | ino the pancreas. | IV antibiotic, antihungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Papulopustular rash | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruritus or tenderness | Papules and/or pustules covering 10-30% BSA, which may or may not be associated with symptoms of prunitus or tenderness, associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness, limiting selFcare ADL; associated with local superinfection with oral antibiotics indicated. | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| | erized by an eruption consisting of pa | | | | , and uppe |
| Paronychia | his rash does not present with whiteh<br>Nail fold edema or erythema:<br>disruption of the cuticle | Localized intervention indicated; oral intervention indicated (e.g., antibiotic, antifungal, antiviral): nail fold edema or erythema with pain; associated with discharge or nail plate separation; limiting instrumental ADL | | Sauti S. | , |
| Definition: A disorder charact | erized by an infectious process involv | ing the soft tissues around the nai | <u> </u> | | |
| Pelvic infection | | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| And the second second second second second | erized by an infectious process involv | | | | |
| Penile infection | | Localized; local intervention<br>indicated (e.g., topical antibiobic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involv | ing the penis | | | |
| Periorbital infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involv | ing the orbit of the eye. | | | |
| Peripheral nerve infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| | erized by an infectious process involv | ing the peripheral nerves. | Asia matta dina dina di | NE a silvera i i i i i i i | |
| Peritoneal infection | | | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process involv | ing the peritoneum. | | | |
| Pharyngitis | | Localized; local intervention<br>indicated (e.g., topical antibiosc,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by inflammation of the throat. | P | | | 1 |
| Phlebitis infective | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |

| | | Infections and infes | tations | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder charact<br>of the infected vein. | erized by an infectious process invo | olving the vein. Clinical manifestation | is include erythema, marked disco | omfort, swelling, and induration alo | ng the cou |
| Pleural infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact<br>Prostate infection | erized by an infectious process invo | Moderate symptoms, oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving the prostate gland. | | | |
| Rash pustular | | Localized; local intervention<br>indicated (e.g., topical antiblotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | • | |
| Definition: A disorder charact | erized by a circumscribed and eleve | ated skin lesion filled with pus. | | · · | |
| Rhinitis infective | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | | | 9 |
| Definition: A disorder charact | erized by an infectious process invo | lving the nasal mucosal. | | | |
| Salivary gland infection | * | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an Infectious process invo | olving the salivary gland | Contract to the same | | |
| Scrotal infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving the scrotum. | 1 | 1 | |
| Sepsis | | | * | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by the presence of pathogen | ic microorganisms in the blood strea | m that cause a rapidly progressin | g systemic reaction that may lead | to shock. |
| Sinusitis | ŧ | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving the mucous membranes of the | paranasal sinuses. | | |
| Skin infection | Localized, local intervention<br>indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving the skin. | | | |
| Small intestine infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving the small intestine. | 1 | | |
| Soft tissue infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an infectious process invo | olving soft tissues. | V | | |
| Splenic infection | | • | IV antibiotic, antifungal, or<br>antiviral intervention indicated:<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |

| Infections and infestations | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | -4 | 5 |
| Definition: A disorder character | ized by an infectious process involv | ing the spleen. | | | |
| Storna site infection | Localized, local intervention indicated | Oral intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a stoma (surgically created op | ening on the surface of the body) | | |
| Tooth infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing a tooth. | _ | | |
| Tracheitis | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the traches | | | _ |
| Upper respiratory infection | | Moderate symptoms; oral<br>intervention indicated (e.g.,<br>antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the upper respiratory tract (no | se, paranasal sinuses, pharynx, la | rynx, or traches). | |
| Urethral infection | * | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic, endoscopic, or<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urethra. | | | |
| Urinary tract infection | | Localized; local intervention<br>indicated (e.g., topical antibiobc,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the urinary tract, most commo | nly the bladder and the urethra. | | |
| Ulerine infection | | Moderate symptoms; oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the endometrium. It may exter | d to the myometrium and parame | trial tissues. | |
| Vaginal infection | | Localized; local intervention indicated (e.g., topical antibiotic, antifungal, or antiviral) | (V antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vagina. | | | |
| Vulval infection | Localized, local intervention indicated | Oral intervention indicated (e.g., antibiotic, antifungal, antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated;<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the vulva. | T. | 1 | |
| Wound infection | | Localized; local intervention<br>indicated (e.g., topical antibiotic,<br>antifungal, or antiviral) | IV antibiotic, antifungal, or<br>antiviral intervention indicated,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by an infectious process involv | ing the wound. | | | |
| Infections and infestations -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | ngery. | , poisoning and procedu | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | 5 |
| Ankle fracture | Mild; non-surgical intervention<br>indicated | Limiting instrumental ADL:<br>operative intervention indicated | Limiting self care ADL; elective<br>surgery indicated | | 1 |
| Definition: A finding of damage to<br>affected leg and foot. | o the ankle joint characterized by | a break in the continuity of the ank | le bone. Symptoms include marke | d discomfort, swelling and difficult | y moving th |
| Aortic injury | | | Severe symptoms; limiting self-<br>care ADL; disabiling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage,<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | o the aorta. | | | | |
| Arterial injury | Asymptomatic diagnostic<br>finding; intervention not<br>indicated | Symptomatic (e.g.,<br>claudication); repair or revision<br>not indicated | Severe symptoms; limiting self<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences:<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | o an artery. | | | | |
| Biliary anastomotic leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage o | f bile due to breakdown of a bilian | y anastomosis (surgical connection | of two separate anatomic structu | res) | P . |
| Bladder anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | furine due to breakdown of a blac | der anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | |
| Bruising | Localized or in a dependent area | Generalized | - | * | 2 |
| Definition: A finding of injury of the | ne soft tissues or bone characteriz | ed by leakage of blood into surrou | nding tissues. | | |
| | - 7 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | Medical intervention; minimal<br>debridement indicated<br>adverse thermal reaction. Burns of<br>ity of exposure and time until provi | | Life-threatening consequences<br>nicals, direct heat, electricity, flam | Death<br>es and |
| Dermatitis radiation | Faint erytherna or dry desquamation | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases, moderate edema | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated | Death |
| Definition: A finding of cutaneous | s inflammatory reaction occurring | as a result of exposure to biologica | ally effective levels of ionizing radio | ation. | |
| Esophageal anastomotic leak | Asymptomatic diagnostic observations only: intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms: radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of an esophagea | al anastomosis (surgical connectio | n of two separate anatomic structu | res). | |
| Fall | Minor with no resultant injuries;<br>intervention not indicated | Symptomatic; noninvasive<br>intervention indicated | Hospitalization indicated | | c |
| Definition: A finding of sudden m | ovement downward, usually resul | ting in injury. | I - | | |
| Fallopian tube anastomotic leak | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a fallopian tub | e anastomosis (surgical connectio | on of two separate anatomic struct | ıres), | |
| Fallopian tube perforation | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| Definition: A finding of rupture of | the fallopian tube wall. | | | | |
| Fracture | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic but non-displaced immobilization indicated | Severe symptoms; displaced or<br>open wound with bone<br>exposure, disabling, operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | | | Civila | | |
|---|---|---|---|---|---|
| And a second decay | | | Grade | | - |
| Adverse Event | | 2 | 3 | 4 | 5 |
| Gastric anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms, radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a gastric anas | tomosis (surgical connection of tw | o separate anatomic structures). | | 1 |
| Gastrointestinal anastomotic<br>leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms, radiologic,<br>endoscopic or elective operative<br>intervention indicated | indicated | Death |
| Definition: A finding of leakage d | ue to breakdown of a gastrointest | nal anastomosis (surgical connec | tion of two separate anatomic stru | ctures). | |
| Gastrointestinal stoma necrosis | 1 | Superficial necrosis;<br>intervention not indicated | Severe symptoms;<br>hospitalization or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of a necrotic | process occurring in the gastroin | estinal tract stoma. | | ANN THE RESERVE TO TH | 1- |
| Hip fracture Definition: A finding of traumatic | injury to the hip in which the conti | Hairline fracture; mild pain;<br>firmiting instrumental ADL; non-<br>surgical intervention indicated<br>nuity of either the femoral head, fe | Severe pain; hospitalization or<br>intervention indicated for pain<br>control (e.g., traction); operative<br>intervention indicated<br>moral neck, intertrochanteric or su | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise<br>btrochanteric regions is broken. | |
| Injury to carotid artery | 2 | | Severe symptoms; limiting self | Life-threatening consequences: | Death |
| injury to carona accery | | | care ADL (e.g., transient<br>cerebral ischemia); repair or<br>revision indicated | urgent intervention indicated | Death |
| Definition: A finding of damage to | the carotid artery. | | | 1 | - |
| Injury to inferior vena cava | | Ť. | | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the inferior vena cava. | | | | |
| Injury to jugular vein | | | Symptomatic limiting self care<br>ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the jugular vein. | | | | |
| Injury to superior vena cava | Asymptomatic diagnostic<br>finding; intervention not<br>indicated | Symptomatic, repair or revision not indicated | Severe symptoms; limiting self-<br>care ADL; disabling; repair or<br>revision indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of damage to | the superior vena cava. | | | ,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,,, | |
| Intestinal stoma leak | Asymptomatic diagnostic | Symptomatic: medical | Severe symptoms: radiologic, | Life-threatening consequences; | Death |
| | observations only; intervention not indicated | intervention indicated | endoscopic or elective operative intervention indicated | urgent operative intervention indicated | |
| Definition: A finding of leakage o | f contents from an intestinal stome | s (surgically created opening on th | e surface of the body) | | 122 |
| Intestinal stoma obstruction | | Self-limited; intervention not<br>indicated | Severe symptoms; IV fluids,<br>tube feeding, or TPN indicated<br>>=24 hrs; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of blockage | of the normal flow of the contents | of the intestinal stoma. | | | |
| Intestinal stoma site bleeding | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of blood leak | age from the intestinal stoma. | | | | |
| Intraoperative arterial injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | o an artery during a surgical proce | dure. | | | |
| Intraoperative breast injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |

| Injury, poisoning and procedural complications | | | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A finding of damage to | the breast parenchyma during | g a surgical procedure. | | | 10- |
| Intraoperative cardiac injury | Tanana wana | | Primary repair of injured<br>organ/structure indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | | | Ter Property | Law and the same of the same o | F |
| Intraoperative ear injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection of injured<br>organ/structure indicated;<br>disabling (e.g., impaired<br>hearing; impaired balance) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the ear during a surgical proc | edure. | | 17 | |
| Intraoperative endocrine injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | | | Lacore and the second | Leaven | |
| Intraoperative gastrointestinal<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the gastrointestinal system di | uring a surgical procedure. | | | |
| Intraoperative head and neck injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated. | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the head and neck during a s | urgical procedure. | | | |
| Intraoperative hemorrhage | | | Postoperative radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of uncontroll | ed bleeding during a surgical p | rocedure. | 1.11.2 | | |
| intraoperative hepatobiliary<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the hepatic parenchyma and/ | or billary tract during a surgical pro | ocedure. | | |
| Intraoperative musculoskeletal<br>injury | Primary repair of injured<br>organ/structure indicated | Pantial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A finding of damage to | the musculoskeletal system o | luring a surgical procedure. | | | |
| Intraoperative neurological<br>injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the nervous system during a | surgical procedure. | | 75 | |
| Intraoperative ocular injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabiling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the eye during a surgical prod | edure. | | | |
| Intraoperative renal injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage to | the kidney during a surgical p | rocedure. | | | |
| Intraoperative reproductive tract injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |

| Injury, poisoning and procedural complications Grade | | | | | |
|---|---|---|---|---|---|
| | | | | 1 2 | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | o the reproductive organs during a | P. C. | | | Z.TVI |
| Intraoperative respiratory injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage t | o the respiratory system during a | surgical procedure. | | 1 | |
| Intraoperative skin injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated:<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage t | o the skin during a surgical proces | fure. | | | |
| Intraoperative splenic injury | | Primary repair of injured<br>organ/structure indicated | Resection or reconstruction of<br>injured organ/structure<br>indicated; disabling | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A finding of damage t | o the spleen during a surgical pro- | cedure. | | | , |
| Intraoperative urinary injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage t | o the urinary system during a surg | ical procedure. | | | |
| Intraoperative venous injury | Primary repair of injured<br>organ/structure indicated | Partial resection of injured<br>organ/structure indicated | Complete resection or<br>reconstruction of injured<br>organ/structure indicated;<br>disabling | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of damage t | o a vein during a surgical procedu | re. | | | |
| Kidney anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | of urine due to breakdown of a kidr | ey anastomosis (surgical connect) | on of two separate anatomic struc | tures). | , |
| Large intestinal anastomotic<br>leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | ue to breakdown of an anastomo: | sis (surgical connection of two sepa | arate anatomic structures) in the la | rge intestine. | |
| Pancreatic anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a pancreatic a | nastomosis (surgical connection c | ftwo separate anatomic structure | s). | |
| Pharyngeal anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms: radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a pharyngeal | anastomosis (surgical connection | of two separate anatomic structure | 95) | |
| Postoperative hemorrhage | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated. | Moderate bleeding; radiologic,<br>endoscopic, or operative<br>intervention indicated | Transfusion indicated of >=2 units (10 cc/kg for pediatrics)<br>pRBCs beyond protocol<br>specification; urgent radiologic,<br>endoscopic, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of bleeding | occurring after a surgical procedur | e. | | | |
| Postoperative thoracic<br>procedure complication | | Extubated within 24 - 72 hrs postoperatively | Extubated >72 hrs<br>postoperatively, but before<br>tracheostomy indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A finding of a previou | sly undocumented problem that or | curs after a thoracic procedure. | | | |
| Prolapse of intestinal stoma | Asymptomatic; reducible | Recurrent after manual<br>reduction; local irritation or stool<br>leakage; difficulty to fit<br>appliance; limiting instrumental | Severe symptoms; elective operative intervention indicated; limiting self-care ADL | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | | , poisoning and procedu | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | in of the intestinal stoma (surgically | | | | , |
| Prolapse of urostomy Definition: A finding of displace | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Local care or maintenance;<br>minor revision indicated | Dysfunctional stoma; elective operative intervention or major stomal revision indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Radiation recall reaction<br>(dermatologic) | Faint erythema or dry<br>desquamation<br>in inflammatory reaction caused by | Moderate to brisk erythema;<br>patchy moist desquamation,<br>mostly confined to skin folds<br>and creases; moderate edema<br>drugs, especially chemotherapeut | Moist desquamation in areas<br>other than skin folds and<br>creases; bleeding induced by<br>minor trauma or abrasion<br>ic agents, for weeks or months fol | Life-threatening consequences;<br>skin necrosis or ulceration of full<br>thickness dermis; spontaneous<br>bleeding from involved site; skin<br>graft indicated<br>lowing radiotherapy. The inflamma | Death |
| is confined to the previously ima | sdiated skin and the symptoms disa | sppear after the removal of the pha | rmaceutical agent. | | |
| Rectal anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a rectal anast | omosis (surgical connection of two | separate anatomic structures). | | |
| Seroma | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; simple aspiration<br>indicated | Symptomatic, elective radiologic<br>or operative intervention<br>indicated | | |
| | e callection of serum in the tissues | | | Las and the same of the same o | -7.00 |
| Small intestinal anastomotic<br>leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of an anastomos | sis (surgical connection of two sepa | rate anatomic structures) in the s | mall bowel. | |
| Spermatic cord anastomotic<br>leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms, radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage | due to breakdown of a spermatic c | ord anastomosis (surgical connecti | on of two separate anatomic struc | tures). | |
| Spinal fracture | Mild back pain; nonprescription<br>analgesics indicated<br>cirjury to the spine in which the co | Moderate back pain:<br>prescription analgesics<br>indicated; limiting instrumental<br>ADL | Severe back pain:<br>hospitalization or intervention<br>indicated for pain control (e.g.,<br>vertebroplasty); limiting self care<br>ADL; disability | Life-threatening consequences;<br>symptoms associated with<br>neurovascular compromise | Death |
| Stenosis of gastrointestinal stoma | - njury to the spine in which the co | | Severely altered GI function:<br>tube feeding. TPN or<br>hospitalization indicated;<br>elective operative intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of narrown | g of the gastrointestinal stoma (sur | gically created opening on the surf | ace of the body). | | |
| Stomal ulcer | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; elective<br>operative intervention indicated | | |
| Definition: A disorder character<br>gastroenterostomy procedure. | ized by a circumscribed, inflammab | ory and necrotic erosive lesion on t | he jejunal mucosal surface close | to the anastomosis site following a | |
| Tracheal hemorrhage | Minimal bleeding identified on<br>clinical or diagnostic exam;<br>intervention not indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition. A finding of bleeding | from the trachea. | | | | |
| Tracheal obstruction | Partial asymptomatic<br>obstruction on examination<br>(e.g., visual, radiologic or<br>endoscopic) | Symptomatic (e.g., noisy airway<br>breathing), no respiratory<br>distress; medical intervention<br>indicated (e.g., steroids); limiting<br>instrumental ADL | Stridor: radiologic or andoscopic intervention indicated (e.g., stent, laser); limiting self care ADL | Life-threatening airway compromise; urgent intervention indicated (e.g., trachectomy or intubation) | Death |

| | mjary | , poisoning and procedu | | | |
|---|---|---|---|---|---|
| | | | Grade | | _ |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Tracheostomy site bleeding | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | kage from the tracheostomy site. | - | | | 1 |
| Ureteric anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| | | stomosis (surgical connection of to | | Annual Control of the | |
| Urethral anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic, medical intervention indicated | Severe symptoms, radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a urethral ana | stomosis (surgical connection of b | vo separate anatomic structures). | | |
| Urostomy leak | Asymptomatic diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | of contents from a urostomy. | | | | |
| Urostomy obstruction | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; dilation or<br>endoscopic repair or stent<br>placement indicated | Attered organ function (e.g.,<br>sepsis or hydronephrosis, or<br>renal dysfunction); elective<br>operative intervention indicated | Life-threatening consequences:<br>organ failure; urgent operative<br>intervention indicated | Death |
| Definition: A finding of blockage | of the urostomy. | | T- | | |
| Urostomy site bleeding | Minimal bleeding identified on<br>clinical exam; intervention not<br>indicated | Moderate bleeding; medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A finding of bleeding | from the prostomy site. | | | | l. |
| Urostomy stenosis | | Symptomatic but no<br>hydronephrosis, no sepsis or no<br>renal dysfunction; dilation or<br>endoscopic repair or stent<br>placement indicated | Symptomatic (e.g., hydronephrosis, or renal dysfunction); elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of narrowing | | Environment of the | 5 | lug at the second | lateral. |
| Uterine anastomotic leak | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a uterine anas | stomosis (surgical connection of tw | o separate anatomic structures). | | |
| Uterine perforation | Asymptomatic diagnostic<br>observations only; intervention<br>not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms: elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a rupture in the uterine wall | <u></u> | r | | |
| Vaginal anastomotic leak | Asymptomatic diagnostic<br>observations only, intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms: radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vaginal ana: | stomosis (surgical connection of tw | o separate anatomic structures). | | |
| Vas deferens anastomotic leak | Asymptomatic diagnostic<br>observations only, intervention<br>not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A finding of leakage of | lue to breakdown of a vas deferen | s anastomosis (surgical connection | of two separate anatomic structu | res). | |
| Vascular access complication | | Device dislodgement, blockage,<br>leak, or malposition; device<br>replacement indicated | Deep vein or cardiac<br>thrombosis; intervention<br>indicated (e.g., anticoagulation,<br>lysis, filter, invasive procedure) | Embolic event including<br>pulmonary embolism or life-<br>threatening thrombus | Death |

| | injury | , poisoning and procedu | - Marie Carlotte Control Control | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event<br>/enous injury | Asymptomatic diagnostic finding; intervention not | Symptomatic (e.g., claudication); repair or revision | Severe symptoms; limiting self care ADL; repair or revision | 4<br>Ufa-threatening consequences;<br>evidence of end organ damage; | 5<br>Death |
| Definition: A finding of damage t | indicated | not indicated | indicated; disabling | urgent operative intervention indicated | |
| Vound complication | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of<br>wound; local care indicated | Hernia without evidence of<br>strangulation; fascial<br>disruption/dehiscence; primary<br>wound closure or revision by<br>operative intervention indicated | Hemia with evidence of<br>strangulation; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| | nent of a new problem at the site of | | 1 | No. | Sec. |
| Vound dehiscence | Incisional separation of <=25% of wound, no deeper than superficial fascia | Incisional separation >25% of<br>yound with local care;<br>asymptomatic hemia or<br>symptomatic hemia without<br>evidence of strangulation | Fascial disruption or dehiscence<br>without evisceration; primary<br>wound closure or revision by<br>operative intervention indicated | Life-threatening consequences;<br>symptomatic hernia with<br>evidence of strangulation;<br>fascial disruption with<br>evisceration; major<br>reconstruction flap, grafting,<br>resection, or amputation<br>indicated | Death |
| Definition: A finding of separatio | n of the approximated margins of a | surgical wound. | | | |
| Wrist fracture | Mild; non-surgical intervention<br>indicated | Limiting instrumental ADL; operative intervention indicated | Limiting self care ADL; elective surgery indicated | 4 | f |
| | injury to the wrist joint in which the | | 1 | ha was a same | Death |
| njury, poisoning and procedural<br>omplications - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening, hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | - County |
| | | | prolongation of existing<br>hospitalization indicated; | | |

| | | Investigations | | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | 5 |
| Activated partial thromboplastin<br>time prolonged | >ULN - 1.5 x ULN | >1,5 - 2.5 x ULN | >2.5 x ULN; hemorrhage | | 1 1 |
| | | romboplastin time is found to be g<br>s and disorders, both primary and | | possible indicator of coagulopa | thy, a prolon |
| Alanine aminotransferase<br>increased | >ULN - 3.0 x ULN | >3.0 - 5.0 x ULN | >5.0 - 20.0 × ULN | >20.0 x ULN | 3 |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of alanine a | minotransferase (ALT or SGPT) in | the blood specimen. | |
| Alkaline phosphatase increased | >ULN - 2.5 x ULN | >2.5 - 5.0 x ULN | >5.0 - 20.0 x ULN | >20.0 x ULN | - |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of alkaline p | phosphatase in a blood specimen. | | - |
| Aspartate aminotransferase increased | >ULN - 3.0 × ULN | >3.0 - 5.0 » ULN | >5,0 - 20,0 x ULN | >20.0 « ULN | 9 |
| Definition: A finding based on lab | oratory test results that indicate a | n increase in the level of aspartate | aminotransferase (AST or SGOT | ) in a blood specimen | |
| Blood antidiuretic hormone<br>abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | | S |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of antidiuratic horn | none in the blood specimen. | | |
| Blood bilirubin increased | >ULN - 1.5 x ULN | >1.5 - 3.0 x ULN | >3.0 - 10.0 x ULN | >10.0 x ULN | 14 |
| Definition: A finding based on lab | poratory test results that indicate a | n abnormally high level of bilirubin | in the blood. Excess bilirubin is a | ssociated with jaundice | |
| Blood corticotrophin decreased | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated | Hospitalization indicated | | 5 |
| Definition: A finding based on lab | oratory test results that indicate a | n decrease in levels of corticotrop | hin in a blood specimen | | |
| Blood gonadotrophin abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | 1 |
| Definition: A finding based on lab | oratory test results that indicate a | bnormal levels of gonadotrophin h | ormone in a blood specimen. | | |
| Blood prolactin abnormal | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | 2 | | 8 |
| Definition: A finding based on lab | | bnormal levels of prolactin hormor | re in a blood specimen. | | |
| Carbon monoxide diffusing<br>capacity decreased | 3 - 5 units below LLN; for follow-<br>up, a decrease of 3 - 5 units<br>(ml/min/mm Hg) below the<br>baseline value | 6 - 8 units below LLN; for follow-<br>up, an asymptomatic decrease<br>of -5 - 8 units (ml/min/mm Hg)<br>below the baseline value | Asymptomatic decrease of >8 units drop; >5 units drop along with the presence of pulmonary symptoms (e.g., > Grade 2 hypoxia or >Grade 2 or higher dyspnes) | | - |
| Definition: A finding based on lun | g function test results that indicate | e a decrease in the lung capacity | to absorb carbon monoxide. | | |
| Cardiac troponin l'increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | | Levels consistent with<br>myocardial infarction as defined<br>by the manufacturer | | - |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin I in a biologica | specimen: | | - |
| Cardiac troponin T increased | Levels above the upper limit of<br>normal and below the level of<br>myocardial infarction as defined<br>by the manufacturer | | Levels consistent with<br>myocardial infarction as defined<br>by the manufacturer | | ę |
| Definition: A laboratory test resul | t which indicates increased levels | of cardiac troponin T in a biologica | al specimen. | | ^ |
| CD4 lymphocytes decreased | <lln -="" 0,5="" 500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200 - 50/mm3; <0.2 × 0.05 -<br>10e9 /L | <50/mm3; <0.05 x 10e9 /L | 19 |
| Definition: A finding based on lab | poratory test results that indicate a | n decrease in levels of CD4 lymph | ocytes in a blood specimen. | | |
| Cholesterol high | >ULN - 300 mg/dL; >ULN - 7.75<br>mmol/L | >300 - 400 mg/dL; >7.75 - 10.34<br>mmol/L | >400 - 500 mg/dL; >10.34 -<br>12.92 mmol/L | >500 mg/dL, >12.92 mmal/L | Ę |
| Definition: A finding based on lab | oratory test results that indicate h | igher than normal levels of cholest | terol in a blood specimen. | | |
| | >ULN - 2.5 x ULN | >2.5 x ULN - 5 x ULN | >5 x ULN - 10 x ULN | >10×ULN | |

| | | Investigations | S | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Creatinine increased | >1 - 1.5 x baseline; >ULN - 1.5<br>x ULN | >1.5 - 3.0 x baseline; >1.5 - 3.0<br>x ULN | >3.0 baseline; >3.0 - 6.0 x ULN | >6.0 x ULN | ÷ |
| Definition: A finding based on lai | poratory test results that indicate in | ncreased levels of creatinine in a b | iological specimen. | | _ |
| Ejection fraction decreased | | Resting ejection fraction (EF) 50<br>- 40%; 10 - 19% drop from<br>baseline | Resting ejection fraction (EF) 39 - 20%; >20% drop from baseline | | |
| Definition: The percentage comp<br>contraction | outed when the amount of blood e | ected during a ventricular contract | ion of the heart is compared to the | amount that was present prior to | the |
| Electrocardiogram QT corrected<br>interval prolonged | OTc 450 - 480 ms | QTc 481 - 500 ms | OTc ≻= 501 ms on at least two<br>separate ECGs | OTc >= 501 or >60 ms change<br>from baseline and Torsade de<br>pointes or polymorphic<br>ventricular tachycardia or<br>signs/symptoms of serious<br>arrhythmia | |
| Definition: A finding of a cardiac | dysrhythmia characterized by an | abnormally long corrected QT inter | val. | | |
| Fibrinogen decreased | <1.0 - 0.75 x LLN or <25%<br>decrease from baseline | <0.75 - 0.5 x LLN or 25 - <50%<br>decrease from baseline | <0.5 - 0.26 x LLN or 50 : <75% decrease from baseline | <0.25 x LLN or 75% decrease<br>from baseline or absolute value<br><50 mg/dL | 8. |
| Definition: A finding based on fal | poratory test results that indicate a | in decrease in levels of fibrinogen | in a blood specimen. | | |
| Forced expiratory volume<br>decreased | FEV1% (percentages of<br>observed FEV1 and FVC<br>related to their respective<br>predicted values) 99 - 70%<br>predicted | FEV1 60 - 89% | 50 - 59% | <= 49% | |
| Definition: A finding based on te | st results that indicate a relative de | ecrease in the fraction of the force | d vital capacity that is exhaled in a | specific number of seconds. | |
| GGT increased | >ULN - 2.5 x ULN | >2.5 - 5.0 × ULN<br>ligher than normal levels of the ena | >5.0 - 20.0 x ULN | >20.0 × ULN | 2 |
| Control of the Contro | and the second s | group from a gamma glutamyl pepi | Salar Anna - Ann | | ma- |
| Growth hormone abnormal | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; medical intervention indicated; limiting instrumental ADL | | | - |
| Definition: A finding based on lai | boratory test results that indicate a | bnormal levels of growth hormone | in a biological specimen. | | |
| Haptoglobin decreased | <lln< td=""><td>19</td><td>-</td><td>1</td><td>14</td></lln<> | 19 | - | 1 | 14 |
| Definition: A finding based on lal | poratory test results that indicate a | in decrease in levels of haptoglobi | n in a blood specimen | | |
| Hemoglobin increased | Increase in >0 - 2 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >2 - 4 gm/dL above<br>ULN or above baseline if<br>baseline is above ULN | Increase in >4 gm/dL.above<br>ULN or above baseline if<br>baseline is above ULN | | ÷.1 |
| Definition: A finding based on lat | coratory test results that indicate in | ncreased levels of hemoglobin in a | biological specimen. | | |
| INR increased | >1 - 1.5 x ULN; >1 - 1.5 times<br>above baseline if on<br>anticoagulation | >1.5 - 2.5 x ULN; >1.5 - 2.5<br>times above baseline if on<br>anticoagulation | >2.5 x ULN; >2.5 times above<br>baseline if or anticoagulation | | 5 |
| Definition: A finding based on la | poratory test results that indicate a | in increase in the ratio of the patier | nt's prothiombin time to a control s | ample in the blood. | |
| Lipase increased<br>Definition: A finding based on lal | >ULN = 1.5 x ULN<br>boratory test results that indicate a | >1.5 - 2.0 x ULN<br>in increase in the level of lipase in | >2.0 - 5.0 x ULN<br>a biological specimen. | >5.0 x ULN | 1 |
| Lymphocyte count decreased | <lln -="" 0.8="" 800="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <800 - 500/mm3, <0.8 - 0.5 x<br>10e9 /L | <500 - 200/mm3; <0.5 - 0.2 x<br>10e9 /L | <200/mm3; <0.2 x 10e9 /L | 6 |
| Definition: A finding based on lal | boratory test results that indicate a | decrease in number of lymphocyt | es in a blood specimen. | | |
| Lymphocyte count increased | | >4000/mm3 - 20,000/mm3 | >20,000/mm3 | | 0 |
| Definition: A finding based on lai | poratory test results that indicate a | in abnormal increase in the number | er of lymphocytes in the blood, effu | sions or bone marrow | r |
| Neutrophil count decreased | <lln -="" 1.5="" 1500="" <lln="" mm3;="" x<br="">10e9 /L</lln> | <1500 - 1000/mm3; <1.5 - 1.0 x<br>10e9 /L | <1000 - 500/mm3; <1.0 - 0.5 x<br>10e9 /L | <500/mm3; <0.5 x 10e9 /L | 7 |
| | poratory test results that indicate a | decrease in number of neutrophil | s in a blood specimen. | | |
| Definition: A finding based on la | | | | | |

| | | Investigations | S | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Platelet count decreased | <lln -="" -<br="" 75,000="" <lln="" mm3;="">75.0 x 10e9 /L</lln> | <75,000 - 50,000/mm3; <75.0 - 50.0 x 10e9 /L | <50,000 - 25,000/mm3; <50.0 - 25.0 x 10e9 /L | <25,000/mm3; <25.0 x 10e9 /L | |
| Definition: A finding based on la | boratory test results that indicate a | decrease in number of platelets in | a blood specimen. | | |
| Serum amylase increased | >ULN - 1.5 x ULN | >1.5 - 2.0 x ULN | >2.0 - 5.0 x ULN | >5.0 × ULN | - |
| Definition: A finding based on la | boratory test results that indicate a | n increase in the levels of amylasi | in a serum specimen. | | |
| Urine output decreased | 2 | • | Oliguria (<80 ml in 8 hr) | Anuria (<240 ml in 24 hr) | + |
| Definition: A finding based on to | est results that indicate urine produc | ction is less relative to previous ou | tput. | | |
| Vital capacity abnormal | 90 - 75% of predicted value | <75 - 50% of predicted value;<br>limiting instrumental ADL | <50% of predicted value,<br>limiting self care ADL | | |
| Definition: A finding based on p | ulmonary function test results that in | ndicate an abnormal vital capacity | (amount of exhaled after a maxin | num inhalation) when compared to | the predi |
| Weight gain | 5 - <10% from baseline | 10 - <20% from baseline | >=20% from baseline | - | - |
| Definition: A finding characteriz | ed by an increase in overall body w | eight; for pediatrics, greater than t | he baseline growth curve. | | |
| Weight loss | 5 to <10% from baseline;<br>intervention not indicated | 10 - ≤20% from baseline;<br>nutritional support indicated | >=20% from baseline; tube<br>feeding or TPN indicated | | S |
| and the second s | ed by a decrease in overall body we | eight; for pediatrics, less than the l | baseline growth curve. | | |
| Definition: A finding characteriz | <lln -="" 3.0="" 3000="" <lln="" mm3:="" td="" x<=""><td>&lt;3000 - 2000/mm3; &lt;3.0 - 2.0 x</td><td>The state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the state of the s</td><td>&lt;1000/mm3; &lt;1.0 x 10e9 /L</td><td>-</td></lln> | <3000 - 2000/mm3; <3.0 - 2.0 x | The state of the s | <1000/mm3; <1.0 x 10e9 /L | - |
| part of the state | 10e9 /L | 10e9 /L | 10e9 /L | | |
| White blood cell decreased | 1 1 2 2 2 0 0 2 2 2 2 2 2 2 2 2 2 2 2 2 | The state of the s | 11111111 | | |

| | | Metabolism and nutrition | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | à |
| Acidosis | pH <normal, <="7.3&lt;/td" but=""><td>2</td><td>pH &lt;7.3</td><td>Life-threatening consequences</td><td>Death</td></normal,> | 2 | pH <7.3 | Life-threatening consequences | Death |
| Definition: A disorder charac | terized by abnormally high acidity (hig | h hydrogen-ion concentration) of t | ne blood and other body tissues. | | |
| Alcohol intolerance | terized by an increase in sensitivity to | Present | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| vomiting, indigestion and he | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | ble adverse ellects of alcohol, will | car can include trasar congestion, | skin libares, tiean dyattytinias, t | iausea( |
| Alkalosis | pH >normal, but <=7.5 | 4 | pH >7.5 | Life-threatening consequences | Death |
| Definition: A disorder charac | terized by abnormally high alkalinity (k | ow hydrogen-ion concentration) of | the blood and other body tissues. | | |
| Anorexia | Loss of appetite without alteration in eating trabits | Oral intake altered without<br>significant weight loss or<br>malnutrition; oral nutritional<br>supplements indicated | Associated with significant weight loss or malnutrition (e.g., inadequate oral caloric and/or fluid intake); tube feeding or TPN indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a loss of appetite. | | | | |
| Dehydration | Increased oral fluids indicated;<br>dry mucous membranes;<br>diminished skin turgor | IV fluids indicated <24 hrs | IV fluids or hospitalization indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by excessive loss of water from | n the body. It is usually caused by | severe diarrhea, vomiting or diapl | horesis. | |
| Glucose intolerance | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; dietary<br>modification or oral agent<br>indicated | Severe symptoms; insulin indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by an inability to properly meta | bolize glucase | | | |
| Hypercalcemia | Corrected serum calcium of<br>>ULN - 11.5 mg/dL; >ULN - 2.9<br>mmol/L; lonized calcium >ULN<br>- 1.5 mmol/L | Corrected serum calcium of >11.5 - 12.5 mg/dL; >2.9 - 3.1 mmol/L; lonized calcium >1.5 - 1.6 mmol/L; symptomatic | Corrected serum calcium of >12.5 - 13.5 mg/dL; >3.1 - 3.4 mmol/L; lonized calcium >1.6 - 1.8 mmol/L; hospitalization indicated | Corrected serum calcium of >13.5 mg/dL, >3.4 mmol/L. lonized calcium >1.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charac | terized by laboratory test results that in | ndicate an elevation in the concen | tration of calcium (corrected for al | bumin) in bload | |
| Hyperglycemia | Fasting glucose value >ULN -<br>160 mg/dL; Fasting glucose<br>value >ULN - 8,9 mmol/L | Fasting glucose value > 160 -<br>250 mg/dL; Fasting glucose<br>value > 8.9 - 13.9 mmol/L | >250 - 500 mg/dL; >13.9 - 27.8<br>mmol/L; hospitalization<br>indicated | >500 mg/dL; >27.8 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charactintolerance. | derized by laboratory test results that in | ndicate an elevation in the concern | tration of blood sugar. It is usually | an indication of diabetes mellitus | ar glucos |
| Hyperkalemia | >UEN - 5.5 mmoVL | >5.5 - 6.0 mmol/L | >6.0 - 7.0 mmol/L;<br>hospitalization indicated | >7.0 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact<br>the use of diuretic drugs. | terized by laboratory test results that in | ndicate an elevation in the concen | tration of potassium in the blood; | associated with kidney failure or so | ometimes |
| Hypermagnesemia | >ULN - 3.0 mg/dL; >ULN - 1.23<br>mmol/L | 3 | >3.0 - 8.0 mg/dL; >1.23 - 3.30<br>mmol/L | >8.0 mg/dL; >3.30 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charac | terized by laboratory test results that in | ndicate an elevation in the concen | tration of magnesium in the blood | L <sub>2</sub> | |
| Hypernatremia | >ULN - 150 mmol/L | >150 - 155 mmol/L | >155 - 160 mmol/L;<br>hospitalization indicated | >160 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charac | terized by laboratory test results that in | | | | |
| Hypertriglyceridemia | 150 mg/dL - 300 mg/dL; 1.71<br>mmol/L - 3.42 mmol/L | mmol/L - 5,7 mmol/L | >500 mg/dL - 1000 mg/dL; >5.7<br>mmol/L - 11.4 mmol/L | life-threatening consequences | Death |
| | ferized by laboratory test results that in | ndicate an elevation in the concen | The second of the second of th | Participation of the second | |
| Hyperuncemia | >ULN - 10 mg/dL (0.59 mmol/L)<br>without physiologic<br>consequences | | >ULN - 10 mg/dL (0.59 mmol/L)<br>with physiologic consequences | >10 mg/dL; >0.59 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charac | terized by laboratory test results that in | ndicate an elevation in the concen | tration of uric acid. | | |
| Hypoalbuminemia | <lln -="" 3="" 30="" <lln="" dl;="" g="" l<="" td=""><td>&lt;3 - 2 g/dL, &lt;30 - 20 g/L</td><td>&lt;2 g/dL; &lt;20 g/L</td><td>Life-threatening consequences; urgent intervention indicated</td><td>Death</td></lln> | <3 - 2 g/dL, <30 - 20 g/L | <2 g/dL; <20 g/L | Life-threatening consequences; urgent intervention indicated | Death |

| | | Metabolism and nutritio | n disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypocalcemia | Corrected serum calcium of<br><lln -="" 2.0<br="" 8.0="" <lln="" dl;="" mg="">mmol/L; lonized calcium <lln -<br="">1.0 mmol/L</lln></lln> | Corrected serum calcium of<br><8.0 - 7.0 mg/dL; <2.0 - 1.75<br>mmol/L; lonized calcium <1.0 -<br>0.9 mmol/L; symptomatic | Corrected serum calcium of<br><7.0 - 6.0 mg/dL; <1.75 - 1.5<br>mmol/L; lonized calcium <0.9 -<br>0.8 mmol/L; hospitalization<br>indicated | Corrected serum calcium of <6.0 mg/dL; <1.5 mmol/L; lonized calcium <0.8 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | idicate a low concentration of cal- | cium (corrected for albumin) in the | blood. | |
| Hypoglycemia | <lln -="" 3.0<br="" 55="" <lln="" dl;="" mg="">mmol/L</lln> | <55 - 40 mg/dL; <3.0 - 2.2<br>mmol/L | <40 - 30 mg/dL; <2.2 - 1.7<br>mmol/L | <30 rng/dL; <1,7 mmol/L; life-<br>threatening consequences;<br>seizures | Death |
| Definition: A disorder charact | erized by laboratory test results that it | ndicate a low concentration of glu- | cose in the blood. | | |
| Hypokalemia | <lln -="" 3.0="" l<="" mmol="" td=""><td><lln -="" 3.0="" mmovl;<br="">symptomatic; intervention<br/>indicated</lln></td><td>&lt;3.0 - 2.5 mmol/L;<br/>hospitalization indicated</td><td>&lt;2.5 mmol/L; life-threatening consequences</td><td>Death</td></lln> | <lln -="" 3.0="" mmovl;<br="">symptomatic; intervention<br/>indicated</lln> | <3.0 - 2.5 mmol/L;<br>hospitalization indicated | <2.5 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that it | ndicate a low concentration of pot | assium in the blood. | | |
| Hypomagnesemia | <lln -="" 0,5<br="" 1.2="" <lln="" dl;="" mg="">mmol/L</lln> | <1,2 - 0.9 mg/dL; <0.5 - 0.4<br>mmol/L | <0.9 - 0.7 mg/dL; <0.4 - 0.3<br>mmal/L | <0.7 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of ma | gnesium in the blood. | 1-2 | 6 |
| Hyponatremia | <lln -="" 130="" l<="" mmol="" td=""><td></td><td>&lt;130 - 120 mmol/L</td><td>&lt;120 mmol/L; life-threatening consequences</td><td>Death</td></lln> | | <130 - 120 mmol/L | <120 mmol/L; life-threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that in | ndicate a low concentration of soc | fium in the blood. | i | |
| Hypophosphatemia | <lln -="" 0.8<br="" 2.5="" <lln="" dl;="" mg="">mmol/L</lln> | <2.5 - 2.0 mg/dL; <0.8 - 0.6<br>mmol/L | <2,0 - 1.0 mg/dL; <0,6 - 0.3<br>mmol/L | <1.0 mg/dL; <0.3 mmol/L; life-<br>threatening consequences | Death |
| Definition: A disorder charact | erized by laboratory test results that is | ndicate a low concentration of pho | sphates in the blood. | | |
| Iron overload | 1 | Moderate symptoms;<br>intervention not indicated | Severe symptoms, intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by accumulation of iron in the t | issues. | | | |
| Obesity | | BMI 25 - 29.9 kg/m2 | BMI 30 - 39.9 kg/m2 | BMI >=40 kg/m2 | 5 |
| Definition: A disorder charact | erized by having a high amount of bo | dy fat. | , | | - |
| Tumor lysis syndrome | erized by metabolic abnormalities tha | - | Present | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Metabolism and nutrition | Asymptomatic or mild | | T | F-94 - 1 - | Death |
| Metabolism and nutrition<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | Muscu | loskeletal and connectiv | e tissue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | - 5 |
| Abdominal soft fissue necrosis | | Local wound care; medical intervention indicated (e.g., dressings or topical medications) | Operative debridement or other invasive intervention indicated (e.g. tissue reconstruction, flap or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | | g in the soft tissues of the abdomin | | | |
| Arthralgia | Mild pain | Moderate pain: limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | 0 |
| Definition: A disorder characteriz | ed by a sensation of marked disci | | | | |
| Arthritis | Mild pain with inflammation, erythems, or joint swelling | Moderate pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>limiting instrumental ADL | Severe pain associated with<br>signs of inflammation,<br>erythema, or joint swelling;<br>irreversible joint damage;<br>disabling, limiting self care ADL | | - |
| Definition: A disorder characteriz | ed by inflammation involving a join | nt. | | | |
| Avascular necrosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by necrotic changes in the bond the destruction of the bone stru | e tissue due to interruption of bloc<br>cture. | d supply. Most often affecting the | epiphysis of the long bones, the n | ecrotic |
| Back pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | - |
| Definition: A disorder characteria | ed by marked discomfort sensation | in the back region. | | | |
| Bone pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | ÷ | S |
| The same section is a second section of the second section is a second section of the section of the second section of the second section of the section of the second section of the section of | ed by marked discomfort sensation | | | | |
| Buttock pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | ľ. | 1 |
| | ed by marked discomfort sensation | | | T | |
| Chest wall pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | 1 |
| | ed by marked discomfort sensation | in in the chest wall region. | | _ | |
| Exostosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; limiting instrumental ADL | Severe symptoms; limiting self<br>care ADL; elective operative<br>intervention indicated | | |
| Definition: A disorder characteriz | ed by non-neoplastic overgrowth | of bone. | | | |
| Fibrosis deep connective tissue | Mild induration, able to move<br>skin parallel to plane (sliding)<br>and perpendicular to skin<br>(pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to<br>slide or pinch skin; limiting joint<br>or orifice movement (e.g.<br>mouth, anus); limiting self care<br>ADL | Generalized; associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Definition: A disorder characteriz | ed by fibrotic degeneration of the | deep connective tissues. | * | | |
| Flank pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 7 |
| Definition: A disorder characterization | ed by marked discomfort sensation | n on the lateral side of the body in | the region below the ribs and abo | ove the hip. | |
| Generalized muscle weakness | Symptomatic: weakness<br>perceived by patient but not<br>evident on physical exam | Symptomatic; weakness evident<br>on physical exam; weakness<br>limiting instrumental ADL | Weakness limiting self care<br>ADL; disabling | - | ÷ |
| Definition: A disorder characteriz | ed by a reduction in the strength ( | of muscles in multiple anatomic sit | 25, | | |
| Growth suppression | Reduction in growth velocity by<br>10 - 29% ideally measured over<br>the period of a year | Reduction in growth velocity by<br>30 - 49% Ideally measured over<br>the period of a year or 0 - 49%<br>reduction in growth from the<br>baseline growth curve | Reduction in growth velocity of >=50% ideally measured over the period of a year | : | + |

| | 400 | | e tissue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Head soft tissue necrosis | | Local wound care, medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g., tissue reconstruction, flap<br>or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by a necrotic process occurring | | | | Ť. |
| Joint effusion | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL, elective operative<br>intervention indicated; disabling | | |
| Definition: A disorder characteriz | ed by excessive fluid in a joint, us | ually as a result of joint inflammati | on. | | |
| Joint range of motion decreased | <=25% loss of ROM (range of<br>motion); decreased ROM<br>limiting athletic activity | >25 - 50% decrease in ROM;<br>limiting instrumental ADL | >50% decrease in ROM; limiting self-care ADL; disabling | | S |
| Definition: A disorder characteriz | ed by a decrease in joint flexibility | of any joint. | | | |
| Joint range of motion decreased<br>cervical spine | Mild restriction of rotation or<br>flexion between 60 - 70 degrees | Rotation <60 degrees to right or<br>left; <60 degrees of flexion | Ankylosed/fused over multiple<br>segments with no G-spine<br>rotation | | |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | cervical spine joint. | | | |
| Joint range of motion decreased<br>lumbar spine | Stiffness; difficulty bending to<br>the floor to pick up a very light<br>object but able to do athletic<br>activity | Pain with range of motion<br>(ROM) in lumbar spine; requires<br>a reaching aid to pick up a very<br>light object from the floor | <50% lumbar spine flexion;<br>associated with symptoms of<br>arikytosis or fused over multiple<br>segments with no L-spine<br>flexion (e.g., unable to reach to<br>floor to pick up a very light<br>object) | 1 | 4 |
| Definition: A disorder characteriz | ed by a decrease in flexibility of a | lumbar spine joint. | .5.0 | | |
| Kyphosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate accentuation, limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self-care ADL | € | ę |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the thoracic portion | of the spine. | | |
| Lordosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate accentuation; limiting instrumental ADL | Severe accentuation; operative intervention indicated; limiting self-care ADL | | - |
| Definition: A disorder characteriz | ed by an abnormal increase in the | curvature of the lumbar portion o | the spine. | | |
| Muscle weakness left-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self-care ADL; disabling | • | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the left side of th | e body | | |
| Muscle weakness lower limb | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | 5 | 5- |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the lower limb muscles. | | | |
| Muscle weakness right-sided | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic: evident on<br>physical exam, limiting<br>instrumental ADL | Limiting self care ADL; disabling | | 7 |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the muscles on the right side of | the body. | | |
| Muscle weakness trunk | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | | - |
| Definition: A disorder characteriz | ed by a reduction in the strength o | f the trunk muscles | | | |
| Muscle weakness upper limb | Symptomatic; perceived by<br>patient but not evident on<br>physical exam | Symptomatic; evident on<br>physical exam; limiting<br>instrumental ADL | Limiting self care ADL; disabling | · | 5 |

| | IMUSCU | loskeletal and connectiv | e ussue dispiders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Musculoskėletai deformity | Cosmetically and functionally insignificant hypoplasia | Deformity, hypoplasia, or<br>asymmetry able to be<br>remediated by prosthesis (e.g.,<br>shoe insert) or covered by<br>clothing | Significant deformity,<br>hypoplasia, or asymmetry,<br>unable to be remediated by<br>prosthesis or covered by<br>clothing; disabling | | ŧ |
| Definition: A disorder characteria | ed by of a malformation of the mu | sculoskeletal system. | 1 | | |
| Myalgia | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | î . | 7 |
| | ed by marked discomfort sensatio | n originating from a muscle or gro | up of muscles. | | |
| Myositis | Mild pain | Moderate pain associated with<br>weakness; pain limiting<br>instrumental ADL | Pain associated with severe<br>weakness; limiting self care<br>ADL | • | 5 |
| Definition: A disorder characteria | zed by inflammation involving the s | keletal muscles. | | | |
| Neck раїп | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 1 |
| Definition: A disorder characteriz | zed by marked discomfort sensatio | n in the neck area. | | | |
| Neck soft tissue necrosis | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g., tissue reconstruction, flap<br>or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | ed by a necrotic process occurring | in the soft tissues of the neck. | | | |
| Osteonecrosis of jaw | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>intervention indicated (e.g.,<br>topical agents); limiting<br>instrumental ADL | Severe symptoms; limiting self-<br>care ADL; elective operative<br>intervention indicated | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a necrotic process occurring | in the bone of the mandible. | | | |
| Osteoporosis | Radiologic evidence of osteoporoxis or Bone Mineral Density (BMD) t-score -1 to -2.5 (osteopenia); no loss of height or intervention indicated | BMD t-score <2.5; loss of<br>height <2 cm; anti-osteoporotic<br>therapy indicated; limiting<br>instrumental ADL | Loss of height >=2 cm:<br>hospitalization indicated; fimiting<br>self care ADL | | P. |
| Definition: A disorder characteristicomposition), resulting in increase | zed by reduced bone mass, with a | decrease in cortical thickness and | in the number and size of the trut | peculae of cancellous bone (but no | ormal chem |
| Pain in extremity | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | ÷ |
| Definition: A disorder characteria | zed by marked discomfort sensatio | n in the upper or lower extremities | | | |
| Pelvic soft tissue necrosis | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g., tissue reconstruction, flap<br>or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteria | zed by a necrotic process occurring | in the soft tissues of the pelvis. | | | |
| Scoliosis | <20 degrees; clinically undetectable | >20 - 45 degrees; visible by<br>forward flexion; limiting<br>instrumental ADL | >45 degrees; scapular<br>prominence in forward flexion;<br>operative intervention indicated;<br>limiting self care ADL; disabling | | - |
| Definition: A disorder characteria | zed by a malformed, lateral curvatu | re of the spine. | | | |
| Soft tissue necrosis lower limb | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g., tissue reconstruction, flap<br>or grafting) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteris | ed by a necrotic process occurring | in the soft tissues of the lower e | (tremity | | |
| Soft tissue necrosis upper limb | | Local wound care; medical<br>intervention indicated (e.g.,<br>dressings or topical<br>medications) | Operative debridement or other<br>invasive intervention indicated<br>(e.g., tissue reconstruction, flap<br>or grafting) | Life-threatening consequences; urgent intervention indicated | Death |

| Adverse Event Superficial soft tissue fibrosis | | iosaciciai dila comiccity | e tissue disorders | | |
|---|---|---|---|---|---|
| Adverse Event<br>Superficial soft tissue fibrosis | | | Grade | | |
| | All Mild induration, able to move skin parallel to plane (sliding) and perpendicular to skin (pinching up) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration; unable to slide or pinch skin; limiting joint or orifice movement (e.g., mouth, anus); limiting self care ADL | 4<br>Generalized, associated with<br>signs or symptoms of impaired<br>breathing or feeding | 5<br>Death |
| Definition: A disorder character | zed by fibrotic degeneration of the | superficial soft tissues. | | | |
| Trismus | Decreased ROM (range of motion) without impaired eating | Decreased ROM requiring small bites, soft foods or purees | Decreased ROM with inability to<br>adequately aliment or hydrate<br>orally | | |
| Definition: A disorder character | ized by lack of ability to open the m | outh fully due to a decrease in the | range of motion of the muscles of | mastication | |
| Unequal limb length | Mild length discrepancy <2 cm | Moderate length discrepancy 2 -<br>5 cm; shoe lift indicated; limiting<br>instrumental ADL | | | Ĺ |
| Definition: A disorder character | ized by of a discrepancy between th | ne lengths of the lower or upper ex | tremities. | | |
| Musculoskeletal and connective<br>lissue disorder - Other, specify | | Moderate; minimal, local of<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening.consequences;<br>urgent intervention indicated | Death |

| Adverse Event 1 2 3 4 5 1 Leukemia secondary to oncology chemotherapy Definition: A disorder characterized by leukemia arising as a result of the mutagenic effect of chemotherapy agents. Myelodysplastic syndrome | Leukemia secondary to oncology chemotherapy Definition: A disorder characterized by leukemia arising as a result of the mutagenic effect of chemotherapy agents. Myelodysplastic syndrome Definition: A disorder characterized by insufficiently healthy hematapoietic cell production by the bornarrow. Treatment related secondary malignancy Definition: A disorder characterized by insufficiently healthy hematapoietic cell production by the bornarrow. Treatment related secondary malignancy Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy; blast crists in leukemia Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Tumor pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Moderate pain; limiting age-appropriate instrumental ADL Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Proposition of existing hospitalization or prolongation of existing hospitalization or prolongation of existing hospitalization or | girant and u | ns beingn, n | n, malignant and | uit and ans | | ai cysts ai | u poly | 49) | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Leukemia secondary to oncology chemotherapy Definition: A disorder characterized by leukemia arising as a result of the mutagenic effect of chemotherapy agents. Myelodysplastic syndrome Life-threatening consequences; urgent intervention indicated Death management related secondary malignancy Treatment related secondary malignancy - Non life-threatening secondary malignancy Non life-threatening secondary malignancy malignancy plast crists in leukemia Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Turnor pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated: limiting age-appropriate instrumental ADL Treatment related secondary malignancy. Acute life-threatening secondary malignancy. Acute life-threatening secondary malignancy. Acute life-threatening secondary malignancy. Severe pain; limiting self care ADL Severe or medically significant but not immediately life-threatening consequences; urgent intervention indicated that not immediately life-threatening secondary malignancy. Death malignancy indicated indicated indicated; limiting age-appropriate instrumental ADL Treatment related secondary malignancy. Turnor pain Mild pain Severe or medically significant but not immediately life-threatening secondary malignancy. Death malignancy malignancy malignancy. Turnor pain Mild pain Severe or medically significant but not immediately life-threatening secondary malignancy. Death malignancy malignancy malignancy. Turnor pain Mild pain Severe or medically significant but not immediately life-threatening secondary malignancy. De | Leukemia secondary to oncology chemotherapy Definition: A disorder characterized by leukemia arising as a result of the mutagenic effect of chemotherapy agents Myelodysplastic syndrome | 100 | | | | Grade | | 1 | - 4 | | 1 |
| Definition: A disorder characterized by leukemia arising as a result of the mutagenic effect of chemotherapy agents | Definition: A disorder characterized by leukernia arising as a result of the mutagenic effect of chemotherapy agents | 2 | - 1- | | 2 | - | 3 | | | | |
| Definition: A disorder characterized by insufficiently healthy hematapoietic cell production by the bone marrow. Treatment related secondary malignancy malignancy Treatment related secondary malignancy malignancy malignancy To production by the bone marrow. Treatment related secondary malignancy malignancy malignancy malignancy malignancy malignancy Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Moderate; minimal, local or noninvasive intervention indicated; limiting age threatening; hospitalization of existing hospitalization indicated; Death under the marked discomfort from metastasis. Life-threatening consequences; Death under the marked or fractured from metastasis. Death under the marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; imiting age threatening; hospitalization indicated; Death under the marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Death under the marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Death under the marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Death under the marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Death under the marked discomfort from a neoplasm that may be pre | Definition: A disorder characterized by insufficiently healthy hematapoietic cell production by the bone marrow. Treatment related secondary malignancy malignancy Treatment related secondary malignancy Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify observations only; intervention indicated indicated; limiting age— threatening; hospitalization or prolongation of existing hospitalization indicated; Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Nooplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify observations only; intervention indicated; limiting age— threatening; hospitalization or prolongation of existing hospitalization indicated; Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Weoplasms benign, malignant and the prolongation of malignancy and the prolongation of existing hospitalization indicated; Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Definition: A disorder characterized by marked discomfort from a neoplasm that | agenic effect of | as a result of the | of the mutagenic effect of | nic effect of cher | notherapy ager | its | , | | | |
| Treatment related secondary malignancy | Prelatment related secondary malignancy malignancy; blast crisis in leukemia Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Tumor pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Ilmiting age— Observations only; intervention indicated indicated; limiting age— Appropriate instrumental ADL prolongation of existing hospitalization indicated; | | | | | li . | | | | | Death |
| Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Severe pain; limiting self care ADL ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Severe or medically significant but not immediately life-threatening; hospitalization or not indicated. Imiting age-appropriate instrumental ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of existing hospitalization indicated; Death propriate instrumental ADL Destriction: ADL Timetring self care and proving self-care and proving self-ca | Definition: A disorder characterized by development of a malignancy most probably as a result of treatment for a previously existing malignancy. Tumor pain Mild pain Moderate pain; limiting instrumental ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Moderate pain; limiting self care ADL Severe pain; limiting self care Loudening self-care and provide indicated or metastasis. Severe or medically significant but not immediately life-threatening; hospitalization or indicated or prolongation of existing hospitalization indicated; limiting age-propriate instrumental ADL prolongation of existing hospitalization indicated; | i production by | ntiny nematapolet | · | saction by the t | Non life-thr | | | malignancy; blast cri | | Death |
| Tumor pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition; A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify observations only; intervention not indicated Moderate pain; limiting self care ADL Severe pain; limiting self care | Tumor pain Mild pain Moderate pain; limiting Severe pain; limiting self care ADL Definition: A disorder characterized by marked discomfort from a neoplasm that may be pressing on a nerve, blocking blood vessels, inflamed or fractured from metastasis. Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify Observations only; intervention not indicated initiated on the properties of instrumental ADL proposite instrument | obably as a resu | a malignancy mo | most probably as a res | oly as a result of | reatment for a | previously ex | | | | |
| Reoplasms benign, malignant of mild symptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Moderate; minimal, local or severe or medically significant but not immediately life—threatening; hospitalization or prolongation of existing hospitalization indicated; limiting age—appropriate instrumental ADL prolongation indicated; | leoplasms benign, malignant of mild symptoms; clinical or diagnostic observations only; intervention not indicated Asymptoms; clinical or diagnostic observations only; intervention not indicated Moderate; minimal, local or noninvasive intervention indicated of threatening; hospitalization or prolongation of existing hospitalization indicated; limiting age-appropriate instrumental ADL | pain; limiting | Mod | Moderate pain; limiting | n; limiting | Severe pai | | | | | 7 |
| and unspecified (incl cysts and observations only; intervention not indicated observations only; intervention not indicated observations only; intervention not indicated observations only; intervention not indicated observations only; intervention not indicated observations only; intervention indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated; | and unspecified (incl cysts and observations only; intervention not indicated observations only; intervention not indicated observations only; intervention not indicated observations only; intervention not indicated observations only; intervention indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated; limiting age-appropriate instrumental ADL prolongation of existing hospitalization indicated. | nat may be press | ort from a neopla: | oplasm that may be pre- | nay be pressing | on a nerve, blo | cking blood ve | ssels, inf | amed or fractured fro | om metastas | sis. |
| | | ive intervention<br>: limiting age- | diagnostic nonit | noninvasive intervention<br>indicated; limiting age- | ntervention<br>iting age- | but not imm<br>threatening<br>prolongation<br>hospitalization | nediately life-<br>y; hospitalizati<br>on of existing<br>tion indicated; | on or | The state of the state of | | Death |
| | | | | | | disabling; | | | | | |
| | | | | | | disabling; | | | | | |
| | | | | | | disabling | | | | | |
| | | | | | | disabling | | | | | |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Abducens nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | Y |
| Definition: A disorder characteri | zed by involvement of the abducen | s nerve (sixth cranial nerve) | | | |
| Accessory nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | 7 | 3 |
| The second secon | zed by involvement of the accessor | | | | |
| Acoustic nerve disorder NOS | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms: limiting self care ADL | | f |
| Definition: A disorder characteri | zed by involvement of the acoustic | nerve (eighth cranial nerve). | | | |
| Akathisia | Mild restlessness or increased motor activity | Moderate restlessness or<br>increased motor activity; limiting<br>instrumental ADL | Severe restlessness or<br>increased motor activity; limiting<br>self care ADL | | ŧ |
| Definition: A disorder characteri | zed by an uncomfortable feeling of | inner restlessness and inability to | T | | _ |
| Amnesia | Mild; transient memory loss | Moderate; short term memory<br>loss; limiting instrumental ADL | Severe; long term memory loss;<br>limiting self care ADL | * | ië i |
| A self- | zed by systematic and extensive lo | ss of memory. | ks and a second and | | |
| Aphonia | | | Voicelessness; unable to speak | | Ä |
| | zed by the inability to speak. It may | | | Land of the second of the seco | Fa. over |
| Arachnoiditis | Mild symptoms | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences:<br>urgent intervention indicated | Death |
| | zed by inflammation of the arachno | In a second | I | | |
| Ataxia | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; mechanical<br>assistance indicated | | ì |
| Definition: A disorder characteri | zed by lack of coordination of musc | le movements resulting in the imp | pairment or inability to perform volu | intary activities. | |
| Brachial plexopathy | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | |
| Definition: A disorder characteri | zed by regional paresthesia of the I | orachial plexus, marked discomfor | t and muscle weakness, and limite | ed movement in the arm or hand. | |
| Central nervous system<br>necrosis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms, corticosteroids indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by a necrotic process occurring | in the brain and/or spinal cord | | | |
| Cerebrospinal fluid leakage | Post-craniotomy: asymptomatic;<br>Post-lumbar puncture: transient<br>headache; postural care<br>indicated | Post-craniotomy: moderate<br>symptoms, medical intervention<br>indicated; Post-lumbar<br>puncture: persistent moderate<br>symptoms; blood patch<br>indicated | Severe symptoms; medical intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteri | zed by loss of cerebrospinal fluid in | to the surrounding tissues. | | | |
| Cognitive disturbance | Mild cognitive disability; not<br>interfering with work/school/life<br>performance; specialized<br>educational services/devices<br>not indicated | Moderate cognitive disability;<br>interfering with work/school/life<br>performance but capable of<br>independent living; specialized<br>resources on part time basis<br>indicated | Severe cognitive disability;<br>significant impairment of<br>work/school/life performance | • | 2 |
| Definition: A disorder characteri | zed by a conspicuous change in co | gnitive function: | | | |
| Concentration impairment | Mild inattention or decreased level of concentration | Moderate impairment in attention or decreased level of concentration; limiting instrumental ADL | Severe impairment in attention<br>or decreased level of<br>concentration; limiting self care<br>ADL | ÷ | 160 |

| | -Y | Nervous system dis | orgers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Depressed level of consciousness | Decreased level of alertness | Sedation; slow response to<br>stimuli: limiting instrumental<br>ADL | Difficult to arouse | Life-threatening consequences | Death |
| Definition: A disorder charact | erized by a decrease in ability to perc | eive and respond. | | | , |
| Dizziness | Mild unsteadiness or sensation of movement | Moderate unsteadiness or<br>sensation of movement; limiting<br>instrumental ADL | Severe unsteadiness or<br>sensation of movement; limiting<br>self care ADL | <b>-</b> 0 | el |
| Definition: A disorder charact | erized by a disturbing sensation of lig | htheadedness, unsteadiness, gidd | liness, spinning or rocking. | | |
| Dysarthria | Mild slurred speech | Moderate impairment of<br>articulation or slurred speech | Severe impairment of<br>articulation or slumed speech | - | 6 |
| Definition: A disorder charact | erized by slow and slurred speech res | sulting from an inability to coordina | te the muscles used in speech. | | |
| Dysesthesia | Mild sensory alteration | Moderate sensory alteration;<br>limiting instrumental ADL | Severe sensory alteration:<br>limiting selfcare ADL | | |
| Definition: A disorder charact | erized by distortion of sensory percep | tion, resulting in an abnormal and | unpleasant sensation | | _ |
| Dysgeusie | Altered taste but no change in<br>diet | Altered taste with change in diet<br>(e.g., oral supplements);<br>noxious or unpleasant taste;<br>loss of taste | | | |
| Definition: A disorder charact | erized by abnormal sensual experienc | e with the taste of foodstuffs; it ca | n be related to a decrease in the | sense of smell. | |
| Dysphasia | Awareness of receptive or<br>expressive characteristics; not<br>impairing ability to communicate | Moderate receptive or<br>expressive characteristics;<br>impairing ability to communicate<br>spontaneously | Severe receptive or expressive<br>characteristics; impairing ability<br>to read, write or communicate<br>intelligibly | | |
| Definition: A disorder charact | erized by impairment of verbal commi | unication skills, often resulting from | n brain damage. | | |
| Edema cerebral | 1 | | | Life-threatening consequences;<br>urgent intervention indicated | 2 |
| Definition: A disorder charact | erized by swelling due to an excessive | e accumulation of fluid in the brain | | | |
| Encephalopathy | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | erized by a pathologic process involvi | La con con constant of the | | | |
| Extrapyramidal disorder | Mild involuntary movements | Moderate involuntary<br>movements; limiting<br>instrumental ADL | Severe involuntary movements<br>or torticollis; limiting self care<br>ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by abnormal, repetitive, involur | ntary muscle movements, frenzied | speech and extreme restlessness | i. | |
| Facial muscle weakness | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms, limiting self care ADL | | - |
| Definition: A disorder charact | erized by a reduction in the strength o | f the facial muscles. | | | |
| Facial nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms, limiting self care ADL | | - |
| Definition: A disorder charact | erized by involvement of the facial ne | | Y- | | 1 |
| Glossopharyngeal nerve<br>disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by involvement of the glossoph | aryngeal nerve (ninth cranial nerv | e). | | |
| Headache | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 2 |
| Definition: A disorder charact | erized by a sensation of marked disco | omfort in various parts of the head. | not confined to the area of distrib | ution of any nerve. | |
| Hydrocephalus | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms;<br>intervention not indicated | Severe symptoms or<br>neurological deficit; intervention<br>indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an abnormal increase of ce | ebrospinal fluid in the ventricles o | f the brain. | | _ |
| Hypersomnia | Mild increased need for sleep | Moderate increased need for sleep | Severe increased need for sleep | - | 4 |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Hypoglossal nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self-<br>care ADL | | ŧ |
| Definition: A disorder characte | rized by involvement of the hypoglo- | ssal nerve (twelfth cranial nerve). | | | |
| intracranial hemorrhage | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Moderate symptoms; medical intervention indicated | Ventriculostomy, ICP<br>monitoring, intraventricular<br>thrombolysis, or operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Ischemia cerebrovascular | Asymptomatic; clinical or<br>diagnostic observations only; | Moderate symptoms | 2 | Ŷ | Ş |
| Definition: A disorder characte<br>damage. | intervention not indicated<br>rized by a decrease or absence of b | lood supply to the brain caused by | obstruction (thrombosis or embo | ism) of an artery resulting in neuro | ological |
| (Vth nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self-<br>care ADL | - | - |
| Definition: A disorder characte | rized by involvement of the trochlea | r nerve (fourth cranial nerve). | | | |
| Lethargy | Mild symptoms; reduced<br>alertness and awareness | Moderate symptoms; limiting instrumental ADL | - | 0 | 3 |
| Definition: A disorder characte | rized by a decrease in consciousne | ss characterized by mental and ph | ysical inertness | | |
| Leukoencephalopathy | Asymptomatic; small focal<br>T2/FLAIR hyperintensities;<br>involving periventricular white<br>matter or <1/3 of susceptible<br>areas of cerebrum +/- mild<br>increase in subarachnoid space<br>(SAS) and/or mild<br>ventriculomegaly | Moderate symptoms; focal<br>T2/FLAIR hyperintensities; involving periventricular white<br>matter extending into centrum<br>semiovale or involving 1/3 to 2/3<br>of susceptible areas of<br>cerebrum +/- moderate increase<br>in SAS and/or moderate<br>ventriculomegaly | Severe symptoms, extensive<br>T2/FLAIR hyperintensities,<br>involving perventricular white<br>matter involving 2/3 or more of<br>susceptible areas of cerebrum<br>+/- moderate to severe increase<br>in SAS and/or moderate to<br>severe ventriculomegaly | Life-threatening consequences; extensive T2/FLAIR hyperintensities, involving periventricular white matter involving most of susceptible areas of cerebrum +/- moderate to severe increase in SAS and/or moderate to severe ventriculomegaly. | Death |
| Definition: A disorder characte | rized by diffuse reactive astrocytosis | with multiple areas of necrotic foo | i without inflammation. | | |
| Memory impairment | Mild memory impairment | Moderate memory impairment;<br>limiting instrumental ADL | Severe memory impairment:<br>limiting selfcare ADL | * | 1 |
| Definition: A disorder characte | rized by a deterioration in memory f | unction. | | | |
| Meningismus | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | rized by neck stiffness, headache, a | nd photophobia resulting from imit | ation of the cerebral meninges. | | |
| Movements involuntary | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | 1 | 7 |
| | rized by uncontrolled and purposele | ss movements. | | | |
| Myelitis | Asymptomatic; mild signs (e.g.,<br>Babinski's reflex or Lhermitte's<br>sign) | Moderate weakness or sensory<br>loss; limiting instrumental ADL | Severe weakness or sensory<br>loss; limiting self-care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by inflammation involving the | spinal cord. Symptoms include wea | kness, paresthesia, sensory loss | marked discomfort and incontine | nce. |
| Neuralgia | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | 7 |
| Definition: A disorder character | rized by intense painful sensation al | 11.7 | | 1 | |
| Nystagmus | | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | 1 | 2 |
| | rized by involuntary movements of t | | | | |
| Oculomotor nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms, limiting<br>instrumental ADL | Severe symptoms, limiting self care ADL | | |
| Definition: A disorder characte | rized by involvement of the oculomo | otor nerve (third cranial nerve) | | | |
| Olfactory nerve disorder | | Moderate symptoms: limiting instrumental ADL | Severe symptoms; limiting self care ADL | - | £ |

| | | Nervous system dis | sorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Paresthesia | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | |
| Definition: A disorder characteriz<br>are experienced in the absence of | | ensory neurons resulting in abnor | mal cutaneous sensations of tingli | ng numbness, pressure cold, and | warmth th |
| Peripheral motor neuropathy | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL; assistive device indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneration | on of the peripheral motor nerves. | | | |
| Peripheral sensory neuropathy | Asymptomatic; loss of deep tendon reflexes or paresthesia | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation or degeneration | on of the peripheral sensory nerve | s. | | |
| Phantom pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | • | |
| Definition: A disorder characteriz | ed by marked discomfort related t | o a limb or an organ that is remov | ed from or is not physically part of | the body | |
| Presyncope | 10. | Present (e.g., near fainting) | 4- | | |
| Application of the property of the contract of | ed by an episode of lightheadedn | | A STATE OF THE PARTY OF THE PAR | Lucia monther and a second | Later and |
| Pyramidal tract syndrome | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by dysfunction of the corticosp<br>nd a decrease in fine motor coord | Charles of the second of the s | al cord. Symptoms include an incre | ease in the muscle tone in the low | er extremiti |
| Radiculitis | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL; medical<br>intervention indicated | Severe symptoms; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz<br>connecting nerve root. | ed by inflammation involving a ne | | ked discomfort radiating along a ne | erve path because of spinal pressu | ire on the |
| Recurrent laryngeal nerve palsy | Asymptomatic; clinical or<br>diagnostic observations only,<br>intervention not indicated | Moderate symptoms | Severe symptoms; medical intervention indicated (e.g., thyroplasty, vocal cord injection) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by paralysis of the recurrent la | ryngeal nerve. | | | |
| Reversible posterior<br>leukoencephalopathy syndrome | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; abnormal<br>imaging studies; limiting<br>instrumental ADL | Severe symptoms; very<br>abnormal imaging studies:<br>limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | | | seizures associated with imaging to and cytotoxic drug treatment. It is | | |
| Seizure | Brief partial seizure: no loss of consciousness | Brief generalized seizure | Multiple seizures despite<br>medical intervention | Life-threatening; prolonged repetitive seizures | Death |
| Definition: A disorder characteriz | ed by a sudden, involuntary skele | tal muscular contractions of cereb | oral or brain stem origin. | | |
| Sinus pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | - |
| Definition: A disorder characteriz | ed by marked discomfort in the fa | ce, between the eyes, or upper te | eth originating from the sinuses. | | |
| Somnolence | Mild but more than usual drowsiness or sleepiness | Moderate sedation; limiting instrumental ADL | Obtundation or stupor | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by characterized by excessive | sleepiness and drowsiness. | | | |
| Spasticity | Mild or slight increase in muscle tone | | Severe increase in muscle tone<br>and increase in resistance<br>through range of motion | Life-threatening; unable to move active or passive range of motion | Death |
| Definition: A disorder characteriz<br>disturbances | ed by increased involuntary musc | | erfering with voluntary movement. | | peach |
| Stroke | Asymptomatic or mild<br>neurologic deficit; radiographic<br>findings only | Moderate neurologic deficit | Severe neurologic deficit | Life-threatening consequences; urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a sudden loss of sensory fu | nction due to an intracranial vasc | ular event. | | 7 |
| Syncope | | - | Fainting; orthostatic collapse | 2 | 200 |

| | | Nervous system dis | orders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| ransient ischemic attacks | Mild neurologic deficit with or<br>without imaging confirmation | Moderate neurologic deficit with<br>or without imaging confirmation | | | ś |
| | erized by a brief attack (less than 24 t | | | neurological deficit. | ř. |
| remor | Mild symptoms | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | |
| | erized by the uncontrolled shaking mo | evernent of the whole body or indi- | | | |
| rigeminal nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms: limiting self-<br>care ADL | 8 | Ē |
| Definition: A disorder characte | erized by involvement of the trigemine | il nerve (fifth cranial nerve). | 1 | | |
| /agus nerve disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Moderate symptoms: limiting instrumental ADL | Severe symptoms, limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | erized by involvement of the vagus ne | rve (tenth cranial nerve). | | | |
| asovagal reaction | | | Present | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | erized by a sudden drop of the blood | pressure, bradycardia, and periph | eral vasodilation that may lead to | loss of consciousness. It results fr | om an |
| ncrease in the stimulation of t<br>Hervous system disorders - | 77 3 17 17 17 | Moderate; minimal, local or | 4 | No. a construction of | Death |
| Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | |

| | Pregn | ancy, puerperium and pe | erinatal conditions | | |
|---|---|---|---|---|---|
| | | | Grade | 1 | |
| Adverse Event | 1 | 2 | 3 | | 5 |
| | rized by death in utero; failure of the | product of conception to show ev | dence of respiration, heartbeat, o | r definite movement of a voluntary | Fetal loss at<br>any<br>gestational<br>age<br>muscle after |
| expulsion from the uterus, with<br>Fetal growth retardation | out possibility of resuscitation. | <10% percentile of weight for gestational age | <5% percentile of weight for gestational age | <1% percentile of weight for gestational age | 3 |
| Definition: A disorder character | rized by inhibition of fetal growth res | ulting in the inability of the fetus to | achieve its potential weight. | | |
| Premature delivery | Delivery of a liveborn infant at >34 to 37 weeks gestation. | Delivery of a liveborn infant at >28 to 34 weeks gestation | Delivery of a liveborn infant at<br>24 to 28 weeks gestation | Delivery of a liveborn infant at<br>24 weeks of gestation or less | C.E. |
| Definition: A disorder characte<br>gestation. | rized by delivery of a viable infant be | efore the normal end of gestation. | Typically, viability is achievable be | etween the twentieth and thirty-sev | enth week of |
| Unintended pregnancy | 1 2 | 4, | Unintended pregnancy | | - |
| N. S. P. S. M. S. P. S. | rized by an unexpected pregnancy s | at the time of conception. | The second secon | 1.0 | |
| Pregnancy, puerperium and<br>perinatal conditions - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderaté, local or noninvasive intervention indicated; limiting instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated; | Life-threatening consequences: urgent intervention indicated | Death |
| | -I | di - | disabling; limiting self care ADL | 1 | |
| | | di - | oisabiling; limining self care AUL | | |
| | | | oisabiling; limining self care AUL | | |
| | | | oisabiling; limining self care AUL | | |
| | | | oisabiling; limining self care AUL | | |
| | | | oisabiling; limining self care AUL | | |
| | | | orsatning; unrining self care AUL | | |
| | | | orsatning; unrining self care AUL | | |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | ħ. |
| Agitation | Mild mood alteration | Moderate mood alteration | Severe agitation; hospitalization not indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charac | terized by a state of restlessness asso | ociated with unpleasant feelings of | irritability and tension. | | |
| Anorgasmia | Inability to achieve orgasm not<br>adversely affecting relationship | Inability to achieve orgasm<br>adversely affecting relationship | | | |
| In case the decision of the first transfer to the contract the contract transfer to the contract transfer | terized by an inability to achieve orgas | Lance of the second | Construction of the construction | Inc. and the second | |
| Anxiety. | Mild symptoms; intervention not<br>indicated | Moderate symptoms; limiting<br>instrumental ADL | Severe symptoms: limiting self<br>care ADL; hospitalization not<br>indicated | Life-threatening; hospitalization indicated | Death |
| Definition: A disorder charac<br>stimulus | terized by apprehension of danger and | d dread accompanied by restlessn | ess, tension, tachycardia, and dy | spries unattached to a clearly ident | ifiable |
| Confusion | Mild disorientation | Moderate disorientation; limiting instrumental ADL | Severe disorientation; limiting self-care ADL | Life-threatening consequences:<br>urgent intervention indicated | Death |
| | terized by a lack of clear and orderly t | hought and behavior | i . | 1- | |
| Delayed orgasm | Delay in achieving orgasm not<br>adversely affecting relationship | Delay in achieving orgasm<br>adversely affecting relationship | | | - |
| | terized by sexual dysfunction characte | | 6 Million and a series and all of the | Ind a service | Descrip |
| Delirium | Mild acute confusional state | Moderate and acute confusional<br>state; limiting instrumental ADL | Severe and acute confusional<br>state; limiting self care ADL;<br>hospitalization indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac<br>reversible condition. | derized by the acute and sudden deve | lopment of confusion, illusions, mo | vement changes, inattentiveness | agitation, and hallucinations. Usu | ally, it is a |
| Delusions | | Moderate delusional symptoms | Severe delusional symptoms;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by false personal beliefs held o | contrary to reality, despite contradi | ctory evidence and common sens | e. | |
| Depression | Mild depressive symptoms | Moderate depressive<br>symptoms; limiting instrumental<br>ADL | Severe depressive symptoms;<br>limiting selfcare ADL;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by melancholic feelings of grie | for unhappiness. | | | |
| Euphoria | Mild mood elevation | Moderate mood elevation | Severe mood elevation (e.g., hypomania) | - | t. |
| Definition: A disorder charac | terized by an exaggerated feeling of w | rell-being which is disproportionate | to events and stimuli. | | |
| Hallucinations | Mild hallucinations (e.g., perceptual distortions) | Moderate hallucinations | Severe hallucinations;<br>hospitalization not indicated | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated | Death |
| Definition: A disorder charac | terized by a false sensory perception i | n the absence of an external stimu | ilus. | | |
| Insomnia | Mild difficulty falling asleep,<br>staying asleep or waking up<br>early | Moderate difficulty falling<br>asleep, staying asleep or<br>waking up early | Severe difficulty in falling<br>asleep, staying asleep or<br>waking up early | | * |
| Definition: A disorder charac | terized by difficulty in falling asleep an | d/or remaining asleep. | | | |
| Libido decreased | Decrease in sexual interest not<br>adversely affecting relationship | Decrease in sexual interest adversely affecting relationship | | ŀ | |
| Definition: A disorder charac | terized by a decrease in sexual desire | · | | 1- | |
| Libido increased | Mild increase in sexual interest<br>not adversely affecting<br>relationship | Moderate increase in sexual<br>interest adversely affecting<br>relationship | Severe increase in sexual<br>interest leading to dangerous<br>behavior | | • |
| Definition: A disorder charac | terized by an increase in sexual desire | 0. | 1 | | |
| Manie | Mild manic symptoms (e.g.,<br>elevated mood, rapid thoughts,<br>rapid speech, decreased need<br>for sleep) | Moderate manic symptoms<br>(e.g., relationship and work<br>difficulties; poor hygiene) | Severe manic symptoms (e.g.,<br>hypomania; major sexual or<br>financial indiscretions);<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; hospitalization indicated | Death |
| Definition, A disorder charac | terized by excitement of psychotic pro | portions manifested by mental and | physical hyperactivity, disorgania | zation of behavior and elevation of | mood. |
| Personality change | Mild personality change | Moderate personality change | Severe personality change;<br>hospitalization not indicated | Life-threatening consequences, threats of harm to self or others; | Death |

| | | Psychiatric disor | ders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | rized by a conspicuous change in a | person's behavior and thinking. | | | |
| Psychosis<br>Definition: A disorder characte | Mild psychotic symptoms rized by personality change, impaire | Moderate psychotic symptoms<br>(e.g., disorganized speach;<br>impaired reality testing)<br>d functioning, and loss of touch vi | Severe psychotic symptoms<br>(e.g., paranoid: extreme<br>disorganization); hospitalization<br>not indicated<br>th reality, it may be a manifestation | Life-threatening consequences,<br>threats of harm to self or others;<br>hospitalization indicated<br>on of schizophrenia, bipolar Gsordi | |
| tumor. | | | | | |
| Restlessness | Mild symptoms; intervention not<br>indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms: limiting self care ADL | | ÷ |
| Definition: A disorder characte | rized by an inability to rest, relax or b | ne still. | | | |
| Suicidal ideation | Increased thoughts of death but<br>no wish to kill oneself | Suicidal ideation with no specific<br>plan or intent | Specific plan to commit suicide<br>without serious intent to die<br>which may not require<br>hospitalization | Specific plan to commit suicide<br>with serious intent to die which<br>requires hospitalization | Χ, |
| | rized by thoughts of taking one's ow | n life. | | | |
| Suicide atternpt | 7 | | Suicide attempt or gesture<br>without intent to die which may<br>not require hospitalization | Suicide attempt with intent to<br>de which requires<br>hospitalization | Death |
| | rized by self-inflicted harm in an atte | | | P-1 | |
| Psychiatric disorders - Other,<br>specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention | Moderate, minimal, local or<br>noninvasive intervention<br>indicated; limiting age- | Severe or medically significant<br>but not immediately life-<br>threatening; disabling; limiting | Life-threatening consequences;<br>hospitalization or urgent<br>intervention indicated | Death |
| + | not indicated | appropriate instrumental ADL | self care ADL | Intervention indicated | |

| | 1 | Renal and urinary di | | | |
|---|---|---|---|---|---|
| | | | Grade | | -2 |
| Adverse Event | - 1 | 2 | 3 | 4 | ħ. |
| Acute kidney injury | Creatinine level increase of >0.3<br>mg/dL; creatinine 1.5 - 2.0 x<br>above baseline | Creatinine 2 - 5 x above baseline | mg/dL; hospitalization indicated | | Death |
| Dennibon: A disorder charac<br>causes (ureleral or bladder o | terized by the acute loss of renal functi<br>outflow obstruction). | on and is traditionally classified a | is pre-renal (low blood flow into kid | ney), renai (kidney damage) and p | ocst-rena! |
| Bladder perforation | terized by a rupture in the bladder wall | Extraperitoneal perforation, indwelling catheter indicated | Intraperitoneal perforation;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>organ failure; urgent operative<br>intervention indicated | Death |
| Bladder spasm | Intervention not indicated | Antispasmodics indicated | Hospitalization indicated | | |
| | terized by a sudden and involuntary co | A STATE OF THE PARTY OF THE PAR | Trospitalization froitated | 1. | |
| Chronic kidney disease | eGFR (estimated Glomerular<br>Filtration Rate) or CrCI<br>(creatinine clearance) <lln -="" 60<br="">ml/min/1.73 m2 or proteinuria<br/>2+ present; urine<br/>protein/creatinine &gt;0.5</lln> | eGFR or CrCl 59 - 30<br>ml/min/1.73 m2 | eGFR or CrCl 29 - 15<br>ml/min/1.73 m2 | eGFR or CrCl-<15 ml/min/1.73<br>m2; dialysis or renal transplant<br>indicated. | Death |
| Definition: A disorder charac | terized by gradual and usually perman | ent loss of kidney function resulti | ng in renal failure. | | |
| Cystitis noninfective | Microscopic hematuria; minimal<br>increase in frequency, urgency,<br>dysuria, or nocturia; new onset<br>of incontinence | Moderate hematuria; moderate increase in frequency, urgency, dysuria, nocturia or incontinence; urinary catheter placement or bladder irrigation indicated; limiting instrumental ADL | Gross hematuria; transfusion, IV<br>medications or hospitalization<br>indicated; elective endoscopic,<br>radiologic or operative<br>intervention indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charac | ferized by inflammation of the bladder | which is not caused by an infection | on of the urinary tract. | | |
| Hematuria | Asymptomatic; clinical or diagnostic observations only, intervention not indicated | Symptomatic; urinary catheter<br>or bladder irrigation indicated;<br>limiting instrumental ADL | Gross hematuria; transfusion, IV<br>medications or hospitalization<br>indicated; elective endoscopic,<br>radiologic or operative<br>intervention indicated; limiting<br>self care ADL | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder charac | terized by laboratory test results that in | dicate blood in the urine. | 1000000 | | |
| Hemoglobinuria | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | | 7 | | r. |
| Definition: A disorder charac | terized by laboratory test results that in | dicate the presence of free hemo | oglobin in the urine. | | |
| Proteinuria | 1+ proteinuria; urinary protein<br><1.0 g/24 hrs. | Adults: 2+ proteinuria: urinary<br>protein 1.0 - 3.4 g/24 hrs:<br>Pediatric urine P/C<br>(Protein/Creatinine) ratio 0.5 -<br>1.9 | Adults: urinary protein >=3.5<br>g/24 hrs;<br>Pediatric: urine P/C >1.9 | | 1 |
| Definition: A disorder charac | terized by laboratory test results that in | dicate the presence of excessive | protein in the urine. It is predomin | antly albumin, but also globulin. | |
| Renal calculi | Asymptomatic or mild<br>symptoms; occasional use of<br>nonprescription analgesics<br>indicated | Symptomatic; oral antiemetics<br>indicated; around the clock<br>nonprescription analgesics or<br>any oral narcotic analgesics<br>indicated | Hospitalization indicated; IV intervention (e.g., analgesics, antiemetics); elective endoscopic or radiologic intervention indicated | Life-threatening consequences;<br>urgent radiologic, endoscopic or<br>operative intervention indicated | Death |
| Definition: A disorder charac | terized by the formation of crystals in t | he pelvis of the kidney. | | | |
| Renal colic | Mild pain not interfering with<br>activity; nonprescription<br>medication indicated | Moderate pain; limiting<br>instrumental ADL; prescription<br>medication indicated | Hospitalization indicated;<br>limiting selfcare ADL | | 4 |
| Definition: A disorder charac | terized by paroxysmal and severe flan | | the inquired area. Often the cause | is the nessame of kidney stones | ti. |

| | Y- | Renal and urinary di | sorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Renal hemorrhage | Mild symptoms; intervention not indicated | Analgesics and hematocrit monitoring indicated | Transfusion, radiation, or<br>hospitalization indicated;<br>elective radiologic, endoscopic<br>or operative intervention<br>indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by bleeding from the kidney. | | | | 1 |
| Urinary fistula | | Noninvasive intervention<br>indicated; urinary or suprapubic<br>catheter placement indicated | Limiting self care ADL; elective<br>radiologic, endoscopic or<br>operative intervention indicated;<br>permanent urinary diversion<br>indicated | Life-threatening consequences;<br>urgent radiologic or operative<br>intervention indicated | Death |
| | ized by an abnormal communication | | system and another organ or anato | omic site. | 1 |
| Urinary frequency Definition: A disorder character | Present ized by unnation at short intervals. | Limiting instrumental ADL;<br>medical management indicated | | | |
| Urinary incontinence | Occasional (e.g., with coughing, sneezing, etc.), pads not indicated | Spontaneous; pads indicated;<br>(imiting instrumental ADL | Intervention indicated (e.g.,<br>clamp, collagen injections);<br>operative intervention indicated;<br>limiting self care ADL | | |
| Definition: A disorder character | ized by inability to control the flow o | furine from the bladder. | | | |
| Urinary retention | Urinary, suprapubic or<br>intermittent catheter placement<br>not indicated, able to void with<br>some residual | Placement of urinary,<br>suprapubic or intermittent<br>catheter placement indicated;<br>medication indicated | Elective operative or radiologic<br>intervention indicated;<br>substantial loss of affected<br>kidney function or mass | Ufe-threatening consequences;<br>organ failure; urgent operative<br>intervention indicated | Death |
| Definition: A disorder character | ized by accumulation of urine within | the bladder because of the inabil | ity to urinate. | | |
| Urinary tract obstruction | Asymptomatic; clinical or diagnostic observations only | Symptomatic but no<br>hydronephrosis, sepsis or renal<br>dysfunction; urethral dilation,<br>urinary or suprapubic catheter<br>indicated | Symptomatic and altered organ function (e.g., hydronephrosis, or renal dysfunction); elective radiologic, endoscopic or operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by blockage of the normal flow | of contents of the urinary tract. | A STATE OF THE PARTY OF THE PAR | | |
| Urinary tract pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 7 |
| The second secon | ized by a sensation of marked disco | | | 6 | |
| Urinary urgency | Present | Limiting instrumental ADL;<br>medical management indicated | | | + |
| Urine discoloration | ized by a sudden compelling urge to<br>Present | aumate. | | 3 | |
| | ized by a change in the color of the | urine. | 15- | | 17 |
| Renal and urinary disorders -<br>Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, local or noninvasive<br>intervention indicated; limiting<br>instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated,<br>disabling; limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Azgospermia | 3 4 6 94 | An extra series at | Absence of sperm in ejaculate | | 4 |
| Definition: A disorder characte | rized by laboratory test results that in | ndicate complete absence of spen | matozoa in the semen. | | |
| Breast atrophy Definition: A disorder characte | Minimal asymmetry; minimal<br>atrophy<br>rized by underdevelopment of the br | Moderate asymmetry; moderate<br>atrophy | Asymmetry >1/3 of breast volume; severe atrophy | 1 | 1 |
| Breast pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | ÷ . | 4 |
| Definition: A disorder characte | rized by marked discomfort sensatio | n in the breast region | 7 | | |
| Dysmenorrhea | Mild symptoms; intervention not indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms, limiting self care ADL | - | 9 |
| Definition: A disorder characte | rized by abnormally painful abdomin | al cramps during menses. | | | |
| Dyspareunia | Mild discomfort or pain<br>associated with vaginal<br>penetration; discomfort relieved<br>with use of vaginal lubricants or<br>estrogen | Moderate discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>partially relieved with use of<br>vaginal lubricants or estrogen | Severe discomfort or pain<br>associated with vaginal<br>penetration; discomfort or pain<br>unrelieved by vaginal lubricants<br>or estrogen | • | |
| Definition: A disorder characte | rized by painful or difficult coitus. | | i- | 1 | |
| Ejaculation disorder | Diminished ejaculation | Anejaculation or retrograde<br>ejaculation | | 1 | |
| Definition: A disorder characte | rized by problems related to ejaculat | tion. This category includes prema | ture, delayed, retrograde and pair | rful ejaculation. | |
| Erectile dysfunction | Decrease in erectile function<br>(frequency or rigidity of<br>arections) but intervention not<br>indicated (e.g., medication or<br>use of mechanical device,<br>penile pump) | Decrease in erectile function<br>(frequency/rigidity of erections),<br>erectile intervention indicated<br>(e.g., medication or mechanical<br>devices such as penile pump) | Decrease in erectile function<br>(frequency/rigidity of erections)<br>but erectile intervention in<br>helpful (e.g., medication or<br>mechanical devices such as<br>penile pump); placement of a<br>permanent penile prosthesis<br>indicated (not previously<br>present) | | |
| Definition: A disorder character | rized by the persistent or recurrent in | nability to achieve or to maintain a | n erection during sexual activity. | 1 | - |
| Fallopian tube obstruction | Diagnostic observations only:<br>intervention not indicated | Mild symptoms: elective<br>intervention indicated | Severe symptoms; elective<br>operative intervention indicated | - | 2 |
| Definition: A disorder characte | rized by blockage of the normal flow | of the contents in the fallopian tub | ie. | | |
| Fallopian tube stenosis | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., organ resection) | Death |
| | rized by a narrowing of the fallopian | | | | |
| Female genital tract fistula | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms, elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communication | n between a female reproductive s | ystem organ and another organ o | r anatomic site | |
| Feminization acquired | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | | | 2 |
| Definition: A disorder characte | rized by the development of seconds | ary female sex characteristics in m | ales due to extrinsic factors. | | |
| Genital edema | Mild swelling or obscuration of<br>anatomic architecture on close<br>inspection | Readily apparent obscuration of<br>anatomic architecture,<br>obliteration of skin folds; readily<br>apparent deviation from normal<br>anatomic contour. | Lymphorrhea; gross deviation<br>from normal anatomic contour<br>limiting self care ADL | - | ÷ |
| Definition: A disorder characte | rized by swelling due to an excessiv | e accumulation of fluid in the genit | als. | | |
| Gynecomastia | Asymptomatic breast enlargement | Symptomatic (e.g., pain or<br>psychosocial impact) | Severe symptoms; elective operative intervention indicated | - | × |
| Definition: A disorder characte | rized by excessive development of the | ne breasts in males. | Y | | |
| Hematosalpīnx | Minimal bleeding identified on<br>imaging study or laparoscopy;<br>intervention not indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | Rep | roductive system and bi | east disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder character | zed by the presence of blood in a fa | allopian tube. | | | |
| Irregular menstruation | Intermittent menses with<br>skipped menses for no more<br>than 1 to 3 months | Intermittent menses with skipped menses for more than 4 to 6 months | Persistent amenorrhea for more than 6 months | | ř. |
| | zed by irregular cycle or duration of | | | | |
| Lactation disorder | Mild changes in Jactation, not<br>significantly affecting production<br>or expression of breast milk | Changes in lactation,<br>significantly affecting breast<br>production or expression of<br>breast milk | | | |
| Definition: A disorder character | zed by disturbances of milk secretic | on. It is not necessarily related to p | pregnancy that is observed in fema | ales and can be observed in male: | |
| Menorrhagis | Mild; Iron supplements indicated | intervention indicated (e.g.,<br>hormones) | Severe; transfusion indicated;<br>surgical intervention indicated<br>(e.g., hysterectomy) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | zed by abnormally heavy vaginal bi | | | 6 | |
| Nipple deformity | Asymptomatic, asymmetry with<br>slight retraction and/or<br>thickening of the nipple areolar<br>complex: | Symptomatic; asymmetry of<br>nipple areolar complex with<br>moderate retraction and/or<br>thickening of the nipple areolar<br>complex | | | |
| Definition: A disorder character | zed by a malformation of the nipple | | | | |
| Oligospermia | Sperm concentration >48 million/mL or mobility >68% | Sperm concentration 13 - 48 million/mL or motility 32 - 68% | Sperm concentration <13 million/mL or motility <32% | ÷ | - |
| Definition: A disorder character | zed by a decrease in the number o | spermatozoa in the semen. | | | - |
| Ovarian hemorrhage | Minimal bleeding identified on<br>imaging study or laproscopy;<br>intervention not indicated | Moderate bleeding, medical<br>intervention indicated | Severe bleeding; transfusion<br>Indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | zed by bleeding from the ovary. | | | | |
| Ovarian rupture | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention not indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | zed by tearing or disruption of the o | varian tissue. | | | |
| Ovulation pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | 1 |
| | zed by marked discomfort sensatio | n in one side of the abdomen bety | veen menstrual cycles, around the | time of the discharge of the ovum | from the |
| ovarian follicle. | Les and a second | | 1 | hading a sold of an arrange | D- ac- |
| Pelvic floor muscle weakness | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic, not interfering<br>with bladder, bowel, or vaginal<br>function; limiting instrumental<br>ADL | Severe symptoms; limiting self care ADL | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder character | zed by a reduction in the strength o | f the muscles of the pelvic floor. | | | |
| Pelvic pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | |
| Definition: A disorder character | zed by marked discomfort sensatio | n in the pelvis. | | | |
| Penile pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | + | - |
| Definition: A disorder character | zed by marked discomfort sensatio | n in the penis. | T | | |
| Perineal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | * | 5 |
| Definition: A disorder character | zed by a sensation of marked disco | mfort in the area between the gen | | | _ |
| Premature menopause<br>Definition: A disorder character | -<br>zed by ovarian failure before the ag | e of 40. Symptoms include hot fla | Present<br>shes, night sweets, mood swings | and a decrease in sex drive | 2 |
| Prostatic hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding, medical intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | Re | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder characte | rized by bleeding from the prostate | gland | | | |
| Prostatic obstruction | Diagnostic observations only;<br>intervention not indicated | Mild symptoms, elective<br>intervention indicated | Severe symptoms, elective operative intervention indicated | | |
| Definition: A disorder characte<br>stream, and incomplete empty | rized by compression of the urethra<br>ing of the bladder). | secondary to enlargement of the | prostate gland. This results in voidi | ng difficulties (straining to void, sl | ow urine |
| Prostatic pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | 5 |
| Definition: A disorder characte | rized by a sensation of marked disc | omfort in the prostate gland. | | | |
| Scrotal pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | - |
| Definition: A disorder characte | rized by marked discomfort sensation | on in the scrotal area. | | | |
| Spermatic cord hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences; urgent operative intervention indicated | Death |
| | rized by bleeding from the spermati | Para and a second | 2 | | T |
| Spermatic cord obstruction | Diagnostic observations only:<br>intervention not indicated | Mild symptoms: elective<br>intervention indicated | Severe symptoms; elective<br>operative intervention indicated | | 7 |
| | rized by blockage of the normal flow | | T | Los - | |
| Testicular disorder | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic but not interfering<br>with urination or sexual<br>activities; intervention not<br>indicated; limiting instrumental<br>ADL | Severe symptoms; interfering<br>with urination or sexual function;<br>limiting self care ADL;<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by involvement of the testis. | | | | ^ |
| Testicular hemorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding: medical intervention indicated | Severé bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by bleeding from the testis. | | | | |
| Testicular pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | * |
| Definition: A disorder characte | rized by a sensation of marked disc | omfort in the testis. | | | , |
| Uterine fistula | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms: elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characte | rized by an abnormal communicatio | n between the uterus and another | organ or anatomic site | | |
| Uterine tremorrhage | Minimal bleeding identified on<br>imaging study; intervention not<br>indicated | Moderate bleeding; medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characte | rized by bleeding from the uterus. | | | | |
| Uterine obstruction | Diagnostic observations only:<br>intervention not indicated | Mild symptoms, elective<br>intervention indicated | Severe symptoms, elective operative intervention indicated | 7 | ĥ |
| Definition: A disorder characte | rized by blockage of the uterine out | et. | | | |
| Uterine pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | | 2 |
| Definition: A disorder characte | rized by a sensation of marked disc | omfort in the uterus. | | | |
| Vaginal dischärge | Mild vaginal discharge (greater than baseline for patient) | Moderate to heavy vaginal<br>discharge; use of perineal pad<br>or tampon indicated | - | | * |
| Definition: A disorder characte | rized by vaginal secretions, Mucus ( | | discharged from the vagina natura | lly, especially during the childbea | ing years |
| Vaginal dryness | Mild vaginal dryness not<br>interfering with sexual function | Moderate vaginal dryness<br>interfering with sexual function<br>or causing frequent discomfort | Severe vaginal dryness<br>resulting in dyspareunia or<br>severe discomfort | | |

| | Rep | productive system and b | reast disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Vaginal fistula | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms, elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the vagina and anothe | r organ or anatomic site. | | |
| Vaginal hemorrhage | Minimal bleeding identified on<br>clinical exam or imaging study;<br>intervention not indicated | Moderate bleeding, medical<br>intervention indicated | Severe bleeding; transfusion<br>indicated; radiologic or<br>endoscopic intervention<br>indicated | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the vagina. | | | | |
| Vaginal inflammation | Mild discomfort or pain, edema,<br>or redness | Moderate discomfort or pain,<br>edema, or redness; limiting<br>instrumental ADL | Severe discomfort or pain,<br>edema, or redness; limiting self<br>care ADL; small areas of<br>mucosal ulceration | Widespread areas of mucosal<br>ulceration; life-threatening<br>consequences; urgent<br>intervention indicated | Death |
| Definition: A disorder characteriz | ed by inflammation involving the v | agina. Symptoms may include re | dness, edema, marked discomfort | and an increase in vaginal dischar | ge. |
| Vaginal obstruction | Diagnostic observations only:<br>intervention not indicated | Mild symptoms; elective<br>intervention indicated | Severe symptoms; elective operative intervention indicated | | 7 |
| Definition: A disorder characteriz | ed by blockage of vaginal canal. | | | | |
| Vaginal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | - |
| Definition: A disorder characteriz | ed by a sensation of marked disco | omfort in the vagina. | | | |
| Vaginal perforation | Asymptomatic clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic and intervention<br>not indicated | Severe symptoms; elective operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a rupture in the vaginal wall | | | | |
| Vaginal stricture | Asymptomatic; mild vaginal shortening or narrowing | Vaginal narrowing and/or<br>shortening not interfering with<br>physical examination | Vaginal narrowing and/or<br>shortening interfering with the<br>use of tampons, sexual activity<br>or physical examination | - | Death |
| Definition: A disorder characteriz | ed by a narrowing of the vaginal c | anal, | | | |
| Vaginismus | Mild discomfort or pain<br>associated with vaginal<br>spasm/tightening; no impact<br>upon sexual function or physical<br>examination | Moderate discomfort or pain<br>associated with vaginal<br>spesm/tightening; disruption in<br>sexual function and physical<br>examination | Severe discomfort or pain<br>associated with vaginal<br>spasm/tightening; unable to<br>tolerate vaginal penetration or<br>physical examination | | ė |
| Definition: A disorder characteriz<br>intercourse. | ed by involuntary spasms of the p | elvic floor muscles, resulting in pr | athologic tightness of the vaginal w | all during penetration such as duri | ng sexu |
| Reproductive system and breast<br>disorders - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate, minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | Keshi | ratory, thoracic and med | lastillal disorders | | |
|---|---|---|---|---|---|
| | 7000 | | Grade | | |
| Adverse Event | 4 | 2 | 3 | 4 | - 1 |
| | ed by progressive and life-threater | ning pulmonary distress in the abs | Present with radiologic findings;<br>intubation not indicated<br>ence of an underlying pulmonary | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated<br>condition, usually following major i | Death<br>trauma or |
| surgery. | And a transport of the second | No. vi. co. Accessor Accessor | | | |
| the product of the same of the same of the same | Mild symptoms; intervention not<br>indicated<br>led by an inflammation of the nasa<br>of the sinuses, eyes, middle ear, a | intervention indicated<br>I mucous membranes caused by | | the state of the s | ay also |
| | or the sinuses, eyes, middle ear, a | line piraryric, Symptoms include si | | The state of the s | Death |
| Арпеа. | | | Present; medical intervention<br>indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by cessation of breathing. | | | | _ |
| Aspiration | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Altered eating habits; coughing<br>or choking episodes after eating<br>or swallowing; medical<br>intervention indicated (e.g.,<br>suction or oxygen) | Dyspnea and pneumonia<br>symptoms (e.g., aspiration<br>pneumonia); hospitalization<br>indicated; unable to aliment<br>orally | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by inhalation of solids or liquids | into the lungs. | | | |
| Atelectasis | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., dyspnea, cough); medical intervention indicated (e.g., chest physiotherapy, suctioning); bronchoscopic suctioning | Oxygen indicated;<br>hospitalization or elective<br>operative intervention indicated<br>(e.g., stent, laser) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by the collapse of part or the e | ntire lung. | | | |
| Bronchial fistula | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL, endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic open<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between the bronchus and anoth | ner organ or anatomic site. | | |
| Bronchial obstruction | Asymptomatic; clinical or diagnostic observations only intervention not indicated | Symptomatic (e.g., mild<br>wheezing), endoscopic<br>evaluation indicated;<br>radiographic evidence of<br>atelectasis/lobar collapse;<br>medical management indicated<br>(e.g., steroids, bronchodilators) | Shortness of breath with stridor; endoscopic intervention indicated (e.g., laser, stent placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by blockage of a bronchus pas | sage, most often by bronchial sec | retions and exudates. | | |
| Bronchial stricture | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., rhonchi or wheezing) but without respiratory distress; medical intervention indicated (e.g., steroids, bronchodilators) | Shortness of breath with stridor;<br>endoscopic intervention<br>indicated (e.g., laser, stent<br>placement) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the bronchial | tube. | | | |
| Bronchopleural fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated, limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>with thoracoplasty, chronic opera<br>drainage or multiple<br>thoracotomies indicated | Death |
| Definition: A disorder characteriz | ed by an abnormal communication | between a bronchus and the ple | ural cavity. | | |
| Bronchopulmonary hemorrhage | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| | Respi | ratory, thoracic and med | | | |
|---|---|---|---|---|---|
| | - | | Grade | | |
| Adverse Event | | 2 | 3 | 4 | 5 |
| Bronchospasm | Mild symptoms; intervention not<br>indicated | Symptomatic: medical<br>intervention indicated; limiting<br>instrumental ADL | Limiting self-care ADL, oxygen<br>saturation decreased | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by a sudden contraction of the | smooth muscles of the bronchial | wall: | | |
| Chylothorax | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; thoracentesis or tube drainage indicated | Severe symptoms; elective operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by milky pleural effusion (abno | rmal collection of fluid) resulting fr | om accumulation of lymph fluid in | the pleural cavity_ | |
| Cough | Mild symptoms; nonprescription<br>intervention indicated | Moderate symptoms, medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self care ADL | | Ĺ |
| Definition: A disorder charact<br>by a distinctive sound, | erized by sudden, often repetitive, spa | asmodic contraction of the thoraci | c cavity, resulting in violent release | e of air from the lungs and usually | accompan |
| Dyspnea | Shortness of breath with moderate exertion | Shortness of breath with<br>minimal exertion; limiting<br>instrumental ADL | Shortness of breath at rest;<br>limiting selfcare ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an uncomfortable sensation | of difficulty breathing. | | | |
| Epistaxis | Mild symptoms; intervention not<br>indicated | Moderate symptoms; medical<br>intervention indicated (e.g.,<br>nasal packing, cauterization;<br>topical vesoconstrictors) | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by bleeding from the nose. | | | | |
| Hiccups | Mild symptoms: intervention not<br>indicated | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; interfering<br>with sleep; limiting self care<br>ADL | r. | |
| Definition: A disorder charact | erized by repeated gulp sounds that r | esult from an involuntary opening | and closing of the glottis. This is a | ttributed to a spasm of the diaphra | igm. |
| Hoarseness | Mild or intermittent voice<br>change; fully understandable;<br>self-resolves | Moderate or persistent voice<br>changes; may require<br>occasional repetition but<br>understandable on telephone;<br>medical evaluation indicated | Severe voice changes including<br>predominantly whispered<br>speech | | |
| Definition: A disorder charact | erized by harsh and raspy voice arisin | g from or spreading to the larynx | | | 4 |
| Hypoxía | | Decreased oxygen saturation<br>with exercise (e.g., pulse<br>oximeter <88%); intermittent<br>supplemental oxygen | Decreased oxygen saturation at rest (e.g., pulse oximeter <88% or PaO2 <=55 mm Hg) | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charact | erized by a decrease in the level of or | rygen in the body. | | | |
| Laryngeal ederne | Asymptomatic: clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical intervention indicated (e.g., dexamethasone, epinephrine, antihistamines) | Stridor, respiratory distress,<br>hospitalization indicated | Life-threatening airway compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charact | erized by swelling due to an excessiv | e accumulation of fluid in the laryr | ix. | | |
| Laryngeal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder charact | erized by an abnormal communication | between the larynx and another | organ or anatomic site. | | |
| Laryngeal hemorrhage | Mild cough or trace hemoptysis;<br>laryngoscopic findings | Moderate symptoms; medical intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening airway compromise; urgent intervention indicated (e.g., tracheotomy or intubation) | Death |
| Definition: A disorder charact | erized by bleeding from the larynx. | | | | |
| Laryngeal inflammation | Mild sore throat; raspy voice | Moderate sore throat; | Severe throat pain; endoscopic | | |

| | | ratory, thoracic and med | The Mark Control of the Control of t | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | | 2 | 3 | 4 | 5 |
| Laryngeal mucositis | Endoscopic findings only; mild<br>discomfort with normal intake<br>ted by an inflammation involving the | Moderate discomfort; altered oral intake | Severe pain; severely altered<br>eating/swallowing; medical<br>intervention indicated | Life-threatening airway compromise; urgent intervention indicated (e.g., trachectomy or intubation) | Death |
| Laryngeal obstruction | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids); limiting instrumental ADL | Limiting self care ADL; stridor; endoscopic intervention indicated (e.g., stent, laser) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by blockage of the laryngeal ai | rway. | | | |
| Laryngeal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., noisy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g.,<br>steroids) | Limiting self-care ADL; stridor;<br>endoscopic intervention<br>indicated (e.g., stent, Jaser) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by a narrowing of the laryngea | l airway. | | | _ |
| Laryngopharyngeal dysesthesia | Mild symptoms; no anxiety;<br>intervention not indicated | Moderate symptoms; mild<br>anxiety, but no dyspnea; short<br>duration of observation and or<br>anxiolytic indicated; limiting<br>instrumental ADL | Severe symptoms; dyspinea and<br>swallowing difficulty; limiting self<br>care ADL | Life-threatening consequences | Death |
| Definition: A disorder characteriz | ed by an uncomfortable persisten | sensation in the area of the laryn | gopharynx. | | |
| Laryngospasm | | Transient episode; intervention not indicated | Recurrent episodes:<br>noninvasive intervention<br>indicated (e.g., breathing<br>technique, pressure point<br>massage) | Persistent or severe episodes<br>associated with syncope; urgent<br>intervention indicated (e.g.,<br>fiberoptic laryngoscopy,<br>intubation, botox injection) | Death |
| The state of the s | ed by paroxysmal spasmodic mus | | T. 10. 1 C. 10. 10 | 22.0 - 172-2 - 172-2 | D-15 |
| Mediastinal hemorrhage | Radiologic evidence only;<br>minimal symptoms; intervention<br>not indicated | Moderate symptoms; medical<br>intervention indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated<br>(e.g., hemostasis of bleeding<br>site) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the mediastin | um. | | | |
| Nasal congestion | Mild symptoms; intervention not indicated | Moderate symptoms; medical<br>intervention indicated | Associated with bloody nasal discharge or epistaxis | 5 | 7 |
| Definition: A disorder characteriz | ed by obstruction of the nasal pas | | | | |
| Pharyngeal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube thoracostomy or medical intervention indicated; limiting instrumental ADL | Severe symptoms; limiting self-<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ed by an abnormal communication | | | | |
| Pharyngeal hemorrhage | Mild symptoms; intervention not<br>indicated | Moderate symptoms; medical<br>intervention indicated | Transfusion, radiologic,<br>endoscopic, or operative<br>intervention indicated (e.g.,<br>hemostasis of bleeding site) | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder characteriz | ed by bleeding from the pharynx. | | | | |
| Pharyngeal mucositis | Endoscopic findings only;<br>minimal symptoms with normal<br>oral intake; mild pain but<br>analgesics not indicated | Moderate pain and analgesics<br>indicated; altered oral intake;<br>limiting instrumental ADL | Severe pain; unable to<br>adequately aliment or hydrate<br>orally, limiting self care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder characteriz | ed by an inflammation involving th | e mucous membrane of the phary | mx. | | |
| Pharyngeal necrosis | | - | Inability to aliment adequately<br>by GI tract; tube feeding or TPN<br>indicated; radiologic,<br>endoscopic, or operative | Life-threatening consequences;<br>urgent operative intervention<br>indicated | Death |

| | | ratory, thoracic and med | | | |
|---|---|---|---|---|---|
| | _ | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Definition: A disorder charact | erized by a necrotic process occurring | in the pharynx. | | | |
| Pharyngeal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., noisy airway<br>breathing), but causing no<br>respiratory distress; medical<br>management indicated (e.g.,<br>steroids); limiting instrumental<br>ADL | Limiting self care ADL; stridor;<br>andoscopic intervention<br>indicated (e.g., stent, laser) | Life-threatening airway compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charact | erized by a narrowing of the pharynge | eal airway. | | | |
| Pharyngo(aryngeal pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | | - |
| Definition: A disorder charact | erized by marked discomfort sensatio | n in the pharyngolaryngeal region | o I | | |
| Pleurál effusion | Asymptomatic: clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; intervention<br>indicated (e.g., diuretics or<br>limited therapeutic<br>thoracentesis) | Symptomatic with respiratory<br>distress and hypoxia; surgical<br>intervention including chest tube<br>or pleurodesis indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by an increase in amounts of fi | uid within the pleural cavity. Symp | toms include shortness of breath, | cough and marked chest discomf | ort. |
| Pleural hemorrhage | Asymptomatic; mild hemorrhage<br>confirmed by thoracentesis | pneumothorax; chest tube<br>drainage indicated | >1000 ml of blood evacuated;<br>persistent bleeding (150-200<br>ml/hr for 2 - 4 hr); persistent<br>transfusion indicated; elective<br>operative intervention indicated | Life-threatening respiratory or<br>hemodynamic compromise;<br>intubation or urgent intervention<br>indicated | Death |
| Definition: A disorder charact | erized by bleeding from the pleural ca | vity. | | | r - |
| Pleuritic pain | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL | 1 | - |
| | erized by marked discomfort sensatio | n in the pleura. | - | | |
| Pneumonitis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical<br>Intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; oxygen indicated | Life-threatening respiratory<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charact | erized by inflammation focally or diffu- | sely affecting the lung parenchym | 3, | | |
| Pneumothorax | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; intervention<br>indicated (e.g., tube placement<br>without sclerosis) | Sclerosis and/or operative<br>intervention indicated;<br>hospitalization indicated | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by abnormal presence of air in | the pleural cavity resulting in the | collapse of the lung. | | |
| Postnasal drip | Mild symptoms; intervention not indicated | An and the second secon | | | ŝ |
| Definition: A disorder charact | erized by excessive mucous secretion | in the back of the nasal cavity or | throat, causing sore throat and/or | coughing. | |
| Productive cough | Occasional/minimal production of sputum with cough | Moderate sputum production;<br>limiting instrumental ADL | Persistent or copious production of sputum; limiting self care ADL | | - |
| Definition: A disorder charact | erized by expectorated secretions upo | on coughing. | · | | |
| Pulmonary edema | Radiologic findings only;<br>minimal dyspnea on exertion | Moderate dyspnea on exertion;<br>medical intervention indicated;<br>limiting instrumental ADL | Severe dyspnea or dyspnea at<br>rest; oxygen indicated, limiting<br>self care ADL | Life-threatening respiratory<br>compromise, urgent intervention<br>or intubation with ventilatory<br>support indicated | Death |
| Definition: A disorder charact | erized by accumulation of fluid in the I | lung tissues that causes a disturbe | ance of the gas exchange that may | lead to respiratory failure. | |
| Pulmonary fibrosis | Mild hypoxemia, radiologic<br>pulmonary fibrosis <25% of lung<br>volume | Moderate hypoxemia; evidence of pulmonary hypertension; radiographic pulmonary fibrosis 25 - 50% | Severe hypoxemia; evidence of right-sided heart failure; radiographic pulmonery fibrosis >50 - 75% | Life-threatening consequences (e.g., hemodynamic/pulmonary complications); intubation with ventilatory support indicated; radiographic pulmonary fibrosis >75% with severe honeycombing | Death |
| | erized by the replacement of the lung | | | | ec con- |
| Pulmonary fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic: tube<br>thoracostomy or medical<br>management indicated; limiting<br>instrumental ADL | Limiting self care ADL:<br>endoscopic stenting or<br>operative intervention indicated | Life-threatening consequences:<br>urgent operative intervention<br>indicated | Death |

| | | ratory, thoracic and med | Grade | | |
|---|---|---|---|---|---|
| Automorphism | 1 | 2 | | 4 | 5 |
| Adverse Event | | | 3 | 4 | 3 |
| Pulmonary hypertension | Minimal dyspnea; findings on<br>physical exam or other<br>evaluation | Moderate dyspnea, cough;<br>requiring evaluation by cardiac<br>catheterization and medical<br>intervention | Severe symptoms, associated with hypoxemia, right heart failure; oxygen indicated | Life-threatening airway consequences; urgent intervention indicated (e.g. tracheotomy or intubation) | Death |
| Definition: A disorder charact | erized by an increase in pressure with | nin the pulmonary circulation due to | lung or heart disorder | 1 | |
| Respiratory failure | | * | | Life-threatening consequences;<br>urgent intervention, intubation;<br>or ventilatory support indicated | Death |
| Definition: A disorder charact<br>with an increase in arterial le | erized by impaired gas exchange by t<br>yels of carbon dioxide. | he respiratory system resulting in | hypoxemia and a decrease in oxy | genation of the tissues that may be | associate |
| Retinoïc acid syndrome | Fiuld retention; <3 kg of weight gain; intervention with fluid restriction and/or diuretics indicated | Moderate signs or symptoms,<br>steroids indicated | Severe symptoms.<br>hospitalization indicated | Life-threatening consequences; ventilatory support indicated | Death |
| Definition: A disorder charact<br>retinoic acid. | erized by weight gain, dyspnea, pleur | al and pericardial effusions, leuko | cytosis and/or renal failure origina | lly described in patients treated wit | h all-trans |
| Sinus disorder | Asymptomatic mucosal crusting;<br>blood-tinged secretions | Symptomatic stenosis or<br>edema/narrowing interfering<br>with airflow; limiting instrumental<br>ADL | Stenosis with significant nasal obstruction; limiting self care ADL | Necrosis of soft tissue or bone;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by involvement of the paranas | al sinuses. | | | |
| Sleep арпеа | Snoring and nocturnal sleep<br>arousal without apnelo periods | Moderate apnea and oxygen<br>desaturation; excessive daytime<br>sleepiness; medical evaluation<br>indicated; limiting instrumental<br>ADL | Oxygen desaturation:<br>associated with hypertension;<br>medical intervention indicated<br>limiting selfcare ADL | Cardiovascular or<br>neuropsychiatric symptoms;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder charact | erized by cessation of breathing for si | | | 1 | |
| Sneezing | Mild symptoms; intervention not indicated | Moderate symptoms; medical intervention indicated | 3 | • | -30 |
| | erized by the involuntary expulsion of | | | | |
| Sore throat | Mild pain | Moderate pain; limiting<br>instrumental ADL | Severe pain; limiting self care<br>ADL; limiting ability to swallow | 1 | - |
| Definition: A disorder charact | erized by of marked discomfort in the | throat | | | |
| Stridor | 0 | | Respiratory distress limiting self<br>care ADL; medical intervention<br>indicated | Life-threatening airway<br>compromise; urgent intervention<br>indicated (e.g., tracheotomy or<br>intubation) | Death |
| Definition: A disorder charact | erized by a high pitched breathing so | und due to laryngeal or upper airw | ay obstruction | | |
| Tracheal fistula | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; tube<br>thoracostomy or medical<br>intervention indicated; limiting<br>instrumental ADL | Severe symptoms; limiting self<br>care ADL; endoscopic or<br>operative intervention indicated<br>(e.g., stent or primary closure) | Life-threatening consequences;<br>urgent operative intervention<br>indicated (e.g., thoracoplasty,<br>chronic open drainage or<br>multiple thoracotomies) | Death |
| Definition: A disorder charact | erized by an abnormal communication | between the traches and another | organ or anatomic site. | | |
| Tracheal mucositis | Endoscopic findings only;<br>minimal hemoptysis, pain, or<br>respiratory symptoms | Moderate symptoms; medical<br>intervention indicated; limiting<br>instrumental ADL | Severe pain; hemorrhage or<br>respiratory symptoms; limiting<br>self care ADL | Life-threatening consequences:<br>urgent intervention indicated | Death |
| Definition: A disorder charact | erized by an inflammation involving th | e mucous membrane of the trache | ea. | | |
| racheal stenosis | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic (e.g., noisy airway breathing), but causing no respiratory distress; medical management indicated (e.g., steroids) | Stridor or respiratory distress<br>limiting self-care ADL;<br>endoscopic intervention<br>indicated (e.g., stent; laser) | Life-threatening airway compromise; urgent intervention indicated (e.g., trachectomy or intubation) | Death |

| | | | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 4 | 2 | 3 | 4 | -10 |
| Alopecia | Hair loss of <50% of normal for<br>that individual that is not<br>obvious from a distance but only<br>on close inspection; a different<br>hair style may be required to<br>cover the hair loss but it does<br>not require a wig or hair piece to<br>camouflage | Hair loss of >=50% normal for that individual that is readily apparent to others; a wig or hair piece is necessary if the patient desires to completely camouflage the hair loss; associated with psychosocial impact | | | T |
| Definition: A disorder charac | terized by a decrease in density of hair | compared to normal for a given i | ndividual at a given age and body | location. | |
| Body odor | Mild odor; physician intervention<br>not indicated; self care<br>interventions | Pronounced odor, psychosocial<br>impact; patient seeks medical<br>intervention | | | 3 |
| Definition: A disorder charac | terized by an abnormal body smell res | ulting from the growth of bacteria | on the body. | | |
| Bullous dermatitis | Asymptomatic; blisters covering <10% BSA | Blisters covering 10 - 30% BSA;<br>painful blisters; limiting<br>instrumental ADL | limiting selfcare ADL | Blisters covering >30% BSA;<br>associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| | terized by inflammation of the skin cha | | The second secon | | 1 |
| Dry skin | Covering < 10% BSA and no associated erythems or pruritus | Covering 10 - 30% BSA and<br>associated with erythema or<br>pruntus; limiting instrumental<br>ADL | Covering >30% BSA and associated with pruritus, limiting self-care ADL | | |
| Definition: A disorder charac | serized by flaky and dull skin; the pores | s are generally fine, the texture is | a papery thin texture. | | |
| Erythema multiforme | Target lesions covering <10%<br>BSA and not associated with<br>skin tenderness | Target lesions covering 10 -<br>30% BSA and associated with<br>skin lenderness | Target lesions covering >30%<br>BSA and associated with oral or<br>genital erosions | Target lesions covering >30%<br>BSA; associated with fluid or<br>electrolyte abnormalities; ICU<br>care or burn unit indicated | Death |
| Definition: A disorder charac<br>Erythroderma | terized by farget lesions (a pink-red rin | g around a pale center). Erythema covering >90% BSA without associated symptoms; limiting instrumental ADL | Erythema covering >90% BSA<br>with associated symptoms (e.g.,<br>prunitus or tenderness); limiting<br>self care ADL | Erythems covering >90% BSA with associated fluid or electrolyte abnormalities; ICU care or burn unit indicated | Death |
| Definition: A disorder charac | terized by generalized inflammatory er | ythema and exfoliation. The inflan | And the second s | | |
| Fat atrophy | Covering <10% BSA and asymptomatic | Covering 10 - 30% BSA and associated with erythema or tendemess; limiting instrumental ADL | Covering >30% BSA;<br>associated with erythema or | - | 2. |
| Definition: A disorder charac | terized by shrinking of adipose tissue. | P | 1 | 1 | |
| Hirsultism | In women, increase in length, thickness or density of hair in a male distribution that the patient is able to camouflage by periodic shaving, bleaching, or removal of hair | in women, increase in length,<br>thickness or density of hair in a<br>male distribution that requires<br>daily shaving or consistent<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial<br>impact | | | 9 |
| Definition: A disorder charac<br>androgen control (beard, mo | terized by the presence of excess hair<br>sustache, chest, abdomen) | growth in women in anatomic site | s where growth is considered to b | e a secondary male characteristic | and under |
| Hyperhidrosis | Limited to one site (palms,<br>soles, or axillae); self care<br>interventions | Involving >1 site; patient seeks<br>medical intervention; associated<br>with psychosocial impact | Generalized involving sites other than palms, soles, or axillae; associated with electrolyte/hemodynamic imbalance | | E. |
| | | | | | A. |

| | | in and subcutaneous tis | Grade | | |
|---|---|---|---|---|---|
| Adverse Event | 1 | 2 | Grade | 4 | 5 |
| Hypertrichosis | Increase in length, thickness or<br>density of hair that the patient is<br>either able to camouflage by<br>periodic shaving or removal of<br>hairs or is not concerned | Increase in length, thickness or<br>density of hair at least on the<br>usual exposed areas of the<br>body [face (not limited to<br>beard/moustache area) | | | |
| | enough about the overgrowth to<br>use any form of hair removal | plus/initius arms] that requires<br>frequent shaving or use of<br>destructive means of hair<br>removal to camouflage;<br>associated with psychosocial<br>impact | | | |
| | ized by hair density or length beyon | | a particular body region, for a part | icular age or race. | |
| Hypohidrosis<br>Definition: A disorder character | and by radiused supplier | Symptomatic; limiting<br>instrumental ADL | Increase in body temperature;<br>limiting self care ADL | Heat stroke | Death |
| Lipohypertrophy | Asymptomatic and covering | Covering 10 - 30% BSA and | Covering >30% BSA and | 2 | is . |
| ырчіўреніорпу | <10% BSA | associated tenderness; limiting | associated tenderness and<br>narcotics or NSAIDs indicated;<br>lipohypertrophy; limiting self<br>care ADL | | |
| Definition: A disorder character | ized by hypertrophy of the subcuter | eous adipose tissue at the site of | multiple subcutaneous injections | of insulin. | |
| Nail discoloration | Asymptomatic; clinical or diagnostic observations only: intervention not indicated | | 7 | | C |
| Definition: A disorder character | zed by a change in the color of the | nail plate. | | | |
| Nail loss | Asymptomatic separation of the nail bed from the nail plate or nail loss | Symptomatic separation of the<br>nail bed from the nail plate or<br>nail loss; limiting instrumental<br>ADL | - | | 1 |
| Definition: A disorder character | ized by loss of all or a portion of the | náil | Li . | | |
| Nail ridging | Asymptomatic; clinical or diagnostic observations only; intervention not indicated | | | | +1 |
| Definition: A disorder character | ized by vertical or horizontal ridges | on the nails | , i | | |
| Pain of skin | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain; limiting self care<br>ADL | É | ş |
| Definition: A disorder character | ized by marked discomfort sensatio | n in the skin. | | | |
| Palmar-plantar<br>erythrodysesthesia syndrome | Minimal skin changes or<br>dermatitis (e.g., erythema,<br>edema, or hyperkeratosis)<br>without pain | Skin changes (e.g., peeling,<br>blisters, bleeding, edema, or<br>hyperkeratosis) with pain;<br>limiting instrumental ADL | Severe skin changes (e.g.,<br>peeling, blisters, bleeding,<br>edema, or hyperkeratosis) with<br>pain; limiting self care ADL | | - |
| Definition: A disorder character | ized by redness, marked discomfort | , swelling, and tingling in the palm | s of the hands or the soles of the | feet. | |
| Periorbital edema | Soft or non-pitting | Indurated or pitting edema;<br>topical intervention indicated | Edema associated with visual disturbance, increased intraocular pressure, glaucoma or retinal hemorrhage, optic neuritis; diuretics indicated; operative intervention indicated | | 9 |
| Definition: A disorder character | ized by swelling due to an excessive | accumulation of fluid around the | orbits of the face. | | |
| Photosensitivity | Paintess erythema and erythema covering <10% BSA | Tender erythema covering 10 -<br>50% BSA | Erythema covering > 30% BSA<br>and erythems with blistering;<br>photosensitivity; oral<br>corticosteroid therapy indicated;<br>pain control indicated (e.g.,<br>narcotics or NSAIDs) | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Pruritus | Mild or localized; topical<br>intervention indicated | Intense or widespread,<br>intermittent; skin changes from<br>scratching (e.g., edema,<br>papulation, excoriations,<br>lichenification, oozing/crusts);<br>oral intervention indicated,<br>limiting instrumental ADL | Intense or widespread;<br>constant; limiting self-care ADL<br>or sleep; oral corticosteroid or<br>immunosuppressive therapy<br>indicated | | |
| Definition: A disorder charac | terized by an intense itching sensation | N | γ- | Т | |
| Purpura | Combined area of lesions covering <10% BSA | Combined area of lesions covering 10 - 30% BSA; bleeding with trauma | Combined area of lesions covering >30% BSA; spontaneous bleeding | | |
| Definition: A disorder character and eventually become a bro | terized by hemorrhagic areas of the skownish-yellow color. | in and mucous membrane, Newe | r lesions appear reddish in color, ( | Older lesions are usually a darker | purple colo |
| Rash acneiform | Papules and/or pustules covering <10% BSA, which may or may not be associated with symptoms of pruntus or tenderness | Papules and/or pustules covering 10 - 30% BSA, which may or may not be associated with symptoms of pruntus or tenderness; associated with psychosocial impact; limiting instrumental ADL | Papules and/or pustules covering >30% BSA, which may or may not be associated with symptoms of pruritus or tenderness; limiting self care ADL; associated with local superinfection with oral antibiotics indicated | Papules and/or pustules covering any % BSA, which may or may not be associated with symptoms of pruritus or tenderness and are associated with extensive superinfection with IV antibiotics indicated; lifethreatening consequences | Death |
| Definition: A disorder charac | terized by an eruption of papules and | pustules, typically appearing in fa- | ce, scalp, upper chest and back. | | |
| Rash maculo-papular Definition: A disorder charac | Macules/papules covering<br><10% BSA with or without<br>symptoms (e.g., prunius,<br>burning, lightness)<br>terized by the presence of macules (fil | Macules/papules covering 10 -<br>30% BSA with or without<br>symptoms (e.g., pruntus,<br>burning, tightness); limiting<br>instrumental ADL<br>at) and papules (elevated). Also k | Macules/papules covering<br>>30% BSA with or without<br>associated symptoms; limiting<br>self care ADL | of the most common cutaneous a | dverse |
| | he upper trunk, spreading centripetally | | | | |
| Scalp pain | Mild pain | Moderate pain; limiting instrumental ADL | Severe pain: limiting self care<br>ADL | - | 2 |
| Definition: A disorder charac | terized by marked discomfort sensatio | n in the skin covering the top and | the back of the head. | 1 | ř |
| Skin atrophy | Covering <10% BSA;<br>associated with telangiectasias<br>or changes in skin color | Covering 10 - 30% BSA;<br>associated with striae or<br>adnexal structure loss | Covering >30% BSA;<br>associated with ulceration | | |
| Definition: A disorder charac | terized by the degeneration and thinni | ng of the epidermis and dermis. | | | |
| Skin hyperpigmentation | Hyperpigmentation covering<br><10% BSA; no psychosocial<br>impact | Hyperpigmentation covering<br>>10% BSA; associated<br>psychosocial impact | | | Ť |
| Definition: A disorder charac | terized by darkening of the skin due to | excessive melanin deposition. | | | |
| Skin hypopigmentation | Hypopigmentation or<br>depigmentation covering <10%<br>BSA; no psychosocial impact | Hypopigmentation or<br>depigmentation covering >10%<br>BSA; associated psychosocial<br>impact | | | |
| Contailing A discoular shares | terized by loss of skin pigment. | | | | |
| Definition: A disorder charac | Mild induration, able to move<br>skin parallel to plane (sliding) | Moderate induration, able to<br>slide skin, unable to pinch skin;<br>limiting instrumental ADL | Severe induration, unable to slide or pinch skin; limiting joint movement or orifice (e.g., | Generalized, associated with<br>signs or symptoms of impaired<br>breathing or feeding | Death |
| Skin Induration | and perpendicular to skin<br>(pinching up) | arming insubmental ADC | mouth, anus); limiting self care<br>ADL | | |
| Skin induration | and perpendicular to skin | | The second secon | | |

| | Sk | in and subcutaneous tis | sue disorders | | |
|---|---|---|---|---|---|
| | Grade | | | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| Stevens-Johnson syndrome | | | Skin sloughing covering <10%<br>BSA with associated signs (e.g.,<br>srythema, purpura, epidermal<br>detachment and mucous<br>membrane detachment) | Skin sloughing covering 10 -<br>30% BSA with associated signs<br>(e.g., erythema, purpura,<br>spidermal detachment and<br>mucous membrane<br>detachment) | Death |
| | ized by less than 10% total body ski | in area separation of dermis. The | syndrome is thought to be a hyper | sensitivity complex affecting the s | kin and the |
| mucous membranes.<br>Telangiectasia | Telangiectasias covering <10%<br>BSA | Telangiectasias covering >10%<br>BSA; associated with<br>psychosocial impact | | | - |
| Definition: A disorder characte | ized by local dilatation of small vess | els resulting in red discoloration of | f the skin or mucous membranes. | | |
| Toxic epidermal necrolysis | | | - | Skin sloughing covering >=30%<br>BSA with associated symptoms<br>(e.g., erythema, purpura, or<br>epidermal detachment) | Death |
| en eller of an order to be a first | | | | | |
| Definition: A disorder character<br>mucous membranes | ized by greater than 30% total body | skin area separation or detinus. ) | ne syndrome is mought to be a ny | persensitivity complex affecting to | e skin and |
| | Unicarial lesions covering <10%<br>BSA; topical intervention<br>indicated | Urticarial lesions covering 10 -<br>30% BSA, oral intervention<br>indicated | Unicarial lesions covering >30%<br>BSA: IV intervention indicated. | | e skin and |
| mucous membranes.<br>Urticaria | Unicanal lesions covering <10%<br>BSA; topical intervention | Urticarial lesions covering 10 -<br>30% BSA; oral intervention<br>indicated | Unicarial lesions covering >30%<br>BSA: /V intervention indicated | | e skin and |

| | | Social circumsta | nces | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 1 |
| Menopause | Menopause occurring at age 46 - 53 years of age | Menopause occurring at age 40 - 45 years of age | Menopause occurring before<br>age 40 years of age | | - |
| Definition: A disorder characteri | zed by the permanent cessation of | menses, usually defined by 12 co | nsecutive months of amenorrhea | | |
| Social circumstances - Other, specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only, intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling; limiting self care ADL | Life-threatening consequences; urgent intervention indicated | Death |

| | | Surgical and medical | | | |
|---|---|---|---|---|---|
| | | 1 | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | - 6 |
| iurgical and medical<br>rocedures - Other, Specify | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disabling: limiting self-care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |

| | | Vascular disorde | ers | | |
|---|---|---|---|---|---|
| | | | Grade | | , |
| Adverse Event | 1 | 2 | 3 | 4 | 4 |
| Capillary leak syndrome | i. | Symptomatic; medical<br>intervention indicated | Severe symptoms; intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | ized by leakage of intravascular flui<br>k syndromes, low-flow states, ische | | | | |
| Flushing | Asymptomatic; clinical or diagnostic observations only, intervention not indicated | Moderate symptoms; medical intervention indicated; limiting instrumental ADL | Symptomatic, associated with<br>hypotension and/or tachycardia;<br>limiting self-care ADL | | 6 |
| Definition: A disorder character | ized by episodic reddening of the fa | ce. | | | - |
| Hematoma | Mild symptoms; intervention not indicated | Minimally invasive evacuation or<br>aspiration indicated | Transfusion, radiologic,<br>endoscopic, or elective<br>operative intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by a localized collection of bloc | d, usually clotted, in an organ, spa | ace, or tissue, due to a break in the | e wall of a blood vessel. | |
| Hot flashes | Mild symptoms; intervention not<br>indicated | Moderate symptoms; limiting instrumental ADL | Severe symptoms; limiting self care ADL | | 2 |
| Definition: A disorder character | ized by an uncomfortable and temp | orary sensation of intense body wa | rmth, flushing, sometimes accom | panied by sweating upon cooling. | |
| Hypertension | Prehypertension (systolic BP<br>120 - 139 mm Hg or diastolic<br>BP 80 - 89 mm Hg) | Stage 1 hypertension (systolic BP 140 - 159 mm Hg or diastolic BP 90 - 99 mm Hg); medical intervention indicated; recurrent or persistent (>=24 hrs); symptomatic increase by >20 mm Hg (diastolic) or to >140/90 mm Hg if previously WNL; monotherapy indicated Pediatric; recurrent or persistent (>=24 hrs) BP >ULN; monotherapy indicated | Stage 2 hypertension (systolic<br>BP >= 160 mm Hg or disatolic<br>BP >= 100 mm Hg); medical<br>the properties indicated; more<br>than one drug or more intensive<br>therapy than previously used<br>indicated<br>Pediatric: Same as adult | Life-threatening consequences (e.g., malignant hypertension, transient or permanent neurologic deficit, hypertensive crisis); urgent intervention indicated Pediatric: Same as adult | Death |
| Definition: A disorder character | ized by a pathological increase in b | ood pressure; a repeatedly elevat | on in the blood pressure exceeding | g 140 over 90 mm Hg. | |
| Hypotension | Asymptomatic, intervention not indicated | Non-urgent medical intervention indicated | Medical intervention or<br>hospitalization indicated | Life-threatening and urgent intervention indicated | Death |
| Definition: A disorder character | ized by a blood pressure that is belo | ow the normal expected for an indi | vidual in a given environment. | | |
| Lymph leakage | | Symptomatic; medical<br>intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | Life-threatening consequences;<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by the loss of lymph fluid into t | ne surrounding tissue or body cavi | ty. | | |
| Lymphedema | Trace thickening or faint discoloration | Marked discoloration; leathery<br>skin texture; papillary formation;<br>limiting instrumental ADL | Severe symptoms; limiting self care ADL | | Ť |
| Definition: A disorder character | ized by excessive fluid collection in | tissues that causes swelling. | | | _ |
| Lymphocele | Asymptomatic; clinical or<br>diagnostic observations only;<br>intervention not indicated | Symptomatic; medical intervention indicated | Severe symptoms; radiologic,<br>endoscopic or elective operative<br>intervention indicated | | - |
| Definition: A disorder character | ized by a cystic lesion containing ly | nph. | | | |
| Peripheral isohemia | 0 | Brief (<24 hrs) episode of<br>ischemia managed non-<br>surgically and without<br>permanent deficit | Recurring or prolonged (>=24<br>hrs) and/or invasive intervention<br>indicated | Life-threatening consequences;<br>evidence of end organ damage;<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by impaired circulation to an ex | tremity. | | | |
| Phlebitis<br>Definition: A disorder character | -<br>ized by inflammation of the wall of s | Present. | - | | = |
| Superficial thrombophlebitis | 8 | Present | - | 4 | - |
| | ized by a blood clot and inflammatic | | TYTEST B | | |

| | | Vascular disord | iers | | |
|---|---|---|---|---|---|
| | | | Grade | | |
| Adverse Event | 1 | 2 | 3 | 4 | 5 |
| | Asymptomatic; incidental finding<br>of SVC thrombosis. | intervention indicated (e.g.,<br>anticoagulation, radiation or<br>chemotherapy) | Severe symptoms; multi-<br>modality intervention indicated<br>(e.g., anticoagulation,<br>chemotherapy, radiation,<br>stenting)<br>and symptoms include swelling an | Life-threatening consequences;<br>urgent multi-modality<br>intervention indicated (e.g.,<br>lysis, thrombectomy, surgery)<br>d cyanosis of the face, neck, and | Death upper arms, |
| ough, orthopnes and headach | 1 | Very service and the | Table 1 | | Iv. |
| Thromboembolic event | Venous thrombosis (e.g., superficial thrombosis) | Venous thrombosis (e.g.,<br>uncomplicated deep vein<br>thrombosis), medical<br>intervention indicated | Thrombosis (e.g.,<br>uncomplicated pulmonary<br>embolism [venous], non-embolic<br>cardiac mural [orterial]<br>thrombus), medical intervention<br>indicated | Life-threatening (e.g.,<br>pulmonary embolism,<br>cerebrovascular event, arterial<br>insufficiency); hemodynamic or<br>neurologic instability; urgent<br>intervention indicated | Death |
| Definition: A disorder character | ized by occlusion of a vessel by a th | rombus that has migrated from a | distal site via the blood stream | | |
| /asculitis | Asymptomatic, intervention not indicated | Moderate symptoms, medical intervention indicated | Severe symptoms, medical intervention indicated (e.g., steroids) | Life-threatening; evidence of<br>peripheral or visceral ischemia,<br>urgent intervention indicated | Death |
| Definition: A disorder character | ized by inflammation involving the w | vall of a vessel. | | | |
| /isceral arterial ischemia | 9 | Brief (<24 hrs) episode of<br>ischemia managed medically<br>and without permanent deficit | Prolonged (>=24 hrs) or<br>recurring symptoms and/or<br>invasive intervention indicated | Life-threatening consequences;<br>evidence of end organ damage:<br>urgent operative intervention<br>indicated | Death |
| Definition: A disorder character | ized by a decrease in blood supply | due to narrowing or blockage of | visceral (mesenteric) artery. | | |
| Vascular disorders - Other, | Asymptomatic or mild<br>symptoms; clinical or diagnostic<br>observations only; intervention<br>not indicated | Moderate; minimal, local or<br>noninvasive intervention<br>indicated; limiting age-<br>appropriate instrumental ADL | Severe or medically significant<br>but not immediately life-<br>threatening; hospitalization or<br>prolongation of existing<br>hospitalization indicated;<br>disablind: limiting self-care ADL | Life-threatening consequences;<br>urgent intervention indicated | Death |
| | not indicated | appropriate instrumental AUL | | | |



# 16.12 Palatability Questionnaire

## LUM001 304 Palatability Questionnaire Caregiver Only

| Clinic Site Staff to capture the patient body weight: | and target dose (µg/kg): |
|---|---|
| Questionnaire to be completed by: | |
| Caregiver only for non-collaborating child (generally) | <4 years of age) |

 On the basis of reaction / facial expression of your child, do you think that the taste of the medication is acceptable?

Mark an X on the box below which best describes your answer.



2. Do you sometimes have problems in giving the medication to your child because he/she refuses to take it <u>because of the taste?</u>

Mark an X on the box below which best describes your answer.

| Yes | Not sure | No |
|-----|----------|----|

3. Based on its taste in the mouth, how easy or difficult it is for your child to take this medicine every day to treat the disease condition?
Mark an X on the box below which best describes your answer.

Very Easy

Easy

Neither Easy or Difficult

Very Difficult

Very Difficult

# LUM001 304 Palatability Questionnaire Child Only or Child and Caregiver

| Clinic Site Staff to capture the | natient body weight: | and target dose (µg/kg): |
|---|---|---|
| Clime Site Stan to capture the | paddit body wording. | and target acce (parky). |

#### Questionnaire to be completed by:

- Child only if >8 years age or
- · Caregiver & collaborating child if 4 to 8 years of age
- How does the medication taste immediately when you swallow it?
   Mark an X on the box below which best describes your answer.

| Very Good | Good | Nor good or<br>bad | Bad | Very Bad |
|-----------|------|--------------------|-----|----------|
| | | | (1) | |

How does the medication taste approximately 5 min after swallowing it? Mark an X on the box below which best describes your answer.



Based on the taste of this medication and how you felt in the mouth, would you take this medication
every day to treat the disease condition?
 Mark an X on the box below which best describes your answer.



### 16.13 Protocol History

| Document | Date | Global/Country/Site Specific |
|-------------------|-------------|------------------------------|
| Original Protocol | 20 Mar 2014 | |
| Amendment 1 | 06 Mar 2015 | Global |
| Amendment 2 | 08 May 2015 | Global |
| Amendment 3 | 13 Nov 2015 | Global |
| Amendment 4 | 28 Mar 2017 | Global |
| Amendment 5 | 06 Nov 2017 | Global |

## 16.13.1 Protocol Amendment 5 Summary of Changes

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BLIND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN APICAL SODIUM-DEPENDENT BILE ACID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 5

**Date:** 06 Nov 2017

The LUM001-304 protocol is being amended to change the study design going forward to an open label study, beyond what was previously described in Protocol Amendment 4. As all subjects have now either reached Week 48 or discontinued prior to Week 48, the interim analysis will be performed and the study will be unblinded.

In addition, in the Appendices, Study Schedule I and J have been updated to include clinician xanthoma scale.

The following changes have been made to the Protocol Amendment 4 (28 March 2017). Note that correction of typographical and grammatical errors are not captured in the below table.

*New text indicated in bold; deleted text indicated in strikethrough.* 

| Section | | | | | De | scripti | on of C | Change | | - | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Synopsis, Statistical | Interim An | alysis | | | | - | | | | | |
| considerations Interim Analysis | There will be an interim analysis (IA) conducted after all subjects complete or discontinue the study after Week 48 to guide the future of the program. At the IA the study will be unblinded. The IA may result in an interim report or publications. The IA will be conducted internally by an unblinded sponsor team as outlined in the unblinded study plan charter. The unblinded sponsor team will not be involved in the day to day clinical study activities | | | | | | | | | | |
| Subject Enrollment<br>6.4 Unblinding of<br>Treatment<br>Assignment | analysis. A schema. All subject the blind of subjects e emergency | ts will during ither where | receive the income the income | e LUM<br>initial<br>itinue<br>identity<br>ity mu | 1001, constant of the state of | or LUM ek per mplete e drug etermir | IOO1 an iod of Week must bed price | intain a d place the stu 48, ex be know | dy should acept in the vn in order omitting a re | his study. not occur e event of to proper | |
| Statistical<br>Considerations<br>Section 12.2.10<br>Interim Analyses | the study a unblinded conducted | fter W . The I interna | eek 48<br><del>A may</del><br><del>illy by</del> | to gui<br><del>result</del><br>an unl | de the<br>in an i | future of the fu | of the p<br><del>report</del><br>or team | rogram.<br><del>or publi</del><br>as outli | ubjects com At the IA cations. The ned in the to the day to | the study<br>e IA will b<br>inblinded s | will be<br>e<br>study plan |
| 16 Appendices | Insertion of clinician xanthoma scale | | | | | | | | | | |
| 16.1.3 Schedule of Procedures I – | Can be Deviced | | | Follo<br>Afterno | w-up Treatn<br>oon Dose Esc | ent Period<br>alation (ADE | ) | | Study activities re<br>after of | epeating in repeatin<br>ompletion of the AE | g 12-week periods<br>E period <sup>h</sup> |
| Long-Term | Study Period<br>FTP Study<br>Week | ADE<br>Day 0 | ADE<br>Week 1 | ADE<br>Week 2 | ADE<br>Week 4 | ADE<br>Week 5 | ADE<br>Week 6 | ADE<br>Week 8 | Week 4 | Week 8 | Week 12 |
| Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, | Scheduling<br>Considerations | To be scheduled as soon as ADE eligibility is confirmed and materials are on-site | | | | | | | The initial Week 4<br>contact will be<br>scheduled 4 weeks<br>following ADE<br>Week 8. | | |
| subject eligible for | Window (in<br>days)<br>Clinician | N/A - see<br>above | (±2) | (±2) | (±2) | | (±2) | (±2) | (±7) | (±7) | (±14)<br>X |
| ADE | Xanthoma Scale Caregiver ItchRO/ Patient ItchRO | X | | | X | | | X | | | X<br>(collected for 2<br>week period<br>following this<br>visit) |
| | PedsQL<br>Palatability | X | | | X | | | X | | | X<br>X |
| | Questionnaire<br>Study Drug | | | | v | | | v | | | X |
| | Supplied <sup>f</sup><br>Assess | X<br>X | | | X<br>X | | | X<br>X | | | X |
| | Compliance<br>Concomitant | X | Х | Х | X | Х | Х | X | X | X | X |
| | Medications Adverse Events Follow-up Phone | X | X | X | X | X | X | X | X | X | Х |
| 16 Appendices 16.1.4 Schedule of Procedures J – Study Termination and End of Treatment | Insertion o | f clinic | eian xa | nthom | a scale | X | Х | | X | X | |

| Section | | Description o | f Change |
|---|---|---|---|
| Procedures | Schedule of Procedures <u>J</u> – End of Treatment (EOT) / Early<br>Termination (ET) Visit and Post-Treatment Safety Follow Up | | |
| | | EOT / ET | Safety Follow Up |
| | Scheduling Considerations | To take place upon<br>completion of study or at<br>the time of early<br>withdrawal | Minimum of 30 days after final<br>dose |
| | Physical Exam | X | |
| | Body Weight & Height | X | |
| | Vital Signs <sup>a</sup> | X | |
| | CBC with Differential <sup>b</sup> | X | |
| | Coagulation <sup>b</sup> | X | |
| | Chemistry Panel <sup>b</sup> | X | |
| | Lipid Panel <sup>b,c</sup> | X | |
| | Cholestasis Biomarkers <sup>b,c</sup> | X | |
| | Fat Soluble Vitaminsb,c,d | X | |
| | Urinalysis <sup>b</sup> | X <sub>F</sub> | |
| | AFP Sample | X | |
| | Serum or Urine Pregnancy<br>Test (if indicated) <sup>e</sup> | X | |
| | Clinician Scratch Scale | X | |
| | Clinician Xanthoma Scale | X | |
| | PedsQL. | X | |
| | Patient/Caregiver<br>Impression of Change | X | |
| | Caregiver Global | X | |
| | Therapeutic Benefit Palatability Questionnaire | X | |
| | Assess Compliance | X | |
| | Concomitant Medications | X | X |
| | Adverse Events | X | X |
| | Follow-up Phone Contact <sup>f</sup> | | X |

### 16.13.2 Protocol Amendment 4 Summary of Changes

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BL<u>I</u>ND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN APICAL SODIUM-DEPENDENT BILE ACID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 4

**Date:** 28 Mar 2017

The changes below were made to Protocol Amendment 3.

The following table provides a summary list of changes that were included in Protocol Amendment 3 (*new text indicated in bold; deleted text indicated in strikethrough*):

| Section | Section Description of Change | |
|---|---|---|
| Cover page, Sponsor; | Changed from: | • |
| Title Page, Sponsor; Sponsor<br>Signature Page<br>Sponsor<br>Protocol Signature page, Sponsor | | Lumena Pharmaceuticals, Inc.<br>12531 High Bluff Drive, Suite 110<br>San Diego, CA 92130<br>USA |
| | То: | Lumena Pharmaceuticals LLC* 300 Shire Way |
| | | Lexington, MA 02421<br>USA |
| | | *Lumena Pharmaceuticals LLC is an indirect wholly-owned subsidiary of Shire North American Group, Inc |
| Title Page, Medical Lead; | Changed from: | |
| Protocol Signature page, Sponsor (Shire) Approval | Medical Lead: | Beatriz Caballero, MD Shire-Human Genetic Therapies, Inc. Zahlerweg 10 6300 Zug Switzerland Phone: +41(0) 41 288 42 30 Email: bcaballero@shire.com |
| | To: | |
| | Medical Lead: | Thomas Jaecklin, MD Shire Zahlerweg 10 6300 Zug Switzerland Phone: +41(0) 79 850 77 18 Email: thomas.jaecklin@shire.com |
| Emergency Contact Information | | nining emergency contact information for terse events (SAEs) to be aligned with Shire |
| Product Quality Complaints | Inserted new page containing product quality complaint information for reporting of investigational product quality complaints to be aligned with Shire protocol template. | |
| Synopsis, Objectives;<br>Section 3, Study Objectives | Objectives of <b>Long-term</b> Optional Follow-up Treatment Period (After Week 48): | |
| | study treatmen occurs: (i) up t or (ii) in the ev subjects are el LUM001 is av stops the prog | le subjects in the LUM001-304 study continued t after Week 48 until the first of the following o 52 weeks of additional treatment (Week 100) rent that a new study opens to enrollment (i) the ligible to enter another LUM001 study, (ii) railable commercially, or (iii) the sponsor gram or development in this indication. |
| | To explore tw<br>daily dosing o | ice a day (BID) dosing regimen and higher f LUM001. |

| Section | Description of Change |
|---|---|
| | • To assess the level of alpha-fetoprotein (AFP), a marker of |
| | hepatocellular carcinoma. |
| | <ul> <li>To assess palatability of the LUM001 formulation.</li> </ul> |
| Synopsis, Study Design; | The study is divided into <b>56</b> parts:a 12-week <b>open-label</b> stable |
| Section 5.1, Study Design | dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period at doses up to 400 µg/kg/day, and an a 52-week optional follow-up treatment period, and a long-term optional follow-up treatment period for eligible subjects who choose to stay on treatment with LUM001. |
| | During this long-term optional follow-up treatment period, subjects may have their dose of LUM001 increased to a maximum of 800 µg/kg/day (400 µg/kg BID), based on efficacy (sBA level and ItchRO [Obs] score) and safety assessment. |
| | Subjects' participation in the long-term optional follow-up treatment period will continue until the first of the following occur: (i) up to 52 weeks of additional treatment (Week 100) or (ii) in the event that a new study opens to enrollment (i) the subjects are eligible to enter another LUM001 study, (ii) LUM001 is available commercially, or (iii) the sponsor stops the program or development in this indication. Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3. |
| Synonsis Inclusion Criteria: | 5. Males and females of child-bearing potential who are |
| Synopsis, Inclusion Criteria;<br>Section 7.1, Inclusion Criteria | sexually active females, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must be prepared to agree and use an effective method ( $\leq 1\%$ failure rate) of acceptable contraception during the trial. Effective methods of contraception are considered to be described in Section 8.6.1. |
| | a. Hormonal (e.g., contraceptive pill, patch, intramuscular implant or injection); or |
| | b. Barrier method, e.g., (a) condom (male or female) or (b) diaphragm, with spermicide; or e. Intrauterine device (IUD). |
| Synopsis, Inclusion Criteria; | Protocol Amendment 4: Eligible Subjects for the long-term optional |
| Section 7.2, Exclusion Criteria | follow-up treatment period: |
| | Inclusion Criteria for subjects with LUM001 dosing interruption <7 days, or ≥7 days: |
| | Subjects will be considered eligible for the long-term optional |
| | follow-up treatment period if they meet the following criteria: |
| | <ol> <li>The subject has either: <ul> <li>completed the protocol through the Week 48 visit with no major safety concerns.</li> </ul> </li> </ol> |
| | OR |
| | o discontinued due to safety reasons judged unrelated to the study drug, and laboratory results have returned to levels acceptable for this patient population or individual and subject does not meet |

| Section | Description of Change |
|---|---|
| | entry into the follow-up period. The decision will<br>be made by the investigator in consultation with<br>the sponsor medical monitor. [Subjects who were<br>discontinued for other reasons will be considered<br>on an individual basis.] |
| | 2. Females of childbearing potential must have a negative urine or serum pregnancy test (β-hCG) at the time of entry into the long-term optional follow-up treatment period. |
| | <ol> <li>Males and females of child-bearing potential who are sexually active, or are not currently sexually active during the study, but become sexually active during the period of the study and 30 days following the last dose of study drug, must agree and use acceptable contraception during the trial.</li> <li>Informed consent and assent (per IRB/EC) as appropriate.</li> <li>Access to phone for scheduled calls from study site.</li> <li>Caregivers (and age appropriate subjects) must be willing and able to use an eDiary device during the study.</li> </ol> |
| | Exclusion Criteria for Subjects with LUM001 dosing interruption≥7 days: All exclusion criteria mentioned for the core study apply upon entry into the long-term optional follow-up period, with the exception of exclusion criterion #18. |
| Synopsis, Treatment Groups;<br>Section 5.5.2, Treatment; | Subjects will be considered for a 52-week optional treatment period, if eligible, receiving up to 400 µg/kg/day, or the highest tolerated dose below the 400 µg/kg/day dose. Subjects will then be considered for the long-term optional 52-week-follow-up treatment, if eligible, to continue on their highest tolerated dose receiving up to 800 µg/kg/day (given as twice daily doses of 400 µg/kg), or to a maximum possible daily dose of 50 mg/day. |
| Synopsis, Study Drug Dosage and<br>Administration; Section 10.1, Study<br>Drug Administration | Study Drug Administration Subjects who weigh 10 kg or more at screening will receive 1.0 mL a grape-flavored solution containing LUM001 or placebo. Subjects who weigh less than 10 kg at screening will receive 0.5 mL grape flavored solution containing LUM001. The volume administered, either 1.0 mL or 0.5 mL will not change during orally once a day (QD) or twice a day (BID) using the the course of the study. Each daily syringe provided. The first dose will should be administered in the morning taken at least 30 minutes prior to dinner (main evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the dose should be taken approximately at the same time every day each day for the duration of the treatment period. |
| | QD Dosing Regimen For QD dosing, the required dose will be delivered in 0.5 mL volume for subjects who weigh less than 10 kg and in 1.0 mL for subjects who weigh 10 kg or more. |

| Section | Description of Change |
|---|---|
| | BID Dosing Regimen For BID dosing, the required dose is delivered in half the dosing volume: 0.25 mL BID for subjects who weigh less than 10 kg and 0.50 mL BID for subjects who weigh 10 kg or more. For subjects weighing less than 10 kg at study entry, once a weight of 10 kg is reached while in the study, the subject will be moved from 0.5 mL maximum daily dosing volume (0.25 mL BID) to 1.0 mL maximum daily dosing volume (0.50 mL BID). |
| Section 5.5.2.1, Dose Escalation<br>Period | Study Drug Dosage Initially, the LUM0001 dose will be administered as a daily morning dose in either a 1.0 mL or 0.5 mL solution. The dose will be increased weekly over a 6-week period up to 400 µg/kg/day QD or a maximum daily dose of 20 mg/day QD as follows |
| Section 5.5.2.4, Long-term Exposure Period | Following the 4-week study drug randomized withdrawal period, subjects who received placebo will receive LUM001 dosed according to a dose escalation schedule that mirrors the initial escalation (ie the LUM001 dose will be increased weekly over a 6-week period to the maximum tolerated dose up to 400 µg/kg/day or a maximum daily dose of 20 mg/day or the highest tolerated dose below the 400 µg/kg/day dose). |
| Section 5.5.2.5, 52-week Optional Follow-up Treatment Period | Optional Follow-up Treatment Period At Week 48, all subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over into the 52 week, optional follow-up treatment period. The 3 following possible scenarios may occur: |
| | <ul> <li>Subjects who are eligible to roll over into the optional follow-up treatment period with a LUM001 dosing interruption of ≥7 days will be dose escalated beginning at 35 μg/kg/day and up to a maximum of 400 μg/kg/day or highest tolerated dose following a 5 week dose escalation beginning at 35 μg/kg/day.</li> <li>Subjects who do not wish to enter the follow-up treatment period will be contacted via telephone by the study site approximately 2830 days after the last dose of study drug.</li> </ul> |
| | During the study, the study drug may be adjusted if there is a change of ≥10% in weight since the screening visit or if there is a change of ≥10% in weight since the last weight based medication adjustment to maintain the target dose (µg/kg/day). |
| Section 5.5.2.6, Long-term Optional Follow-up Treatment Period | Long-term Optional Follow-up Treatment Period Upon completion of the 52-week follow-up treatment period and/or implementation of this amendment, whichever occurs first, subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over (or enter) into the long-term optional, |

| Section | Description of Change |
|---|---|
| | follow-up treatment period. The 3 following possible scenarios may |
| | occur: |
| | Scenario 1: Subjects eligible to roll over into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days: |
| | <ul> <li>Subjects with normal sBA level AND ItchRO(Obs) score</li> <li>&lt;1.5 will be maintained at the same dose level and will continue morning dosing only.</li> </ul> |
| | <ul> <li>Subjects with sBA level above normal AND/OR<br/>ItchRO(Obs) score ≥1.5 will start BID dosing (afternoon<br/>dose escalation; ADE) as follows:</li> </ul> |
| | <ul> <li>The morning dose will be continued at the same<br/>dose level, but the volume of the morning dose will<br/>be reduced by half at the same time that the<br/>afternoon dose is initiated.</li> </ul> |
| | O The afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a |
| | period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 µg/kg. |
| | Scenario 2: Subjects eligible to roll over into the long-term optional |
| | follow-up treatment period with a LUM001 interruption of ≥7 days: |
| | <ul> <li>First, the morning dose is escalated up to 400 μg/kg/day or<br/>highest tolerated dose following a 5-week dose escalation<br/>beginning at 35 μg/kg/day.</li> </ul> |
| | <ul> <li>Once the morning dose of 400 μg/kg or maximum tolerated</li> </ul> |
| | dose is achieved, sBA and ItchRO(Obs) score will be |
| | evaluated. Subjects with normal sBA AND ItchRO(Obs) score <1.5 after morning dose escalation will be maintained at the same dose level and will continue morning dosing only. Subjects with sBA above normal AND/OR |
| | ItchRO(Obs) score ≥1.5 will begin BID dosing |
| | (ADE) as follows: |
| | The morning dose will be continued at the<br>same dose level, but the volume of the<br>morning dose will be reduced by half at<br>the same time that the afternoon dose is<br>initiated. |
| | ■ The afternoon dose will be initiated at |
| | dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this |
| | dose level is tolerated, the afternoon dose |
| | will then be escalated to 400 μg/kg. |
| | The following parameters apply to both dosing scenarios outlined above: |
| | <ul> <li>The afternoon dose will only be initiated once the subject<br/>has been treated on stable morning doses for at least 4<br/>weeks.</li> </ul> |
| | The sBA value used for determination of ADE eligibility<br>will be the most recent available value collected within the |
| | will be the most recent available value confected within the |

| Section | Description of Change |
|---|---|
| | <ul> <li>prior 16 weeks. The ItchRO(Obs) score used for ADE eligibility will be derived from the most recent available 7-day interval of ItchRO(Obs) collected within the prior 16 weeks.</li> <li>The maximum daily dose will be 400 μg/kg BID, ie,</li> </ul> |
| | 800 μg/kg/day (up to a maximum possible daily dose of 50 mg/day). |
| | Scenario 3: Subjects who do not consent to Protocol Amendment 4 will continue their treatment as outlined in Protocol Amendment 3. |
| Synopsis, Rationale for Dose and Schedule Selection | During the study, the study drug may be adjusted if there is a change of ≥10% in body weight since the screening visit or if there is a change of ≥10% in weight since the last weight based medication adjustment to maintain the target dose. |
| | If a subject experiences intolerance due to gastrointestinal symptoms (eg, diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the sponsor medical monitor may lower the dose to a previously tolerated dose; later attempts to escalate the dose are permitted. If the subject is on a BID dosing regimen, dose lowering should first be attempted with the afternoon dose |
| | The dose may be down titrated, at the investigator's discretion and in consultation with the Sponsor Medical Monitor, for subjects experiencing intolerance to a given dose. |
| | Under Protocol Amendment 4, an afternoon dose is introduced for eligible subjects in the long-term optional follow up treatment period. LUM001 doses will be escalated over a period of 4-8 weeks up to a maximum dose of 400 µg/kg BID (or maximum tolerated dose). The afternoon dose is only initiated and escalated in subjects with elevated sBA and/or ItchRO(Obs) ≥1.5 on the maximum (or maximum tolerated) morning dose. |
| | This escalation regimen is supported by the safety profile observed in completed and ongoing clinical studies of LUM001. Twice daily dosing is used in this study based on the findings of a healthy volunteers study in adult males (Study SHP625-101), which demonstrated that bile acid levels in feces increase with escalating doses and twice-daily regimen of LUM001 (up to 100 mg QD and 50 mg BID). In this study, subjects who were randomized to LUM001 treatment, received 1 of 4 doses of LUM001 (10, 20, 50, 100 mg) during 7 days. No titration was used in this study. There was a dose-dependent increase in total fecal BA excretion. In addition, BID dosing (ie, 50 mg BID) led to a further increase in fecal BA excretion as compared to QD dosing (ie, 100 mg QD). It is therefore hypothesized that twice-daily dosing has the potential to allow for more complete target engagement throughout the day at the level of the distal ileum. |
| | The higher dosing level is also supported by favorable results from a juvenile toxicity study conducted in rats administered LUM001 for 43 days (post-natal day, PND21 through PND63). As expected |

| Section | Description of Change |
|---|---|
| | for a drug intentionally designed to be minimally absorbed, systemic LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies in adult rats. No adverse effects were observed on postnatal growth and development of offspring at the highest doses tested (200 mg/kg/day in males, 1000 mg/kg/day in females). This study was initiated in juvenile animals at PND21, which from a whole animal development perspective, is typically representative of a 2-year old child. However, given the fact that LUM001 is a minimally absorbed drug, of particular importance is the age at which the GI tract is considered functionally mature. In humans this is considered to have occurred by 12 months of age; likewise, postnatal maturation of the GI tract in rats occurs during the first 3 weeks of life. Therefore, results from this study can be used to support the dosing levels proposed here for children 12 months of age and older. |
| Synopsis, Study Visit Schedule and Procedures; Section 5.5 | Clarified titles of study design schemes and updated figures to reflect<br>the addition of the extended follow-up treatment period beyond what<br>was previously described in Protocol Amendment 3. |
| Synopsis only | For an individual subject, the study participation period will consist of a screening period of up to 4 weeks, a 48 week treatment period (a 6 week open-label, dose escalation period, a 12-week open-label stable dosing period, a 4 week randomized, double blind, placebo controlled drug withdrawal period, and a 26 week long term exposure period), and a follow-up period of up to 4 weeks. Subjects who complete 48 weeks of treatment and those subjects who were previously treated with LUM001 may be eligible to receive treatment for up to 52 weeks during the optional follow-up treatment period. |
| Synopsis, Study Visit Schedule and<br>Procedures;<br>Section 8.1.1, Screening Period (Day -<br>28 to -1) | Screening Period (Day -28 to Day -1): For subjects who do not have documentation of a JAGGED-1 or <b>NOTCH2</b> mutation, a blood sample will may be obtained for genotyping. |
| Synopsis, Study Visit Schedule and Procedures; Section 8.1.9, Long-term Optional Follow-up Treatment Period | In addition the following assessments should be completed: the ItehRO (Pt and Obs), the clinician scratch scale, the clinician xanthoma scale, the PedsQL, the Patient Impression of Change (PIC), the CIC, the Caregiver Impression of Change, the CGTB, Caregiver Global Therapeutic Benefit assessments, and the palatability questionnaire, as defined for ET Early Termination. Efforts must be made to follow. For subjects for at least 4 weeks following their last dose of who complete the study drug, an EOT visit will be completed; the assessments performed at this visit will be identical to the assessments performed at the ET visit. |
| Section 8.1.8 (only, not synopsis), 52-<br>week Optional Follow-up Treatment<br>Period | 52-week Optional Follow-up Treatment Period post Week 48 to Week 100): Subjects who are eligible to roll over onto into the 52-week optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7days will be maintained at the same dose level within the 52-week optional follow-up treatment period (Figure 4). |

| Section | Description of Change |
|---|---|
| Synopsis, Study Visit Schedule and Procedures; | will continue to receive study drug at the dose they were receiving at Week 48 for up to 52 weeks of additional treatment or in the event that a new study opens to enrollment, whatever occurs first. |
| | Subjects who are eligible to roll over into the follow up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level. During the this-follow-up treatment period, subjects will return to the clinic at Weeks 60, 72, 84, 96, and 100; and telephone contacts to will occur at Weeks 52, 56, 64, 68, 76, 80, 88, and 92. |
| | Long-term Optional Follow-up Treatment Period Upon completion of the additional 52-week follow up treatment period and/or implementation of this amendment, whichever occurs first, subjects who are eligible to roll over onto the long-term optional follow-up treatment period will continue to receive study drug until the first of the following occurs: i. The subjects are eligible to enter another LUM001 study, ii. LUM001 is commercially available, or iii. The sponsor stops the program or development of this indication. |
| Section 8.1.9 (only, not synopsis),<br>Long-term Optional Follow-up<br>Treatment Period | Once Protocol Amendment 4 is implemented at the site, a determination about ADE will be made. Subjects who are eligible to roll over from the 52-week follow-up treatment period into the long-term optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days prior to implementation of Protocol Amendment 4 will be consented and evaluated for eligibility for ADE. Once a determination about ADE has been made, the subject will then either initiate the ADE (Synopsis Figure 6) or continue receiving the same dose of LUM001 once a day (Synopsis Figure 5), depending on whether they meet criteria for initiating ADE. Screening evaluations for subjects with ≥7 days since last dose of LUM001 prior to implementation of Protocol Amendment 4 will be performed from Day -14 to Day -1. After obtaining informed consent (and/or assent when appropriate), subjects will undergo a physical examination including body weight, height, and vital signs, and have blood and urine samples taken for clinical laboratory testing. Females who are of childbearing potential will have a serum pregnancy test. Eligibility criteria will be confirmed prior to the Baseline Visit. The clinician scratch scale and clinician xanthoma scale will be completed. Concomitant medications and any adverse events will be recorded. Rescreening: If a subject is unable to complete the screening procedures and meet eligibility criteria within the 14-day screening period, consideration may be given to rescreening at a later date. Screening procedures should be repeated at that time. Subject data pertaining to screening will be collected after the subject has been rescreened and determined to meet eligibility. |

| Section | Description of Change |
|---|---|
| | Subjects with ≥7 days since last dose of LUM001 prior to |
| Synopsis, Study Visit Schedule and | implementation of Protocol Amendment 4 will be dose escalated up |
| Procedures; Section 8.1.9, Long-term | to 400 µg/kg/day or to the highest tolerated dose beginning at Dose |
| Optional Follow-up Treatment Period | Level 2 (35 μg/kg/day), as outlined in Synopsis Figure 4 (or Figure 6 |
| | for body of protocol). The dose escalation (DE) period will proceed as follows: |
| | Protocol Amendment 4 DE-2 Clinic Visit: obtain consent, |
| | weight, and draw blood for laboratory analyses |
| | Protocol Amendment 4 DE Day 0 Clinic Visit: investigator |
| | evaluates laboratory results, study drug is dispensed, and |
| | subject begins at 35 μg/kg/day dose level (if no safety |
| | concerns) |
| | <ul> <li>Protocol Amendment 4 DE Week 1 Telephone Contact:</li> </ul> |
| | subject escalates to 70 μg/kg/day dose level |
| | Protocol Amendment 4 DE Week 2 Telephone Contact: |
| | subject escalates to 140 µg/kg/day dose level if prior dose level was tolerated |
| | • Protocol Amendment 4 DE Week 3 Telephone Contact:<br>subject escalates to 280 µg/kg/day dose level if prior dose |
| | level was tolerated |
| | Protocol Amendment 4 DE Week 4 Clinic Visit: laboratory |
| | tests and dose escalates to 400 μg/kg/day dose (maximum |
| | daily dose of 20 mg), if prior dose level was tolerated |
| | <ul> <li>Protocol Amendment 4 DE Week 8 Telephone Contact:</li> </ul> |
| | eligibility for ADE will be determined. |
| | Subjects not eligible for ADE (subjects with normal sBA level AND ItchRO(Obs) score <1.5), will be maintained at the same dose level and will continue morning dosing only. Subjects will have study activities repeated in repeating 12-week periods as follows, until study completion or termination: |
| | Repeating Period Week 4 Telephone Contact (ie, beginning 4 weeks after consent to Protocol Amendment 4): Collection of concomitant medications and any adverse events. |
| | • Repeating Period Week 8 Telephone Contact: Collection of concomitant medications and any adverse events. |
| | Repeating Period Week 12 Clinic Visit: Physical exam, body weight and height, vital signs, and blood samples for clinical laboratory testing including fasting lipid panel. Blood will also be collected for determination of baseline fat-soluble vitamins. Urine samples for clinical laboratory testing will be collected at every other visit. ItchRO compliance will be assessed, the electronic diary will be issued, the clinician scratch scale and clinician xanthoma scale will be administered, and the PedsQL questionnaire will be administered. Additionally, a palatability questionnaire will be completed. Female subjects who are of childbearing potential will have a urine pregnancy test |
| | prior to dispensing study drug. Study drug compliance will |

| Section | Description of Change |
|---|---|
| | be assessed and study drug will be dispensed. Concomitant |
| | medications and adverse events will be collected. |
| | • Subjects who do not qualify for ADE may be assessed at a later time point on a case by case basis following discussions between the investigator and medical monitor. Such re-evaluations may only occur at the Week 12 visit of any Repeating Period beginning with RP2. If in the course of the ADE re-evaluation, a subject is found to qualify for ADE, then the subject will move into Schedule F or G, as outlined in Section 16.1. During the follow-up treatment period, subjects will return to the clinic every 3 months. |
| | Subjects eligible for ADE,( ie, who have sBA level above normal AND/OR ItchRO(Obs) score ≥1.5), will begin BID dosing (afternoon dose escalation; ADE) as follows (see Figure 8): |
| | • On ADE Day 0, morning dosing will continue at 400 µg/kg or the maximum tolerated dose. However, the volume of the morning dose will be reduced by half. Of note: Morning dosing must have been stable for ≥4 weeks prior to initiation of ADE. |
| | • On ADE Day 0, the afternoon dose will be initiated at dose level 140 μg/kg and will continue at this dose for a period of 4 weeks. If this dose level is tolerated, the afternoon dose will then be escalated to 400 μg/kg. |
| | The following procedures will occur during the ADE period: |
| | ADE Day 0 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The clinician scratch scale, clinician xanthoma scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and any adverse events will be collected. |
| | <ul> <li>ADE Week 1 and Week 2 Telephone Contact: Collection of<br/>concomitant medications and any adverse events.</li> <li>Subject/caregiver will be reminded of dosing instructions.</li> </ul> |
| | ADE Week 4 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The clinician scratch scale, clinician xanthoma scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be |

| Section | Description of Change |
|---|---|
| | assessed and study drug will be dispensed. Concomitant |
| | medications and any adverse events will be collected. |
| | ADE Week 5 and Week 6 Telephone Contact: Collection of |
| | concomitant medications and any adverse events. |
| | Subject/caregiver will be reminded of dosing instructions. |
| | ADE Week 8 Clinic Visit: Physical exam, body weight and height, vital signs, and blood and urine samples for clinical laboratory testing, including fasting lipid panel. Blood will also be collected for determination of fat-soluble vitamins. Plasma sample will be obtained for LUM001 pharmacokinetics. The clinician scratch scale, clinician xanthoma scale, and the PedsQL questionnaire will be administered. Female subjects who are of childbearing potential will have a urine pregnancy test prior to dispensing study drug. Study drug compliance will be assessed and study drug will be dispensed. Concomitant medications and any adverse events will be collected. |
| | If any subject experiences intolerance, the investigator, in consultation with the sponsor medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period; later attempts to escalate the dose are permitted. At the investigator's discretion, and in consultation with the sponsor medical monitor subjects who were previously down titrated may be rechallenged during the follow-up treatment period. If the subject is on a twice daily dosing regimen, dose lowering should be first attempted with the afternoon dose. |
| | Safety and clinical laboratory evaluations, and PedsQL will be administered and study drug compliance will be assessed (PedsQL will not be performed at DE-2 or DE52).certain clinic visits – please refer to schedule of procedures). The Patient and Caregiver Impression of Change (PIC & CIC), and the Caregiver Global Therapeutic Benefit assessments will be completed at Weeks 84, 96, and 100. Subjects/caregivers will receive follow up phone calls at Weeks 64, 68, 76, 80, 88, and 92.100, and the End of Treatment (EOT)/Early Termination (ET) visit. Palatability data will be collected at each clinic visit during the long-term optional follow up treatment period (including the EOT/ET visit), with the exception of the PA4 DE, and ADE visits. Plasma samples will be obtained for LUM001 pharmacokinetics at the ADE Day 0, ADE Week 4, and ADE Week 8 visits, and at the 3 scheduled clinic visits following completion of the ADE period. Subjects/caregivers will receive follow-up phone calls at Weeks 64, 68, 76, 80, 88, 92, as well as those outlined within the PA4 DE, ADE, and repeating 12-week periods. |
| | Twice daily completion of the electronic diary will be required by caregivers and age appropriate subjects during the 2 weeks following the Week 60, 72, 84, and 96 clinic visits, at PA4 DE Week 4, and every clinic visit within the repeating 12-week periods. |
| | With the exception of the Week 96 and Week 100-EOT/ET visit (Study |

| Section | Description of Change |
|---|---|
| | Termination), |
| | Subjects will be encouraged to complete all study activities and visits. Any subject who withdraws from the study prior to completion of all treatment period clinic visits should undergo safety and clinical laboratory evaluations, including <b>pharmacokinetic sampling of LUM001</b> , determination of serum bile acids, other cholestasis biochemical markers, fat soluble vitamins, and plasma drug level. AFP. In addition the following assessments should be completed: the ItehRO (Pt and Obs), the clinician scratch scale, clinician xanthoma scale, the PedsQL, the Patient Impression of ChangePIC, the CIC, the Caregiver Impression of Change CGTB, and the Caregiver Global Therapeutic Benefit palatability questionnaire, as defined for Early Termination. Efforts must be made to follow (ET). For subjects for at least 4 weeks following their last dose of who complete the study drug., an EOT visit will be completed; the assessments performed at this visit will be identical to the assessments performed at the ET visit. At Following completion of the Follow-up Treatment Period or early discontinuation: a safety follow-up phone call will be made 4 weeks 30 days after the last dose of study drug (Week 100). |
| Synopsis, Safety and Tolerability; | Alpha-fetoprotein (AFP), a marker of hepatocellular carcinoma, will be measured every 6 months throughout the optional extension period. |
| Synopsis, Study Visit Schedule and Procedures; Section 8.1.9, Long-term Optional Follow-up Treatment Period | Plasma samples will be obtained for LUM001 pharmacokinetics at the ADE Day 0, ADE Week 4, and ADE Week 8 visits, and at the 3 scheduled clinic visits following completion of the ADE period. |
| Synopsis, Safety Evaluations | <ul> <li>The following assessments will be used to evaluate safety:</li> <li>Adverse events (AEs) and serious adverse events (SAEs).</li> <li>Clinical laboratory results, including alpha-fetoprotein (AFP) as a screening for hepatocellular carcinoma.</li> <li>Vital signs.</li> <li>Physical exam findings, including body weight and height.</li> <li>Concomitant medication usage.</li> </ul> |
| Synopsis, Efficacy Evaluations;<br>Section 12.2.5.1, Efficacy Variables | The primary efficacy-evaluation endpoint will be the mean change in from Week 18 to 22 of fasting serum bile acid levels from Week 18 to Week 22 for those who in subjects who previously responded to LUM001 treatment, which is as defined as subjects who had by a >50% reduction serum bile acid levels sBA>70% from baseline to Week 12 or Week 18. A sensitivity analysis will also be conducted using subjects who experienced a reduction from baseline in serum bile acids of ≥50% at the Week 48 measurement. □ Pruritus as measured by ItchRO (Observer ItchRO/patient ItchRO).) in subjects who previously responded to LUM001 |
| | treatment, as defined by a reduction in ItchRO scale >1 point from baseline to Week 12 or Week 18. Change from baseline to Weeks 18, 22 48, and 48 then every |

| Section | Description of Change |
|---|---|
| | 12 weeks in: |
| | Evaluations will be the mean-Change from Baseline (Day 0) to Week 18, prior to randomization, and the change from Week 18 to Week 48 and Week 18 to Week 100 in: Biochemical markers of cholestasis and liver disease [alanine aminotransferase (ALT), alkaline phosphate (ALP), gamma-glutamyltransferase (GGT) and bilirubin (total and direct)]. |
| | <ul> <li>Pruritus as measured by the electronic diary ItchRO instruments (ItchRO(Obs), caregiver instrument/ItchRO(Pt) patient instrument).</li> </ul> |
| | The change from Baseline (Day 0) to Week 48 in xanthomas, as measured by clinician xanthoma scale will also be evaluated. |
| | Additional assessments of efficacy variables will occur during the 52-week optional treatment period. For subjects entering the 52-week optional treatment period with $\geq 7$ days since last dose of LUM001, in 12 weekly intervals. Any of the above evaluations may also occur at clinic visits during the DE-period, PA4 DE, and ADE periods. |
| Synopsis, Palatability Data; | Palatability data will be collected at each clinic visit in the follow up |
| Section 12.2.9, Palatability Analyses | treatment period, with the exception of the DE, PA4 DE, and ADE visits. A palatability questionnaire will be completed by the subject and/or caregiver (dependent on age). Assessment of change over |
| Section 16.12, Palatability<br>Questionnaire | time will be evaluated. Baseline will be defined as the first recorded evaluation. |
| | Added palatability questionnaire |
| Section 8.5.8, Palatability | A palatability questionnaire (see Section 16.12) will be completed by the subject and/or caregiver (dependent on age) at clinic visits at time points as outlines in the Schedule of Procedure in Section 16.1 |
| Synopsis, Statistical Considerations | Safety measures including AEs, clinical laboratory tests, vital signs, physical exams, and concomitant medication usage will be summarized descriptively by study period and over the entire study duration (Weeks 0-48). <b>EOT Visit</b> ). |
| Section 12.2.10, Statistical Considerations | Interim Analysis There will be an interim analysis (IA) conducted after all subjects complete or discontinue the study after Week 48 to guide the future of the program. The IA may result in an interim report or publication. The IA will be conducted internally by an unblinded sponsor team as outlined in the unblinded study plan charter. The unblinded sponsor team will not be involved in the day-to-day clinical study activities. |
| Section 4.4.1.3, Toxicology | The results from this study were very favorable. As expected for a drug intentionally designed to work in the intestinal lumen and to be minimally absorbed, LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies with adult rats. |
| Section 4.5, Rationale for Dose and | Updated Sample Daily Exposure (mg/day) in Pediatric Subjects table. |

| Section | Description of Change |
|---|---|
| Schedule of Administration | In the current study, safety and efficacy of LUM001 will be assessed in children with ALGS and cholestatic liver disease, 12 months of age and older. The highest dose is equivalent to less than the well tolerated 1 mg dose used in Study 014 (~17 µg/kg, 60 kg body weight), where only two subjects reported moderate or severe GI associated AEs during 14 days. On a weight basis, 23 subjects received a dose approximately $\geq$ 14 µg/kg/day. The highest starting dose in Study 014 was 168 µg/kg/day. To reduce the risk of loose stools and diarrhea in subjects in study LUM001-304, the LUM001 dose will be escalated over an up to 6-week period; dosing will start at 14 µg/kg/day, and will then be increased at 7 day intervals to 35 µg/kg/day, 70 µg/kg/day, 140 µg/kg/day, 280 µg/kg/day, and 400 µg/kg/day (equivalent to 20 mg daily dose in a 50 kg subject). |
| | The doses explored in the current study (up to 400 µg/kg/day BID) in subjects with ALGS are supported by the safety profile observed in completed and ongoing clinical studies of LUM001. Twice daily dosing is used in this study based on the findings of a healthy volunteers study in adult males (Study SHP625-101), which demonstrated that bile acid levels in feces increase with escalating doses and twice-daily regimen of LUM001 (up to 100 mg QD and 50 mg BID, respectively). In this study, subjects who were randomized to LUM001 treatment, received 1 of 4 doses of LUM001 (10, 20, 50, 100 mg) during 7 days. No titration was used in this study. There was a dose-dependent increase in total fecal BA excretion. In addition, BID dosing (i.e. 50 mg BID) led to a further increase in fecal BA excretion as compared to QD dosing (i.e. 100 mg QD). It is therefore hypothesized that higher doses and twice-daily dosing both have the potential to allow for more complete target engagement throughout the day at the level of the distal ileum. The higher dosing level is also supported by favourable results from a juvenile toxicity study conducted in rats administered LUM001 for 43 days (PND21 through PND63). As expected for a drug intentionally designed to be minimally absorbed, systemic LUM001 exposure was very low and consistent with levels that were previously determined in several oral gavage studies in adult rats. No adverse effects were observed on postnatal growth and development of offspring at the highest doses tested (200 mg/kg/day in males, 1000 mg/kg/day in females). This study was initiated in juvenile animals at PND21, which from a whole animal development perspective, is typically representative of a 2-year old child. However, given the fact that LUM001 is a minimally absorbed drug, of particular importance is the age at which the GI tract is considered functionally mature. In humans this is considered to have occurred by 12 months of age; likewise, postnatal maturation of the GI tract in rats occurs during the first 3 w |
| Section 5.1, Study Design | At Week 48, all subjects will be assessed by the investigator to determine their willingness and eligibility to roll over into the 52 week, optional follow up treatment period. The 3 following possible scenarios |

| Section | Description of Change |
|---|---|
| | may occur: |
| | For subjects who are eligible to roll over into the follow up |
| | treatment period, those with <7 days since the last dose of |
| | LUM001 will be maintained at the highest tolerated dose at Week 48. |
| | • For subjects who are eligible to roll over into the follow up treatment period, those with ≥7 days since the last dose of LUM001 will be dose escalated up to 400 μg/kg/day or highest tolerated dose following a 5 week dose escalation beginning at 35 μg/kg/day. |
| | For subjects who do not wish to enter the follow up treatment |
| | period, or are not eligible to enter the follow up treatment |
| | period, a safety follow up phone call will be made by the study |
| | site 28 days after the last dose of study drug |
| Section 5.5, Overall Study Duration and Follow-up | For an individual subject, the duration of the study, including subject participation period will consist of a screening, period of up to 4 weeks, a 48-week treatment period (including a 6-week, open-label, dose escalation period, a 12-week open-label stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, safety a 26-week long-term exposure period) as well as a 52-week optional follow-up treatment period, and a long-term optional treatment period. A safety follow-up is expected to phone call will be approximately 56 weeks. made by the study site |
| | 30 days after the last dose of study drug. |
| Section 5.5.2, Treatment | Study drug will be dispensed to subjects/caregivers at the study. During the course of the study, it may be necessary to instruct the subject/caregiver to return to the site—for an unscheduled dispensation of study drug. |
| | Subjects who weigh 10 kg or more at screening will receive a 1.0 mL grape flavored solution per day containing LUM001 Subjects who weigh less than 10 kg at screening will receive a 0.5 mL grape flavored solution per day containing LUM001. The daily volume administered will not change during the course of the study. Dosing will occur over a 48 week treatment period. Each daily dose will be administered in the morning at least 30 minutes before breakfast (qAM, ac). Study drug should be administered approximately at the same time every day. |
| | Subjects will receive a grape-flavored solution containing LUM001 administered orally once a day (QD) or twice a day (BID) using the syringe provided. The first dose should be taken at least 30 minutes prior to the first meal of the day and the second dose, where applicable, should be taken at least 30 minutes prior to dinner (main evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the dose should be taken approximately at the same time each day for the duration of the treatment period. |
| | All subjects will receive LUM001, up to 400 μg/kg/day or a maximum daily dose of 20 mg/day during the initial open-label |

| Section | Description of Change |
|---|---|
| | treatment period of the study. After completion of the 12-week stable dosing period, subjects will be randomized 1:1 to either a 4-week double-blind study drug withdrawal period during the study or will remain on study drug. Subjects will then enter a 26-week long-term stable dosing period and all subjects will receive LUM001, up to 400 $\mu g/kg/day$ or a maximum daily dose of 20 mg/day during the initial open-label treatment period of the study. Subjects will then be considered for an optional follow-up treatment, if eligible, to continue on their highest tolerated dose receiving up to 800 $\mu g/kg/day$ (given as twice daily doses of 400 $\mu g/kg$ ), or a maximum possible daily dose of 50 mg/day. |
| Section 5.5.2.1, Dose Escalation<br>Period | Initially, the LUM001 dose will be <b>administered as a daily morning dose in either a 1.0 mL or 0.5 mL solution. The dose will be</b> increased weekly over a 6-week period up to 400 g/kg/day <b>QD</b> or a maximum daily dose of 20 mg/day <b>QD</b> as follows |
| Section 5.5.2.4, Long-term Exposure<br>Period | During the long-term exposure period, the dose may be adjusted to account for a change of ≥10% in weight since the screening visit (e.g. the amount of drug dosed may be increased to reflect the subject's weight increase). |
| Section 5.5.2.6, Long-term Optional Follow-up Treatment Period | Subjects who are eligible to roll over into the <b>optional</b> follow-up treatment period, those with <7 days since the last dose of will continue treatment under dosing scenarios based on whether their LUM001 will be maintained at the highest tolerated dose at Week 48 dosing will continue 1) without interruption/interruption of <7 continuous days, or 2) with interruption ≥7 days. Eligibility for BID dosing will be determined based on efficacy as measured by sBA level and ItchRO score. The 2 following dosing scenarios may occur. |
| Section 5.5.3, Safety Follow-up Period | A safety follow-up phone call will be made by the study site 2830 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and any AEs noted during this phone call will be recorded. Subjects who complete the study or who discontinued early due to reasons other than safety may be eligible for participation in the optional follow-up treatment period under Protocol Amendment 4. If any subject experiences intolerance, the investigator, in consultation with the Sponsor Medical Monitor, may lower the dose to a previously tolerated dose at any time during the entire follow up treatment period. At the investigator's discretion, and in consultation with the Sponsor Medical Monitor, subjects who were previously down titrated may be re-challenged during the follow up treatment period. During the follow up treatment period, subjects will return to the clinic at Weeks 60, 72, 84, 96, and 100. Safety and clinical laboratory evaluations and a physical exam (including collection of vital signs, height and weight measurements) will be completed at each clinic visit. In addition, the clinician scratch scale, clinician xanthoma scale, and PedsQL (clinician xanthoma scale and Peds QL will not be evaluated at DE 2 and DE 52) will be administered and study drug compliance will be assessed. The Patient and Caregiver Impression of Change (PIC & CIC), and the Caregiver Global Therapeutic Benefit assessments will be completed at Weeks 84, 96, and 100. Subjects/caregivers will receive follow up phone calls at Weeks 64, 68, 76, 80, 88, and 92. Concomitant medications and any |

| Section | Description of Change |
|---|---|
| | AEs will be evaluated and recorded at all clinic visits and at scheduled telephone contacts. |
| | Twice daily completion of the electronic diary will be required by |
| | caregivers and age appropriate subjects during the 2 weeks following |
| | the Week 60, 72, 84, and 96 clinic visits. Electronic diaries will be |
| | provided to subjects and caregivers at these visits and re training on the use of the diary will occur, as appropriate. |
| | At the physician investigator's discretion, withdrawal of concomitant |
| | medications used for the treatment of pruritus may occur during the long term exposure period. |
| | With the exception of the Week 96 and Week 100 visit (Study |
| | Termination), Additional study drug will be supplied at each clinic visit |
| | during the follow-up treatment period. Used and unused study drug will |
| | be collected at every each clinic visit and dosing compliance will be assessed. |
| Section 5.6, End of Study | For subjects who do not consent to the long-term optional follow-up treatment period, a subject is considered to have completed |
| | treatment if treatment was not permanently discontinued prior to |
| | the Week 48 visit. A follow-up phone contact is required for all |
| | subjects should the final visit occur earlier than 30 days from the final dose. |
| | The subject is considered to have completed treatment and study |
| | period for the corresponding follow-up treatment period (when |
| | consented under Protocol Amendment 3 or Protocol Amendment 4) |
| | if study treatment was not discontinued prior to completing Week<br>96 for Protocol Amendment 3 or completing the EOT visit in |
| | Schedule J under Protocol Amendment 4. Temporary drug |
| | interruption is not considered treatment discontinuation. A follow- |
| | up contact is required for all subjects should the final visit occur earlier than 30 days from the final dose. |
| | The end of study for the purposes of regulatory reporting is the point at |
| | which the last contact with the last subject during the protocol-specified |
| | scheduled follow-up period is made. |
| Section 6.1, Screening | Subjects will be enrolled in the optional follow-up treatment period based on the investigator's determination of meeting eligibility |
| | criteria outlined in Section 7. A subject will be considered enrolled |
| | in the long-term optional follow-up period under Protocol |
| | Amendment 4 after the subject consents and the investigator has |
| | determined the subject meets study entry eligibility criteria per<br>Protocol Amendment 4. However, any subject who consents to |
| | Protocol Amendment 4 and does not meet criteria per the |
| | investigator is considered a screen failure for the long-term optional |
| | follow-up period under Protocol Amendment 4. Screen failures are eligible for rescreening (Section 8.1.1). |
| Section 8.1.1, Screening Period (Day - | In the absence of documented JAGGED1 or NOTCH2 mutation prior to |
| 28 to Day -1) | screening, genetic testing may be performed for JAGGED1 and/or NOTCH2 (Spinner et al., 2000). |
| | For subjects who do not have documentation of a JAGGED-1 or |
| | NOTCH2 mutation, a blood sample may be obtained for genotyping |
| | Rescreening: Subject data pertaining to screening will be collected after the subject has been rescreened and determined to |
| Section | Description of Change |
|---|---|
| × + | meet eligibility. |
| Section 8.1.10, End of Treatment of Early Termination | Any subject subject who completes or withdraws from the study prior to completion of all treatment period clinic visits should undergo all procedures specified for the EOT/ET visit (see Schedule J). The following assessments are to be completed at the EOT/ET visit: safety and clinical laboratory evaluations, including determination of serum bile acids, lipid panel, other cholestasis biochemical markers, fat soluble vitamins, and plasma drug level. In addition and AFP. Female subjects who are of childbearing potential will have a urine pregnancy test. Study drug compliance will be assessed. Concomitant medications and adverse events will be collected. In addition, the following assessments Efforts must be made to follow subjects for at least 4 weeks following their last dose of study drug. |
| Section 8.1.11, Safety Follow-up<br>Period | A safety follow-up phone call will be made 30 days after the last dose of study drug. This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and adverse events noted during this phone call will be recorded. |
| Section 8.5.1, Itch Reported Outcome (ItchRO <sup>TM</sup> ); Section 8.5.2, Clinician Scratch Scale; Section 8.5.3, Clinician Xanthoma Scale; Section 8.5.4, Pediatric Quality of Life Inventory (PedsQL); Section 8.5.5, Patient Impression of Change; Section 8.5.6, Caregiver Impression of Change; Section 8.5.7, Caregiver Global Therapeutic Benefit | Edited text to indicate all assessments will be performed as outlined in the Schedule of Procedures in Section 16.1. |
| Section 8.6.1, Contraception Requirements | Sexually active female subjects of childbearing potential must continue to use acceptable contraception with their partners, or refrain from sexual activity, from the time of screening until the end of the study, throughout the study period and for 30 days following the last dose of the study drug. If hormonal contraceptives are used they should be administered according to the package insert. Females of child-bearing potential who are not currently sexually active must agree to use acceptable contraception, as defined below, if they become sexually active during the period of the study and 30 days following the last dose of the IP. Acceptable methods of contraception are: Acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized. a. Hormonal contraceptives (eg, oral contraceptive pill, depot, patch, intrauterine device, diaphragm with spermicidal ring), stabilized for at least 30 days if first use, plus condoms; and/or b. Barrier method, eg, (i) condom (male or female) or (ii) diaphragm, with spermicide; or c. Intrauterine device (IUD). d. or a sexual partner who is surgically sterilized. |

| Section | Description of Change |
|---|---|
| | Male Contraception: Contraception is required for all sexually-active male subjects and their partners. All male subjects agree not to donate sperm, and to use 1 of the following approved methods of contraception until 30 days following study discharge: |
| | <ul> <li>a. Male condom with spermicide</li> <li>b. Intrauterine device with spermicide (use by female sexual partner)</li> <li>c. Female condom with spermicide (use by female sexual</li> </ul> |
| | partner) d. Contraceptive sponge with spermicide (use by female sexual partner) e. Intravaginal system (eg, vaginal ring with spermicide, a |
| | diaphragm with spermicide, or a cervical cap with spermicide) (use by female sexual partner) f. Oral, implantable, transdermal, or injectable hormonal contraceptive (use by female sexual partner). |
| Section 8.6.2, Fasting Requirements | On these visit days study drug should be administered as usual (1 mL, 5 mL, or 0.5 mL 25 qAM, ac), in the morning 30 minutes before breakfast. |
| Section 9.1.1, LUM001 | Added new composition of LUM001 1.0 mL, 0.5 mL, and 0.25 mL Oral Solution tables. |
| Section 9.1.2, Placebo | Added new composition of placebo 1.0 mL, 0.5 mL, and 0.25 mL Oral Solution tables. |
| Section 10.1, Study Drug<br>Administration | The dose may also be down-titrated, at the investigator's discretion and in consultation with the sponsor medical monitor, for subjects experiencing intolerance (eg, gastrointestinal symptoms such as diarrhea, abdominal pain, cramping) to a given dose. If the subject is on twice daily dosing regimen, dose reduction should first be attempted with the afternoon dose. Subjects who were previously down-titrated may be rechallenged during the long-term exposure period. |
| | Study drug will be dispensed to subjects/caregivers at the study site. Each subject dose for subjects who weigh 10 kg or more-Subjects will be administered orally as a receive a grape-flavored solution containing study drug (LUM001 or placebo) using the syringes provided. Each subject dose for subjects who weigh less than 10 kg will be administered orally as once a 0.5 mL solution containing study drug (LUM001day (QD) or placebo twice a day (BID) using the syringes syringe provided. The daily volume administered will not change during the course of the study. Study drug first dose should be taken at least 30 minutes prior to the first meal of the day (qAM, ae) and should and the second dose, where applicable, should be taken at least 30 minutes prior to dinner (evening meal). The doses will not be administered q12h in order to better cover the luminal bile acid release associated with dinner and to minimize the risk of disturbing sleep due to the potential for abdominal pain and diarrhea at night. It is recommended that the doses should be taken approximately at the same time each day for the duration of the |

| Section | Description of Change |
|---|---|
| Section | treatment period. |
| Section 10.2, Treatment Compliance | Subjects and/or caregivers will be asked to complete a paper diary indicating when they took their study medication and when they ate breakfast and, for subjects who receive a BID regimen, when they ate dinner (evening meal). |
| Section 10.5.1, General Monitoring<br>Rules | If an individual subject exhibits a CTCAE Grade 3 treatment emergent toxicity laboratory abnormality, with the exception of the specific rules outlined below (Sections 10.5.2), dosing will can be suspended. Continued dosing with study drug may be considered or continued as per the investigator's judgement and following discussion with the sponsor medical monitor. If suspended the |
| | The Data Monitoring Committee (DMC) will be notified of any SAE as specified in the DMC charter. |
| Section 10.5.2, Safety Monitoring<br>Rules | Of note: the INR re-test should be conducted by the central laboratory, but may also be conducted at a local laboratory on an as needed basis In this case, the subjects should be retested locally, but normal laboratory ranges should be recorded, results should be made available to study investigators and medical monitors immediately |
| | The investigator should also assess the need to capture an AE, its severity according to the CTEAE directives and potential causality. These assessments should also include an evaluation of whether criteria for an SAE are fulfilled (see Section 11.2.3), in particular whether the event should be considered as an important medical event, ie. an event that would have met one of the other seriousness criteria in the absence of appropriate medical interventions. |
| Section 10.6, Adjustment of Dose | If an individual subject exhibits a treatment emergent CTCAE Grade 2 or greater drug-related GI toxicity, study drug dose may be lowered to a previously well tolerated dose; later attempts to escalate the dose are permitted. If the subject is on twice daily dosing regimen, dose lowering should first be attempted with the afternoon dose. |
| Section 11.3, Monitoring and<br>Recording of Adverse Events | In addition, AEs that occur while the subject is not enrolled in the study during a gap period will be collected as medical history unless the AE started within 30 days of last dose. |
| Section 11.3.1, Serious Adverse<br>Events | The collection of SAEs will begin after the subject signs the informed consent/assent form and stop at the end of the subject's follow up period which is defined as Week 52 for subjects who do not roll over into the optional treatment follow-up period, Week 100 for subjects who do roll over into the optional treatment follow up period, or 28 days after the last dose of study drug for those subjects that terminate prior to the Week 96 visit 30 days after the last dose of study drug. |
| Section 11.3.2, Non-serious Adverse<br>Events | The recording of non-serious AEs will begin after the subject signs the informed consent/assent form and will stop at the end of the subject's follow up period, which is defined as Week 52 for subjects who do not roll over into the optional treatment follow-up period, Week 100 for subjects who do roll over into the optional treatment follow up period, or 30 days after the last dose of study drug for those subjects that terminate prior to the Week 96 visit-30 days after the last dose of study drug. |
| Section, 11.3.3.2 Severity | Please also refer to Section 10.5.2 regarding specific safety |

| Section | Description of Change |
|---|---|
| | monitoring for liver chemistry tests given that subjects with ALGS may have abnormal liver enzyme levels at baseline. |
| Section 12.2.2, Efficacy Populations | The main population for efficacy will be the modified intention-to-treat population (MITT), defined as all subjects who were enrolled, received study medication through Week 18, had a reduction from baseline in serum bile acids of ≥50% at the Week 12 <b>or Week 18</b> measurement. |
| Section 12.2.5.1, Efficacy Variables | A sensitivity analysis will also be conducted using subjects who experienced a reduction from baseline in serum bile acids of ≥50% at the Week 48 measurement. in subjects who previously responded to LUM001 treatment, as defined by a reduction in ItchRO scale >1 point from baseline to Week 12 or Week 18. In addition, an analysis for a daily score defined as an average of morning and evening scores will be conducted. |
| Section 12.2.6.1, Safety Assessments | Serum alpha-fetoprotein (AFP) |
| Section 12.2.8.2, Laboratory Tests | Changes within a treatment group for selected safety measures will be assessed at Weeks 3, 6, 12, 18, 22, 28, 38, 48, 60, 72, 84, 96, and at additional time points during the 52-week and long-term optional treatment periods |
| Section 12.2.8.6, Serum Alpha-<br>fetoprotein | (new section) Assessments of serum AFP will be listed for individual subjects and summarized using descriptive statistics by study visit. |
| Section 16.1.2, Schedule of Procedures E-F | Added Overall Scheme and Corresponding Schedule of Procedures Added Schedule of Procedures E-F: Rollover under Protocol Amendment 4: Schedule of Procedures E – Extension of Long-term Optional Follow- up Treatment Period, for subjects ineligible for ADE, applicable as follows: • Subject did not yet complete the optional follow up treatment period as outlined under Protocol Amendment 3 and is able to consent to Protocol Amendment 4 activities without an interruption in LUM001 dosing, OR • Subject completed long-term optional follow up treatment period as outlined under PA3 and dosing interruption was <7 days. • Subject deemed ineligible for ADE. Schedule of Procedures F – Extension of Long-term Optional Follow-up Treatment Period, for subjects eligible for ADE, applicable as follows: • Subject did not yet complete the long-term optional follow up treatment period as outlined under Protocol Amendment 3. and is able to consent to Protocol Amendment 4 activities without an interruption in LUM001 dosing, OR • Subject completed the optional follow up treatment period as outlined under PA3 and dosing interruption was <7 days. • Subject deemed eligible for ADE. |
| Section 16.1.3, Schedule of Procedures G-I | Added Schedule of Procedures G-I: Rollover under Protocol<br>Amendment 4: |

| Section | Description of Change |
|---|---|
| | Schedule of Procedures <u>G</u> – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, applicable as follows: |
| | <ul> <li>Subject previously completed (or early terminated from) the<br/>optional follow up treatment period as defined under Protocol<br/>Amendment 3 and has subsequently experienced an<br/>interruption in LUM001 dosing ≥7days</li> </ul> |
| | <ul> <li>Subject is considered eligible for study re-entry under Protocol<br/>Amendment 4</li> </ul> |
| | <ul> <li>Subject eligibility will be assessed for afternoon dose<br/>escalation at Protocol Amendment 4 DE Week 8 shown in the<br/>table below.</li> </ul> |
| | o If subject is found to be <u>ineligible</u> for ADE, subject will move from Schedule G to Schedule H. If which is found to be aligible for ADE, which will |
| | O If subject is found to be <u>eligible</u> for ADE, subject will move from Schedule G to Schedule I. O In the ADE of the ADE, subject will move from Schedule I. |
| | Schedule of Procedures <u>H</u> – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, subject <u>ineligible</u> for ADE |
| | Schedule of Procedures <u>I</u> – Long-term Optional Follow-up Treatment Period: Re-entry under Protocol Amendment 4, subject <u>eligible</u> for ADE |
| | Added Schedule of Procedures $\underline{J}$ - Study Termination and End of Treatment Procedures |
| Section 16.2, List of Laboratory<br>Analytes | Added alpha-fetoprotein (AFP) under Marker of hepatocellular carcinoma |
| Section 16.7, Pediatric Quality of Life Inventory (PedsQL <sup>TM</sup> ) | Subjects will continue to fill out the same questionnaire used at baseline for continuity of data collection, regardless of subsequent birthdays after the baseline visit. |

## 16.13.3 Protocol Amendment 3 Summary of Changes

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BLIND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN API<u>C</u>AL S<u>O</u>DIUM-DEPE<u>N</u>DENT B<u>I</u>LE A<u>C</u>ID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 3

**Date:** 13 Nov 2015

The changes below were made to Protocol Amendment 2.

The following table provides a summary list of changes that were included in Protocol Amendment 3 (*new text indicated in bold; deleted text indicated in strikethrough*):

| Section | Description of Change |
|---|---|
| Title Page,<br>Sponsor<br>Medical<br>Monitor | Added: Sponsor Medical Monitor: Susanne Schmidt, MD, PhD Premier Research Office: +1 215 282 5406 Cell: +1 267 838 2380 Email: medmonitorLUM304@premier-research.com |
| Title Page,<br>Medical Lead | Changed from: Ciara Kennedy, PhD Lumena Pharmaceuticals, Inc. Phone: 00-1-858-337-7922 Email: cikennedy@shire.com To: Beatriz Caballero, MD Shire, Inc. Zahlerweg 10 6300 Zug Switzerland Phone: +41(0) 41 288 42 30 Email: bcaballero@shire.com |
| Study<br>Synopsis,<br>Objectives;<br>Section 3,<br>Study<br>Objectives | <ul> <li>To evaluate the effect of LUM001 on serum bile acid levels in children with ALGS.</li> <li>To evaluate the effect of LUM001 on biochemical markers of cholestasis and liver disease in children with ALGS.</li> <li>To evaluate the effect of LUM001 on pruritus in children with ALGS.</li> <li>To evaluate the long-term durability of effect of LUM001 in children with ALGS 48-weeks of treatment.</li> <li>To evaluate the long-term safety and tolerability of LUM001 in children with ALGS.</li> <li>Objectives of Optional Follow-up Treatment Period (After Week 48):</li> <li>To offer eligible subjects treated in the LUM001-304 study continued study treatment after Week 48 until the first of the following occur: (i) up to 52 weeks of additional treatment (Week 100), or (ii) in the event that a new study opens to enrollment.</li> <li>To obtain safety and efficacy data in patients treated long term on LUM001 including genotyping characteristics.</li> </ul> |
| Synopsis (Section 1), Study Design and Overall Study Duration and Follow-up (Sections 5.1 and 5.4), Schedule of Procedures (Appendix 16.1) | This is a long-term, open-label study with a double-blind, placebo-controlled, randomized drug withdrawal period in children with ALGS designed to evaluate the safety and efficacy of LUM001. The study is divided into 5 parts: a 6-week open-label, dose escalation period at doses up to 400 µg/kg/day, a 12-week stable dosing period, a 4-week randomized, double-blind, placebo-controlled drug withdrawal period, a 26-week long-term stable dosing period at doses up to 400 µg/kg/day, and an optional 52-week follow-up treatment period for eligible subjects who choose to stay on treatment with LUM001. Subjects' participation in the optional follow-up treatment period will continue until the first of the following occur: (i) completion of 52 weeks of additional treatment (Week 100), or (ii) in the event that a new study of LUM001 opens to enrollment. |
| | This is a long term, open label study with a double blind, placebo controlled, randomized drug withdrawal period in children with ALGS designed to evaluate the safety and efficacy |

| Section | Description of Change |
|---|---|
| | of LUM001. The study is divided into 4 parts: a 6 week open label, dose escalation period at doses up to 400 μg/kg/day, a 12 week stable dosing period, a 4 week randomized, double blind, placebo controlled drug withdrawal period, and a 26 week long term stable dosing period at doses up to 400 μg/kg/day. |
| Synopsis (Section 1), | Exclusion Criteria |
| Study | Subjects will be excluded from the study if they meet any of the following criteria: |
| population<br>(Section 7) | <ol> <li>Chronic diarrhea requiring ongoing intravenous fluid or nutritional intervention.</li> <li>Surgical interruption of the enterohepatic circulation.</li> </ol> |
| | 3. Previous liver transplant. |
| | 4. Decompensated cirrhosis [ALT >15 x ULN, INR >1.5 (unresponsive to vitamin K therapy), albumin <3.0 g/dL, history or presence of clinically significant ascites, variceal hemorrhage, and/or encephalopathy]. |
| | 5. History or presence of other concomitant liver disease. |
| | 6. History or presence of any other disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs, including bile salt metabolism in the intestine (eg, inflammatory bowel disease). |
| | 7. History or presence of gallstones or kidney stones. |
| | 8. Known diagnosis of human immunodeficiency virus (HIV) infection. |
| | 9. Cancers, except for in situ carcinoma, or cancers treated at least 5 years prior to Screening with no evidence of recurrence. |
| | 10. Recent medical history or current status that suggests that the subject may be unable to complete the study. |
| | 11. Any female who is pregnant or lactating or who is planning to become pregnant during the study period. |
| | 12. Known history of alcohol or substance abuse. |
| | 13. Administration of bile acid or lipid binding resins within 28 days prior to screening and throughout the trial. |
| | 14. Known hypersensitivity to LUM001or any of its components. |
| | 15. Receipt of investigational drug, biologic, or medical device within 28 days prior to Screening, or 5 half-lives of the study agent, whichever is longer. |
| | 16. History of non-adherence to medical regimens, unreliability, mental instability or incompetence that could compromise the validity of informed consent or lead to non-adherence with the study protocol based upon investigator judgment. |
| | 17. Any other conditions or abnormalities which, in the opinion of the investigator or <b>sponsor</b> medical monitor, may compromise the safety of the subject, or interfere with the subject participating in or completing the study. |
| | 18. Subjects weighing over 50 kg at screening. |
| | Fligible cubicate for the 52 week follow up wasiads |
| | Eligible subjects for the 52-week follow-up period: Subjects will be considered eligible for the optional 52-week follow-up treatment period if they have: |
| | Completed the protocol through the Week 48 visit with no safety concerns. Subjects who were discontinued due to safety reasons can be rechallenged if blood tests are back to relatively normal values for this patient population and subject does not meet any of the protocol's stopping rules. The decision will be made by the investigator in |

| Section | Description of Change |
|---|---|
| | consultation with the sponsor medical monitor. |
| | • Subjects who have undergone a surgical disruption of the enterohepatic circulation will not be eligible to enter into the follow up treatment period. |
| | • Subjects who were discontinued for other reasons will be considered for the optional 52-week follow-up treatment period on an individual basis. The decision will be made by the investigator in consultation with the sponsor medical monitor. |
| Synopsis<br>(Section 1) | All subjects will receive LUM001, up to 400 µg/kg/day or a maximum daily dose of 20 mg/day. After completion of the 12-week stable dosing period, subjects will be randomized 1:1 to either a 4-week study drug withdrawal period during the study or will remain on study drug. Subjects will then enter a 26-week long-term stable dosing period and all subjects will receive LUM001, up to 400 µg/kg/day or a maximum daily dose of 20 mg/day. Subjects will then be considered for an optional 52-week follow-up treatment, if eligible, to continue on their highest tolerated dose. |
| Synopsis | Optional Follow-up Treatment Period |
| (Section 1),<br>Study Design<br>(Section 5.1) | At Week 48, all subjects will be assessed by the investigator to determine their willingness and eligibility to roll-over into the 52-week, follow-up treatment period. The 3 following possible scenarios may occur: |
| | • Subjects who are eligible to roll over into the optional follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level. |
| | • Subjects who are eligible to roll over into the optional follow-up treatment period with a LUM001 dosing interruption of ≥7 days, will be dose escalated up to 400 μg/kg/day or highest tolerated dose following a 5-week dose escalation beginning at 35 μg/kg/day. |
| | • Subjects who do not wish to enter the follow-up treatment period will be contacted via telephone by the study site approximately 28 days after the last dose of study drug. |
| | During the study, the study drug may be adjusted if there is a change of $\geq 10\%$ in weight since the screening visit or if there is a change of $\geq 10\%$ in weight since the last weight-based medication adjustment to maintain the target dose ( $\mu g/kg/day$ ). |
| | The anticipated adverse reaction or intolerance is gastrointestinal in nature (e.g., diarrhea, abdominal pain, cramping, etc.). During the respective escalation periods, in the absence of intolerance, escalation to the next dose level for an individual subject will occur following a scheduled phone call or visit (see Schedule of Procedures, Section 16.1). |
| | If a subject experiences intolerance due to gastrointestinal <b>symptoms</b> (eg, diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the sponsor medical monitor may lower the dose to a previously tolerated dose. At the investigator's discretion, subjects who had their dose reduced due to intolerability may have a one time dose re challenge during the long term exposure period with a higher dose. |
| Synopsis | Added to synopsis: |
| (Section 1),<br>Overall Study<br>Duration and<br>Follow-up | For subjects in the 52-week optional follow-up treatment period with ≥7 days since the last dose of LUM001, dosing will start at 35 µg/kg/day, and will then be increased over the first 5 weeks up to 400 µg/kg/day or to the maximum tolerated dose. This escalation |
| (Section 5.4) | regimen is supported by the safety profile observed in completed and ongoing clinical studies of LUM001 and allows for subjects to reach 400 µg/kg/day or a maximum tolerated dose within a 5-week period. The dose may be down-titrated, at the investigator's discretion and in consultation with the sponsor medical monitor, for |







| Section | Description of Change |
|---|---|
| | event that a new study opens to enrollment, whatever occurs first. |
| | Subjects who are eligible to roll over into the follow-up treatment period with no LUM001 dosing interruption or an interruption of <7 days will be maintained at the same dose level. Telephone contacts to occur at Week 52 and Week 56. During the follow-up treatment period, subjects will return to the clinic at Weeks 60, 72, 84, 96, and 100; and telephone contacts to occur at Weeks 64, 68, 76, 80, 88, and 92. |
| | Subjects with ≥7 days since last dose of LUM001 will be dose escalated up to 400 μg/kg/day or to the highest tolerated dose with 35 μg/kg/day. This escalation regimen is supported by the safety profile observed in completed and ongoing clinical trials of LUM001 and allows for subjects to reach 400 μg/kg/day or highest tolerated dose within a 5-week period. The dose escalation (DE) period will proceed as follows: |
| | <ul> <li>Week DE-2 Clinic Visit: obtain consent, weight, and draw blood for laboratory<br/>analyses.</li> </ul> |
| | <ul> <li>Week DE 0 Clinic Visit: PI evaluates laboratory results, study drug is dispensed, and<br/>subject begins at 35 μg/kg/day dose level (if no safety concerns).</li> </ul> |
| | • Week DE 49 Telephone Contact: subject escalates to 70 μg/kg/day dose level. |
| | <ul> <li>Week DE 50 Telephone Contact: subject escalates to 140 μg/kg/day dose level if prior<br/>dose level was tolerated.</li> </ul> |
| | <ul> <li>Week DE 51 Telephone Contact: subject escalates to 280 μg/kg/day dose level if prior<br/>dose level was tolerated.</li> </ul> |
| | <ul> <li>Week DE 52 Clinic Visit: laboratory tests and dose escalates to 400 μg/kg/day dose<br/>(maximum daily dose of 20 mg), if prior dose level was tolerated.</li> </ul> |
| | If any subject experiences intolerance, the investigator, in consultation with the sponsor medical monitor, may lower the dose to a previously tolerated dose at any time during the entire follow-up treatment period. At the investigator's discretion, and in consultation with the sponsor medical monitor subjects who were previously down titrated may be rechallenged during the follow-up treatment period. |
| | Safety and clinical laboratory evaluations and a physical exam (including collection of vital signs, height and weight measurements) will be completed at each clinic visit. In addition, the clinician scratch scale, clinician xanthoma scale, and PedsQL will be administered and study drug compliance will be assessed (PedsQL will not be performed at DE-2 or DE52). The Patient and Caregiver Impression of Change (PIC & CIC), and the Caregiver Global Therapeutic Benefit assessments will be completed at Weeks 84, 96, and 100. Subjects/caregivers will receive follow-up phone calls at Weeks 64, 68, 76, 80, 88, and 92. Concomitant medications and any AEs will be evaluated and recorded at all clinic visits and at scheduled telephone contacts. |
| | Twice daily completion of the electronic diary will be required by caregivers and age appropriate subjects during the 2 weeks following the Week 60, 72, 84, and 96 clinic visits. Electronic diaries will be provided to subjects and caregivers at these visits and re-training on the use of the diary will occur, as appropriate. |
| | At the physician investigator's discretion, withdrawal of concomitant medications used for the treatment of pruritus may occur during the long-term exposure period. |
| | With the exception of the Week 96 and Week 100 visit (Study Termination), additional study drug will be supplied at each clinic visit during the follow-up treatment period. Used and unused study drug will be collected at every visit. |

| Section | Description of Change |
|---|---|
| | Subjects will be encouraged to complete all study activities and visits. Any subject who withdraws from the study prior to completion of all treatment period clinic visits should undergo safety and clinical laboratory evaluations, including determination of serum bile acids, other cholestasis biochemical markers, fat soluble vitamins, and plasma drug level. In addition the following assessments should be completed: the ItchRO (Pt and Obs), the clinician scratch scale, clinician xanthoma scale, the PedsQL, the Patient Impression of Change, the Caregiver Impression of Change, and the Caregiver Global Therapeutic Benefit assessments, as defined for ET (see Schedule of Procedures, Section 16.1) Efforts must be made to follow subjects for at least 4 weeks following their last dose of study drug. |
| | At completion of the Follow-up Treatment Period: a safety follow-up phone call will be made 4 weeks after the last dose of study drug (Week 100). This call will be made for all subjects who complete the study, as well as any subject who terminates from the study early. Concomitant medications and adverse events noted during this phone call will be recorded. |
| Synopsis | From the synopsis: |
| (Section 1),<br>Pruritus and<br>Quality of Life | Evaluations for the durability of the therapeutic effect will be the mean change from Baseline (Day 0) to Week 18, prior to randomization, and the change from Week 18 to Week 48 in: |
| Assessments (Section 8.5), Efficacy | Biochemical markers of cholestasis and liver disease [alanine aminotransferase (ALT), alkaline phosphate (ALP), gamma-glutamyltransferase (GGT) and bilirubin (total and direct)]. |
| Variables<br>(Section<br>12.2.5.1) | Pruritus as measured by the electronic diary ItchRO instruments (ItchRO(Obs), caregiver instrument/ItchRO(Pt) patient instrument). |
| | The change from Baseline (Day 0) to Week 48 in xanthomas, as measured by clinician xanthoma scale will also be evaluated. |
| | Additional assessments of efficacy variables will occur during the 52-week optional treatment period. For subjects entering the 52-week optional treatment period with ≥7 days since last dose of LUM001, any of the above evaluations may also occur at clinic visits during the DE period. |
| | Additional exploration of evaluations of safety and the durability of the therapeutic effect will be specified in the statistical analysis plan. |
| | Section 8.5: |
| | 8.5 Pruritus and Quality of Life Assessments |
| | 8.5.1 Itch Reported Outcome (ItchRO <sup>TM</sup> ) |
| | ALGS subjects/caregivers will be required to submit twice daily assessments using the electronic diary for the duration of the study. Electronic diaries will be returned to the study site at the Week 48 clinic visit (or sooner if the subject has withdrawn from the study before the Week 48 visit). For subjects who enter the optional follow-up treatment period, daily completion of the diary will also occur during the 2 weeks following the Week 60, 72, 84, and 96 clinic visits. |
| | 8.5.2 Clinician Scratch Scale |
| | A clinician's assessment of pruritus made by the principal investigator or appropriate designee using the clinician scratch scale (Section 16.5) will be recorded at screening, Day 0 (baseline), Weeks 3, 6, 12, 18, 22, 28, 38, and 48. For subjects who enter the optional follow-up treatment period the clinician scratch scale will be recorded at Weeks 60, 72, 84, 96, and 100. For subjects with interruptions in LUM001 dosing of ≥7 days, assessments will also |

| Section | Description of Change |
|---|---|
| | be conducted during the DE period at DE -2, DE Day 0, and DE 52. |
| | 8.5.3 Clinician Xanthoma Scale |
| | A clinician's assessment of xanthomatosis will be made by the principal investigator or appropriate designee using the clinician xanthoma Scale (Section 16.6). This assessment will be completed at Baseline (Day 0) and at Weeks 18, and 48. For subjects who enter the optional follow-up treatment period the clinician xanthoma scale will be recorded at 60, 72, 84, 96, and 100. For subjects with interruptions in LUM001 dosing of ≥7 days, assessments will also be conducted during the DE period at DE Day 0, and DE 52. |
| | 8.5.4 Pediatric Quality of Life Inventory (PedsQL) |
| | The PedsQL™ is a questionnaire that will be administered to subjects and/or caregivers at the Week 0 (baseline), 18, 22, and 48. For subjects who enter the optional follow-up treatment period, the PedsQL will be administered at Weeks 60, 72, 84, 96, and 100 using the age-appropriate PedsQL module (see Section 16.7). For subjects with interruptions in LUM001 dosing of ≥7 days, the PedsQL will also be administered at DE Day 0. The PedsQL is a validated, modular instrument designed to measure health-related quality of life (HRQoL) in children and adolescents (Varni, Seid, & Kurtin, 2001). In addition to the core generic PedsQL module, the multidimensional fatigue and family impact questionnaire will also be administered at the Week 0 (baseline), 18, 22, and Week 48 using the age-appropriate module (see Section 16.7). Age at baseline will be used as the age for the determination of the appropriate module to be used for the study and this same module will be used for the duration of the study (regardless of subsequent birthdays after the baseline visit). |
| | 8.5.5 Patient Impression of Change |
| | The Patient Impression of Change (PIC) is designed to assess the subject's perception of his/her itching after various points of study drug treatment compared to his/her itching prior to the start of treatment with study drug. The PIC will be completed, by subjects who were 9 years of age or older at the Week 18, 22, and 48 visits. For subjects who enter the optional follow-up treatment period, the PIC will be completed by subjects who were 9 years of age or older at the Week 60, 72, 84, 96, and 100 visits (see Section 16.8). |
| | 8.5.6 Caregiver Impression of Change |
| | The Caregiver Impression of Change (CIC) is designed to assess the caregiver's perception of the subject's itch related symptoms and xanthoma severity after various points of study drug treatment compared to his/her itch related symptoms and xanthoma severity prior to the start of treatment with study drug. The CIC will be completed by all caregivers at the Week 18, 22, and 48 visits. For subjects who enter the optional follow-up treatment period the CIC will be completed at Week 84, 96, and 100 visits (see Section 16.9). |
| | 8.5.7 Caregiver Global Therapeutic Benefit |
| | The Caregiver Global Therapeutic Benefit (CGTB) questionnaire is designed to assess the caregiver's perception of the treatment benefits on the subject's itching compared to the side effects experienced with study drug. The CGTB will be completed by all caregivers at the Week 18, 22, and 48 visits. For subjects who enter the optional follow-up treatment period the CGTB will be completed at Week 84, 96, and 100 visits (see Section 16.10). |
| | Section 12.2.5.1: |
| | The following additional efficacy evaluations will be assessed: |
| | Change from baseline to Weeks 18, 22, 48, <b>60, 72, 84, 96, and 100</b> in: o Fasting serum bile acid levels. |

| Section | Description of Change |
|---|---|
| Section | Liver enzymes (ALT, ALP) and bilirubin (total and direct). |
| | <ul> <li>Pruritus as measured by the average daily ItchRO (Observer ItchRO/patient ItchRO).</li> </ul> |
| | Other biochemical markers of cholestasis [total cholesterol, low-density lipoprotein cholesterol (LDL-C)]. |
| | <ul> <li>Bile acid synthesis [serum 7α-hydroxy-4-cholesten-3-one (7αC4)].</li> </ul> |
| | Responder analysis at Weeks 18, 48, <b>60, 72, 84, 96, and 100</b> in: |
| | <ul> <li>Pruritus response rates as measured by ItchRO (Observer ItchRO/patient ItchRO)</li> </ul> |
| | Clinician scratch scale |
| | Change from baseline for PedsQL at Week 18, 22, 48, 60, 72, 84, 96, and 100 and change from Week 18 to Week 22. |
| | <ul> <li>Patient Impression of Change (PIC) at Week 18, 22, 48, 84, 96, and 100 and change from Week 18 to Week 22.</li> </ul> |
| | <ul> <li>Caregiver Impression of Change (CIC) at Week 18, 22, 48, 84, 96, and 100 and change from Week 18 to Week 22.</li> </ul> |
| | <ul> <li>Caregiver Global Therapeutic Benefit (CGTB) assessment at Weeks 18, 22, 48, 84,</li> <li>96, and 100 and change from Week 18 to Week 22.</li> </ul> |
| | Evaluations for the durability of the therapeutic effect will be the mean change from Baseline (Day 0) to Week 18, prior to randomization, and the change from Week 18 to Week 48 and Week 18 to Week 100 in: |
| | <ul> <li>Biochemical markers of cholestasis and liver disease [alanine aminotransferase (ALT), alkaline phosphate (ALP), gamma-glutamyltransferase (GGT) and bilirubin (total and direct)].</li> <li>Pruritus as measured by the electronic diary ItchRO instruments (ItchRO(Obs),</li> </ul> |
| | caregiver instrument/ItchRO(Pt) patient instrument). The change from Baseline (Day 0) to Week 48 and to Week 100 in xanthomas, as measured by clinician xanthoma scale will also be evaluated. |
| | For subjects entering the 52-week optional treatment period with ≥7 days since last dose of LUM001, any of the above evaluations may also occur at clinic visits during the DE period. Additional exploration of evaluations of durability of therapeutic effect will be specified in the statistical analysis plan. |
| Dose<br>Escalation<br>Period<br>(Section 5.5.2.1 | The anticipated adverse reaction or intolerance is gastrointestinal in nature (e.g., diarrhea, abdominal pain, cramping, etc.). In the absence of intolerance as determined by the physician investigator, escalation to the next dose level for an individual subject will occur following a scheduled phone call or visit (see Schedule of Procedures, Section 16.1). |
| ) | If a subject experiences intolerance due to gastrointestinal symptoms (eg, diarrhea, abdominal pain, cramping) at any time during the study, the physician investigator in consultation with the sponsor medical monitor may lower the dose to a previously tolerated dose. In these circumstances an unscheduled visit will occur and the appropriate replacement study medication will be issued to the subject as quickly as possible. |
| Genetic Testing (Section 8.2) and List of Laboratory Analytes | JAGGED1 and NOTCH2 mutations can be predictive of ALGS. For ALGS subjects who meet clinical diagnostic criteria for ALGS (see Section 16.3) but do not have documentation of a JAGGED1 or NOTCH2 mutation, the clinical diagnosis of ALGS may be confirmed by genotyping. Genetic counseling, as appropriate, will be provided to subjects and their legal caregivers. Subjects for whom prior genotyping was performed may need to have an optional repeat analysis performed if the original information collected at screening was |

| Section | Description of Change | |
|---|---|---|
| (Appendix 16.2) | insufficient for complete documentation of the diagnosis of ALGS including the type of mutation recorded. For those participants for which the type of the mutation cannot be documented, genetic testing may be conducted and the results recorded. | |
| Study Drug | Table 1: Composition of LUM001 1.0 mL Oral Solution | |
| Description (Section 9.1) | Component | Quantity per 1.0 mL |
| (300001711) | LUM001 | <b>0.02</b> <del>0.05</del> to 20 mg |
| | Propylene Glycol | 250 mg |
| | Sucralose | 7.5 mg |
| | Grape Flavoring Agent | 5 mg |
| | Water | q.s. to 1.0 mL |
| | Table 2: Composition of LUM001 0.5 mL Oral Solution | |
| | Component | Quantity per 0.5 mL |
| | LUM001 | <b>0.02</b> 0.05 to 20 mg |
| | Propylene Glycol | 125 mg |
| | Sucralose | 3.75 mg |
| | Grape Flavoring Agent | 2.5 mg |
| Monitoring and | Water | q.s. to 0.5 mL<br>gns and/or symptoms present in a subject prio |
| Recording<br>Adverse Events<br>(Section 11.3) | the study (i.e., before informed consent) should be recorded as Medical History and not recorded as AEs unless the pre-existing condition worsened. Symptoms of the disease under study should not be classed as AEs as long as they are within the normal day-to-day fluctuation or expected progression of the disease and are part of the efficacy data to be collected in the study; however, significant worsening of the symptoms should be recorded as an AE. The investigator should always group signs and symptoms into a single term that constitutes a single unifying diagnosis if possible. 11.3.1 Serious Adverse Events | |
| | In the interest of subject safety, and in order to fulfill regulatory requirements, all SAEs (regardless of their relationship to study drug) should be reported to the sponsor or designee within 24 hours of the study center's first knowledge of the event. The collection of SAEs will begin after the subject signs the informed consent/assent form and stop at the end of the subject's follow-up period which is defined as Week 52 for subject who do not roll over into the optional treatment follow-up period, Week 52 100 for subjects who do roll over into the optional treatment follow-up period, or 28 days after the last dose of study drug for those subjects that terminate the prior to the Week 48 100 visit. 11.3.2 Non-serious Adverse Events | |
| | The recording of non-serious AEs will begin after the subject signs the informed consent/assent form and will stop at the end of the subject's follow-up period, which is defined as Week 52 for subjects who do not roll over into the optional treatment follow-up period, Week 100 for subjects who do roll over into the optional treatment follow-up period, or 30 days after the last dose of study drug for those subjects that terminate prior to the Week 100 visit. The investigator will monitor each subject closely and record all observed or volunteered | |

| Section | Description of Change |
|---|---|
| | AEs on the Adverse Event Case Report Form. |
| Subject<br>Disposition<br>(Section<br>12.2.4.1) | Subject disposition will be summarized descriptively. The number and percentage of subjects enrolled, completed, and withdrawing, along with reasons for withdrawal, will be tabulated overall, and by study phase and treatment group. For purposes of analysis there will be 3 study phases: Dose escalation/stable dose (Weeks 0-18), Randomized Withdrawal (Weeks 19-22) and Long-Term Exposure (Weeks 23-48 and 23-100). |
| Laboratory<br>Tests (Section<br>12.2.8.2) | A separate listing will present laboratory values of all subjects who change from normal to abnormal or from abnormal to normal during the course of the study, where normal ranges for this population are outlined in the SAP. Changes within a treatment group for selected safety measures will be assessed at Weeks 3, 6, 12, 18, 22, 28, 38, 48, 60, 72, 84, 96, and final study evaluation visit using methods to be specified in the SAP prior to unblinding the data. |
| Schedule of | Added to Screening – Week 22 (footnote): |
| Procedures<br>(Section 16.1) | Optional genotype sample will be performed to provide a full characterization and the associated documentation of the mutation in support of the diagnosis of ALGS. |
| | Schedule of Procedures (cont'd) – Long-term Exposure: Week 23–Week 48: "Study Termination" removed. |
| | Schedule of Procedures – Follow-up Treatment Period (FTP) for Those Subjects <7 Days from the Last Dose of LUM001 and Schedule of Procedures – Follow-up Treatment Period for Those Subjects ≥ 7 Days from the Last Dose of LUM001added. |
| List of | NOTCH2 added. |
| Laboratory<br>Analytes<br>(Section 16.2) | |
| Overall change | Throughout the protocol, reference evaluating durability of effect of LUM001 was removed. Durability of effect may not be assessed in this study, as a treatment effect has not yet been established, and the randomized withdrawal design is not statistically powered. |

## 16.13.4 Protocol Amendment 2 Summary of Changes

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BL<u>I</u>ND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN APICAL SODIUM-DEPENDENT BILE ACID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 2

**Date:** 08 May 2015

The changes below have been made to Protocol Amendment 1.

The following table provides a summary list of changes to Protocol Amendment 2:

| Section | Description of Change |
|---|---|
| Study Synopsis and Section 7 | Exclusion criteria added: 18. Subjects weighing over 50 kg at screening. |
| Study Synopsis | "26-week <u>open label</u> period" changed to "enter a 26-week <u>long-term stable dosing</u> period" |
| Study Synopsis, Section 4.5 | "equivalent to approximately 30 mg daily dose in a 70 kg adult" changed to "equivalent to approximately 20 mg daily dose in a 50 kg subject" |
| Study Synopsis; Sections 5.5.2.1, 5.5.2.4, and 8.1.5 | Maximum daily dose changed from 30 mg/day to 20 mg/day. |
| Study Synopsis, Section 8.1.3, Table 6 and Table 7 | Time of usage of placebo corrected to the following: |
| | "Study drug (or placebo) will be supplied at Weeks 12 and study drug (or placebo) supplied at Week 18." |
| | changed to: |
| | "Study drug will be supplied at Week 12 and study drug (or placebo) supplied at Week 18." |
| Study Synopsis and Sections 6.2, 12.2.2, and 12.2.5.1 | Responder definition corrected from Week 18 to Week 12:serum bile acid levels from baseline to Week 12 serum bile acids ≥50% at the Week 12 measurement |
| Study Synopsis; Section 8.1.3; Section 16.1:<br>Schedule of Procedures – Screening – Week 22,<br>Footnote d;<br>Section 16.1: Schedule of Procedures – Long-Term<br>Exposure: Week 23 – Week 48 / Study Termination,<br>Footnote c | "2 to 4 hours post-dosing" changed to "approximately 4 hours post-dosing" |
| Study Synopsis, Section 12.2.3 | Language added to address the randomization and statistical management of data generated from siblings |

| Section | Description of Change |
|---|---|
| | enrolled in the study: |
| | Siblings The enrollment of siblings is allowed. During the placebocontrolled, randomized drug withdrawal period, siblings will be assigned in a blinded manner to the same treatment arm. The data from all enrolled participants (including siblings) will be used for the safety analysis. For the efficacy analysis, data from only one of the siblings will be used. The choice of which subject's data to use in the efficacy analysis will be done in a random fashion before the LUM001-304 study is unblinded. Details of the analysis methods will be outlined in the SAP. |
| Section 5.5.3, Section 8.1.8 | Language added to describe a planned extension study: Subjects who complete the study may be eligible for participation in an extension study of LUM001. |
| Section 6.2 | Language added to address the randomization of siblings enrolled in the study: During the placebo-controlled, randomized drug withdrawal period, siblings will be assigned in a blinded manner to the same treatment arm. |
| Section 6.4, Section 12.2.4.1 | Randomized withdrawal period corrected from "Weeks <u>18</u> -22" to "Weeks <u>19</u> -22" |
| Section 8.5.4 | "Age at screening" changed to "Age at baseline" "birthdays after the screening visit" changed to "birthdays after the baseline visit" |
| Section 10.1 | "at least <u>8 weeks</u> " changed to"at least <u>12 months</u> " |
| Sections 10.5.2.4, Section 16.2 | "tocopherol $[(\alpha)]$ , total lipids" changed to "tocopherol $[\alpha]$ " Total lipids removed from 16.2 table. |
| Section 16.1, Schedule of Procedures – Long-Term Exposure: Week 25 – Week 48 / Study Termination | Header changed to: Long-Term Exposure: Week 23 – Week 48 |
| Section 16.1, Schedule of Procedures – Long-Term Exposure: Week 23 – Week 48 / Study Termination | Study days corrected to: 161, 168, 175, 182, 189, 196, 231, 266, 301 |

## 16.13.5 Protocol Amendment 1 Summary of Changes

**Protocol Number:** LUM001-304

**Protocol Title:** LONG-TERM, OPEN-LABEL STUDY WITH A DOUBLE-BL<u>I</u>ND,

PLACEBO-CONTROLLED, RANDOMIZED DRUG WITHDRAWAL PERIOD OF LUM001, AN API<u>C</u>AL S<u>O</u>DIUM-DEPE<u>N</u>DENT B<u>I</u>LE A<u>C</u>ID TRANSPORTER INHIBITOR (ASBTi), IN PATIENTS WITH

ALAGILLE SYNDROME

Amendment: 1

**Date:** 06 Mar 2015

The changes below were made to the original protocol.

The following table provides a summary list of changes that were included in Protocol Amendment 1:

| Section | Description of Change |
|---|---|
| Exclusion Criteria (Section 1, Synopsis and Section 7, Subject Eligibility) | Additional exclusion criteria were added: • History or presence of gallstones or kidney stones. |
| | Known hypersensitivity to LUM001 or any of its components. |